#### Statistical Analysis Plan

Main Study ID: 201584

Main Study Official Title: A Phase III, Randomized, Multicenter, Parallel-group, Open-Label Study Evaluating the Efficacy, Safety, and Tolerability of Long-Acting Intramuscular Cabotegravir and Rilpivirine for Maintenance of Virologic Suppression Following Switch from an Integrase Inhibitor Single Tablet Regimen in HIV-1 Infected Antiretroviral Therapy Naive Adult Participants

NCT ID for Main Study: NCT02938520

**Sub-Study ID:** 201584-001

**Sub-Study Official Title:** An Amendment to the FLAIR Study to Evaluate the Pharmacokinetics, Safety, Tolerability, Maintenance of Virological Suppression and Patient Reported Outcomes for Participants Receiving Cabotegravir (CAB 200 mg/mL) and Rilpivirine (300 mg/mL) Long-Acting Injections Following Subcutaneous (SC) Administration in the Anterior Abdominal Wall SC Tissue Compared With Intramuscular (IM) Administration in the Gluteus Medius Muscle in Adult Participants Living With HIV-1 Infection in the FLAIR Study

NCT ID for Sub-Study: NCT05896748

Date of Document of Sub-Study: 03-Aug-2023

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : 201584: A Phase III, Randomized, Multicenter, Parallel-group, Open-Label Study Evaluating the Efficacy, Safety, and Tolerability of Long-Acting Intramuscular Cabotegravir and Rilpivirine for Maintenance of Virologic Suppression Following Switch from an Integrase Inhibitor Single Tablet Regimen in HIV-1 Infected Antiretroviral Therapy Naive Adult Participants

Compound Number : GSK1265744

Effective Date : 03-AUG-23

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Subcutaneous Sub-study Clinical Study Report for Protocol 201584. Reporting details pertaining to the primary Week 48 and the earlier analyses (Week 96 and Week 124) have been retained for completeness.
- This version of the RAP includes amendments to the originally approved RAP.

#### **RAP Author(s):**

| 02 ALIC 22 |
|------------|
| 03-AUG-23 |

Copyright 2023 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

# **RAP Team Review Confirmations (Method: E-mail)**

| Approver | | Date |
|---|---|---|
| PPD | | 03-AUG-23 |
| _ ` | evelopment Scientist, ViiV Healthcare) | |
| PPD | | 03-AUG-23 |
| Clinical Study Manager (Global Clinical Sciences & Delivery, | | |
| GSK) | | |
| PPD | | 03-AUG-23 |
| Principle Pr | | |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | | Date |
|----------|----------------------------------------|-------------|
| PPD | | 03-AUG-23 |
| PPD | , Statistics (GSK Clinical Statistics) | |
| PPD | | 03-AUG-23 |
| PPD | | V3 116 G 25 |
| PPD | | 03-AUG-23 |
| PPD | , ViiV Healthcare) | |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | | DUCTIONRAP Amendments | |
| 2. | CLIMANA | ARY OF KEY PROTOCOL INFORMATION | 17 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | |
| | ۷.۷. | 2.2.1. Subcutaneous Sub-study Objectives and Endpoints | 11 |
| | 2.3. | Study Design | |
| | 2.5. | 2.3.1. Subcutaneous Sub-Study Design | 3/ |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | | IED ANALYSES | 26 |
| ა. | | Interim Analyses | |
| | 3.1. | 3.1.1. Subcutaneous Sub-Study Interim Analyses | |
| | 3.2. | | |
| | 3.2. | Final Analyses | 31 |
| 4. | ΛΝΛΙ ∨ | SIS POPULATIONS | 38 |
| 4. | 4 1 | Protocol Deviations | |
| | 4.1. | FIGURE Deviations | 4 I |
| 5. | CONSI | DERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONVE | ENTIONS | 41 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | 41 |
| | 5.2. | Baseline Definitions | |
| | | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups/Covariates | |
| | | Multiple Comparisons and Multiplicity | |
| | | 5.5.1. Primary Comparison of Interest | |
| | | 5.5.2. Other Comparisons of Interest | |
| | | 5.5.3. Secondary Comparisons | 49 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | | Conventions | 50 |
| 6. | STUDY | POPULATION ANALYSES | 52 |
| | 6.1. | Overview of Planned Study Population Analyses | 52 |
| | 6.2. | Subcutaneous Sub-Study Population Analyses | 53 |
| 7. | FFFICA | ACY ANALYSES | 55 |
| • | | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | |
| | | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |

| വ | 1 | 1584 |
|----|---|------|
| 20 | ш | 1004 |

| | | 7.2.4.<br>7.2.5. | Strategy for Intercurrent (Post-Randomization) Events Statistical Analyses / Methods | |
|---|---|---|---|---|
| 8. | SAFE | TY ANALY | /SES | 65 |
| | 8.1. | | Events Analyses | |
| | 8.2. | | Events of Special Interest Analyses | |
| | 8.3. | | _aboratory Analyses | |
| | 8.4. | | afety Analyses | |
| | 8.5. | | Safety Analysis | |
| | | 8.5.1. | Injection Site Reactions | |
| | | 8.5.2. | Statistical Analyses/Methods | |
| | 8.6. | | neous Sub-Study Safety Analyses | |
| 9. | | | NETIC AND PHARMACOKINETIC/PHARMACODYNAMIC | 70 |
| | | | Di | |
| | 9.1. | | Pharmacokinetic Analyses | |
| | | 9.1.1.<br>9.1.2. | Endpoint / Variables | |
| | | 9.1.2.<br>9.1.3. | Planned Analyses | |
| | 9.2. | | Statistical Analyses/Methods | |
| | 9.2. | 9.2.1. | neous Sub-Study<br>Endpoint / Variables | |
| | | 9.2.1. | Planned Analyses | |
| | | 9.2.3. | Statistical Analyses/Methods | |
| 10. | PHAR | MACOKIN | NETIC ANALYSES (DAY 1 JAPAN) | 81 |
| | 10.1. | | Pharmacokinetic Analyses | |
| | | 10.1.1. | | |
| | | 10.1.2. | Summary Measure | |
| | | 10.1.3. | Population of Interest | |
| | | 10.1.4. | Strategy for Intercurrent (Post-Randomization) Events | 82 |
| | | 10.1.5. | Statistical Analyses / Methods | |
| 11. | | | OMES ANALYSES | |
| | 11.1. | • | t / Variables | |
| | | 11.1.1. | | |
| | | | Population of Interest | |
| | | 11.1.3. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 11.1.4. | Planned Health Outcomes Analyses | |
| | 44.0 | 11.1.5. | Statistical Analyses/Methods | |
| | 11.2. | | neous Sub-Study Endpoint / Variables | |
| | | 11.2.1.<br>11.2.2. | • | 88 |
| 12. | VIROL | _OGY | | 90 |
| 13. | REFE | RENCES. | | 92 |
| 14. | | | | 94 |
| | 14.1. | | x 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | |
| | | | Exclusions from Per Protocol Population | |
| | 14.2. | | x 2: Schedule of Activities | |
| | | 14.2.1. | Protocol Defined Schedule of Events | 97 |

| | 14.2.2. | Protocol Defined Schedule of Events for the | |
|---|---|---|---|
| | | Subcutaneous Sub-Study | |
| 14.3. | Appendi | x 3: Assessment Windows | |
| | 14.3.1. | Definitions of Assessment Windows | 115 |
| | 14.3.2. | Definitions of Assessment Windows for Data Other than | |
| | | Health Outcomes and PK | 116 |
| | 14.3.3. | Assessment Window for Study Conclusion | 126 |
| | 14.3.4. | Assessment Window for Health Outcome Data | 126 |
| | 14.3.5. | Assessment Window for PK concentration Data | 130 |
| | 14.3.6. | Multiple assessments within an Analysis Window | 131 |
| 14.4. | Appendi | x 4: Study Phases and Treatment State | |
| | 14.4.1. | Study Phases | 133 |
| | 14.4.2. | Treatment State | 145 |
| | 14.4.3. | Combining Treatment Phases and States | 147 |
| 14.5. | Appendi | x 5: Data Display Standards & Handling Conventions | |
| | 14.5.1. | Reporting Process | 148 |
| | 14.5.2. | Reporting Standards | 148 |
| | 14.5.3. | Reporting Standards for Pharmacokinetic | |
| 14.6. | Appendi | x 6: Derived and Transformed Data | |
| | 14.6.1. | General | |
| | 14.6.2. | Study Population | |
| | 14.6.3. | Safety | |
| | 14.6.4. | Efficacy | |
| | 14.6.5. | Pharmacokinetic | |
| | 14.6.6. | Health Outcome | |
| | | Viral Genotype and Phenotype | |
| 14.7. | Appendi | x 7: Reporting Standards for Missing Data | 177 |
| | 14.7.1. | | 177 |
| | 14.7.2. | Handling of Missing Data | |
| 14.8. | | x 8: Values of Potential Clinical Importance | |
| 14.9. | | x 9: Population Pharmacokinetic (PopPK) Analyses | |
| 14.10. | | x 10: Pharmacokinetic / Pharmacodynamic Analyses | |
| | | x 11: Snapshot Algorithm Details | |
| | | x 12: AESI identification | |
| | | Hepatic Safety Profile | |
| | | Hypersensitivity Reactions | |
| | | Rash including severe cutaneous adverse reactions | |
| | | Prolongation of the Corrected QT Interval of the ECG in | |
| | | Supra Therapeutic Doses | 195 |
| | 14.12.5. | Suicidal Ideation/Behaviour | |
| | | Depression | |
| | | Bipolar Disorder | |
| | | Psychosis | |
| | | Mood Disorders | |
| | | ). Anxiety | |
| | | Sleep Disorders | |
| | | 2. Injection site Reactions | |
| | | 3. Seizures | |
| | | l Weight Gain | |
| | | 5.Rhabdomyolysis | |
| | | 5. Pancreatitis | |
| | | /.Impact on Creatinine | |
| | — | | |

| | 14.12.18 | Safety During Pregnancy | .222 |
|---|---|---|---|
| 14.13. | | x 13: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 14.14. | | x 14: List of Data Displays for Week 48/Week 96 | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Pharmacokinetic Tables | |
| | | .Pharmacokinetic Figures | |
| | | .Pharmacokinetic / Pharmacodynamic Tables | |
| | 14.14.12 | .Pharmacokinetic / Pharmacodynamic Figures | 279 |
| | 14.14.13 | .Health Outcomes Tables | .284 |
| | 14.14.14 | .Health Outcomes Figures | .289 |
| | 14.14.15 | .Virology Tables | .290 |
| | 14.14.16 | .ICH Listings | .293 |
| | | .Non-ICH Listings | |
| 14.15. | Appendix | x 15: List of Data Displays for Week 124 | .301 |
| | 14.15.1. | Data Display Numbering | .301 |
| | 14.15.2. | Mock Example Shell Referencing | .301 |
| | | Deliverables | |
| | 14.15.4. | Study Population Tables | .302 |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables – Extension Switch Population | |
| | | Safety Tables – Maintenance + Extension Phase | |
| | | (Randomized Q4W Only) | 328 |
| | 14.15.9. | Safety Tables – Long Term Follow Up | |
| | | Safety Figures – Extension Switch Population | |
| | | Safety Figures – Maintenance + Extension Phase | |
| | | (Randomized Q4W) | |
| | 14 15 12 | Pharmacokinetic Tables | |
| | | .Pharmacokinetic Figures | |
| | | .Virology Tables | |
| | | .ICH Listings | |
| | | Non-ICH Listings | |
| 14 16 | | x 16: IDMC | |
| 11.10. | | CVF Monitoring (Adhoc IDMC review) | |
| 14 17 | | x 17: Variables Defined for Time to Event Analysis | |
| | | x 18: Japan-Specific Requirements | |
| 17.10. | | Study Population Tables - Japan | |
| | | Efficacy Tables - Japan | |
| | | Safety Tables - Japan | |
| | | Pharmacokinetic Tables - Japan | |
| | | Pharmacokinetic Figures - Japan | |
| | | Health Outcomes Tables - Japan | |
| | | • | |
| | 14.10.1. | ICH Listings - Japan | . 505 |

| | 14.18.8. | Non-ICH Listings - Japan | 364 |
|---|---|---|---|
| 14.19. | Appendix | 19: List of Data Displays for Subcutaneous Sub-study | |
| | Analysis | | 365 |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | 14.19.4. | Study Population Tables | 366 |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Pharmacokinetic Tables | |
| | | .Pharmacokinetic Figures | |
| | | .Health Outcomes Tables | |
| | | .Virology Tables | |
| | | .ICH Listings | |
| | | Non-ICH Listings | |
| 14.20. | | c 20: Example Mock Shells for Data Displays | |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for protocol 201584.

| GlaxoSmithKline<br>Document Number | Date | Version |
|------------------------------------|-------------|-----------------|
| 2015N248866_00 | 2016-MAY-26 | Original |
| 2015N248866_01 | 2016-DEC-13 | Amendment No. 1 |

The reasons for this amendment were to: added new primary Medical Monitor contact information; added lipid objective and endpoint back in to the table within the Synopsis section; added clarification of text for patient reported outcome endpoints; added additional clarification regarding provision of CAB LA and RPV LA until available through public/government health sectors; new text added to allow use of local labs to determine eligibility in exceptional circumstances; updated Time and Events Table to provide more clarity around assessments conducted during the Extension Phase, added 'X' to include collection of cardiovascular risk information at Screening, added temperature to Vital Signs row, added row for randomization, and clarified timings for completion of patient reported questionnaires relative to other clinical assessments in the table footnotes; clarified timing of dosing for abacavir/dolutegravir/lamivudine (ABC/DTG/3TC, Triumeq) for the Day 1 visit; added additional clarification that participants of child bearing potential must continue contraception for at least 52 weeks after the last injection; revised text to say that Investigators may provide 'bridging' supply after consultation with Medical Monitor (vs Medical Monitor authorizing bridging supply); provided clarification that cabotegravir and rilpivirine exposure may persist for more than one year in some participants after intramuscular administration (with added references); minor edits to prohibited medication information; added statement that drugs that cause Torsade de Pointes should be used with caution when taking rilpivirine; additional clarification that background NRTI therapy is not considered Investigational Product and accountability will not be done for NRTI background; changed film coat color for Tivicay (dolutegravir) from white (clinical trial material supply) to yellow (commercial supply) and removed statement to "protect from light" (for both Triumeq and Tivicay); sentence added for collection of additional details for the injection device used for IM administration; additional information included regarding randomization schedule; added text stating the investigator must discuss long-term commitment for the study with potential participants; added statement regarding serofast RPR results; allowed serum pregnancy testing where required locally (e.g. when urine testing is not available); removed duplicate text regarding monitoring for suicidal related events; added option for patient reported outcomes to be collected on paper instrument if needed; removed information in Appendix requiring collection of pregnancy information for female partners of male study participants; definition of ACCEPT, HIVTSQc, and HIVTSQs added to abbreviations table, duplication of ICH

abbreviation removed; other minor corrections (e.g., updated references, adding cross reference to sections, correction of hyperlink to one table).

2015N248866\_02 2017-JUL-19 Amendment No. 2

The reasons for this amendment are as follow: update of contact information for secondary Medical Monitor; modify text to allow dose reduction for participants who have a decline in creatinine clearance to <50 mL/min; clarify that for participants not eligible to continue into the Maintenance Phase, only samples with HIV-1 RNA > 400 c/mL will be sent for resistance testing; add mitigation for ECG pad removal; clarify  $\pm 3$  day window is for all oral dosing (both Induction and Maintenance Phase); add "LA Arm" back to columns for Week 68, 76, 84, 92 on Time and Events Schedule (hidden when column was narrowed); clarify Week 104b visit is specific to those participants transitioning from oral IP to CAB LA + RPV LA; clarification added to footnote 'p' that genetics sample can be collected at any visit after signing informed consent, but Week [-20] preferred; correct footnote on Week 5 visit to reflect footnote 't'; add footnote 'y' back to Time and Events column for Withdrawal Visit (for Induction Phase); add clarification to Time and Events column that ISR assessments are only conducted for participants receiving injections; remove text from Section 12.2: 'In addition, all deaths related to an AE are to be classified as grade 5.' Administrative typographical errors corrected (e.g. clarification provided regarding genetics sample taken after participants are enrolled into the study [vs when participants are randomized]), and investigator brochure references updated.

| 2015N248866_03 | 2018-JUN-25 | Amendment No. 3 |
|----------------|-------------|-----------------|

Changes for Amendment 3 were made to the protocol to manage and mitigate risks following identification of a potential safety issue related to neural tube defect in infants born to women with exposure to dolutegravir (DTG) at the time of conception.

A Risk Assessment table was added to include language regarding risk and mitigation of neural tube defects seen with DTG.

- The withdrawal criteria were updated to include a reminder that females of reproductive potential who change their minds and desire to be pregnant should also be withdrawn from the study.
- The Time and Events table was updated to include a reminder for investigators to check at every visit that females of reproductive potential are avoiding pregnancy. Additionally, clarifications were provided for the following:
  - the DTG IB should be referenced for additional risks, safety information, drug interactions, etc.;
  - 'suspected' was added to the text prior to the bulleted definition of suspected virologic failure in Section 5.4.5.3.;
  - specific storage conditions were removed from the protocol for IP, and a statement added to store according to product label;
  - insulin was removed from the section regarding clinical assessments performed during the study;

• timeframe for pregnancy reporting and follow-up were updated to 24 hours to align with current reporting process;

• prescribing information and IB references were updated.

2015N248866\_04 | 2018-SEPT-24 | Amendment No. 4

The primary reason for protocol amendment 04 is to allow an optional (vs mandatory) oral lead-in for participants randomized to the ABC/DTG/3TC arm who choose to continue into the Extension Phase of the study and receive CAB LA + RPV LA. The Appendix for contraceptive guidance and collection of pregnancy information was updated to be consistent with current protocol template text. Other minor clarifications were made as needed, e.g., the eCSSRs timing in the footnote for the Time and Events Table, updated abbreviations, etc.

2015N248866\_05 2020-MAY-20 Amendment No. 5

The reason for protocol amendment 05 is to include an Appendix with Covid-19 guidance for clinical trial continuity (participant and study management) during the pandemic. This appendix will replace the previous Appendix 9, and Appendix 9 "Protocol Amendment History," will be included as Appendix 10.

TMF-13030701 2021-AUG-21 Amendment No. 6

The primary purposes of this amendment are:

- To allow participants who become pregnant while in the study to remain in the study and not be withdrawn due to pregnancy. Allowing pregnant participants to continue in the study will negate any additional and subsequent fetal exposures to new antiretroviral agents that would occur if the pregnant participant was withdrawn from the study and placed on an oral SOC regimen. An appendix, "Information and Guidance for Managing Pregnant Participants" was inserted as Appendix 10 and all subsequent appendices were renumbered accordingly.
- Contraceptive methods have been updated to permit the use of progestogenonly implantable and injectable contraceptives without the requirement of a second highly effective method.
- Removal of the optional collection of cord blood and/or breast milk after delivery.
- Removal of the option for study treatment rechallenge following suspected drug-induced liver injury (DILI).
- Clarification of which participants enter the LTFU phase when CAB+RPV LA marketed product is locally available.
- Medical Device reporting requirement added.
- Co-enrolment (only applicable for eligible female participants in South Africa in the ACTG A5392 study).
- Updates to primary and secondary Medical Monitors.

| Other additional edits were made, for clarity and/or correction. | | |
|---|---|---|
| TMF-147-28112 | 2022-JUN-17 | Amendment No. 7 |

The primary purposes of this amendment are:

- To include the Sub-Cutaneous Abdominal Injection Sub-Study appendix (only applicable for countries participating in the Sub-Study).
- Clarification added: In Russia, subjects who become pregnant while on study
  may not elect to remain on study treatment and must withdraw and enter the
  LTFU Phase.

Inclusion of Appendix 13: Mitigations for Geopolitical Situation in Russia/Ukraine

| TMF-15038148 | 2022-OCT-21 | Amendment No. 8 |
|--------------|-------------|-----------------|

This amendment is considered to be substantial based on the criteria defined in EU Clinical Trial Regulation No 536/2014 of the European Parliament and the Council of the European Union.

Overall Rationale for the Amendment:

The primary purposes of this amendment are:

- To include the Sub-Study Interim Analysis 1: ISR Monitoring Criteria into the Sub-Cutaneous Abdominal Injection Sub-Study appendix (only applicable to for countries participating in the Sub-Study).
- To include the Sub-Study Interim Analysis 2: Week 9 Safety and PRO Review into the Sub-Cutaneous Abdominal Injection Sub-Study appendix (only applicable for countries participating in the Sub-Study).

| TBD | TBD | Amendment No. 9 |
|-----|-----|-----------------|

This amendment is considered to be substantial based on the criteria in EU Clinical Trial Regulation No 536/2014 of the European Parliament and the Council of the European Union.

The primary purposes of this amendment are to update the Potential Risk of Clinical Significance of Hypersensitivity Reactions (HSR) when using integrase inhibitors, such as CAB.

#### 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Plan_201584_Final_V1 [17-AUG-2018] | |
| Reporting and Analysis Plan_201584_Amendment_Final_V1 [17-SEPT-2018] | |

| RAP Section | Amendment Details | | |
|---|---|---|---|
| Reporting and Analysis Plan_201584_Amendment_2_Final_V1 | | | |
| Japan Specific Reporting Requirements for Regulatory Submission | | • | Added data displays to be generated for Japan participants: study population, efficacy, safety, and pk. Added details for the analysis of PK samples for participants in Japan, including estimation of PK parameters by non-compartmental methods using concentration-time day on Day 1. Added analysis population for Japan PK. |
| Adverse Events of Special In | nterest | • | Harmonized list of Adverse Events of Special Interest with that used in the Week 48 integrated analysis of safety summaries (with |
| · | | | grouping based on clinical review of preferred<br>terms and Standardized MedDRA Queries<br>(SMQs)) |
| | | • | Removed Last CAB/RPV Trough Concentration as a candidate predictor of efficacy outcomes at Week 96 (as this covariate is confounded with accumulation overtime). |
| | | • | Removed PK/PD efficacy displays related to Last CAB/RPV Trough Concentration (as this covariate is confounded with accumulation overtime). |
| Updated PK/PD analysis pla | n for Week 96 | • | Added condition that PK/PD efficacy analysis/displays will only be produced if the Week 96 dataset includes at least one new CVF since the Week 48 analysis |
| | | • | Clarified that the following PK/PD safety figures will not be produced at Week 96 given limited PK collection post W48: |
| | | | <ul> <li>Scatter Plot of Maximum Change<br/>from Maintenance Baseline (Day 1) in<br/>ALT/Bilirubin versus Last Trough<br/>CAB/RPV PK Concentrations</li> </ul> |
| | | | <ul> <li>Box Plot of Maximum Toxicity Grades<br/>of Most Frequently Reported Non-<br/>ISR AEs versus Last Trough<br/>CAB/RPV PK Concentrations</li> </ul> |
| Data Handling | | • | Minor update to the algorithm used to assign data to the Extension phase to account for direct to inject vs. start with oral lead-in. |
| | | • | Minor correction to W96 visit window for CD4+ cell count data and NRS questionnaire data. |

| RAP Section | Amendment Details | |
|---|---|---|
| | • | Added Region (country grouping) and Baseline Integrase L74I mutation as subgroup variables Clarified definition of Hepatitis B and C status |
| | • | at Baseline Updated imputation rule for adverse events with partial end dates (to use last contact date instead of treatment stop date). Clarified analysis visit assignment for LTFU PK samples. Update the rationale for the prespecified list of mutations associated with resistance to integrase strand transfer inhibitors based on |
| | | 2019 IAS-US guideline. |
| | • | The following data displays were added for Week 96: |
| | • | Summary of Change from Plasma HIV-1 RNA (log10 c/mL) by Visit (Maintenance Phase) |
| | | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA >= 50 c/mL (and <50 c/mL) at Week 96 by Selected Demographic Subgroups (Maintenance Phase) - Snapshot Analysis |
| | • | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA >= 50 c/mL (<50 c/ml) at Week 96 by Selected HIV Disease Characteristic Subgroups (Maintenance Phase) - Snapshot Analysis |
| Data Displays | • | Summary of Plasma CAB/RPV PK<br>Concentration -Time Data by Treatment and<br>Visit (Maintenance Phase) – Included Log-<br>transformed Statistics by Hepatitis C Status at<br>Induction Baseline |
| | • | Individual Plasma CAB/RPV Concentration-<br>Time Plots (Semi-Log) Post Last Injection<br>for Subjects in LTFU |
| | | Listing of Plasma CAB/RPV PK Concentration-Time Data (LTFU Phase) |
| | | Listing of Concomitant Medications for<br>Subjects with Confirmed Virologic Failure |
| | • | Summary of Shift in BMI Categories at Week 96 |
| | • | Summary of Shift in BMI from Induction<br>Baseline (Week -20) to Maximum Post-<br>baseline Category (Maintenance Phase) |

| RAP Section | Amendment Details | |
|---|---|---|
| RAP Section | Amendment Details | <ul> <li>Scatter Plot of Maximum vs. Extension Baseline (Week 100) for ALT (Extension Phase) – Switch Q4W IM</li> <li>Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin (Extension Phase) – Switch Q4W IM</li> <li>Matrix Plot of Maximum Liver Chemistries (Extension Phase) – Switch Q4W group</li> <li>Summary tables for Adverse Events of Special Interest</li> <li>Listing of All Adverse Events</li> <li>Listing of all Subjects Meeting Liver Stopping Criteria</li> <li>Summary of HIVTSQs - Change from Maintenance Baseline (Day 1) in Individual</li> </ul> |
| | | <ul> <li>Item Score by Visit - LOCF (Maintenance Phase)</li> <li>Listing of All Genotypic Data</li> <li>Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure (Maintenance + Extension Phase) — Randomized Q4W arm</li> <li>Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria (Extension Phase) — Switch Q4W IM</li> </ul> |
| | | Updated the following table to present minimum NCEP Category instead of Maximum: Summary of Changes in Maintenance Baseline (Day 1) NCEP Fasting Lipid Category to Minimum Maintenance Phase Category – HDL Cholesterol |
| | | Added further stratification by 'any history' vs. 'no history' for the following table: Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety and Suicidal Ideation/Behaviour at Screening Updated some display titles in Appendix 14: List of Data Displays. |
| Reporting and Analysis Pla | Reporting and Analysis Plan_201584_Amendment_3_Final_V1 | |
| Data Handling and Data Di | | Clarified extension phase analyses window for AE data in Table 16 |

| RAP Section | Amendment Details | | |
|---|---|---|---|
| | | • | Clarified derivation of Extension Phase extent of exposure in Section 14.6.2. |
| | | • | Added treatment group descriptors for Switch Q4W (Direct to Inject) and Switch Q4W (Oral Lead-In) in Table 3. |
| | | • | Added list of specific data displays to be produced for the Week 124 analysis to Section 14.15. |
| Reporting and Analysis Pla | an_201584_Amendmer | nt_4 | |
| | | • | Updated visit/phase slotting algorithms to handle the newly added sub-study assessments and time points in the protocol. |
| Data Handling and Data Dis | plays for Sub-study | • | Added new analysis populations for sub-study analysis. |
| | | ana | ned a separate list of displays for sub-study<br>lysis including a cut set of listings due to use of<br>RAPIDO DV. |
| | | • | Added details of sub-study interim analyses including monitoring for ISRs of interest. |
| | | • | Added calculation methods for extent of exposure in sub-study. |
| Safety Analysis | | • | Extended lipid LOCF approach to include both SC Injection and Return to Gluteal Injection phases in sub-study. |
| | | • | Added display shells for summaries of COVID-<br>19 assessments including accommodation of<br>possible scenarios of multiple COVID-19 case<br>diagnoses per participant. |
| PK Analysis | | • | Added analysis methods for PK parameters derived from sub-study concentration-time data including interim analyses |
| T (Villalysis | | • | Extended evaluability criteria to include substudy PK concentration data. |
| | | • | Added windows for evaluating concomitant ART/non-ART medications in sub-study. |
| Study Population Analysis | | • | Added a/listings for data collected from the Transition to CAB + RPV LA Marketed Product Status eCRF form. |
| Libralith Outramas Analysis | | • | Clarified that LOCF will no longer be used for HO analyses |
| | | • | Added analysis for the newly added questionnaires: |
| Health Outcomes Analysis | 1. | Preference Subcutaneous Injection vs Gluteal Injection questionnaire. | |
| | | 2. | Reason for switch questionnaire |
| | | • | Interest in self administration questionnaire |

| RAP Section | Amendment Details | |
|---|---|---|
| General Updates | | <ul> <li>Added Endpoint &amp; Estimand text for the Substudy endpoints</li> <li>Added sub-study Schedule of Activities per new protocol.</li> <li>Added additional minor clarifications and corrections to typographical errors/formatting to RAP text.</li> </ul> |
| Reporting and Analysis Plan_201584_Amendment_5 | | |
| Data Handling for Sub-s | study | Updated visit/phase slotting algorithms to appropriately handle Adverse Events within the sub-study and clarified algorithm to ensure all records are associated with the correct visit. |
| General Updates | | Added additional minor clarifications and corrections to typographical errors/formatting to RAP text. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There is a single deviation planned from protocol amendment #8 [(Dated: 21-OCT-2022)]. Due to delay in study enrolment for implementation of protocol amendment 8, interim analysis 2 will include PK summaries while the protocol indicates that no PK analyses will be included.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Interim analysis 2 is planned to only summarize safety, tolerability, and HO data. | PK data available around<br>the Week 9 Safety<br>timepoint will also be<br>analyzed | Delay in study start due to protocol amendment 8 necessitated the need for an earlier reporting of PK data. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| To demonstrate the non-inferior antiviral activity of switching to intramuscular CAB LA + RPV LA every 4 weeks (monthly) compared to continuation of ABC/DTG/3TC over 48 weeks in HIV-1 antiretroviral naïve participants. | Proportion of participants with a 'virologic failure' endpoint as per FDA Snapshot algorithm at Week 48 (Missing, Switch, or Discontinuation = Failure, Intent-to-Treat Exposed [ITT-E] population). |
| Secondary | |
| To demonstrate the antiviral and immunologic activity of switching to intramuscular CAB LA + RPV LA every 4 weeks (monthly) compared to continuation of ABC/DTG/3TC. | <ul> <li>Proportion of participants with plasma<br/>HIV-1 RNA &lt;50 copies/mL (c/mL) at<br/>Week 48 using the FDA Snapshot<br/>algorithm (Intent-to-Treat Exposed [ITT-E]<br/>population).</li> </ul> |
| | <ul> <li>Proportion of participants with plasma<br/>HIV-1 RNA &lt;200 c/mL at Week 48 using<br/>the FDA Snapshot algorithm (ITT-E<br/>population).</li> </ul> |
| | Proportion of participants with plasma<br>HIV-1 RNA <200 c/mL and HIV-1 RNA<br><50 c/mL at Week 96 using the FDA<br>Snapshot algorithm (ITT-E population). |
| | Proportion of participants with a 'virologic failure' endpoint as per FDA Snapshot algorithm at Week 96. |
| | Proportion of participants with confirmed |

| Objectives | Endpoints |
|---|---|
| | virologic failure at Week 48 and Week 96. |
| | <ul> <li>Absolute values and change from Baseline<br/>in plasma HIV-1 RNA (log<sub>10</sub> copies/mL) at<br/>Week 48 and Week 96.</li> </ul> |
| | Absolute values and changes from Baseline in CD4+ cell counts over time including Week 48 and Week 96. |
| | Incidence of disease progression (HIV-<br>associated conditions, acquired<br>immunodeficiency syndrome [AIDS] and<br>death). |
| To evaluate the safety and tolerability of switching to CAB LA + RPV LA every 4 weeks (monthly) compared to continuation of | Incidence and severity of adverse events (AEs) and laboratory abnormalities over time including Week 48 and Week 96. |
| ABC/DTG/3TC over time. | <ul> <li>Proportion of participants who discontinue<br/>treatment due to AEs over time including<br/>Week 48 and Week 96.</li> </ul> |
| | Absolute values and changes in laboratory parameters over time including Week 48 and Week 96. |
| To evaluate the effects of CAB LA + RPV LA every 4 weeks on fasting lipids over time compared to continuation of ABC/DTG/3TC over time. | Change from Baseline in fasting lipids over time including Week 48 and Week 96. |
| To assess the development of viral resistance in participants experiencing protocol-defined virologic failure. | Incidence of treatment emergent genotypic<br>and phenotypic resistance to CAB, RPV,<br>and other on-study ART at Week 48 and<br>Week 96. |
| To characterize CAB and RPV concentrations and population pharmacokinetics (PK) and identify important determinants of variability. | Plasma PK parameters for CAB LA and RPV LA (when evaluable, C <sub>trough</sub> , concentrations post dose [~Cmax], and area under the curve [AUC]). |
| | Demographic parameters including, but<br>not limited to, age, sex, race, body weight,<br>body mass index (BMI), and relevant<br>laboratory parameters will be evaluated as<br>potential predictors of inter- and intra-<br>participant variability for pharmacokinetic<br>parameters. |
| To assess the acceptance of pain and injection site reactions following injections. | Change from Week 5 in Dimension scores<br>(e.g., "Bother of ISRs", "Leg movement", |

| Objectives | Endpoints |
|---|---|
| | "Sleep", and "Injection Acceptance") and individual item scores assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time using the Perception of iNjection questionnaire (PIN). |
| | Proportion of participants considering pain<br>and local reactions following injection to be<br>extremely or very acceptable based on the<br>acceptability score over time using the<br>Perception of iNjection questionnaire<br>(PIN). |
| To assess treatment satisfaction of CAB LA + RPV LA compared to continuation of ABC/DTG/3TC. | Change from baseline in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Questionnaire (status version) (HIVTSQs) at Week 4b, Week 24, Week 44, Week 96 (or Withdrawal). |
| | Change in treatment satisfaction over time<br>(using the HIVTSQc change version<br>[HIVTSQc]) at Week 48 (or Withdrawal). |
| To assess degree of health-related quality of life (HR QoL). | Change from Baseline in HR QoL using<br>the HIV/AIDS targeted quality of life<br>questionnaire (HAT-QoL) short format<br>Week 24, Week 48, Week 96 (or<br>Withdrawal). |
| To assess health status. | Change from Baseline in health status at<br>Week 24, Week 48, and Week 96 (or<br>Withdrawal) using the 12-item Short Form<br>Survey (SF-12). |
| To assess treatment acceptance. | Change from Baseline in treatment acceptance at Week 8, Week 24, Week 48, Week 96 (or Withdrawal) using the "General Acceptance" dimension of the Chronic Treatment Acceptance (ACCEPT) questionnaire. |
| To assess tolerability of injections. | Change from Week 4b in tolerability of injections at Week 5, Week 40, Week 41, and Week 96 using the Numeric Rating Scale (NRS) within the CAB LA + RPV LA |

| Objectives | Endpoints |
|---|---|
| | arm. |
| To evaluate the antiviral and immunologic effects, safety and tolerability, and development of viral resistance to CAB LA + RPV LA at Week 124 and over time for participants switching from ABC/DTG/3TC in the Extension Phase, with and without optional | <ul> <li>Proportion of participants with HIV-1 RNA ≥ 50 c/mL at Week 124, with and without oral lead-in (FDA Snapshot algorithm, Extension Switch population).</li> <li>Proportion of participants with plasma HIV-</li> </ul> |
| oral lead-in. | 1 RNA <50 c/mL and HIV-1 RNA <200 c/mL time over. |
| | Proportion of participants with confirmed virologic failure over time. |
| | <ul> <li>Incidence of treatment emergent genotypic<br/>and phenotypic resistance to CAB and<br/>RPV over time.</li> </ul> |
| | Absolute values and change from Baseline in CD4+ cell counts over time. |
| | Incidence and severity of AEs and laboratory abnormalities over time. |
| | Proportion of participants who discontinue treatment due to AEs over time. |
| | Absolute values and change in laboratory parameters over time. |
| To evaluate the pharmacokinetics of CAB and RPV in the setting of no oral lead-in for participants switching from ABC/DTG/3TC in the Extension Phase. | To evaluate plasma CAB and RPV concentrations over time (Week 100 [direct to inject without oral lead-in] and Week 104 [both direct to inject and optional oral lead-in participants]) |
| Exploratory | |
| To explore the effect of participant characteristics on the virologic and immunologic response of CAB LA and RPV LA compared to continuation of ABC/DTG/3TC. | Proportion of participants by patient subgroup(s) (e.g., by age, gender, BMI, race, HIV-1 subtype, Baseline CD4+) with Virologic Failure over time including Week 48, and 96 using the Snapshot algorithm for the ITT-E population. |
| | Proportion of participants by subgroup(s) (e.g. by age, gender, BMI, race, HIV-1 subtype, Baseline CD4+) with plasma HIV-1 RNA <50 c/mL at Week 48 and Week 96. |
| | Change from Baseline in CD4+ cell counts |

| Objectives | Endpoints |
|---|---|
| | by subgroups at Week 48 and Week 96. |
| To explore relationship(s) between plasma concentrations of CAB and RPV and pharmacodynamic endpoints. | Relationship between plasma PK concentrations and virologic, immunologic responses, and/or occurrence of adverse events [AEs] over time may be explored. |
| To evaluate renal and bone biomarkers in participants receiving CAB LA and RPV LA compared to continuation of ABC/DTG/3TC over time. | Absolute values and change from Baseline in renal (in urine and blood) and bone (in blood) biomarkers over time including Week 48 and Week 96. |
| To assess preference for CAB LA + RPV LA compared to oral antiretroviral (ARV) therapy using a single dichotomous preference question. | <ul> <li>For participants randomized to the "CAB<br/>LA + RPV LA" arm, preference for CAB<br/>LA + RPV LA compared to oral ARV<br/>regimen, at Week 48.</li> </ul> |

# 2.2.1. Subcutaneous Sub-study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Pharmacokinetic | |
| To evaluate PK of monthly dosing of CAB LA (200 mg/mL) with RPV LA (300 mg/mL) following SC administration in the anterior abdominal wall SC tissue compared with intramuscular administration in the gluteus medius muscle in HIV-1 infected participants currently enrolled in the FLAIR Phase 3 study | Plasma PK parameters for CAB LA 200 mg/mL and RPV LA 300 mg/mL (Ctau, concentrations 1-week post dose [~Cmax], and area under the curve [AUC (0-tau)]) for SC injections during the SC injection phase compared with similar PK parameters for gluteal IM injections |
| Secondary Objectives | Secondary Endpoints |
| Safety and tolerability | |
| To assess safety and tolerability of monthly dosing of CAB LA (200 mg/mL) administered with RPV | Incidence and severity of ISRs and AEs of special interest during the SC injection phase. |
| (300 mg/mL) LA following SC administration in the anterior abdominal wall SC tissue compared with intramuscular injections in the gluteus medius muscle in HIV-1 | Proportion of participants who discontinue treatment due to ISRs and AEs of special interest during the SC injection phase. |
| infected participants currently enrolled in the FLAIR Phase 3 study To assess additional safety events including other AEs, SAEs, and safety labs of monthly dosing of CAB LA and RPV LA following SC injections in the | Incidence of other AEs not of special interest, SAEs and change in laboratory parameters from the last IM gluteal injection (prior to the SC abdominal Injection Phase) to the end of the SC injection phase (week 12). |

| Objectives | Endpoints |
|---|---|
| abdominal wall SC tissue in HIV-1 | |
| infected participants currently enrolled in the FLAIR sub-study | |
| Virologic Response | <u> </u> |
| To assess the ability to maintain virologic suppression (HIV-RNA <50 copies) in participants who transition from IM to SC administrations of CAB LA (200 mg/mL) plus RPV LA (300 mg/mL) in the FLAIR sub-study. To assess virologic non-response (HIV-RNA ≥50 c/mL and ≥200 c/mL) in participants who transition from IM to SC administrations of CAB LA (200 mg/mL) plus RPV LA (300 mg/mL) in the FLAIR sub-study. | Proportion of participants with plasma HIV-1 RNA <50 copies at week 12 during the SC abdominal injection phase using the FDA Snapshot algorithm. Proportion of participants with plasma HIV-RNA ≥50 c/mL as per Food and Drug Administration (FDA) Snapshot algorithm at week 12 during the SC abdominal injection phase. Proportion of participants with protocol-defined confirmed virologic failure (CVF) of ≥200 c/mL at week 12 during the SC injection phase. |
| To assess viral resistance in participants experiencing protocoldefined confirmed virologic failure. | Incidence of treatment emergent genotypic and phenotypic resistance to CAB, RPV during the SC injection phase. |
| Health Outcomes | |
| To assess patient reported outcomes during the SC injection phase by administering the following health outcome measurements: NRS, | Numerical Rating Scale (NRS): To assess the tolerability of injections during both the SC abdominal and IM Gluteal Injection Phases, separate for CAB LA and RPV LA. |
| HIVTSQ (both s and c versions), and PIN. | HIVTSQ (both s and c versions): To measure levels of satisfaction and detect change in satisfaction when switching from IM gluteal to SC abdominal injections in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Questionnaire (HIVTSQ) during the SC Injection Phase as well as change from SC during the Return to IM Gluteal Phase. |
| | Perception of injection questionnaire (PIN): To assess the acceptance of pain and injection site reactions following SC abdominal and IM gluteal injections separate for CAB LA and RPV LA. |
| To assess participant's preference of SC injections during the SC abdominal injection phase compared to IM gluteal injections. | Preference Questionnaire: To assess patient's preference, and reasons for preference, for injections received during the SC Injection Phase compared with prior IM gluteal injections as well as for injections received during the Return to Gluteal phase compared with prior SC injections. |

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To assess reasons for switch to SC | Reasons for switch and interest for home |
| from IM injection and interest in a | administration options questions: To assess the |
| potential option for self-administration | reasons participants agreed to switch to a SC |
| of SC injections | abdominal injection from a IM gluteal injection and their |
| | interest in a potential option for self-administration of |
| | SC injections. |

# 2.2.1.1. Subcutaneous Sub-study Estimands

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| administration in the ant | erior abdomina<br>pants currently | al wall SC ty enrolled i | sing of CAB LA (200 mg/mL) with RP tissue compared with intramuscular adn the FLAIR Phase 3 study | V LA (300 mg/mL) following SC ministration in the gluteus medius muscle |
| • Plasma PK parameters for CAB LA 200 mg/mL and RPV LA 300 mg/mL (Ctau, concentrations 1-week post dose [~Cmax], and area under the curve [AUC (0-tau)]) for SC injections during the SC injection phase compared with similar PK parameters for gluteal IM injections | Pharmacok inetic Parameter & Pharmacok inetic Concentration | CAB+R<br>PV LA<br>IM vs.<br>CAB+R<br>PV LA<br>SC | Ratio of geometric least squares (GLS) means of PK parameters between SC and IM injections and the corresponding 90% CI estimated via a linear mixed-effects model PK Concentration: Arithmetic mean, median, sd, min, max, 90% Confidence Interval (CI) for the mean (or 95% CI) PK parameters: Arithmetic mean, median, sd, min, max, 90% CI for the arithmetic mean, geometric mean, sd (log), | Study treatment discontinuation due to any reason: While-on-treatment strategy Rationale: Discontinuation of planned study treatment may bias the evaluation of Pharmacokinetic behaviour of study treatment so only samples collected while on treatment will be summarized. |

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| | | | geometric %CV, 90% for the geometric mean | |
| | | | Steady State: | |
| | | | Point estimate and 90% CI of slope of log(concentration) vs. timepoint estimated via a linear mixed-effects model | |
| | | | List summary statistics as needed | |

Secondary Objective: To assess safety and tolerability of monthly dosing of CAB LA (200 mg/mL) administered with RPV (300 mg/mL) LA following SC administration in the anterior abdominal wall SC tissue compared with intramuscular injections in the gluteus medius muscle in HIV-1 infected participants currently enrolled in the FLAIR Phase 3 study

To assess additional safety events including other AEs, SAEs, and safety labs of monthly dosing of CAB LA and RPV LA following SC injections in the abdominal wall SC tissue in HIV-1 infected participants currently enrolled in the FLAIR sub-study

| • | severity of ISRs and AEs of special | CAB+R<br>PV LA<br>(SC & | Frequency, descriptive sta | percentages,<br>itistics | and | • Study treatment discontinuation due to any reason: <b>Treatment policy strategy</b> |
|---|---|---|---|---|---|---|
| | interest during the SC injection phase. | IM) | | | | Rationale: Safety data will be monitored throughout the study after the start of treatment. There is interest in evaluating |

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| <ul> <li>Proportion of participants who discontinue treatment due to ISRs and AEs of special interest during the SC injection phase.</li> <li>Incidence of other AEs not of special interest, SAEs and change in laboratory parameters from the last IM gluteal injection (prior to the SC abdominal Injection Phase) to the end of the SC injection phase (week 12).</li> </ul> | | | | and reporting safety events regardless of whether participants have completed treatment course or not. Safety events will be appropriately labeled as occurring during the IM or SC phases based on injections dates and summarized accordingly. |

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |

Secondary Objective: To assess the ability to maintain virologic suppression (HIV-RNA <50 copies) in participants who transition from IM to SC administrations of CAB LA (200 mg/mL) plus RPV LA (300 mg/mL) in the FLAIR sub-study.

To assess virologic non-response (HIV-RNA  $\geq$ 50 c/mL and  $\geq$ 200 c/mL) in participants who transition from IM to SC administrations of CAB LA (200 mg/mL) plus RPV LA (300 mg/mL) in the FLAIR sub-study.

To assess viral resistance in participants experiencing protocol-defined confirmed virologic failure.

| <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 copies at week 12 during the SC abdominal injection phase using the FDA Snapshot algorithm.</li> <li>Proportion of participants with plasma HIV-RNA ≥50 c/mL as per Food and Drug Administration (FDA) Snapshot algorithm at week 12 during the SC</li> </ul> | I | CAB+R<br>PV LA<br>SC | The proportion of participants with plasma HIV-RNA >= or < 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at SC Injection Phase Week 12. The proportion of participants with confirmed virologic failure while on CAB+RPV LA SC. | <ul> <li>Study treatment discontinuation due to lack of efficacy or other reasons that impact the viral load outcome: Composite strategy Rationale: "The presence of missing data due to lack of efficacy or discontinuation for other reasons on the primary endpoint is adequately accounted for in the FDA Snapshot Algorithm which frames the outcome around these events. Please see Section 14.11 for details."</li> <li>Rescue medication use/Change in Background ART strategy: Composite strategy Rationale: "The presence of missing data due to a change in background</li> </ul> |
|---|---|---|---|---|
|---|---|---|---|---|

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| abdominal injection phase. • Proportion of participants with protocol-defined confirmed virologic failure (CVF) of ≥200 c/mL at week 12 during the SC injection phase. | | | | medication is adequately accounted for in the FDA Snapshot Algorithm which employs a composite strategy in this regard, conservatively assuming that any participants who changed background ART without a current viral load and without discontinuing are classified as having HIV-1 RNA >50c/mL. Please see Section 14.11 for details." |
| • Incidence of treatment emergent genotypic and phenotypic resistance to CAB, RPV during the SC injection phase. | Safety | CAB+R<br>PV LA<br>SC | Prevalence of (% of participants with) Treatment Emergent Resistance Mutations (frequency count) Prevalence of (% of participants with) Phenotype, Replication Capacity (frequency count) | Missing data for any ICE including unevaluable sampling: While-ontreatment strategy Rationale: "Should there be missing genetic data, it would be expected that any data collected while a participant is off study IP would be impacted differently that when they are on study IP. Therefore, only data collected and available while the participant was on study IP will be analyzed." |

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |

Secondary Objective: To assess patient reported outcomes during the SC injection phase by administering the following health outcome measurements: NRS, HIVTSQ (both s and c versions), and PIN.

To assess participant's preference of SC injections during the SC abdominal injection phase compared to IM gluteal injections.

Exploratory Objective: To assess reasons for switch to SC from IM injection and interest in a potential option for self-administration of SC injections

| Numerical Rating Scale (NRS): To assess the tolerability of injections during both the SC abdominal and IM Gluteal Injection Phases, separate for CAB LA and RPV LA. HIVTSQ (both s and c versions): To measure levels of satisfaction and detect change in satisfaction when switching from IM gluteal to SC abdominal injections | CAB+R<br>PV LA<br>IM vs.<br>CAB+R<br>PV LA<br>SC | Scale scores where prescribed, change from Baseline in repeated measures, frequency counts, and descriptive statistics | Missing data for any ICE including study treatment discontinuation: Treatment policy strategy Rationale: "HO assessments are administered to align at treatment specific timepoints (SC vs LA). They also account for differences in treatment by design and thus, significant deviation from the administration window is not expected to impact the outcome and data can be assumed to be missing at random. There is interest in evaluating and reporting HO data regardless of whether participants have completed treatment course or not. Imputation is |
|---|---|---|---|
|---|---|---|---|

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Questionnaire (HIVTSQ) during the SC Injection Phase as well as change from SC during the Return to IM Gluteal Phase. • Perception of injection questionnaire (PIN): To assess the acceptance of pain and injection site reactions following SC abdominal and IM gluteal injections separate for CAB LA and RPV LA. • Preference Questionnaire: To | | | | not considered appropriate for any of these measures. " |

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| assess patient's | | | | |
| preference, and | | | | |
| reasons for | | | | |
| preference, for | | | | |
| injections received | | | | |
| during the SC | | | | |
| Injection Phase | | | | |
| compared with prior | | | | |
| IM gluteal | | | | |
| injections as well as | | | | |
| for injections | | | | |
| received during the | | | | |
| Return to Gluteal | | | | |
| phase compared | | | | |
| with prior SC | | | | |
| injections. | | | | |
| • Reasons for switch | | | | |
| and interest for | | | | |
| home | | | | |
| administration | | | | |
| options questions: | | | | |
| To assess the | | | | |
| reasons participants | | | | |
| agreed to switch to a | | | | |
| SC abdominal | | | | |

| | Estimand | | | |
|---|---|---|---|---|
| Endpoint | Population | Treatm<br>ent | Summary Measure | Intercurrent event (IE) / strategy / rationale |
| injection from a IM gluteal injection and their interest in a potential option for self-administration of SC injections. | | | | |

#### 2.3. Study Design



| Overview of S | tudy Design and Key Features |
|---|---|
| Interim | IDMC analyses: |
| Analysis | <ul> <li>Futility analysis at 50% of participants completing Week 24 Continuous<br/>time monitoring of confirmed virologic withdrawal (CVF) until all<br/>participants complete Week 24</li> </ul> |
| | No study summary data according to actual randomized treatment groups will be available to sponsor staff prior to the planned Week 48 analysis. |
| Planned<br>Sponsor | The main analysis will be conducted to evaluate the primary objective of the study at Week 48. |
| Analyses | <ul> <li>An additional planned analysis at Week 96 will be conducted to evaluate<br/>long-term antiviral activity, safety, and tolerability and participant<br/>satisfaction of the regimens.</li> </ul> |
| | Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications. |

#### 2.3.1. Subcutaneous Sub-Study Design

The FLAIR amendment (sub-study) will consist of three phases including a Screening/IM Gluteal injection Phase (T-4 weeks with 1 gluteal injection interval of 4 weeks), a Sub-Cutaneous Abdominal Injection Phase (12 weeks with 3 injection intervals of 4 weeks each) and a Return to Intramuscular Gluteal Injection Phase (8 weeks with 2 injection intervals of 4 weeks each). 80 participants will be targeted for enrollment in order to reach the 30-50 necessary to assess the primary PK endpoint as well as to achieve a more robust safety conclusion. At the conclusion of the sub-study, participants will have the option to continue on the FLAIR parent study or if commercial access is available, the participant can transition off the sub-study, complete their participation in the FLAIR study and proceed directly to commercially sourced CAB/RPV LA treatment.

Figure 1 Sub-Cutaneous Sub-Study Amendment Design (included as part of the Parent FLAIR Study)



Single arm, non-randomized to CAB 200mg/mL (2mL) + RPV 300mg/mL (2mL). HCP administered

Primary objectives: to describe the safety, PK and acceptability of SC CAB+RPV; Secondary objectives: VL outcomes, proportion remaining <50 cpm; PROs to include PIN, NRS and preference questionnaire and acceptance questionnaire to self-administer</li>

#### 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to show that the antiviral effect of oral ABC/DTG/3TC followed by intramuscular CAB LA + RPV LA regimen is non-inferior to continuation of ABC/DTG/3TC at Week 48 of maintenance treatment. Non-inferiority in the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL at Week 48 for Intent-to-Treat Exposed (ITT-E) population (per FDA's snapshot algorithm) can be concluded if the upper bound of a two-sided 95% confidence interval for the difference in the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL between the two treatment arms (CAB – ABC/DTG/3TC) is less than 6%.

If  $f_{la}$  is the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL for the Q4W IM arm and  $f_c$  is the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL (per FDA snapshot algorithm) for the ABC/DTG/3TC arm, then the hypotheses can be written as follows:

$$H_0$$
:  $f_{la} - f_c \ge 6\%$   $H_1$ :  $f_{la} - f_c < 6\%$
### 3. PLANNED ANALYSES

At least three analyses will be conducted to evaluate the objectives of the protocol: after all randomized participants have completed their visits at Week 48 and Week 96, respectively, and after all Extension switch participants have completed the Week 124 visit. The Week 48 analysis will be primary. Additional analysis will be conducted to evaluate the objectives of the sub-study after all participants have completed their EOS visit at Sub-study Week 20. A final End-of-Study analysis will be conducted when all participants have completed the study.

## 3.1. Interim Analyses

An Independent Data Monitoring Committee (IDMC) will be instituted to ensure external objective medical and/or statistical review of efficacy and safety in order to protect the ethical interests and well-being of participants and to protect the scientific validity of this study and study 201585.

An IDMC will evaluate accumulating efficacy, tolerability / safety, and PK of CAB LA + RPV LA at predetermined times during the study. An interim futility analysis will be performed with the intent of having approximately 50% of participants reaching Week 24 and providing sufficient lead time to allow the IDMC to review the data prior to any participants reaching the Week 48 visit. A futility rule based on Bayesian posterior predictive probability approach will be applied to assess the probability that CAB LA + RPV LA injectable regimen demonstrates non-inferiority to the continued ABC/DTG/3TC arm given the partial data set. The Sponsor will remain blinded to this analysis.

In addition, the IDMC may also monitor the incidence of participants meeting confirmed virologic failure criteria until all participants complete Week 24 to ensure that participants are not being sub-optimally treated in the CAB + RPV arm.

Full details of the analyses, estimated timing and the decision criteria that will be used to determine regimen performance will be pre-specified in the IDMC Charter.

## 3.1.1. Subcutaneous Sub-Study Interim Analyses

The SC Sub-study will contain two interim analyses. Interim analysis 1 for ISR monitoring criteria will take place after 50% of participants (equating to 25 out of an expected 50) have experienced their first SC injection with a follow-up Week 1 visit. An in-stream safety data cut will be performed for ISR data including site reports of details of ISRs of interest which include grade 4 ISRs and grade 3 ISRs that include ulceration, secondary infection, phlebitis, sterile abscess, or drainage. The posterior probability that the rate of ISRs of interest will be calculated based on ISRs of interest collected through SC Week1 for each participant. If the Bayesian posterior probability that the true rate of ISRs of interest is >0.05 (equating to > 1 participant out of 25) is low (< 5%), then individual ISRs will undergo standard safety review. However, if the Bayesian posterior probability that the true rate of ISRs of interest is >0.05 is high (≥5%), then a formal review of all ISR safety data will take place by the VSLC with the potential consideration to pause SC injections. As enrollment will be staggered by country, if 3 participants

experience an ISR of interest prior to 25 participants reaching the SC Week 1 visit, VSLC review will automatically be triggered as 3 out of 25, or a sub-study rate of 0.12, would lead to the posterior probability of the rate of ISRs of interest >0.05 being >5%. Otherwise, VSLC will only be triggered based on the interim posterior probability being >5%. An evidence threshold of 5% gives us 95% confidence that the true rate of ISRs of interest is not >0.05 should our interim posterior probability not trigger a decision to bring forth formal VSLC review. For further analysis details, see Section 8.6.

Interim analysis 2 will take place within the subcutaneous sub-study once 50% of enrolled participants have completed their sub-study Week 9 visit. The 50% threshold will have been considered reached once 15-20 participants have completed their Week 9 visit as aligned with the targeted population of 30-50 to assess the primary endpoint. The analysis will consist of an internal review of key PK, safety/tolerability, and preference endpoints in order to assist in compound development. No formal stopping decisions will be made. No formal data cleaning activities will occur. Data will be processed in stream with what is available at the time of the data cut. Queries will be issued in extreme circumstances.

## 3.2. Final Analyses

The primary analysis will be conducted to evaluate the primary objective of the protocol at Week 48. These analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed Week 48 and had a re-test if necessary.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomization codes have been distributed according to Ramos NG procedures.

Further analyses will be conducted at Week 96, Week 124, a sub-study analysis, and a final End-of-Study analysis will be conducted when all participants have completed the study.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects Screened Population | <ul> <li>Comprised of all participants screened for inclusion in the study.</li> <li>Participants may be re-screened once, for which they will receive a new subject number.</li> <li>Only the latest re-screening data will be included in the screening population summaries/analyses.</li> </ul> | Study Population |
| All Participants<br>Enrolled | All enrolled participants who receive at least one dose of study drug in the Induction Phase. | Secondary population for some analyses |
| Intent-to-Treat<br>Exposed Population<br>(ITT-E) | <ul> <li>All randomized participants who receive at least one dose of IP during the Maintenance Phase of the study (on or after Day 1 visit).</li> <li>Participants will be analyzed according to the randomized treatment regardless of what treatment was actually received.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Per-Protocol Exposed (PP) | <ul> <li>Consist of all participants in the ITT-E Population with the exception of major protocol violators.</li> <li>Protocol deviations that would exclude participants from the PP-E population are defined in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population).</li> </ul> | Efficacy (Sensitivity Analysis) |
| | This population is not applicable for the W124 analysis. | |
| Safety | <ul> <li>All randomized participants who receive at least one dose of IP during the Maintenance Phase of the study (on or after Day 1 visit).</li> <li>Participants will be assessed according to actual treatment received.</li> </ul> | Safety |
| PK Population | All participants who receive CAB and / or RPV and undergo PK sampling during the study and provide evaluable CAB and /or RPV plasma concentration data (i.e., at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values)). | • PK |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Confirmed Virologic Failure (CVF) | Comprised of all participants in the ITT-E population who met Confirmed Virologic Failure (CVF) *CVF during the Maintenance and Extension Phases is defined as: Rebound as indicated by two consecutive plasma HIV-1 RNA levels ≥200 c/mL after prior suppression to <200 c/mL | <ul><li>Genotypic</li><li>Phenotypic</li><li>IDMC CVF<br/>Analysis</li></ul> |
| All Participants<br>Randomized<br>Population | All randomized participants | Secondary population for some analyses |
| Extension Switch<br>Population (ES) | <ul> <li>All randomized subjects from ABC/DTG/3TC arm who receive at least one dose of CAB and/or RPV during the Extension Phase of the study.</li> <li>Participants will be assessed according to actual treatment received during the Extension Phase.</li> </ul> | Safety and efficacy of switching to CAB LA + RPV LA, with and without oral lead-in. |
| Long-Term Follow-up<br>Population (LTFU) | All subjects receiving at least one dose of<br>CAB LA and/or RPV LA who have<br>discontinued the CAB LA+ RPV LA regimen<br>and have a least one Long-Term Follow-up<br>Phase clinic visit. | Safety and PK during LTFU |
| Futility analysis population | Comprised of all participants in the ITT-E population who started study treatment at least 168 days prior to the IDMC cut-off date (in order to account for participants who withdrew early but would have achieved Week 24). | IDMC futility<br>analysis |
| Japan PK Population | All Japanese heritage participants (living in Japan) who receive CAB and / or RPV and undergo PK sampling and provide evaluable CAB and /or RPV plasma concentration data (i.e., at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values)). PK assay results from samples collected from a subject with emesis occurring within 4 hours of the dose will not be considered as evaluable. | Japan PK<br>displays |
| Sub-study Screened | Comprised of all participants screened for inclusion in the sub-study. | Study Population |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | All screened participants will continue using<br>their subject numbers received in the main<br>study. | |
| Sub-study Enrolled | All participants who sign informed consent into the sub-study, excluding screen failures. | Study Population |
| Sub-study Safety | All enrolled participants who received at least | Study Population |
| | one CAB and/or RPV SC injection. | Safety |
| | | Efficacy |
| | | Health Outcomes |
| Sub-study Pharmacokinetic Concentration (PC) | All participants who received at least one CAB and/or RPV SC injection and provided at least one non-missing CAB and/or RPV plasma concentration value during the substudy value (non-quantifiable values will be considered as non-missing values). | PK Concentration<br>and individual<br>figures |
| Sub-study<br>Pharmacokinetic<br>Parameter (PP) | All participants who received at least one CAB and/or RPV SC injection and had at least one evaluable PK parameter estimated during the sub-study. | PK Parameters |

- Please refer to Appendix 14: List of Data Displays for Week 48/Week 96, Appendix 15: List of Data Displays for Week 124, Appendix 19: List of Data Displays for the Subcutaneous Sub-Study, and Appendix 18: Japan-Specific Requirements which details the population to be used for each display being generated.
- In all documents, datasets and data displays the term "Subject" and "Participant" are interchangeable.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population)].

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

Randomized treatment groups will be displayed as shown in Table 2.

Table 2 Data Display Treatment Descriptors for Randomized Arms

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Randomization System Data Displays for Reporting | | | |
| Code | Description | Description | Order in TLF |
| Α | CAB LA + RPV LA | Q4W IM | 1 |
| В | ABC/DTG/3TC | ABC/DTG/3TC | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

• Q4W IM vs. ABC/DTG/3TC

In data displays of Induction Phase data for the All Enrolled Population and Extension Phase data for the Extension Switch population, respectively, study treatment will be displayed as shown in Table 3.

Table 3 Data Display Treatment Descriptors for All Enrolled Population and Extension Switch Population

| Data Type | Descriptor |
|---|---|
| Induction Phase Data for All Enrolled Population | Induction Phase ABC/DTG/3TC |
| Extension Phase Data for Extension Switch Population | Switch Q4W IM (Direct to Inject) |
| | Switch Q4W IM (Oral Lead-In) |

## 5.2. Baseline Definitions

For all assessments evaluated at Screening and/or Week -20 (including labs, vital signs, ECGs, virology assessments, etc.), the Induction Baseline (Week -20) value will be the latest valid (e.g., fasting for lipids) Pre-treatment value observed. This is generally expected to be from the Week -20 visit, although such values may be missing, or unscheduled assessments may be performed before treatment start; however, for virology data, this is generally expected to be from the Screening visit (except in the case of CVF for which virology data is expected at Week -20).

Electrocardiograms (ECGs) are to be performed in triplicate on Week -20 visit. The Induction Baseline (Week -20) value for an ECG parameter will be the mean of the last pre-treatment set of assessments from the same date.

If pre-treatment genotypic/phenotypic results are available from both the central laboratory and Monogram Biosciences, then Induction Baseline (Week -20) genotype/phenotype will be determined based only upon the data provided by Monogram assays.

The baseline value for each phase of the study is defined as the last valid (e.g., fasting for lipids) value observed, up to and including date of first dose of study treatment in the respective phase as described in Table 4.

Baseline values for the sub-cutaneous sub-study will be assigned as the last observation prior to the first CAB and/or RPV SC injection in the subcutaneous abdominal phase.

Table 4 Baseline Definitions for Each Study Phase

| Definition | Reporting Details |
|---|---|
| Induction Baseline (Week -20) | Last available recorded value up to and including the date of first Induction Phase dose of IP |
| Maintenance Baseline (Day 1) | Last available recorded value up to and including the date of first Maintenance Phase dose of IP |
| Extension Baseline (Week 100) | Last available maintenance phase recorded value up to and including the date of first Extension Phase dose of IP (Oral CAB/RPV or CAB/RPV LA) |

| Definition | Reporting Details |
|---|---|
| | <ul> <li>only applicable to the Extension Switch population participants.</li> </ul> |
| | population participants. |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

Data will be summarized for all centres combined. Country will be treated as an exploratory subgroup for analyses of the primary efficacy endpoint as described in Section 7.1.5.1. and secondary efficacy endpoint (HIV-1 RNA <50 c/mL) as described in Section 7.2.5.1. Some countries may be combined for exploratory subgroup analyses with consideration due to the number of participants enrolled.

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Strata | Randomization Strata: |
| | For the proportion of participants with plasma HIV-RNA greater than or equal to 50 c/mL per FDA Snapshot algorithm at Week 48 (primary endpoint), a stratified analysis with Cochran-Mantel Haenszel weights will be used to adjust the primary treatment comparison for the randomization strata corresponding to sex at birth and Induction Baseline (Week -20) HIV-1 RNA (<100,000, ≥100,000 c/mL). A similar approach will be used to adjust the analysis of the proportion of participants with HIV-1 RNA <50 c/mL (per the FDA's Snapshot algorithm) at Week 48 (key secondary endpoint) and repeat analyses of these endpoints at Week 96. |
| | See Section 7.1.5 for more details on the statistical analysis methodology. |
| Other Subgroups/Covariates | See details in Section 5.4.2 |
| Subcutaneous Sub-Study | |
| Covariate | Sub-study Baseline BMI The primary endpoint comparison between the SC and IM PK parameters as well as ISR incidence between SC and IM will be calculated considering Baseline BMI taken at the start of sub-study SC dosing as a covariate to account for potential individual differences in compound distribution. The |
| | following levels will be used: ■ BMI ≥ 30 kg/m² ■ BMI < 30 kg/m² |

## 5.4.2. Examination of Subgroups/Covariates

The following is a list of subgroups that may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of participants is small within a particular subgroup, then the subgroup categories may be combined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.
- For subgroup analysis, per European Medicines Agency Guideline on the investigation of subgroups in confirmatory clinical trials (EMA, 2013), factors defining a subgroup population may be put in three categories:

EMA Subgroup Category 1: Factors with strong reason to expect a heterogeneous response to treatment. In this case separate trials should usually be planned. There are no factors falling into this category in this study.

EMA Subgroup Category 2: Factors with at least some biological plausibility or external evidence such that a heterogeneous response might be hypothesized. In this study, stratified randomisation strata, key demographic and baseline characteristic factors, will fall into this category. For these factors, subgroup analyses will be performed but likely underpowered so that a formal proof of efficacy will not be available individually in all subgroups. If consistent findings across multiple comparisons were observed, then these analyses would still be suggestive of a generalizable finding from the overall population.

EMA Subgroup Guideline Category 3: Factor with good argumentation why homogeneity of response to treatment is plausible. The impact of factors falling into this category will be explored.

Additional covariates of clinical interest may also be considered.

| Category | Covariates and / or Subgroups |
|---|---|
| EMA Subgroup Category 2: | |
| Stratified Randomisation Strata | <ul> <li>Induction Baseline (Week -20) HIV-1 RNA (&lt;100,000, ≥100,000 c/mL)</li> <li>Gender at birth (Male, Female)</li> </ul> |
| | For analysis purposes, randomization strata will be derived using eCRF data, even if this differs from the strata captured in RAMOS NG. |
| | All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| Demographic and Baseline<br>Characteristic Subgroups | Age: |

| Category | Covariates and / or Subgroups |
|---|---|
| | <35; 35-<50; ≥50 (for statistical modelling analysis, the first two groups will be combined, i.e., <50, ≥50) |
| | Race: |
| | <ul> <li>White; Non-White (for statistical modelling analysis)</li> <li>Black/ African American; Non- Black/ African American</li> </ul> |
| | <ul> <li>Country (not used for statistical modelling)</li> <li>Canada;</li> <li>France;</li> <li>Germany;</li> <li>Italy;</li> <li>Japan</li> <li>The Netherlands;</li> <li>Russian Federation;</li> <li>South Africa;</li> <li>Spain;</li> <li>United Kingdom;</li> <li>United States</li> </ul> |
| | <ul> <li>Region <ul> <li>Western/Central Europe and North America (grouping of Canada, France, Germany, Italy, The Netherlands, Spain, United Kingdom, United States)</li> <li>Japan;</li> <li>Russian Federation;</li> <li>South Africa.</li> </ul> </li> <li>Induction Baseline (Week -20) HIV-1 RNA c/mL <ul> <li>&lt;1000;</li> <li>1000 to &lt;10,000;</li> <li>10,000 to &lt;50,000;</li> <li>50,000 to &lt;100,000;</li> <li>≥100,000 to &lt;200,000;</li> <li>≥200,000 c/mL</li> </ul> </li> </ul> |
| | The above subgroup with granular categories for viral load will not be used in statistical modelling. |
| | <ul> <li>Visit of First Suppression (HIV-1 RNA &lt;50 c/mL)<sup>a</sup>:</li> <li>Week -20</li> <li>Week -16;</li> <li>Week -12;</li> <li>Week -8;</li> </ul> |

| Category | Covariates and / or Subgroups |
|---|---|
| | ○ Week -4 |
| | <ul> <li>Maintenance Baseline (Day 1) HIV-1 RNA:</li> <li> <ul> <li>&lt;50;</li> <li>≥ 50 c/mL.</li> </ul> </li> </ul> |
| | <ul> <li>Induction Baseline (Week -20) CD4+ cell count:</li> <li>&lt;200;</li> <li>200 to &lt;350;</li> <li>350 to &lt;500;</li> <li>≥ 500 cells/mm³.</li> </ul> |
| | <ul> <li>Maintenance Baseline (Day 1) CD4+ cell count:</li> <li>&lt;200;</li> <li>200 to &lt;350;</li> <li>350 to &lt;500;</li> <li>≥ 500 cells/mm³.</li> </ul> |
| | <ul> <li>Derived Maintenance Baseline (Day 1) Centers for Disease Control and Prevention (CDC) category: <ul> <li>Stage I;</li> <li>Stage II;</li> <li>Stage III</li> </ul> </li> </ul> |
| | <ul> <li>HIV-1 Subtype at Induction Baseline (Week -20)</li> <li>A;</li> <li>A1;</li> <li>AE;</li> <li>AG;</li> <li>B;</li> <li>C;</li> <li>Other</li> </ul> |
| | <ul> <li>Missing</li> <li>K103N Mutation at Induction Baseline (Week -20):</li> </ul> |
| | ○ Yes vs. No |
| | <ul> <li>Induction Baseline (Week -20) BMI (&lt;30, ≥ 30 kg/m<sup>2</sup>)</li> </ul> |
| | <ul> <li>L74I Integrase Mutation at Induction Baseline (Week - 20):</li> <li>Yes vs. No (Note: do not derive is baseline integrase genotype is not available)</li> </ul> |
| EMA Subgroup Category 3: | |
| Additional subgroup/covariates for PK/PD efficacy analysis | Week 48 Analysis Only: Last CAB/RPV Trough (predose) PK concentration by Week 48 (i.e., If pre-dose PK concentration at nominal Week 48 is missing, then last pre-dose PK concentration prior to Week 48 will be used) |

| Category | Covariates and / or Subgroups |
|---|---|
| | Week 8 CAB/RPV Trough PK concentration (i.e., pre-<br>dose PK concentration at nominal visit of Week 8 |
| | The above two covariates will be dichotomized into two subgroup factors as follows: |
| | <ul> <li>Needle length for CAB injection at Week 4b: (&lt;2, ≥2 inch);</li> <li>Needle length for RPV injection at Week 4b: (&lt;2, ≥2 inch);</li> <li>See Section 8.5.1 for additional details regarding attribution of ISRs to causal agent (CAB/RPV) and Needle Length.</li> </ul> |
| | <ul> <li>Induction Baseline (Week -20) BMI (&lt;30, ≥ 30 kg/m<sup>2</sup>)</li> </ul> |
| Additional subgroup/covariates for PK/PD safety analysis – | Last CAB/RPV trough PK concentration |
| Week 48 Analysis Only | For the plot of "Maximum Change from Maintenance Baseline (Day 1), CBF, in ALT/Total Bilirubin versus Last Trough CAB/RPV PK Concentrations", Last CAB/RPV Trough PK concentration is the most recent trough PK concentration prior or equal to the date of the earliest Lab assessment corresponding to the maximum CFB during the Maintenance Phase. |
| | For the Plot of "Maximum Toxicity Grades of Most Frequently Reported AEs versus Last Trough CAB/RPV PK Concentrations", Last CAB/RPV Trough PK concentration is the most recent trough PK concentration prior or equal to the earliest onset date of maximum graded AE (for each preferred term among non-ISR AEs occurring in ≥5% of participants in the Q4W arm during the Maintenance Phase). If a participant does not experience the corresponding preferred term event during the Maintenance Phase, then the last trough value during the Maintenance Phase will be used for the plot. |
| Additional subgroup for Bone<br>Marker analysis | <ul> <li>Induction Baseline (Week -20) BMI (kg/m^2) <ul> <li>&lt;30;</li> <li>≥30</li> </ul> </li> <li>Smoking status at Screening: <ul> <li>Never;</li> <li>Current;</li> <li>Former</li> </ul> </li> </ul> |

| Category | Covariates and / or Subgroups |
|---|---|
| | <ul> <li>Tenofovir Disoproxil Fumarate (TDF) Use at Maintenance Baseline (Day 1)</li> <li>Yes;</li> <li>No</li> </ul> |
| Additional subgroup for ISR | <ul> <li>For each common ISR preferred term (pain, induration, nodules and any other ISR with &gt;=5% participants during the Maintenance Phase, Maintenance + Extension Phase (for Randomized Q4W), and Extension Phase (for Switch Q4W), respectively:</li> <li>Needle Length for Last CAB Injection prior to and including the onset date of the earliest corresponding drug-related CAB ISR with maximum toxicity grade during the phase(s) of interest: (&lt;2, ≥2 inch);</li> <li>Needle Length for Last RPV Injection prior to and including the onset date of the earliest corresponding drug-related RPV ISR with maximum toxicity grade during the phase(s) of interest: (&lt;2, ≥2 inch);</li> <li>The above subgroup variables will be produced for each common ISR preferred term.</li> <li>Note: If there is no ISR of interest reported during the phase(s) of interest for a participant, these subgroup variables will be derived using the needle length of the participant's last injection during the phase(s) of interest.</li> </ul> |
| Subcutaneous Sub-Study subg | roups |
| Demographic, Efficacy, Safety, PK, & HO Subgroups | <ul> <li>Age:</li> <li>&lt;35; 35-&lt;50; ≥50</li> <li>Sex at birth</li> <li>Male, Female</li> <li>Race/Ethnicity</li> <li>White: Non-Hispanic, White: Hispanic, Black, Asian, Other</li> <li>Sub-study Baseline BMI</li> <li>&lt;30 kg/m², ≥30kg/m²</li> </ul> |

a) Based on any HIV-1 RNA <50 c/mL within the assessment window defined in Table 14.

# 5.5. Multiple Comparisons and Multiplicity

## 5.5.1. Primary Comparison of Interest

The primary analysis will be based on the ITT-E population. The primary comparison will be made at a one-sided 2.5% level of significance. Treatment with Q4W IM will be declared non-inferior to ABC/DTG/3TC if the upper end of a two-sided 95% confidence interval for the difference between the two groups (Q4W IM– ABC/DTC/3TC) in the

proportion of participants with HIV-RNA ≥50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) lies below 6%.

The primary comparison of interest is the comparison between Q4W IM and ABC/DTC/3TC for the primary endpoint in the ITT-E population. This analysis will be adjusted for by the stratification factor applied at randomization.

If the primary analysis shows non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring CAB LA + RPV LA will be declared if the upper end of the confidence interval is below 0% for the ITT-E population analysis. If superiority is declared, the p-value for superiority will also be calculated.

#### 5.5.2. Other Comparisons of Interest

The analysis described above will also be performed using the PP population and the results will be compared for consistency with the results from the ITT-E population.

#### 5.5.3. Secondary Comparisons

If the primary comparison of interest (Section 5.5.1) using the ITT-E population demonstrates non-inferiority of Q4W compared to ABC/DTG/3TC then the following key secondary comparisons using the ITT-E population will be tested:

- Treatment with Q4W IM will be declared non-inferior to ABC/DTG/3TC with respect to the proportion of participants with HIV-1 RNA < 50 copies/mL at Week 48 (defined by the US FDA snapshot algorithm) if the lower end of a two-sided 95% confidence interval for the difference in response rates (Q4W IM– ABC/DTG/3TC) lies above -10%.
- Superiority of Q4W IM compared to ABC/DTG/3TC with respect to change from maintenance baseline (Day 1) HIVTSQs total score at Week 44 using a two-sided 5% level of significance.
- Changes in the PIN acceptance score within the Q4W arm over time using separate two-sided 5% level of significance tests for the change from Week 5 to Week 41 and change from Week 5 to Week 48, respectively.

There are no planned adjustments for multiple comparisons or multiplicity.

For the primary endpoint treatment comparison at Week 48, no multiple comparison adjustment is necessary for testing non-inferiority followed by superiority (conditional on achieving a significant test for non-inferiority) since testing follows a pre-specified sequence of hypothesis such that if the first hypothesis tested is not significant, all subsequent tests will not be performed. This fixed sequence procedure controls the type I error rate at the nominal level.

In addition to the primary and the key secondary comparisons, the comparisons between two treatment arms for ACCEPT (general acceptance score), SF-12 (health status), and HAT-QoL (Life satisfaction) at timepoints through Week 48 will also be performed as supportive analyses.

Lastly, for the IDMC interim analyses, since the statistical stopping guidelines will not result in early stopping for positive efficacy findings, these interim treatment comparisons will not inflate the Type I error rate for the primary treatment comparison.

#### 5.5.3.1. Week 124 Extension Switch Analysis

For the Week 124 Extension Switch population analysis, antiviral response will be assessed according to the proportion of participants with and without oral lead-in, respectively, who have HIV-1 RNA ≥50 c/mL at Week 124 (i.e., 24 weeks from initiation of CAB LA + RPV LA, +/- 6 week analysis window, using the FDA Snapshot algorithm), with corresponding 95% confidence interval. The primary efficacy endpoint of interest for this analysis is the proportion of participants without oral lead-in who have HIV-1 RNA ≥50 c/mL at Week 124. No formal statistical comparisons with respect to safety and efficacy outcomes will be performed.

#### 5.5.3.2. Subcutaneous Sub-Study Analysis

For the Subcutaneous sub-study analysis, select pharmacokinetic parameters from both the gluteal phase and the subcutaneous phase will be informally compared with a geometric mean ratio and corresponding 90% confidence interval. No formal statistical comparisons with respect to safety and efficacy outcomes will be performed.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

### CONFIDENTIAL

| Section | Component |
|---------------|--------------------------------------------------------------|
| Section 14.2 | Appendix 2: Schedule of Activities |
| Section 14.3 | Appendix 3: Assessment Windows |
| Section 14.4 | Appendix 4: Study Phases and Treatment State |
| Section 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 14.6 | Appendix 6: Derived and Transformed Data |
| Section 14.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 14.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 14.9 | Appendix 9: Population Pharmacokinetic (PopPK) Analyses |
| Section 14.10 | Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses |
| Section 14.11 | Appendix 11: Snapshot Algorithm Details |
| Section 14.14 | Appendix 14: List of Data Displays for Week 48/Week 96 |
| Section 14.15 | Appendix 15: List of Data Displays for Week 124 |
| Section 14.16 | Appendix 16: IDMC |
| Section 14.17 | Appendix 17: Variables Defined for Time to Event Analysis |
| Section 14.18 | Appendix 18: Japan-Specific Requirements |
| Section 14.19 | Appendix 19: List of Displays for the Subcutaneous Sub-study |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

Details of the planned study population displays for the Week 124 analysis are provided in Appendix 15: List of Data Displays for Week 124. The study population analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and treatment accountability will be based on GSK Core Data Standards.

Table 5 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 5 Overview of Planned Study Population Analyses

| Display Type | Data Disp | lays Generated |
|---|---|---|
| | Table | Listing |
| Randomisation | | |
| Randomisation [1] | | <b>Y</b> [2] |
| Subject Disposition | | |
| Study Populations [3] | Y | |
| Study Recruitment [3] | Υ | |
| Reasons for Screening Failures [3] | Y | Y |
| History of Rescreened Participants [3] | | |
| Age categories | Υ | |
| Subject Disposition | <b>Y</b> [4][5] | |
| Reasons for Withdrawal by Visit | <b>Y</b> [4][5] | Y |
| IP discontinuation | Υ | Y |
| Important Protocol Deviations | Y | Y |
| Deviations leading to exclusion from PP | Y | Υ |
| Inclusion and Exclusion Criteria Deviations | Y | Υ |
| Demography and Baseline | | |
| Demographics Characteristics [6] | Y | Υ |
| Race & Racial Combinations [7] | Y | Υ |
| Hepatitis Status at Induction Baseline (Week -20) | Y | |
| CDC Classification of HIV infection (2014) at Maintenance<br>Baseline (Day 1) | Y | |
| Cardiovascular Risk Assessments at Induction Baseline (Week - 20) | Y | |

| Display Type | Data Dis | plays Generated |
|---|---|---|
| | Table | Listing |
| Distribution of CD4+ Cell Counts at Maintenance Baseline (Day 1) | Υ | |
| Distribution of Quantitative Plasma HIV-1 RNA and CD4+ Cell Counts at Screening and Induction Baseline (Week -20) | Y | |
| HIV-1 Subtype at Induction Baseline (Week -20) | Y | |
| Medical Conditions, Concomitant Medications & Antiretrov | riral Therapy | |
| Medical Conditions (Current/Past) [8] | Y | |
| Medical Conditions: Sub-conditions (Current/Past) [9, 10] | Y | |
| Concomitant Medications (non-ART) | Υ[10] | |
| Prior Antiretroviral Therapy | | Y |
| Concomitant Antiretroviral Therapy during Induction and Maintenance Phase, respectively | | Y |
| ART Regimen at Randomization | Y | Y |
| Lipid Modifying Agents (Maintenance Baseline (Day 1) and During Maintenance Phase) | Υ | |
| Substance use at Screening | Y | |
| Medical History of Seizure | | Y |
| Other | | |
| Study Treatment Accountability [11] | | Υ |
| Transition to CAB+RPV LA Marketed Product | | Y |

- T = Tables, L = Listings, Y = Display Generated,
- a. All Participants Randomized population
- b. One listing of participants randomized but not treated, and one listing of planned and actual treatment strata.
- c. All Subjects screened population.
- d. Participants who have not been recorded as either completing or withdrawing from the study will be categorized as "Ongoing at time of the analysis" for summary purposes.
- e. Analysis of subject disposition will be performed for each study Phase separately, as well as for overall study
- f. Age and ethnicity collected at Screening; weight and height collected at Baseline (Week -20)
- g. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high-level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- h. Medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
- Sub conditions are Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions
- i. summarised by Ingredient combinations
- k. Dispensation information (dates and number of tablets dispensed and returned).

# 6.2. Subcutaneous Sub-Study Population Analyses

Participant sub-study enrollment, protocol deviations, concomitant medications, and sub-study disposition for the SC injection phase, return to gluteal phase, and overall will be summarized for the sub-study screening, enrolled, and safety populations where

#### **CONFIDENTIAL**

201584

appropriate. Time on prior CAB+RPV treatment though the start of the SC abdominal injection phase will be summarized. Oral Bridging will not be summarized as participants requiring oral bridging will discontinue the sub-study per the protocol. Transition either back to the parent study or to commercial product will be summarized as applicable for sub-study participants. See <a href="Appendix 19">Appendix 19</a>: List of Data Displays for Subcutaneous Sub-Study Analysis for further details.

#### 7. EFFICACY ANALYSES

Details of the planned efficacy displays for the Week 124 analysis are provided in Appendix 15: List of Data Displays for Week 124.

## 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoint / Variables

Proportion of participants with plasma HIV-RNA greater than or equal to 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Week 48 (Intent-to-Treat Exposed [ITT-E] population); see <u>Section 14.11</u> for additional details.

## 7.1.2. Summary Measure

Difference in the proportion of participants with HIV-RNA ≥50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) between each treatment group (Q4W IM – ABC/DTG/3TC).

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Intent-To-Treat Exposed population, unless otherwise specified.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the Snapshot algorithm, HIV-RNA  $\geq$  50 c/mL is determined by the last available HIV-1 RNA measurement while the participant is on treatment within the analysis visit window of interest.

Participants without evaluable HIV-RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq 50$  c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-RNA  $\geq 50$  c/mL.

### 7.1.5. Statistical Analyses / Methods

Table 6 provides an overview of the planned efficacy analyses. Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK data standards and statistical principles.

Table 6 Overview of Planned Primary Efficacy Analyses

| Endpoints | St | Stats Analysis Summary | | | | Indivi | dual |
|---|---|---|---|---|---|---|---|
| | T | F | L | T | F | F | L |
| Proportion of Participa | nts with ' | HIV-1 ≥ \$ | 50 c/mL' a | at Week 48 – \$ | Snapshot | | |
| Primary analysis comparison between the two groups (Q4W IM – ABC/DTG/3TC) in 'HIV-1 RNA≥50 c/mL' rates at Week 48 | <b>Y</b> [1] | | | <b>Y</b> [1,2] | <b>Y</b> [4] | | <b>Y</b> [2] |
| Treatment Heterogeneity across randomization strata | Y | | | | | | |
| By Subgroup [3]<br>(Exploratory analysis<br>to support primary<br>analysis) | | | | <b>Y</b> [5] | <b>Y</b> [4] | | |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Generated using the 'Intent-to-Treat Exposed' (primary) and 'Per-Protocol' (sensitivity) populations.
- 2. Study outcomes (i.e., response below 50 c/mL, 'HIV-1 RNA≥50' or reason for no data in the window) based on the snapshot algorithm.
- 3. Randomisation Strata, Demographic and Baseline Characteristics (refer to Section 5.4.2).
- 4. Plot of the difference in proportion of participants with HIV-1 RNA ≥50 c/mL (Snapshot algorithm) and its 95% confidence intervals for 'overall' (on the top of the figure) and by subgroup at Week 48.
- 5. Study outcomes based on the Snapshot algorithm by subgroup at Week 48 will also be produced.

#### 7.1.5.1. Statistical Methodology Specification

## **Primary Statistical Analyses**

#### **Endpoint**

 Proportion of Participants with Plasma HIV-1 ≥ 50 c/mL at Week 48 using the Snapshot algorithm for the ITT-E population. 'HIV-1 RNA≥50' are based on the Snapshot algorithm includes participants who had plasma HIV-1 RNA ≥ 50 c/mL at Week 48, who discontinued for lack of efficacy, who discontinued for other reasons while not <50 c/mL, or who changed ART).</li>

#### **Snapshot Dataset**

- Virologic outcome ('HIV-RNA <50' or '≥ 50 c/mL') per Snapshot algorithm is determined by the
  last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest
  (please refer to analysis window defined in Table 17). In addition, participants who discontinue
  for reasons not related to adverse event with on-treatment HIV-1 RNA result at the time of
  discontinuation ≥ 50 c/mL or who change study treatment not permitted per protocol during
  Maintenance Phase before the analysis visit are classified as 'HIV-RNA ≥ 50 c/mL'.</li>
- Full details of the Snapshot algorithm are provided in Section 14.11.

#### **Primary Statistical Analyses**

#### **Model Specification**

- The primary efficacy endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for Induction Baseline (Week -20) HIV-1 RNA (<100,000, ≥100,000 c/mL) and gender at birth.</li>
- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each of the following four analysis strata:
  - o Induction Baseline (Week -20) HIV-1 RNA < 100 000 c/mL AND Male gender at birth
  - Induction Baseline (Week -20) HIV-1 RNA < 100 000 c/mL AND Female gender at birth
  - o Induction Baseline (Week -20) HIV-1 RNA ≥ 100 000 c/mL AND Male gender at birth
  - o Induction Baseline (Week -20) HIV-1 RNA ≥ 100 000 c/mL AND Female gender at birth
- If n<sub>k</sub> is the number of CAB LA + RPV LA treated participants, m<sub>k</sub> is the number of ABC/DTG/3TC control arm treated participants, and N<sub>k</sub> = n<sub>k</sub> + m<sub>k</sub> is the total number of participants in the kth stratum, then the CMH estimate is given by

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and  $\hat{d}_k$  are estimates of the differences in proportions between the two treatment arms,  $f_{la}$  -  $f_c$  for the *kth* stratum.

The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\hat{\text{var}}(\hat{d}_{cmh})}$$

where the variance estimator [Sato, 1989] is consistent in both sparse data and large strata and is given below

$$\operatorname{var}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

#### **Primary Statistical Analyses**

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

with  $x_k$  and  $y_k$  corresponding to the number of participants with Plasma HIV-1 RNA  $\geq$  50 c/mL at Week 48 per FDA Snapshot for CAB LA + RPV LA and ABC/DTG/3TC control arm, respectively, for the *kth* stratum.

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of participants with 'HIV-1 RNA≥50' between each treatment group (CAB LA + RPV LA ABC/DTG/3TC) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval
  (CI) for the CMH adjusted difference in proportion of participants with 'HIV-1 RNA≥50' in the
  CAB LA + RPV LA group minus proportion of participants with 'HIV-1 RNA≥50' in the
  ABC/DTG/3TC group is less than 6%.
- If the analysis shows non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring CAB LA + RPV LA will be declared if the upper end of the confidence interval is below 0% for the ITT-E population analysis. If superiority is declared, the p-value for superiority will also be calculated.

#### **Subgroup Analyses**

- 1. Treatment Heterogeneity across randomization strata:
  - The weighted least squares chi-squared statistic [Fleiss, 1981] will be used to test for one-way homogeneity across the levels of each categorical variable, with each categorical variable considered separately.
  - Following Lui and Kelly [Lui, 2000] ½ will be added to each cell in any strata for which
    the stratum-specific rate estimates of either fla or fc are zero or one, and tests will be
    one-sided.
  - Any heterogeneity found to be statistically significant will be explored and if necessary
    results will be reported for each level of the categorical variable. Investigation of
    heterogeneity will be confined to the primary. Tests of homogeneity will be assessed at
    the one-sided 10% level of significance.

## 2. Exploration of Subgroups

- An analysis for demographic and baseline characteristic subgroups listed in Section 5.4.2 will be performed. This will show the proportion of participants with plasma HIV-1 RNA ≥50 c/mL at the time of analysis (Week 48) based on the Snapshot algorithm and will be presented by treatment group.
- Unadjusted difference in proportions between treatment groups and corresponding two-sided 95% CI will also be presented by subgroups. The confidence interval will be calculated using an unconditional exact method (Chan, 1999) with two inverted onesided tests based on the score statistic. These results will also be presented graphically.
- Summary of study outcomes (i.e., response below 50 c/mL, 'HIV-1 RNA≥50'or reason for no data in the window) by subgroup will be produced.

## **Primary Statistical Analyses**

Note: These subgroup analyses will be exploratory and likely underpowered so that interpretation may therefore focus on point estimates as well as the upper bounds of 95% CIs for the treatment differences and response rates. Additionally, multiple comparisons are being made which inflates the risk of false positive findings. Therefore, if consistent findings across the multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding of non-inferiority.

#### **Sensitivity and Supportive Analyses**

1. Per-protocol population analysis:

To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis.

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

Proportion of participants with plasma HIV-1 RNA <50 c/mL at Week 48 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population).

Subcutaneous sub-study efficacy endpoints for the study are listed below:

- Proportion of participants with plasma HIV-1 RNA < 50 c/mL at Week 12 using the FDA Snapshot algorithm during the Sub-study Subcutaneous Abdominal Injection phase (Sub-study Safety population)
- Proportion of participants with plasma HIV-1 RNA ≥ 50 c/mL at Week 12 using the FDA Snapshot algorithm during the Sub-study Subcutaneous Abdominal Injection phase
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) of ≥200 c/mL through Week 12 of the Sub-study Subcutaneous Abdominal Injection phase
- Incidence of treatment emergent genotypic and phenotypic resistance to CAB, RPV during the SC injection phase.

The incidence of observed genotypic and phenotypic resistance to NRTIs and INIs, PIs, and NNRTIs will be summarized for subjects meeting confirmed virologic failure criteria.

The proportion of participants with HIV-1 RNA ≥50 c/mL and HIV-1 RNA <50 c/mL at Week 12 of the SC injection phase will be summarized using FDA Snapshot algorithm for the Safety population in the sub-study. Proportion of participants with protocol-defined confirmed virologic failures at Week 12 will also be summarized. Summaries will be presented by subgroup as needed where data allow.

### 7.2.2. Summary Measure

Difference in the proportion of participants with HIV-RNA < 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) between each treatment group (Q4W IM – ABC/DTC/3TC).

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

## 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Participants with last available HIV-1 RNA measurement less than 50 c/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA < 50 c/mL.

### 7.2.5. Statistical Analyses / Methods

Table 7 provides an overview of the planned efficacy analyses. Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK data standards and statistical principles.

# Table 7 Overview of Planned Secondary Efficacy Analyses

| Endpoints | St | ats Analy | sis | Sum | mary | Indiv | /idual |
|---|---|---|---|---|---|---|---|
| | Т | F | L | Т | F | F | L |
| Proportion of Participa | nts with ' | HIV-1 ≥ 5 | 50 c/mL' a | at Week 96 – 9 | Snapshot [1] | | |
| | <b>Y</b> [2] | | | <b>Y</b> [2,3] | <b>Y</b> [5] | | <b>Y</b> [3] |
| Treatment<br>Heterogeneity across<br>randomization strata | Y | | | | | | |
| By Subgroup [4] (Exploratory analysis) | | | | <b>Y</b> [6] | <b>Y</b> [5] | | |
| Proportion of Participa | nts with I | Plasma H | IV-1 < 50 | c/mL at Weel | k 48/Week 96 | – Snapshot [1 | ] |
| Key Secondary<br>Analysis (Week 48) | <b>Y</b> [2] | | | <b>Y</b> [2, 3] | Y | | <b>Y</b> [3] |
| Treatment<br>Heterogeneity across<br>randomization strata | Y | | | | | | |
| Proportion of Participal discontinuation (TRDF) | | | | | | r treatment-re | elated |
| Kaplan-Meier estimate | | | | Υ | | | |
| Proportion of Participal Snapshot | nts with I | Plasma H | IV-1 RNA | ≥ 50 copies/ | mL over time | (Maintenance | e Phase)– |
| by Visit | | | | Υ | <b>Y</b> [7] | | |
| by Visit and<br>Subgroup <sup>[4]</sup> | | | | Υ | <b>Y</b> [9] | | |
| Proportion of Participal Snapshot | nts with I | Plasma H | IV-1 RNA | < 50 copies/ | mL over time | (Maintenance | Phase)- |
| by Visit | | | | Υ | <b>Y</b> [8] | | |
| by Visit and Subgroup | | | | Υ | <b>Y</b> [9] | | |
| Proportion of Participal Snapshot | nts with I | Plasma H | IV-1 RNA | < 200 copies | /mL over time | e (Maintenand | ce Phase)- |
| by Visit | | | | <b>Y</b> [10] | Υ[11] | | |
| Proportion of Participal | nts with I | Plasma H | IV-1 RNA | ≥ 200 copies | s/mL over time | e – Snapshot | |
| by Visit | | | | <b>Y</b> [10] | Υ[11] | | |
| Proportion of Participal | | | IIV-1 RNA | < 50 copies/ | mL at Week 4 | 8 by delay in | IP injection |
| by Delay in IP injection | - | | | Y | | | |
| Proportion of Participa | nts with I | Plasma H | IV-1 RNA | < 2 copies/m | L (explorator | y analysis) | |
| by Visit - Observed<br>Case Analysis | | | | <b>Y</b> [13] | | | |

| Endpoints | St | ats Analys | sis | Sum | mary | Indiv | ridual |
|---|---|---|---|---|---|---|---|
| | T | F | L | T | F | F | L |
| Time from First HIV-1 R | NA < 50 | copies/m | L until In | itiation of Ma | intenance Ph | ase Treatmen | t |
| | | | | Υ | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. This analysis will be performed using the same approach as described for the primary analysis in Section 7.1.
- 2. Generated using the 'Intent-to-Treat Exposed' (primary) and 'Per-Protocol' (sensitivity) populations.
- 3. Study outcomes (i.e., response below 50 c/mL, 'HIV-1 RNA≥50' or reason for no data in the window) based on the snapshot algorithm.
- 4. Randomisation Strata, Demographic and Baseline Characteristics (refer to Section 5.4.2).
- 5. Plot of the difference in proportion of participants with HIV-1 RNA ≥50 c/mL (Snapshot algorithm) and its 95% confidence intervals for 'overall' (on the top of the figure) and by subgroup at Week 96.
- 6. Study outcomes based on the Snapshot algorithm by subgroup at Week 96 will also be produced.
- 7. Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation.
- 8. Line plots, with 95% confidence intervals, for the proportion of participants with HIV-1 RNA<50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 100%; otherwise, they are derived using the normal approximation.
- 9. Plot of the unadjusted treatment difference and its 95% confidence intervals (Snapshot algorithm) overall and by subgroup at Week 48/Week 96.
- 10. Study outcomes (i.e., HIV-1 RNA< 200 c/mL, HIV-1 RNA≥200c/mL, or reason for no data in the window) based on the snapshot algorithm by subgroup for Week 48/Week 96 will also be produced.
- 11. Line plots, with 95% confidence intervals, for the proportion of participants with HIV-1 RNA <200c/mL and ≥200 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0% or 100%; otherwise, they are derived using the normal approximation
- 12. Delay in IP injection (days) is defined in Section 14.6.4
- 13. Using observed case (OC) data which contains the data that is available at a particular time point, with no imputation for missing values and expanded  $\pm$  6-week window for W48/W96 and last value in window (see Section 14.6.4).

#### Table 8 Overview of Additional Secondary Efficacy Analyses

| Endpoints | Absolute | | | | | | | | Change from Maintenance Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | Ш | Т | F | F | Ш |
| Plasma HIV-1 RNA Ove | r Tim | е | | | | | | | | | | | | |
| Observed [1] | | | | <b>Y</b> [8] | | <b>Y</b> [2] | <b>Y</b> [3] | | | | Υ | | | |
| Detected vs Non-<br>detected by Visit [1,5] | | | | Υ | | | <b>Y</b> [6] | | | | | | | |
| Confirmed Virologic Fa | ilure | (CVF) | | | | | | | | | | | | |
| CVF Overall | | | | Υ | | | | | | | | | | |
| CVF by Visit | | | | Υ | | | Υ | | | | | | | |

| Endpoints | | | A | Absolu | ite | | | Change from Maintenance Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | ridual |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| HIV-1 RNA at time of<br>suspected and<br>confirmed Virologic<br>Failure | | | | Υ | | | | | | | | | | |
| CD4+ & CD8+ Cell Cou | nts O | ver Ti | me | | | | | | | | | | | |
| CD4+ observed | | | | <b>Y</b> [7] | | | | | | | <b>Y</b> [7] | | | |
| CD8+ observed | | | | <b>Y</b> [7] | | | | | | | <b>Y</b> [7] | | | |
| CD4+/CD8+ ratio observed | | | | <b>Y</b> [7] | | | | | | | | | | |
| HIV-1 Conditions and D | )iseas | e Pro | gress | ion | | | | | | | | | | |
| HIV Conditions including/excluding Recurrences as recorded in eCRF | | | | Υ | | | Υ | | | | | | | |
| HIV Disease<br>Progressions [4] | | | | Υ | | | | | | | | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Using observed case (OC) data which contains the data that is available at a particular time point, with no imputation for missing values and expanded  $\pm$  6 week window for W48/W96 and last value in window (see Section 14.6.4).
- 2. Individual plasma HIV-1 RNA only for participants who are in the category of 'viral load ≥50 c/mL' at Week 48 per Snapshot algorithm or who are CVF participants. The figures will display all HIV-1 RNA values collected.
- 3. For CVF participants (during the Induction and Maintenance Phase, respectively, and participants with viral load ≥ 50 c/mL at any time during the Maintenance Phase).
- 4. HIV disease progressions (Section 14.6.4)
- 5. See Section 14.6.4 for a definition of "Target Detected" and "Target Non-detected".
- 6. Included in the Observed HIV-1 RNA listing
- 7. Using observed case (OC) data which contains the data that is available at a particular time point, with no imputation for missing values
- 8. Using log10 transformed values

## 7.2.5.1. Statistical Methodology Specification

#### **Key Secondary Statistical Analyses**

#### **Endpoint**

 Proportion of participants with plasma HIV-1 RNA <50 c/mL at Week 48 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population)

## **Snapshot Dataset**

As described in Section 7.1.5.1 and Section 14.11

#### **Model Specification**

 As specified in Section 7.1.5.1 but with Snapshot HIV-1 RNA <50 c/mL replacing Snapshot HIV-1 ≥ 50 c/mL

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of participants with plasma HIV-1 RNA <50 c/mL at Week 48 between each treatment group (Q4W IM – ABC/DTG/3TC) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval for the CMH adjusted treatment difference (Q4W IM – ABC/DTG/3TC) is greater than -10%.

## **Subgroup Analyses**

- Treatment Heterogeneity across randomization strata:
  - $\circ$  As specified in Section 7.1.5.1 but with Snapshot HIV-1 RNA <50 c/mL replacing Snapshot HIV-1 RNA  $\geq$  50 c/mL.

#### **Sensitivity and Supportive Analyses**

Per-protocol population analysis:

To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis.

## 8. SAFETY ANALYSES

Details of the planned safety displays for the Week 124 analysis are provided in Appendix 15: List of Data Displays for Week 124.

The safety analyses will be based on the Safety population, unless otherwise specified.

For the Week 48 primary analysis, a set of separate outputs will also be presented for the oral lead-in period at Maintenance Phase, including summary of adverse events, SAE, AE leading to withdrawal, emergent chemistry/haematology abnormality, participants with hepatobiliary abnormality criteria.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 14: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify Adverse Events of Special Interest (AESI). [Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.] The details of the current planned grouping, including Standardized MedDRA Query (SMQ) values (as applicable), and planned displays are provided in Appendix 12: AESI identification and Appendix 14: List of Data Displays.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 14: List of Data Displays.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 14: List of Data Displays.

ECG Values of Potential Clinical Interest are defined as a QTc of > 550ms.

# 8.5. Planned Safety Analysis

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 9 Overview of Planned Safety Analyses

| Endpoint | Absolute | | | | Mair | | je from<br>ce Bas | | Max Post Maintenance<br>BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | /idual | Sum | mary | Indiv | idual | Sum | mary | Indiv | idual |
| | T | F | F | L | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | | | | | |
| Extent of Exposure[1] | Υ | | | <b>Y</b> [2] | | | | | | | | |
| Adherence to Q4W Dosing Schedule [1] | Y | | | | | | | | | | | |
| Injection Needle | | | | | | | | | | | | |
| Length and Gauge | Υ | | | | | | | | | | | |
| Adverse Events[3] | | | • | • | • | | • | | | • | | |
| All AEs by SOC | Y | | | | | | | | | | | |
| All AEs by SOC and Toxicity <sup>[3]</sup> | <b>Y</b> [24] | | | <b>Y</b> [4] | | | | | | | | |
| Common AEs by freq [5] | Υ | <b>Y</b> [6] | | | | | | | | | | |
| Common Grade 2-5<br>AEs [5] by freq | Y | | | | | | | | | | | |
| All Drug-Related AEs by SOC and toxicity <sup>[3]</sup> | Y | | | | | | | | | | | |
| Common Drug-related<br>Grade 2-5 AEs [5] | Y | | | | | | | | | | | |
| All AEs | | | | Υ | | | | | | | | |
| Serious and other signi | ficant a | dvers | e even | ts | • | | • | | | • | | |
| All SAEs by SOC | <b>Y</b> [24] | | | | | | | | | | | |
| Reason for Considering<br>as a Serious Adverse<br>Event (FDA) | | | | Υ | | | | | | | | |
| All Drug-Related SAEs by SOC | Υ | | | | | | | | | | | |
| Fatal SAEs | | | | Υ | | | | | | | | |
| Non-Fatal SAEs | Υ | | | Υ | | | | | | | | |
| Drug-related non-fatal SAEs | Υ | | | | | | | | | | | |
| Withdrawal AEs | <b>Y</b> [24] | | | Υ | | | | | | | | |
| Common Non-Serious<br>AEs (FDAAA) | Υ | | | | | | | | | | | |
| Number of occurrences<br>of Common Non-serious<br>AEs by SOC (EudraCT) | Υ | | | | | | | | | | | |
| Number of occurrences of SAEs, Fatal SAEs, | Υ | | | | | | | | | | | |

| Endpoint | | Abs | solute | | | | e from | | Max | | lainten<br>BL | laintenance<br>L |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | /idual | Sum | mary | Indiv | idual | Sum | mary | Indiv | idual |
| | Т | F | F | L | Т | F | F | L | Т | F | F | L |
| and Drug-related SAEs (EudraCT) | | | | | | | | | | | | |
| Cumulative AEs by visit | Υ | | | | | | | | | | | |
| Depression, Suicidal<br>and Self-Injury AEs by<br>Prior History | Υ[25] | | | | | | | | | | | |
| Suicidality assessment | | | | | | | | | | | | |
| PSRAE | | | | <b>Y</b> [7] | | | | | | | | |
| Columbia suicidality (C-SSR) | Y | | | | | | | | | | | |
| Injection Site Reaction | Advers | e Ever | its <sup>[12]</sup> | | | | | | | | | |
| ISR AEs (Event-Level) | Y | | | | | | | | | | | |
| ISR AEs (Subject-Level) | Y | Y | | | | | | | | | | |
| ISR AEs (Subject-Level) by Visit and Severity | Y | <b>Y</b> [19] | | | | | | | | | | |
| Maximum ISR AE<br>Grade by Needle<br>Length [21] | Υ | | | | | | | | | | | |
| Laboratory: Chemistry a | and He | matolo | gy | | | | | | | | | |
| Clinical Chemistry & Renal Biomarkers [11] | Y | | | | Y | | | | Y [23] | | | |
| %Lipids <sup>[22]</sup> | | | | | Υ | | | | | | | |
| NCEP shifts in lipids | | Υ | | | | | | | Υ | | | |
| Hematology | Υ | | | | Υ | | | | <b>Y</b> [23] | | | |
| Laboratory: Urinalysis ( | regard | less of | fastin | g statu | s) | | l | I. | l | | | |
| Urine Dipstick | <b>Y</b> [8] | | | | | | | | | | | |
| Urine Concentration & Renal biomarkers <sup>[12]</sup> | | | | | Y | | | | | | | |
| Laboratory: Hepatobilia | ry | | | | | | | | | | | |
| Liver Assessment | | | | Y [14] | | | | | | | | |
| Hepatobiliary<br>Abnormality criteria | <b>Y</b> [15] | | | Y | | | | | | | | |
| Liver Chemistries | | | | <b>Y</b> [16] | | | | | | <b>Y</b> [9] | | |
| Laboratory: Markers | | | | | | | | | | | | |
| Bone markers | | | | | <b>Y</b> [10] | | | | | | | |
| | | • | | • | | | | • | | | | |

| Endpoint | Absolute | | | | Mair | Chang | | | Max Post Maintenance<br>BL | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | /idual | Sum | Summary | | Individual | | Summary | | ridual |
| | Т | F | F | L | Т | F | F | L | Т | F | F | L |
| ECG | | | | | | | | | | | | |
| ECG findings | Υ | | | Υ | | | | | | | | |
| ECG values | | | | | Υ | | | | | | | |
| QTC values by Category | Υ | | | | Y | | | | Y | | | |
| Other | | | | | | | | | | | | |
| Vital Signs | | | | | Υ | | | | | | | |
| Weight & BMI | | | | | Y[24] | | | | | | | |
| Abacavir HSR | | | | <b>Y</b> [13] | | | | | | | | |
| Participants who became Pregnant | | | | Y | | | | | | | | |
| Patient Profiles | | | | <b>Y</b> [20] | | | | | | | | |
| Dosing Errors and IP<br>Device Malfunctions | | | | Y | | | | | | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Refer to Section 14.6.2 for defining Extent of Exposure and adherence to Q4W dosing intervals,
- 2. Includes reason for any dose change/interruption.
- 3. For AEs reported more than once by a participant, the most severe intensity will be included. Separate summary tables including and excluding injection site adverse reactions.
- 4. One listing of all AEs including verbatim text and preferred term, one showing the relationship between verbatim text, preferred term and SOC and another giving subject numbers for individual all treatment emergent AEs.
- 5. Common AEs are those with ≥5% incidence in either treatment group summarised by frequency.
- 6. Plots of incidence rates and relative risk with 95% CI for Q4W IM vs. ABC/DTG/3TC.
- Four PSRAE listings: Event and Description (Section 1 and Section 2), Possible Cause (Section 3), Section 4 and Section 5 - Section 8.
- 8. Shift table summarising Maintenance Baseline (Day 1) vs. maximum Maintenance Phase result for urine dipstick protein.
- 9. Scatter plot of baseline vs. maximum post-baseline for ALT. Scatter plot of maximum ALT vs. maximum Bilirubin. Matrix plot of maximum liver chemistries.
- 10. Bone markers including: Bone-specific alkaline phosphatase, procollagen type 1 N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin, 25 hydroxy-Vitamin D.
- 11. Renal markers: Urine Retinol Binding Protein, Retinol Binding Protein, Cystatin C. CKD-EP1 GFR using Cystatin C (derived in Section 14.6.3) will also be summarized
- 12. Repeat for CAB/RPV, CAB, RPV respectively.
- 13. Separate listings for exposure to abacavir, history of drug allergies, family conditions, skin rash, symptoms, vital signs, individual symptoms, and diagnostic category assignment.
- 14. Separate listings for time of event, RUCAM score, biopsy, imaging, past/ current conditions and follow up
- 15. One summary of participants and another table showing Subject lds. Table of participants meeting hepatobiliary abnormally criteria during the maintenance oral lead-in Phase will also be produced.
- 16. Patient profiles for participants meeting protocol defined liver stopping criteria and for patients with virologic failure. Patient profiles can also be provided for any other participants, as necessary for medical review.
- 17. Event-level summary: Percentages based on total number of ISR events within each treatment group including distribution of grade, duration, and event characteristics;

- 18. Subject-Level summary: Characteristics of ISR AE (Overall and by Common ISRs); Percentage based on number of participants within each treatment group; Includes distribution of grade and max grade, event characteristics, number of events per subject, rate of number of events per injection visit;
- 19. A corresponding plot of all grades and a separate plot of grade 3-5 events will be produced
- 20. Patient profiles are not planned. But it can be produced post hoc, as necessary.
- 21. Please refer to Section 5.4.2 "Additional subgroup for ISR" for derivation of needle length used in this summary
- 22. Please refer to Section 14.6.3 for defining percentage change from Maintenance Baseline (Day 1) in Lipids
- 23. Separate tables will be produced for Maintenance Phase data and Oral Lead-in period data (see Table 28 and Table 29)
- 24. Change from Induction Baseline (Week -20) for BMI and Weight.
- 25. By SOC and Maximum Toxicity, and history based on prior/current medical conditions collected at Screening

## 8.5.1. Injection Site Reactions

For the summary of Injection Site Reaction Adverse Events by Visit and Maximum Severity (Overall and by Common ISRs): ISRs will be assigned based on onset date to the most recent planned IM injection visit prior or equal to the AE onset date.

Maximum grade at each visit will be derived as the maximum grade among ISRs assigned to the particular visit, with consideration for whether the summary applies to a particular preferred term (vs. across preferred terms), or drug-related associated to CAB and/or RPV.

Drug-related ISRs (based on investigator discretion) will be attributed to the causal agent (CAB vs. RPV) when this can be determined specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the causal agent in those cases where both drugs are given on one side and the ISR is reported non-specifically, then the attribution to a specific causal agent will remain unknown.

ISRs will be attributed to the needle length when this can be determined specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the needle length in those events where both drugs are given on one side and their needle lengths are different, then the attribution to a needle length will remain unknown.

Common ISR includes injection site pain, injection site induration, injection site nodules and any other ISR occurring in ≥5% of participants (for Q4W arm only). The same set of common terms will be applied to 'overall' (CAB and/or RPV), CAB alone, RPV alone.

## 8.5.2. Statistical Analyses/Methods

#### Statistical Analyses

#### **Endpoints**

Change from Maintenance Baseline (Day 1) in Bone Markers at Week 48

#### Covariates

- Treatment (Q4W IM, ABC/DTG/3TC)
- Induction Baseline (Week -20) HIV-1 RNA (<100,000, ≥100,000 c/mL), Gender at Birth, TDF use at Maintenance Baseline (Day 1), Age, body mass index category at Induction Baseline (Week -20), smoking status, and Log-transformed bone marker value at Maintenance Baseline (Day 1) (as defined in Section 5.4.2)</li>

## **Data Handling**

All data remains as is (observed).

## **Model Specification**

- Bone marker results will be log-transformed. The change in the log-transformed data at week 48 from Maintenance baseline (i.e., log of ratio of post-baseline value over Maintenance baseline value) for each bone marker will be analysed for the comparison between the two treatment arms.
- Analysis of covariance (ANCOVA) model will be used with the above covariates/subgroups.
  Age and Log-transformed bone marker value at Maintenance Baseline (Day 1) will be
  included as continuous variables in the model and all other covariates will be included as
  categorical variables.

#### **Model Results Presentation**

- The estimated coefficients of the ANCOVA model will be transformed back (exponential transform) to reflect the change in the ratio of post-baseline value over Maintenance Baseline (Day 1) value rather than the change in the log ratio. The change in the ratio can then be translated into percent change from maintenance baseline (Day 1) (e.g., the ratio bb48/bbbl = 1.3 can be translated into 30% increase from baseline).
- For each treatment, adjusted (geometric) means of ratio and corresponding confidence intervals will be presented. Adjusted point estimates will be derived as LSMEAN S using the observed margins (OM) option within PROC MIXED in SAS.
- The adjusted (geometric mean) difference of the ratio (post-baseline value)/(baseline value) between the two treatments with the corresponding confidence interval and p-value will be presented
- Interactions between treatment and each of the covariates will be investigated but not
  included in the main model. If interactions are found to be significant (p-value <0.10), results
  will be presented separately by subgroup.</li>

 Statistical analysis will only be performed when all expected data through Week 48 has been received from the laboratory.

## 8.6. Subcutaneous Sub-Study Safety Analyses

The proportion of participants reporting AEs will be tabulated for each injection type. This will include the following AE summaries:

- Incidence and severity of ISRs and AEs of special interest during the SC injection phase
  - This includes incidence of Grade 4 ISRs and Grade 3 ISRs including ulceration, secondary infection, phlebitis, sterile abscess, or drainage affecting Interim 1 monitoring criteria.
- Proportion of participants who discontinue treatment due to ISRs and proportion of AEs of special interest during the SC injection phase
- Incidence and severity of AEs not of special interest
- Incidence of SAEs
- Dimensional characteristics (length & width in mm) of SC ISRs of erythema, redness, induration, and swelling
- Change from baseline (latest non-missing value prior to the first SC injection) in laboratory parameters will be summarized by visit through the end of the SC phase.

AE and ISR summaries will be repeated for the following subgroups: Age (<50 vs >=50), Sex at Birth (Female vs Male), Race/Ethnicity (White: Non-Hispanic, White: Hispanic, Black, Asian, Other), Sub-study Baseline BMI (<30, >=30).

Incidence Rate ratios and their 95% CIs for the incidence of ISRs between SC and IM will also be calculated using a Poisson regression model that accounts for within-subject variation by using a repeated effect of subject. Categorical Baseline BMI (<30, >=30) will be included as a covariate in the model. These informal comparisons will be graphically displayed overall and for each subgroup. Results will be repeated for Grade 1+ ISRs as well as for Grade 2+ ISRs. Sub-study participant data will be matched to their individual IM data via the following comparisons:

- 1. The first 2 SC injections vs. the two IM injections post-SC dosing
- 2. All 3 SC injections vs. the first 3 IM injections in the parent study

ISRs of interest will be simply tabulated (i.e., Grade 3+ ulceration, secondary infection, phlebitis, abscess, drainage or a Grade 4 ISR) at interim analysis 1 for ISR monitoring. Once counted, the posterior probability that the true rate of ISRs of interest is >0.05 will be calculated using a Bayesian Beta-Binomial model to produce posterior hyperparameters  $\alpha'$  successes and  $\beta'$  failures as indicated below.
$$a' = a + \sum_{i=1}^{n} x_{i}$$
$$\beta' = \beta + \sum_{i=1}^{n} N_{i} - \sum_{i=1}^{n} x_{i}$$

Where prior  $\alpha = 0.001$  and prior  $\beta = 79$  based on previous and ongoing studies mentioned in protocol amendment 8, Section 12.12.1.3,  $x_i$  is the total number of participants with an event, and  $N_i$  is the total number of participants with an SC injection at the interim.

The posterior probability that the true rate of ISRs of interest is >0.05 will then be calculated from a Beta Distribution CDF using the posterior hyperparameters  $\alpha'$  and  $\beta'$  and summarized for determination of formal VSLC review of all data for ISRs of interest.

# 9. PHARMACOKINETIC AND PHARMACOKINETIC/PHARMACODYNAMIC ANALYSES

Details of the planned PK displays for the Week 124 analysis are provided in Appendix 15: List of Data Displays for Week 124.

The GSK Division of Clinical Pharmacology Modelling and Simulation (CPMS) will be responsible for the PK analysis of CAB. The Division of Global Clinical Pharmacology at Janssen Research and Development will be responsible for conduct or oversight of the PK analysis for RPV.

All PK and PK/PD displays will be based on the PK Population.

## 9.1. Primary Pharmacokinetic Analyses

## 9.1.1. Endpoint / Variables

## 9.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 14.5.3 Reporting Standards for Pharmacokinetic)

#### 9.1.1.2. Derived Pharmacokinetic Parameters

A population-based PK analysis will be described under separate Population-PK Reporting and Analysis Plans for CAB LA and RPV LA.

## 9.1.2. Planned Analyses

Table 10 provides an overview of the planned analyses based on observed plasma CAB/RPV concentration data only with full details being presented in Section Appendix 14: List of Data Displays.

Unless otherwise specified, drug concentration and pharmacodynamic measures will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Table 10 Overview of Planned Pharmacokinetic Analyses

| | Stats Analysis | | | Summai | 'n | Individual | |
|---|---|---|---|---|---|---|---|
| | Т | F | L | Т | F | F | L |
| Pharmacokinetic [5] | | | | | | | |
| Plasma CAB concentration by Visit | | | | <b>Y</b> [1][2 | <b>Y</b> [1][3][4] | <b>Y</b> [3] | Υ |
| Plasma RPV concentration by Visit | | | | <b>Y</b> [1][2] | <b>Y</b> [1][3][4] | <b>Y</b> [3] | Υ |
| Steady state concentration [8] | | | | <b>Y</b> [1] | | | |

| Pharmacokinetic/Pharmacodynamic | | | | |
|------------------------------------------|---|---|----|---|
| CAB/RPV last trough and Week 8 | | | | |
| concentrations by Snapshot virologic | | Υ | Υ | |
| Response at Week 48 | | , | Į. | |
| CAB/RPV Week 8 concentrations by | | | | |
| Snapshot virologic Response at Week | | Υ | Υ | |
| 96 [7] | | ' | | |
| Analysis of Snapshot 'HIV-1 RNA≥50' at | | | | |
| Week 48 by last trough CAB/RPV | | | | |
| concentration, Week 8 trough | | | | |
| concentration, and subgroups [6] – | Υ | | | |
| Univariable analysis /multivariable | | | | |
| analysis | | | | |
| Analysis of Snapshot 'HIV-1 RNA≥50' at | | | | |
| Week 96 by Week 8 CAB/RPV trough | | | | |
| concentration, and subgroups [6] – | Υ | | | |
| Univariable analysis /multivariable | - | | | |
| analysis [7] | | | | |
| Individual CAB/RPV Concentration-Time | | | | |
| Profiles for Participants with HIV-1 RNA | | | Υ | |
| ≥ 50 c/mL at Week 48 (or Week 96) | | | | |
| Change from Maintenance Baseline | | | | |
| (Day 1) in 2hr post-dose QTc and 2-hour | | | | Υ |
| post-dose CAB & RPV concentration at | | | | ı |
| Week 4b, Week 48, Week 96 | | | | |
| Maximum Change from Maintenance | | | | |
| Baseline (Day 1) in ALT/Total Bilirubin | | | | Υ |
| versus Last Trough CAB/RPV | | | | ' |
| Concentrations [8] | | | | |
| Maximum Toxicity Grades of Most | | | | |
| Frequently Reported AEs versus Last | | | | Υ |
| Trough CAB/RPV PK Concentrations [8] | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 3. For both 'all' concentration and the 'evaluable' concentration. The evaluable concentration is derived from samples collected within pre-specified Time window (Section 14.6.5) and not affected by dosing errors or oral bridging.
- 2. For both 'untransformed' and 'log –transformed' statistics.
- 3. The plots will be produced for the untransformed scale (i.e., a linear plot) and the log transformed scale (i.e., log-linear plot), separately.
- 4. Separate plots will be produced for Mean (SD) and Median concentration.
- 5. Standard summary statistics for concentration data will be calculated (i.e., mean, standard deviation, median, minimum, and maximum). For Logarithmically transformed data, the summary statistics (i.e., geometric mean, coefficient of variation on geometric mean, 95% confidence interval for the geometric mean and standard deviation) will also be calculated.
- 6. Please refer to Section 5.4.2. i.e., randomisation strata, baseline and demographic factors, and additional subgroups for PK/PD analyses
- Will be produced only if at least one new CVF has occurred since Week 48 (randomized Q4W arm).
- 8. Produced for Week 48 only.

## 9.1.3. Statistical Analyses/Methods

#### Planned PK statistical analysis

## **Steady State Concentration**

#### **Endpoints**

 log<sub>e</sub>-transformation of the Trough/Pre-dose plasma concentrations (CAB/RPV) on Week 16-48

#### **Covariates**

Study Week

## **Data Handling**

All data remains as is (observed).

## **Model Specification**

A mixed effects ANOVA model will be fitted with Week (continuous variable) as a fixed effect and subject as a random effect for each analysis separately. The Kenward & Roger (KR) degrees of freedom approach will be used. The coefficient for the slope of the day effect on the loge-scale will be used to evaluate steady state for each drug (CAB/RPV). The 90% confidence intervals for the slope for each treatment will be calculated. If it does not appear that steady-state has been demonstrated, early weeks (e.g., Week 16, 20, 24, etc...) results will be dropped and the analysis repeated.

## **Model Checking & Diagnostics**

• The Steady state will be claimed (the coefficient for the slope of the Week effect on the (natural) log scale was close to 0 or the 90% CI for the slope estimate included zero. If steady-state is not demonstrated, concentrations from early weeks (e.g., Week 16, 20, 24, etc.) dropped in sequence and the analysis repeated until either steady state is shown or only two timepoints remain.

#### **Model Results Presentation**

The coefficient for the slope of the day effect on the log<sub>e</sub>-scale, its Standard error and 90% interval will be presented.

## **Population PK Analysis**

 A population-based PK analysis will be done under separate Population-PK Reporting and Analysis plans.

#### Exposure - antiviral activity analysis (PK/PD)

#### **Endpoints**

Snapshot 'HIV-1 RNA≥50' at Week 48 (or W96)

#### **Covariates**

- Randomisation strata, demographic, and baseline characteristics (as specified in Section 5.4.2), and the following additional subgroup/covariates for PK/PD efficacy analysis
  - last CAB/RPV trough concentration (Week 48 analysis only)
  - CAB/RPV trough concentration at the nominal Week 8 visit, Induction Baseline (Week -20) BMI, needle length for CAB/RPV injections at Week 4b)
  - See "Additional subgroup/covariates for PK/PD efficacy analysis" in Section 5.4.2 for derivation details.
- For the W96 CSR, this exploratory analysis will be performed only if at least one new CVF has occurred since Week 48.

## **Data Handling**

All data remains as is (observed).

## **Model Specification**

 Logistic regression will be used to exam the correlation between the endpoint (Snapshot 'HIV-1 RNA≥50') at Week 48 and the covariates/subgroups. This logistic regression analysis will be performed for each covariate, separately (univariable analysis), and will also be performed with one multivariable analysis using Backward stepwise selection approach to identify the covariates potentially affecting virologic response.

## Model Checking & Diagnostics

- For the multivariable analysis, a logistic regression model that best predicts the dependent variable (i.e., 'HIV-1 RNA≥50') from the independent variables (i.e., covariates/factors with P <0.15 from univariable analysis) will be determined using the backward stepwise selecting approach. The last trough and Week 8 trough PK concentration will be logarithmically transformed with base of 2 (i.e., one-unit increase of the point estimate of log2 PK concentration is equivalent to 'doubling the concentration' in the original value). The analysis will start with all covariates in the model and remove a covariate with the largest p-value (i.e., the least statistically significant) each time and continue until the stopping rule is reached when all remaining covariates have p-value <15%.</p>
- If problems with model convergence occur due to zero event counts or complete/quasicomplete separation, then alternative methods such as Fisher's exact test (univariate analysis) and exact logistic regression (multivariable analysis) may be used.

#### **Model Results Presentation**

• The odds ratio, 95% confidence interval, and p-value will be presented. Estimated effect represents the change in log odds for a two-unit increase in PK concentration.

# 9.2. Subcutaneous Sub-Study

## 9.2.1. Endpoint / Variables

• Plasma PK parameters for CAB LA 200 mg/mL and RPV LA 300 mg/mL (Ctau, concentrations 1-week post dose [~Cmax], and area under the curve [AUC (0-tau)])

for SC injections during the SC injection phase compared with similar PK parameters for gluteal IM injections

Plasma CAB and RPV concentration values will be summarized with descriptive statistics by dosing interval and planned timepoint for the PK Concentration Population (PC). These concentration values will be determined directly from concentration-time data from each analyte. Descriptive statistics including the n, mean with associated 95% CI, standard deviation, median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of logarithmically transformed data, 5<sup>th</sup>/95<sup>th</sup> percentiles and the geometric coefficient of variation (CV%).

Individual concentration-time profiles and median/mean profiles from each analyte in each dosing interval will be plotted for the PK Concentration (PC) Population. Each of the figures will contain one plot on the untransformed scale (i.e., a linear plot) and one plot on the log transformed scale (i.e., semi-log plot). Actual assessment times will be used in the individual concentration-time plots. Nominal times will be used for the purposes of summarization and in mean and median plots. See <u>Appendix 4</u>: Data Display Standards & Handling Conventions. for details on pharmacokinetic figure and table displays

Pharmacokinetic parameters will be derived by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or higher (Pharsight, Inc., Cary, NC). All calculations of non-compartmental PK parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits. Ct will be taken from CAB and RPV concentration data at the prescribed timepoint. The following PK parameters will be derived and displayed for the PP Population as data permits:

Table 11a Derived PK Parameters

| Paramete r | Parameter Description | Gluteal<br>Injection | SC Injection 1 | SC Injection 2 | SC Injection 3 |
|---|---|---|---|---|---|
| C <sub>max</sub> | Maximum observed concentration during the dosing interval | Week-4 -<br>Day 1 | Day 1 –<br>Week 4 | Week 4 –<br>Week 8 | Week 8 –<br>Week 12 |
| t <sub>max</sub> | Time of occurrence of C <sub>max</sub> | | | | |
| AUC <sub>0-</sub> τ | Area under the concentration time curve from time zero to the end of the dosing interval | | | | |
| Сτ | Trough concentrations (Cτ) at the end of the dosing interval | Day 1 | Week 4 | Week 8 | Week 12 |

NOTES: NA: Not Applicable

Additional parameters may be included as required.

All the derived pharmacokinetic parameters will be summarized and listed for the PP population by study phase and treatment. For each of these PK parameters, with the exception of t<sub>max</sub>, the following descriptive summary statistics will be calculated for each treatment: n, arithmetic mean with associated 95% CI, standard deviation, median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of

logarithmically transformed data, and the geometric coefficient of variation (CV<sub>b</sub>(%)). For  $t_{max}$ , the n, median, minimum, and maximum summary statistics will be provided. Where AUC<sub>0- $\tau$ </sub> is collected out of the appropriate window, AUC<sub>0- $\tau$ </sub> (the last quantifiable concentration) will be used in place of AUC<sub>0- $\tau$ </sub>.

Interim analysis 2 will include descriptive summaries and graphs of PK concentration and parameters as data permit. PK summaries will be presented by subgroup as needed where data allow. Data display specifications for derived PK parameter summaries and listings are given in <u>Appendix 19</u> of this RAP

PK samples collected outside the protocol defined time-windows and/or other protocol deviations will be reviewed by the study team to determine whether the sample will be excluded from PK analyses.

## 9.2.2. Planned Analyses

The primary objective of this sub-study is to evaluate the pharmacokinetics of cabotegravir LA (200 mg/mL) and rilpivirine (RPV) LA (300 mg/mL) for monthly dosing as a SC injection in the anterior abdominal Wall SC Tissue versus an IM injection into the gluteal muscle in HIV-1 infected participants currently enrolled in the FLAIR study.

An estimation approach will be taken and point estimates and confidence intervals will be constructed for the ratio of the geometric mean of SC abdominal injection PK parameters to the geometric mean of the IM gluteal injection PK parameters.

The primary analysis is to compare the abdominal SC injection with gluteal IM injection using the ratio of the geometric mean of SC injection to the geometric mean of IM injection for a PK parameter within each analyte (CAB, RPV). The primary PK parameters of interest include concentrations at the end of the dosing interval [Ctau], concentrations 1-week post dose [~Cmax], and area under the curve for the dosing interval [AUC (0-tau)] (Table 24). CAB and RPV concentrations and parameters will be summarized descriptively.

Following log-transformation, C<sub>max</sub>, C<sub>tau</sub> and AUC(0-<sub>tau</sub>) will be separately analyzed by analyte using a mixed effects model with fixed effect term for type of injection (SC, gluteal) and BMI (≥30 Kg/m², <30 Kg/m²) in addition to a random effect term for subject. As it is suspected that varying participant BMI may impact the PK concentration distribution, BMI is being included in the model as a covariate to control for any potential impact beyond the effect of injection type. In each model, only participants with PK parameter estimates from corresponding both SC and gluteal injections are included. For example, in the model for comparing C<sub>max</sub> between the first CAB SC injection vs gluteal CAB injection, only participants with C<sub>max</sub> estimates from both first CAB SC injection and CAB gluteal injection are included.

Point estimates and their associated 90% confidence intervals will be constructed for the differences between the SC injection and the gluteal injection. The point estimates and their associated 90% confidence intervals from the log-transformed analysis will then be backtransformed to provide point estimates and 90% confidence intervals for the ratios between

the SC injection and the gluteal injection on the original scale. This analysis will be performed using the PK Parameter (PP) population for the dosing intervals given in Table 11b using the Gluteal parameters as the reference variables and each SC injection-based set of parameters as the test variables. While no formal bioequivalence testing will be performed, parameters can be assumed to be similar if the geometric mean ratio and its 90% CI fall within 0.80 - 1.25.

Table 11b Parameters and dosing

| Parameters (CAB<br>200mg/mL +<br>RPV 300mg/mL) | Q Monthly Dosing | | |
|---|---|---|---|
| Cmax (1-week post injection),<br>Ctau (end of dosing interval)<br>AUC(0-tau) | SC Injection 1:<br>gluteal injection | SC Injection 2: gluteal injection | SC Injection 3: gluteal injection |

The point estimate of the slope of  $C\tau$  following the last IM injection through 3rd SC injection will also be determined to assess changes in steady state conditions established previously. This will be performed using another mixed-effects model with concentration timepoint as a predictor variable of concentration and a random effect of subject. The model will initially include all concentration values from Day 1 – Week 12 and will then be repeated, removing the earliest timepoint in each run until the last two timepoints remain, Week 9 – Week 12. Point estimates and 90% confidence intervals for the slope will be presented in tabular format.

## 9.2.3. Statistical Analyses/Methods

#### **Endpoints**

**PK Parameters** 

## Geometric Mean Ratio:

 As data permit, Log<sub>e</sub>-transformation of the PK parameters (Ctau, Cmax and AUC(0-tau) for each sub-study dosing interval for participants in the sub-study PK Concentration Population

#### Steady State:

 log<sub>e</sub>-transformation of the Trough/Pre-dose plasma concentrations (CAB/RPV) on all appropriate dosing intervals

#### Model Specification

#### Geometric Mean Ratio:

Following Log<sub>e</sub>-transformation, PK parameters will be separately analyzed by treatment arm and analyte using a mixed effects model with dosing interval (gluteal injection vs 1<sup>st</sup>, 2<sup>nd</sup>, and 3rd SC injection) and Sub-study Baseline BMI (<50 kg/m², ≥ 30 kg/m²) as fixed effects and subject as a random effect. In each model, only subjects with evaluable PK parameter</li>

estimates in both dosing intervals are included. For example, in the model for comparing Cmax estimated from the first CAB SC injection interval with Cmax estimated from the gluteal injection interval, only the subjects with evaluable Cmax estimates from both first CAB SC injection interval and gluteal injection interval are included.

## Steady State:

• A mixed effects ANOVA model will be fitted with Day / Week (categorical variable) as a fixed effect and subject as a random effect for each analyte. The Kenward & Roger (KR) degrees of freedom approach will be used. The coefficient for the slope of the day effect on the logescale will be used to evaluate steady state for each drug (CAB/RPV). The 90% confidence intervals for the slope for each treatment will be calculated. The model will be initially run with all timepoints from Day 1 – Week 12, removing the earliest timepoint at each iteration until the last two timepoints remain, Week 9 - Week 12. Only evaluable concentrations will be included in the analysis.

## **Model Checking & Diagnostics**

#### Geometric Mean Ratio:

 Model assumptions will be applied, but appropriate adjustments may be made based on the data. Parameters can be assumed to be similar if the geometric mean ratio and its 90% CI fall within 0.80 – 1.25

#### Steady State:

 The Steady state will be claimed (the coefficient for the slope of the Week effect on the (natural) log scale was close to 0 or the 90% CI for the slope estimate included zero.
 Concentrations from earlier timepoints (e.g., Day 1, Week 1 etc.) will be dropped in sequence and the analysis repeated until only two timepoints remain.

#### **Model Results Presentation**

## Geometric Mean Ratio:

The estimated difference and 90% CI obtained on the log<sub>e</sub> scale will be exponentiated to
provide an estimate of geometric mean ratio and its associated 90% CI. The estimate of
within-subject variability (%CVw) will also be provided.

#### Steady State:

 The coefficient for the slope of the day / week effect on the log<sub>e</sub>-scale, its Standard error and 90% interval will be presented

## 10. PHARMACOKINETIC ANALYSES (DAY 1 JAPAN)

For Japanese participants in the study, blood samples for CAB will be taken at the Day 1 visit at each of the sampling times shown in Table 11c, in addition to sparse samples collected at other visits as specified in the protocol for all CAB LA + RPV LA randomized participants.

Table 11c Additional PK Visit and Sample Times for Japanese Participants

| Day | Time (Related to Dosing of Study agent) |
|---|---|
| Oral Cabotegravir | |
| Day 1 (following first oral dose during lead-in phase) | Pre-dose, 1, 2, 3, 4, 8, and 24 hours post-dose |

## 10.1. Primary Pharmacokinetic Analyses

Pharmacokinetics of CAB following a single 30 mg dose using the Phase 3 formulation in Japanese in 201584 (FLAIR) will be evaluated. Approximately 20 Japanese participants will be enrolled and randomized 1:1 to CAB or ABC/DTG/3TC to achieve ~10 participants who receive oral CAB.

The GSK Division of Clinical Pharmacology Modelling and Simulation (CPMS) will be responsible for the PK analysis of CAB. The Division of Global Clinical Pharmacology at Janssen Research and Development will be responsible for conduct or oversight of the PK analysis for RPV.

## 10.1.1. Endpoint / Variables

#### 10.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 14.5.3 Reporting Standards for Pharmacokinetic).

Assay results from Day 1 samples collected from a subject with emesis occurring within 4 hours of the dose will not be considered as evaluable and will be excluded from all data displays and PK analyses.

#### 10.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters for Japanese participants randomized to CAB LA + RPV LA will be calculated using plasma concentration-time data on Day 1 by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | The area under the plasma concentration-time curve from time zero to the last quantifiable concentration following the first dose, determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations |
| Cmax | The first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. |
| C24 | Concentration observed at 24-hours post dose (±30 mins) determined directly from the raw concentration-time data. |
| tlag | The time of sample preceding first quantifiable concentration, determined directly from the raw concentration-time data. |
| tmax | The time at which Cmax is observed, determined directly from the raw concentration-time data. |
| tlast | The time of last quantifiable concentration |

#### NOTES:

Additional parameters may be included as required.

## 10.1.2. Summary Measure

For plasma CAB concentrations, the following summary statistics will be calculated by planned sampling time: n, mean, standard deviation (SD), coefficient of variation (%CV), median, minimum and maximum, geometric mean, 95% confidence interval and the between-subject CV (%CVb) based on the geometric mean for the loge-transformed values.

For PK parameters, except for tmax, tlag, and tlast, the following summary statistics will be calculated: n, mean, standard deviation (SD), coefficient of variation (%CV), median, minimum and maximum, geometric mean, 95% confidence interval and the between-subject CV (%CVb) based on the geometric mean for the loge-transformed values. For tmax, tlag, and tlast, the following summary statistics will be calculated: median, maximum, minimum, arithmetic mean, and standard deviation.

#### 10.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Japan Pharmacokinetic population, unless otherwise specified.

## 10.1.4. Strategy for Intercurrent (Post-Randomization) Events

Data following the intercurrent event of randomized treatment discontinuation will not be used in the analysis as the concentrations and PK parameters to be estimated is while ontreatment.

## 10.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 1: Japan-Specific Requirements and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

PK parameters that have mass in the units should be reported in μg/mL and μg•h/mL.

Deviations from planned times will be examined for scheduled assessments. PK parameters will be calculated using actual assessment times. Actual assessment times will be used in the individual concentration-time plots. Nominal times will be used for the purposes of summarization and in mean and median plots. Concentration-time data will be listed using actual assessment times.

All available data will be summarized, with no imputation for missing data.

#### 10.1.5.1. Statistical Methodology Specification

No formal hypothesis will be tested. Descriptive statistics will be used to summarize data.

## 11. HEALTH OUTCOMES ANALYSES

## 11.1. Endpoint / Variables

- Change from Maintenance Baseline (Day 1) in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs);
- Change in treatment satisfaction over time (using the HIVTSQc change version) at Week 48:
- Change from Week 5 in Dimension Scores and proportion of participants considering pain and local reactions following injection using PIN (Perception of Injection Questionnaire) (Q4W arm only);
- Change from Maintenance Baseline (Day 1) in Subscale of Life satisfaction, HIV medication, and disclosure worries using HAT-QoL;
- Change from Maintenance Baseline (Day 1) in Mental health component (MCS) and physical component summary (PCS) using SF-12;
- Change from Maintenance Baseline (Day 1) in treatment acceptance using ACCEPT;
- Change from Week 4b in tolerability of injections using NRS (Q4W arm only)

## 11.1.1. Summary Measure

Mean treatment difference (Q4W IM – ABC/DTG/3TC) at visits of interest through to Week 96 (i.e., the assessment visits detailed in Table 12), excluding PIN and NRS endpoints.

Mean change at visits of interest through to Week 96 (i.e., the assessment visits detailed in Table 12), for PIN and NRS endpoints.

## 11.1.2. Population of Interest

The primary health outcomes analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

## 11.1.3. Strategy for Intercurrent (Post-Randomization) Events

If a participant discontinues treatment prior to the timepoint of interest such that there is no evaluable on-treatment assessment for the timepoint of interest (see Table 30 for definition of on-treatment), the data will be computed or imputed (see Section 14.6.6).

## 11.1.4. Planned Health Outcomes Analyses

Table 12 provides an overview of the planned analyses. Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Table 12 Overview of Planned Health Outcome Analyses

| Endpoints | | | P | Absolu | ite | | | Change from Maintenance Baseline | | | | | eline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | T | F | L | Т | F | F | L | Т | F | L | T | F | F | L |
| Perception of Injection | າ (PIN | ) at W | /eek 5 | 5, 41, 4 | 18, 96 | , Withd | rawal | (Q4V | / arm | only) | | | | |
| Individual Item<br>Scores | | | | Y | | | | | | | | | | |
| Domain of 'Bother from injection site reactions', 'Leg movement', 'Sleep', 'Acceptability' | Y[4] | | | Y | | | | | | | <b>Y</b> [5] | | | |
| Health-related quality | Health-related quality of life (HATQoL) at Day 1, Week 24, 48, 96, Withdrawal | | | | | | | | | | | | | |
| Individual Item<br>Scores | | | | Υ | | | | | | | | | | |
| Subscale of Life satisfaction, HIV medication, and disclosure worries | | | | Y | | | | Υ | <b>Y</b> [1] | | Y | | | |
| Health Status (SF-12) | <b>at</b> Day | / 1, W | eek 2 | 4, 48, | 96, W | ithdrav | val | | | | | | | |
| Individual Item<br>Scores | | | | Υ | | | | | | | | | | |
| Mental health component (MCS) and physical component summary (PCS)[2] | | | | Y | | | | Υ | <b>Y</b> [1] | | Υ | | | |

| Endpoints | | | A | Absolu | ite | | | Cha | nge f | Change from Maintenance Base | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | Τ | F | L | Т | F | F | L | T | F | L | Τ | F | F | L |
| Treatment Satisfaction | ı Sco | re (HI | VTSC | <b>(s)</b> at [ | Day 1, | Week | 4b, 24 | 4, 44, | 96, W | /ithdra | wal | | | |
| Individual Item<br>Scores | | | | Y | | | | | | | | | | |
| Individual Item Scores by Subgroup <sup>[3]</sup> | | | | Y | | | | | | | | | | |
| Treatment Satisfaction Score | Υ | | | Υ | | | | Υ | <b>Y</b> [1] | | Υ | | | |
| Treatment Satisfaction | ı Sco | re Ch | ange | (HIVT | SQc) | at Wee | ek 48, | Withd | Irawal | | | | | |
| Individual Item<br>Scores | | | | Υ | | | | | | | | | | |
| Treatment Satisfaction Score Change | Υ | | | Y | | | | | | | | | | |
| Treatment Acceptance | AC( | CEPT | ) at D | ay 1, V | Veek 8 | 8, 24, 4 | 18, 96 | , With | drawa | ıl | | | | |
| Proportion of Individual item score | | | | Υ | | | | | | | | | | |
| Acceptance/General Dimension Score | | | | Υ | | | | Υ | <b>Y</b> [1] | | Υ | | | |
| Tolerability of injectio | n (NR | S) at | Week | 4b, 5, | 40, 4 | 1, 96 ( | Q4W a | arm o | nly) | | | | | |
| Proportion of Individual item score | | | | Y | | | | | | | | | | |
| Tolerability Score<br>(Q4W IM only) | | | | Υ | | | | | | | Y | | | |
| Treatment Preference | at We | ek 48 | (Q4V | V arm | only) | 1 | 1 | 1 | 1 | 1 | | 1 | | |
| Treatment: Monthly injection vs Daily oral ART | | | | Υ | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Line Plot of Adjusted Mean (95% CI) for each treatment arm, as well as the adjusted mean difference (95% CI) between the two treatment arms (if questionnaire was used for both arms during Maintenance Phase).
- 2. Component scores will be calculated form Computer Software purchased from QualityMetric.
- 3. Subgroups: Induction Baseline (Week -20) HIV-1 RNA (<100,000, ≥100,000 c/mL), gender at birth, age (<35; 35-<50; ≥50), Maintenance Baseline (Day 1) CD4+ cell count <200; 200 to <350; 350 to <500; ≥ 500 cells/mm3), and race (i.e., white, non-white).
- 4. Statistical analysis (i.e., p-value) produced only for the acceptance score comparing Week 40/41/96 to Week 5.
- 5. Change versus Week 5 for PIN.

## 11.1.5. Statistical Analyses/Methods

#### **Statistical Analyses**

## **Endpoints**

- Change from Maintenance Baseline (Day 1) in
  - HIVTSQs total treatment satisfaction score 24, 44, and 96
  - ACCEPT general acceptance score at Week 8, 24, 48, and 96
  - SF-12: physical component summary (PCS) and mental component summary (MCS) at week 24, 48, and 96
  - HATQoL (Life satisfaction, HIV medications, disclosure worries) at Week 24, 48, and 96.

## **Model Specification**

- An analysis of covariance (ANCOVA) model will be used at each visit at Maintenance Phase with covariates: treatment, age (<50, ≥ 50 years old), Induction Baseline (Week -20) HIV-1 RNA (<100,000, ≥100,000 c/mL), gender at birth, race (i.e., white, non-white) and Maintenance Baseline (Day 1) score value (as a continuous variable).</li>
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM) option within PROC MIXED in SAS.
- No adjustment for multiplicity will be applied as these analyses will be considered supportive.
- Interactions between treatment and each of the covariates will not be assessed unless the
  exploratory subgroup analyses on the primary endpoint highlights significant interactions. In
  this situation, the interaction(s) of interest will be assessed and, if necessary, results will be
  reported in the clinical study report. Interactions between treatment and the baseline score
  will be investigated but not included in the model. If interactions are found to be significant
  (p<0.10), results may be presented separately by subgroup.</li>

#### **Dataset**

LOCF dataset will be used.

#### **Model Results Presentation**

- Adjusted treatment difference (Q4W IM ABC/DTG/3TC), its 95% CI and the associated p-value. The interaction between treatment and the baseline score will be included in a footnote.
- Plots of adjusted mean change from Maintenance Baseline (Day 1) (95% CI) for each treatment group, and the adjusted mean difference (95% CI) between the two treatment arms from the model will be generated across visit.

#### **Statistical Analyses**

#### **HIVTSQc**

Treatment Satisfaction Score (Change) at Week 48

## **Model Specification**

- An analysis of variance (ANOVA) model will be used with covariates: treatment, age (<50, ≥ 50 years old), Induction Baseline (Week -20) HIV-1 RNA (<100,000 c/mL, ≥ 100,000 c/mL), Gender at birth, and Race (white, non-white)</li>
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM) option within PROC MIXED in SAS.
- Interactions between treatment and each of the covariates will not be assessed unless the
  exploratory subgroup analyses on the primary endpoint highlights significant interactions. In
  this situation, the interaction(s) of interest will be assessed and, if necessary, results will be
  reported in the clinical study report. If interactions are found to be significant (p<0.10), results
  may be presented separately by subgroup.</li>
- No adjustment for multiplicity will be applied as these analyses will be considered supportive.

#### **Dataset**

• The observed case (OC) dataset uses only the data that is available at Week 48, with no imputation for missing values.

#### **Model Results Presentation**

 Adjusted means, 95% CI, and associated p-value will be presented for the treatment difference (Q4W IM – ABC/DTG/3TC).

## **Statistical Analyses**

#### PIN

• Change from Week 5 in the PIN acceptance score at Week 41 and Week 48 (Q4W arm only)

#### Statistical Test

• The Wilcoxon Signed-Rank Test will be used to evaluable whether the change from Week 5 to Week 41 and to Week 48, respectively, is statistically different than zero based on a two-sided p<0.05. Separate tests will be performed for the change from Week 5 to Week 41 and for the change from Week 5 to Week 48.

#### **Dataset**

LOCF dataset will be used

#### **Results Presentation**

 Summary statistics at each timepoint (Week 5, Week 41 and W48) and p-value for each comparison (W48/W41) versus scores at Week 5

# 11.2. Subcutaneous Sub-Study Endpoint / Variables

- Change from gluteal to SC in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) during the SC Injection phase as well as the change from SC to gluteal during the Return to Gluteal Injection phase
- Change from gluteal to SC using the HIV Treatment Satisfaction Change (HIVTSQc) questionnaire at Sub-study Week 9

- Changes in the tolerability of injections (NRS) over time during the sub-study, separate for CAB LA and RPV LA
- Changes in the perception of injections (PIN) over time during the sub-study, separate for CAB LA and RPV LA
- Preference for SC injections compared with prior gluteal injections and the injections received during the Return to Gluteal Injection phase respectively.
- Reasons for switch to SC from IM
- Interest for home administration options

## 11.2.1. Summary Measure

The health outcomes analyses include analyses of data collected from the following questionnaires, HIVTSQ (both s and c versions), NRS, PIN, and Preference between SC and gluteal injections. The reasons for switch to SC from IM injections will be assessed, as well as the interest in a potential option for self-administration of SC injections. Health Outcomes assessments will be summarized, where applicable, by study drug (CAB and RPV), domain, and item. Summaries will be presented by subgroup as needed where data allow.

For the sub-study, the change from sub-study Baseline in Total Treatment Satisfaction and Individual Item scores as well as the mean difference between SC injections and gluteal injections from visits of interest will be presented for the HIVTSQs (Baseline vs. Week 9 and Week 17). Change from sub-study Baseline will be presented for the NRS and the PIN (Domain and Individual Item scores). Descriptive statistics and frequency counts will be presented as appropriate for all measures.

Results for the Preference questionnaire, the HIVTSQs, the PIN, and the NRS will be displayed by subgroup (age group, sex, race/ethnicity, Baseline BMI).

Descriptive NRS and Preference score statistics will also be presented at interim analysis 2.

## 11.2.2. Statistical Analyses/Methods

#### **Statistical Analyses**

## NRS/PIN/HIVTSQs

- Change from Sub-study Baseline in the NRS, PIN domain and item scores, and HIVTSQs total treatment satisfaction score at all available subsequent sub-study timepoints
- The mean difference between SC injections and IM injections from all visits in a phase will be calculated between all SC results and all return to IM results for the NRS, PIN, and HIVTSQs.

#### **Statistical Test**

• The Wilcoxon Signed-Rank Test will be used to evaluate:

For HIVTSQs, whether the change from Sub-study Baseline to each post-baseline sub-study visit is statistically different from zero based on a two-sided p<0.05. Separate tests will be

### **Statistical Analyses**

performed for the change from Baseline to Week 9, for the change from Baseline to Week 17, and for the change from Week 9 (SC phase) to Week 17 (return to IM phase).

For the PIN domains, whether the change from Sub-study Baseline to each post-baseline sub-study visit is statistically different from zero based on a two-sided p<0.05. Separate tests will be performed for the change from Baseline to Week 1, Baseline to Week 9, and Baseline to Week 13, and for the change from Week 9 (SC phase) to Week 13 (return to IM phase) by treatment (CAB vs RPV).

#### **Dataset**

Observed values will be used for all measures

#### **Results Presentation**

- For HIVTSQs, summary statistics at Sub-study Baseline, Sub-study Week 9, and Sub-study Week 17 a p-value for the comparison between scores at each post-baseline sub-study visit with scores at Sub-study Baseline will be presented.
- For the PIN domains, summary statistics at Sub-study Baseline, Sub-study Weeks 1, 9, and 13 a p-value for the comparison between scores at each post-baseline sub-study visit with scores at Sub-study Baseline will be presented.

## 12. VIROLOGY

Details of the planned virology displays for the Week 124 analysis are provided in Appendix 15: List of Data Displays for Week 124.

Virology displays for the subcutaneous sub-study will be produced when data is available. Further details available in <u>Appendix 19</u>: List of Data Displays for Subcutaneous Sub-Study Analysis.

The virology analyses will be for the CVF populations using genotype and phenotype data based on population sequencing assay, unless otherwise specified.

Table 13 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 13 Overview of Planned Virology Analyses

| Endpoint | Absolute | | | |
|---|---|---|---|---|
| | Sum | mary | Indivi | dual |
| | Т | F | F | L |
| Genotypic resistance at time of CVF[1] | T | T | | |
| Prevalence of Resistance Mutations | <b>Y</b> [2] | | | Y [4] |
| Prevalence of Emergent Resistance Mutations – Relative to Genotype at Baseline (Week -20) [5] | <b>Y</b> [2] | | | |
| Phenotypic resistance at time of CVF[1] | | | | |
| Prevalence of Phenotype | Υ[3] | | | Y [4] |
| Fold Change for CAB, RPV, DTG | Y | | | |
| Change from Induction Baseline (Week -20) in Fold Change to CAB, RPV, DTG. | Y | | | |
| IN, PR/RT Replication Capacity | | | | Y |
| Other | | | | |
| Viral load, Genotypic and Phenotypic data for Participants with genotype and/or phenotype data for CVF and non-CVF participants | | | | Υ[4] |
| Prevalence of Resistance Mutations at Induction Baseline (Week -20) | <b>Y</b> [2] | | | |
| All Genotypic Data | | | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e., modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e., descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.

- 1. For the CVF as indicated by two consecutive plasma HIV-1 RNA levels ≥200 c/mL after prior suppression to <200 c/mL, the first visit of these two consecutive visits is defined as 'the suspected visit', and the 2nd one is the confirmed visit. Sample used for resistance testing is taken at the suspected visit date, and only tested once a participant confirms virological failure at a subsequent visit. If the test fails with the sample at the suspected visit, we will just report it as 'no data'. The sample from the confirmed visit will not be tested for resistance.</p>
- 2. No. and percentage of participants with IN resistance mutations or major mutations in the classes of NNRTI, NRTI, PI, respectively, as defined in 14.6.7
- 3. Separate outputs by phenotypic cut-off and by number of drugs to which participants are resistant.
- 4. Includes the following at all available timepoints (including screening, Week -20, and all post-baseline samples): HIV-1 subtype (Induction Baseline (Week -20)), resistance mutations and fold change to EFV/ETR/RPV, DTG/RAL/EVG/CAB and ARTs (for the ABC/DTG/3TC arm) received during the Maintenance Phase. Non-CVF participants may include those with genotype/phenotype data upon withdrawal from treatment with last ontreatment HIV-1 RNA ≥200 c/mL.
- 5. Emergent Mutations defined in Section 14.6.7

Additional analyses for HIV-1 resistance may be carried out on peripheral blood mononuclear cell (PBMC) samples collected at Day 1 and Week 96 (or withdrawal if prior to Week 96).

If pre-treatment genotypic/phenotypic results are available from both the central laboratory and Monogram Biosciences, then Baseline genotype/phenotype will be determined based only upon the data provided by Monogram assays.

## 13. REFERENCES

Chan, I. S. F. and Zhang, Z. (1999), "Test-Based Exact Confidence Intervals for the Difference of Two Binomial Proportions," Biometrics, 55, 1202–1209.

Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection questionnaire. Health Qual Life Outcomes. 2008 mar 4; 7:21

D'Agostino RB, Vasan RS, Pencina MJ, et al. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

EMA/CHMP/539146/2013, Guideline on the investigation of subgroups in 4 confirmatory clinical trials, 23 January 2014

Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.

Gilet H, Arnould B. Acceptance by the patients of their treatment (ACCEPT) Questionnaire, 2014.

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA. 2001;285 (19):2486-2497.

HIVTSQ user guidelines, Health Psychology Research Unit, Royal Holloway, University of London, 2016

Holmes WC, HIV/AIDS-Targeted Quality of Life Instrument 1999.

Kalbfleisch J.D., Prentice R.L. *The Statistical Analysis of Failure Time Data*. 1st ed. New York: John Wiley & Sons; 1980.

Levey AI, Christopher HS, Hocine T, John HE, Harold IF, Tom G, et al. Estimating Glomerular Filtration Rate from Serum Creatinine and Cystatin C. N Engl J Med 2012, 367: 20-29.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, Biometrics, 2000;56:309-315.

Mary E. Nilsson, Shailaja Suryawanshi, Cristiana Gassmann-Mayer, Sarah, Dubrava, Paul McSorley, and Kaihong Jiang. Columbia–Suicide Severity Rating Scale, Scoring and Data Analysis Guide, 2013

Nilsson ME, Suryawanshi S, Gassmann-Mayer C et al, Columbia–Suicide Severity Rating Scale, Scoring and Data Analysis Guide, 2013.

Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. *Am J Psychiatry*. 2007;164:1035–1043.

Ralph B. D'Agostino, Ramachandran S. Vasan, Michael J. Pencina, Philip A. Wolf, Mark Cobain, Joseph M. Massaro, William B. Kannel. 2008. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989;42:311-323.

SF-12 (v2) Health Survey 1994, 2002 Medical Outcomes Trust and QualityMetric Incorporated, 2018

Wensing AM et al, 2019 Update of the Drug Resistance Mutations in HIV-1, Volume 27 Issue 3 July/August 2019.

# 14. APPENDICES

| Section | Appendix |
|---|---|
| Analysis Popu | lations |
| Section 14.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| General Considerations for Data Analyses & Data Handling Conventions | |
| Section 14.2 | Appendix 2: Schedule of Activities |
| Section 14.3 | Appendix 3: Assessment Windows |
| Section 14.4 | Appendix 4: Study Phases and Treatment State |
| Section 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 14.6 | Appendix 6: Derived and Transformed Data |
| Section 14.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 14.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 14.9 | Appendix 9: Population Pharmacokinetic (PopPK) Analyses |
| Section 14.10 | Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses |
| Section 14.11 | Appendix 11: Snapshot Algorithm Details |
| Section 14.12 | Appendix 12: AESI identification |
| Section 14.17 | Appendix 17: Variables Defined for Time to Event Analysis |
| Other RAP App | pendices |
| Section 14.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 14.14 | Appendix 14: List of Data Displays for Week 48/Week 96 |
| Section 14.15 | Appendix 15: List of Data Displays for Week 124 |
| Section 14.16 | Appendix 16: IDMC |
| Section 14.18 | Appendix 18: Japan-Specific Requirements |
| Section 14.19 | Appendix 19: List of Displays for Subcutaneous Sub-study |
| Section 14.20 | Appendix 20: Example Mock Shells for Data Displays |

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 14.1.1. Exclusions from Per Protocol Population

Important protocol deviations leading to exclusion from the Per Protocol population are those deviations which may

- directly impact the efficacy endpoint of HIV-1 RNA; or
- lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the protocol deviations which, if they occur prior to an analysis timepoint of interest (e.g., Week 48/96), will lead to exclusion of a participant from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. A final review will occur before the clinical database has been frozen for analysis.

A participant meeting any of the following criteria will be excluded from the Per Protocol population based on case-by-case clinical determination:

| Number | Exclusion Description |
|---|---|
| 01 | Participant deviates from inclusion or exclusion criteria that may significantly affect exposure, response to therapy or participant safety or that are fundamentally inconsistent with the intended study population, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 02 | Participant has non-compliance with IP (including IM dosing errors) or took/received incorrect IP (i.e., other than the one to which they were randomized) up to an analysis timepoint of interest (i.e., Week 48/96), meeting the following conditions: |
| | <ul> <li>Maintenance Phase: <ul> <li>Two or more injection intervals affected by over dosage deviations (e.g., extra injection or excessive volume administered, length of time between injections less than 3 weeks, excluding split doses) up to the analysis visit of interest; or</li> </ul> </li> <li>Week 96 analysis only: <ul> <li>For participants discontinuing injections by Week 52: Two or more injection intervals affected by over dosage deviations (e.g., extra injections less than 3 weeks, excluding split doses) up to the analysis visit of interest.</li> <li>For participants receiving injections beyond Week 52: Three or more injection intervals affected by over dosage deviations (e.g., extra injection or excessive volume administered, length of time</li> </ul> </li> </ul> |

| Number | Exclusion Description |
|---|---|
| | between injections less than 3 weeks, excluding split doses) up to the analysis visit of interest; or |
| | 3. At least 10% of total time on-treatment with under dosing deviations in the Maintenance Phase up to the analysis visit of interest (i.e. Week 48/96), where the % with non-compliance is derived the ratio of the total number of non-compliant under dosing days occurring as of the date of the last analysis timepoint snapshot viral load (i.e. last on-treatment viral load during the Maintenance Phase up to Study Day 378 for W48 and up to Study Day 714 for W96) divided by the number of days on-treatment from start of Maintenance Phase treatment to the date of the last analysis timepoint snapshot viral load, and non-compliance days are defined as follows: |
| | ABC/DTG/3TC Arm: a. Duration of interruptions in ABC/DTG/3TC arm ART for reasons other than treatment-related adverse events/laboratory abnormalities (based on Exposure eCRF forms); |
| | Q4W IM Arm: |
| | <ul> <li>a. Length of time (in days) until next injection from date of<br/>dosage/administration deviation potentially resulting in under dosage<br/>(e.g., 1ml administered instead of 2ml)</li> </ul> |
| | <ul> <li>b. Length of time (in days) in excess beyond 35 days between injections post Week 12 and in excess beyond 28 days for Week 8 and Week 12 (e.g., missed or late injection visit)</li> </ul> |
| | <ul> <li>Length of time (in days) in excess beyond 35 days from last injection<br/>until start of oral bridging post Week 12 and exceeding 4 weeks for<br/>Week 8 and Week 12</li> </ul> |
| 03 | Prohibited medications: receiving ART medication other than that prescribed/allowed by the study (excluding permanent changes in ART regimen; such cases will be retained as 'HIV1-RNA≥50 c/mL' in the per protocol snapshot analysis) or receiving prohibited concomitant medication that would impact exposure or response to therapy with duration and route of administration taken into consideration, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination) |
| 04 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF Conclusion form). |
| 05 | Other important protocol deviations that exclude participant from Per protocol population as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |

# 14.2. Appendix 2: Schedule of Activities

## 14.2.1. Protocol Defined Schedule of Events

| Proced ures | | Inc | luctic | on Ph<br>Veek | | by | | | | | | M | lainte | enan | ce Pl | hase | by W | /eek | | | | | | | | | | n Ph<br>Veek | | | | | • |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- I A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal | Long-Term Follow-Up |
| | | | | | | | | | | | | | Clin | ical a | and ( | Other | Ass | essm | ents | | | | | | | • | | | | | | | |
| Written<br>Informed<br>Consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Eligibility<br>Verificatio<br>n<br>(Inclusion<br>/<br>Exclusion<br>Criteria) | X | X | | | X<br>b | | | | | | | | | | | | | | | | | X<br>b | | | | | | | | | | | |
| Randomiz ation | | | | | | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Demogra<br>phy | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

| Proced ures | | Ind | | on Pl<br>Week | | by | | | | | | N | lainte | enan | ce Pl | nase | by W | /eek | | | | | | | | Ext | ensic<br>by V | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- I A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal <sup>y</sup> | Long-Term Follow-Up |
| Medical<br>History <sup>c</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medicatio<br>n History /<br>Prior ART<br>History | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Symptom<br>Directed<br>Physical<br>Exam and<br>Medical<br>Assessme<br>nt d | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight,<br>BMI, and<br>Height e | | Х | | | | Х | | | | | | | | | | X | | | | | | X | | | | | X | | | | | Х | |
| Cardiovas<br>cular Risk<br>Assessme<br>nt | X | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

| Proced ures | | Inc | | on Pł<br>Week | | by | | | | | | N | lainte | enan | ce Pł | nase | by W | /eek | | | | | | | | | | on Ph<br>Veek | | | | | <b>c</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- 1 A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal <sup>y</sup> | Long-Term Follow-Up |
| Vital<br>Signs<br>(BP, HR,<br>temperatu<br>re) f | Х | Х | | | | Х | Х | | | | | | | | | Х | | | | | | X | | | | | Х | | | | 0 | X | |
| 12-Lead<br>ECG <sup>9</sup> | X | X<br>pr<br>e-<br>do<br>se<br>x3 | | | | X | X | | X<br>g | | | | | | | X<br>g | | | | | | X | | | | | Х | | | | | X | |
| CDC<br>Classificat<br>ion | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| HIV<br>Associate<br>d<br>Condition<br>s | | | X | Х | X | Х | X | X | Х | X | X | X | X | X | X | Х | X | X | X | Х | Х | X | Х | X | Х | Х | X | X | Х | Х | X | Х | X |

| Proced ures | | Ind | | on Pł<br>Week | | by | | | | | | N | lainte | enan | ce Pl | nase | by W | /eek | | | | | | | | | | on Ph<br>Veek | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- 1 A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal | Long-Term Follow-Up |
| AE and<br>SAE<br>Assessme<br>nt, Con<br>Meds | X | Х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | X | Х | X | X | X | Х | Х | X | Х | Х |
| ISR<br>Assessme<br>nt (LA<br>Arm Only) | | | | | | | | | X | X | X | X | X | X | Х | X | X | X | X | Х | Х | X | Х | X | Х | Х | X | X | X | Х | X | X | X<br>If<br>ap<br>pli-<br>ca<br>ble |
| Columbia<br>Suicide<br>Severity<br>Rating<br>Scale<br>(eC-<br>SSRS) | X | Х | | | X | X | X | | X | | X | X | X | X | | X | | | X | W<br>72 | W8<br>4 | X | | | | | | | | | | X | |
| Clinical<br>Chemistry<br>and | Х | Х | Х | Х | Х | Х | Х | Х | | | Х | Х | Х | Х | | Х | Х | Х | Х | Х | | Χ | Х | | Х | Х | | Х | Х | | Х | Х | Х |

| Proced ures | | Inc | | on Pł<br>Week | | by | | | | | | N | laint | enan | ce Pl | nase | by W | /eek | | | | | | | | | | on Ph<br>Veek | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- 1 A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal | Long-Term Follow-Up |
| Hematolo<br>gy | | | | | | | | | | | | | | | | | | | | | | | | | | 1 | | | | | G | | |
| Rapid<br>Plasma<br>Reagin<br>(RPR) | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnanc<br>y Testing <sup>j</sup> | S | U | S | S | S | S | U | S | U | | S | S | S | S | | S | S | S | S | S | S | S | S<br>U | | S | S | U | S | S | S -<br>Q4<br>W | | S | S |
| HIV-1<br>RNA and<br>sample<br>for<br>storage <sup>k</sup> | X<br>k | Х | X | X | X | Х | X | | Х | | X | X | Х | X | | Х | S k | X | X | Х | | X | S <sup>k</sup> | | Х | | X | X | X | | X | X | Х |
| CD4+ | Х | Х | Χ | Х | Χ | Х | Х | | Х | | Χ | Χ | Х | Χ | | Х | | Χ | Χ | Х | | Χ | | | | | Χ | Χ | Χ | | Х | Χ | Χ |
| CD8+ | | Х | | | Х | | Х | | Х | | | Χ | | | | Х | | | | | | Χ | | | | | Χ | | | | | Χ | |
| Urinalysis <sup>I</sup> | | Х | | | | | Х | Χ | | | | Χ | | | | Х | | | | | | Х | | | | Χ | | | | | | Χ | |

| Proced ures | | Inc | | on Pl<br>Week | | by | | | | | | N | lainte | enan | ce Pl | nase | by W | /eek | | | | | | | | | ensic<br>by V | | | | | | c |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- I A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal <sup>y</sup> | Long-Term Follow-Up |
| Fasting Lab Assessme nts: Glucose, Cholester ol (Total, HDL and LDL) and Triglycerid es m | | X | | | | | X | | | | | | | | | Х | | | | | | X | | | | | X | | | | | X | |
| Hepatitis<br>B<br>(HBsAg),<br>Anti-HBc,<br>and Anti-<br>HBsAG<br>Hepatitis<br>C<br>(anti-HCV<br>Ab) | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

| Proced ures | | Inc | | on Pl<br>Neek | hase | by | | | | | | N | lainte | enan | ce Pł | nase | by W | /eek | | | | | | | | | ensio<br>by W | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- I A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal <sup>y</sup> | Long-Term Follow-Up |
| HLA-<br>B*5701 | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| PT/PTT/I<br>NR | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Renal and<br>Bone<br>marker<br>analytes<br>(blood/uri<br>ne) <sup>n</sup> | | | | | | | X | | | | | | | | | X | | | | | | Х | | | | | | | | | | X | |
| Peripheral<br>Blood<br>Mononucl<br>ear Cells<br>(PBMCs) ° | | | | | | | Х | | | | | | | | | | | | | | | Х | | | | | | | | | | Х | |
| Genetic<br>Sample <sup>p</sup> | | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |

| Proced ures | | Inc | | on Pl<br>Neek | nase | by | | | | | | N | /laint | enan | ce Pl | nase | by W | /eek | | | | | | | | | ensio<br>by W | | | | | | C |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- I A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal <sup>y</sup> | Long-Term Follow-Up |
| | | | | | | | | | | | | | Phar | maco | kinet | ics (C | CAB - | ⊦ RP\ | / only | y) | | | | | | | | | | | | | |
| PK<br>Sample<br>(S)=<br>Storage<br>sample | | | | | | | | | X<br>v<br>w | X <sup>t</sup> | X | X | Х | X | X | X<br>v | X | X | X | S | | X | Х | X | X | | X<br>v<br>w | S | | | | X | S |
| OI CAD | | | | | | | <sub>V</sub> | V | | | | | | Inve | stiga<br> | tiona | I Pro | duct | S | | | | V× | | | Vv | | | | | | | |
| Oral CAB<br>and Oral<br>RPV<br>Dispensat<br>ion | | | | | | | X | X | | | | | | | | | | | | | | | X <sup>x</sup><br>O LI<br>O nl<br>y | | | X <sup>x</sup><br>OL<br>On<br>Iy | | | | | | | |
| ABC/DTG<br>/3TC<br>Dispensat<br>ion (or<br>DTG<br>alternate) | | Х | X | X | X<br>qr | | Х | Х | | | X | X | Х | Х | | Х | | Х | | X | | Х | | | | | | | | | | | |

| Proced ures | | Ind | | on Ph<br>Neek | | by | | | | | | N | lainte | enan | ce Pł | nase | by W | /eek | | | | | | | | | | on Ph<br>Veek | | | | | O |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (-4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- I A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal <sup>y</sup> | Long-Term Follow-Up |
| Study<br>Treatment<br>Accounta<br>bility<br>(pill<br>counts) | | | X | X | Xr | X | X | Х | X<br>u | | X | X | Х | X | | X | | X | | X | | X | X O LI O nl y | | | X<br>O<br>LI<br>O<br>nl<br>y | X<br>u | | | | | | |
| IM Study Treatment Administr ation – Q4W throughou t Maintena nce and Extension Phase | | | | | | | | | X | | X | X | X | X | t Rep | X | X | X | X | X | Х | X | X | | X | X | Xs | X | X | X – co nt do s-ing Q4 W | | | |
| HAT-QoL<br>(short<br>form) | | | | | | | Х | | | | | Х | | atieiii | . Kep | X | Jou | COM | E3- | | | Х | | | | | | | | | | Х | |

| Proced ures | | Ind | | on Pl<br>Neek | hase | by | | | | | | N | laint | enan | ce Pl | nase | by W | /eek | | | | | | | | Exte | | on Ph<br>Veek | | | | | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening a | Baseline (-20) | (-16) | (-12, -8) | (4) | WDy | Day 1 | 4a | 4b – LA arm | 5t – LA arm | 8, 12, 16, 20 | 24 | 28, 32, 36 | 40, 44 | 41 – LA arm | 48 | 52 - LA Arm | 56 | 60 – LA Arm | 64, 72, 80, 88 | 68,76, 84, 92<br>- 1 A Arm | 96 | 100 | 101 – Direct to Inject Arm | 104a - Direct to Inject Arm | 104a LA and Oral Lead-In Arm | 104b - Oral Lead-In Arm | 108 | 112, 116, 120,124 | Q4W after 108 (LA Arm) or | Q12W beginning 112 (LA Arm) | Withdrawal | Long-Term Follow-Up |
| SF-12 | | | | | | | Х | | | | | Χ | | | | Х | | | | | | Х | | | | , | | | | | | Χ | |
| ACCEPT | | | | | | | Х | | | | W<br>8 | Χ | | | | Х | | | | | | Х | | | | | | | | | | Χ | |
| HIVTSQ(s | | | | | | | Х | | Χ | | | Х | | W4<br>4 | | | | | | | | Х | | | | | | | | | | Х | |
| HIVTSQ(c) | | | | | | | | | | | | | | | | Х | | | | | | | | | | | | | | | | Х | |
| PIN (LA<br>Arm<br>Only)aa | | | | | | | | | | Х | | | | | Х | Х | | | | | | Х | | | | | | | | | | Х | |
| NRS (LA<br>Arm Only) | | | | | | | | | Х | Х | | | | W4<br>0 | Х | | | | | | | Х | | | | | | | | | | | |
| Preferenc<br>e (LA Arm<br>Only) | | | | | | | | | | | | | | | | Х | | | | | | | | | | | | | | | | | |

Follow Up Visit: Conduct ~4 weeks after the last dose of oral IP. Required only if the participant has ongoing AEs / lab abnormalities at the last on-study visit. This visit may be conducted by telephone.

Direct to Inject: Participants transitioning into the Extension Phase who do not use the optional CAB + RPV oral lead-in beginning at Week 100.

Oral Lead-In: Participants transitioning into the Extension Phase who do use the optional CAB + RPV oral lead-in beginning at Week 100.

LA Arm: Participants who were originally randomized to CAB LA + RPV LA at Day 1.

Switch Arm: All participants who transition into the Extension Phase from ABC/DTG/3TC (or DTG + 2 NRTI's) at Week 100 – e.g., both direct to inject and oral lead-in participants.

Note: BMI- Body mass Index, BP – Blood pressure, HR – Heart Rate, HDL – High Density Lipoprotein, LDL – Low Density Lipoprotein, PT – Prothrombin Time / PTT – Partial Thromboplastin Time / INR – International Normalized Ratio

- a. Complete all Screening assessments within 35 days. Participants may begin the Induction Phase as soon as all Screening assessments are complete. Participants may be rescreened once and will be assigned a new participant number. Confirmation of eligibility to enter the Maintenance Phase, eligibility to enter the Extension Phase.
- b. Collect full routine medical history plus (report at Baseline visit): HIV risk factors (may be collected at a later study visit), cardiovascular risk factors (assessments include smoking status and history, family history of cardiac events), recent [≤6 months] illicit drug use, intravenous drug use, gastrointestinal disease, metabolic, psychiatric, renal and neurologic disorders.
- c. Physical exams should be conducted as part of normal routine clinical care but data will not be collected in the eCRF. Medical assessments include any decisions the study staff must make for participant management and / or care.
- d. Height collected at Baseline only.
- e. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- f. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. Perform ECG at Baseline (Week [-20]) in triplicate prior to dosing. For participants randomized to CAB LA + RPV LA, at Week 4b and Week 48, a second ECG will be obtained approximately 2 hours after the last injection and just prior to the 2 hour post dose PK sampling.
- g. Collect SAEs at Screen only if associated to study participation.
- h. On Day 1, the eC-SSRS is to be administered prior to randomization. During the Maintenance Phase, the eC-SSRS will be administered at each Q4W visit through the Week 48 primary endpoint, and then followed by Q12W assessments for CAB LA + RPV LA arm, thereafter through Week 96 (LA: Week 60, 72, 84, 96). The ABC/DTG/3TC arm will have assessments at Week 72 and Week 96). Preferably completed at the beginning of the visit following administration of other patient reported questionnaires required prior to injections.
- i. Conduct pregnancy tests for only women of childbearing potential at every visit throughout the study, including Q4W during the Extension Phase. Remind females of reproductive potential of the need to avoid pregnancy while in study and adherence to the study's contraception requirements. A negative urine pregnancy test is required prior to beginning the Induction Phase (Week [-20]), on Day 1 (preferably prior to randomization), and at Week 4b (or Week 104b for participants transitioning from ABC/DTG/3TC) prior to the first injection. Serum pregnancy test can substitute for urine pregnancy test if locally required but must be appropriately timed to confirm pregnancy status prior to e.g. randomization and first IM administration. S=Serum/U=Urine.
- j. Plasma for storage will be used: to determine genotypic eligibility at Screen, for possible future analyses, as back- up in case samples are lost or damaged in transit to the lab and for genotypic and phenotypic analyses in cases of virologic failure. HIV-1 RNA will not be collected for analysis at Week 52 and Week 100 (Week 48 or Week 96 retest will be captured as unscheduled visit). Plasma for storage will be collected at Week 52 and Week 100.
- k. A morning specimen is preferred. To assess biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate.
- I. Overnight fast is preferred; however, a minimum of a 6 hour fast is acceptable.
- m. Blood sample for renal and bone biomarker assessments: **Renal:** Cystatin C; Retinol Binding Protein (RBP); **Bone:** bone specific alkaline phosphatase, procollagen type 1-N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin, 25 hydroxy-Vitamin D
- n. Whole blood/Peripheral Blood Mononuclear Cell collection samples may be used for virologic analyses. PBMCs will be collected at Day 1, Week 96, Withdrawal visits.
- o. Informed consent for genetic research must be obtained before sample collection. Sample may be collected at any visit after signing informed consent, but preferably at the Week [-20] visit.
- p. Instruct participants to continue to take the ABC/DTG/3TC regimen until Day 1 of the Maintenance Phase. Participants will be randomized at Day 1 to continue on ABC/DTG/3TC arm or begin oral CAB + oral RPV. Day 1 dosing should occur after randomization to determine defined treatment for the Maintenance Phase.
- q. Remind participants of the potential change in study treatment and visit frequency beginning at Day 1.
- r. Visit Week 104b is only required for participants transitioning from the ABC/DTG/3TC arm.
- s. The Week 5 visit should be performed approximately 7 days after the first injections at Week 4b (3 to 10-day window allowed).
- t. For oral CAB + RPV only.
- u. Take PK samples pre-dose. At Week 4b (and Week 104b for participants transitioning to LA from ABC/DTG/3TC using the optional oral lead-in), the pre-dose PK sample should be taken after review of the PK diary and prior to the final oral CAB + RPV dose. A sample will be also be taken at Week 4b, Week 48, and Week 96 (and Week 100 [direct to inject] or Week 104b [using CAB + RPV oral lead-in]), approximately 2 hours post-injections. The Week 5, Week 41, and Week 101 visit can be performed at any time from 3 to 10 days after the Week 4b, Week 40, and Week 100 injection, respectively. PK samples at Week 5, Week 41, and Week 101 can be taken at any time during the visit.
- v. Participants should take the last dose of oral CAB+RPV at Week 4b (and Week 104b for participants transitioning to LA from ABC/DTG/3TC if using the optional oral lead-in) in the clinic after PK sampling. Participants should take the last dose of ABC/DTG/3TC at Week 100 if transitioning directly to injections at Week 100. Injections should be administered within 2 hours of the last oral dose where possible.
- w. For participants transitioning to CAB LA + RPV LA from ABC/DTG/3TC only.
- x. Follow Up Visit: Conduct approximately 4 weeks after the last dose of oral IP. Required only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. This visit may be conducted by telephone.
- y. With the exception of the NRS questionnaire, patient reported questionnaire/surveys are recommended to be administered at the beginning of the visit before any other clinical assessments are conducted, and prior to completion of the eCSSRs assessments. Only conduct questionnaires/surveys at Withdrawal if occurring prior to Week 96 (The NRS will not be collected at Withdrawal).
- z. The PIN, Preference, and NRS questionnaires are to be administered only to participants receiving CAB LA + RPV LA injections. The NRS should be collected 30 to 60 minutes post-injection (and at Week 5 and Week 41, one-week post-injections) the participant should record the maximum level of pain experienced with the most recent injections.

14.2.2. Protocol Defined Schedule of Events for the Subcutaneous Sub-Study

| Procedures | Screenin | g Phase <sup>d</sup> | | SC / | Abdominal lı | njection Pha | ise <sup>d</sup> | | F | Return to IM | Gluteal Inje | ction Phase | d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>Week -4 | Week -3 | Day 1 | Week 1 | Week 4 | Week 5 | Week 8 | Week 9 | Week 12 | Week 13 | Week 16 | Week 17 | Week 20 |
| IM Gluteal<br>Administration | Х | | | | | | | | X k | | Х | | |
| SC Abdominal<br>Administration <sup>k</sup> | | | Х | | Х | | Х | | | | | | |
| Written<br>Informed<br>Consent | Х | | | | | | | | | | | | |
| Eligibility<br>Verification | Х | | | | | | | | | | | | |
| Inclusion /<br>Exclusion<br>Criteria | | | | | | | | | | | | | |
| Symptom<br>directed<br>physical exam<br>and medical<br>assessment <sup>a</sup> | Х | | Х | | X | | Х | | Х | | Х | | |
| Height, Weight and BMI | | | Х | | | | | | Х | | | | |

| Procedures | Screening Phase d | | | SC / | Abdominal I | njection Pha | ase d | | F | Return to IM | Gluteal Inje | ction Phase | , d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>Week -4 | Week -3 | Day 1 | Week 1 | Week 4 | Week 5 | Week 8 | Week 9 | Week 12 | Week 13 | Week 16 | Week 17 | Week 20 |
| Vital Signs, BP,<br>HR, temp <sup>b</sup> | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| 12 EKG ° | Х | | Х | | | | | | Х | | | | |
| HIV associated conditions | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| AEs, SAEs, concomitant medications | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| ISR<br>assessments<br>for IM injections | Х | Х | Х | | | | | | Х | Х | Х | Х | |
| ISR<br>assessments<br>for SC<br>injections | | | Х | Х | Х | Х | Х | Х | Х | | | | |
| Clinical<br>Chemistry and<br>Hematology | Х | | Х | | Х | | Х | | Х | | Х | | |
| Pregnancy testing, serum <sup>e</sup> | Х | | Х | | Х | | Х | | Х | | Х | | |

| Procedures | Screening | g Phase d | | SC A | Abdominal li | njection Pha | ise <sup>d</sup> | | F | Return to IM | Gluteal Inje | ction Phase | d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>Week -4 | Week -3 | Day 1 | Week 1 | Week 4 | Week 5 | Week 8 | Week 9 | Week 12 | Week 13 | Week 16 | Week 17 | Week 20 |
| HIV-1 RNA and sample for storage (S) | X | | X | | Х | | X | | X | | X | | |
| CD4+ cell count | Х | | Х | | Х | | Х | | Х | | Х | | |
| CD8+ cell count | | | Х | | | | | | Х | | | | |
| Urinalysis f | Х | | Х | | | | | | Х | | | | |
| Fasting lab<br>assessments:<br>glucose,<br>cholesterol<br>(total, HDL and<br>LDL) and<br>triglycerides <sup>9</sup> | X | | X | | | | | | Х | | | | |
| | | | | | PK | Sample Co | llection <sup>j</sup> | | | | | | |
| Pre dose PK<br>samples for<br>CAB and RPV | X | | X | | X | | X | | Х | | X | | |
| Post dose PK sampling (~C <sub>max</sub> ) | | Х | | X | | Х | | Х | | Х | | Х | |

| Procedures | Procedures Screening Phase d | | | SC A | Abdominal I | njection Pha | ase d | | F | Return to IM | Gluteal Inje | ction Phase | d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>Week -4 | Week -3 | Day 1 | Week 1 | Week 4 | Week 5 | Week 8 | Week 9 | Week 12 | Week 13 | Week 16 | Week 17 | Week 20 |
| PROs <sup>m</sup> | | | | | | | | | | | | | |
| HIVTSQc | | | | | | | | Х | | | | | |
| HIVTSQs1 | | X m | | | | | | Х | | | | Х | |
| NRS h | Х | Х | Х | Х | | | Х | Х | Х | Х | | | |
| PIN i | | Х | | Х | | | | Х | | Х | | | |
| Preference SC<br>Abdominal<br>injection vs IM<br>Gluteal injection | | | | | | | | Х | | | | Х | |
| Reason for switch | | Х | | | | | | | | | | | |
| Interest for home administration | | | | | | | | Х | | | | | |

- a. Physical exams should be conducted as part of normal routine clinical care.
- b. Measure vital signs about 5 minutes of rest in a semi-supine position.
- c. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose.

- d. All injection visits during the sub-study should be kept to the same projected visit schedule as in the parent study.
- e. Women of childbearing potential only. SR = serum, UR = urine. Urine pregnancy test can be performed at study visits where other blood draws are not required in order to limit needle sticks.
- f. A morning specimen is preferred.
- g. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- h. Should be collected 30 to 60 minutes post injection. To be assessed separately for CAB LA and RPV LA
- i. To be assessed separately for CAB LA and RPV LA.
- j. PK window allowed for sample collection: For 1-week post dose sample (3 to 10 days post dose).
- k. During the SC phase (and for the first IM injection in the return to IM injection phase), the dosing window can be -7 days, however, it cannot be +7 days from the projected visit date. Once SC injections begin, the next SC administration can be 3-4 weeks later, however, SC administration may not take place 5 weeks later. See details in Section 12.12.1.2. and Section 12.12.4.3.
- 1. All Patient Reported Outcome Questionnaires/Surveys will be administered via paper instrument (in exception circumstances, the questionnaires could be completed via telephonic interview, please refer to the COVID19 appendix for additional details) at the beginning of the visit before any other assessments are conducted, with the exception of the NRS.
- m. For HIVTSQs, we want to measure satisfaction with IM gluteal injection prior to switch to sub-cutaneous. This will be assessed at week -3 (questionnaire can be administered at any time during the visit).

## 14.3. Appendix 3: Assessment Windows

#### 14.3.1. Definitions of Assessment Windows

AEs, SAEs and concomitant medications to be assessed pre-dose. IM administration itself and all other assessments will be considered part of the parent study, and should be completed as per the study time and events tables in Section 14.2.

Laboratory data, vital signs, ECGs, NRS questionnaire (health outcomes) assessments, protocol deviations, and genotypic/phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

In most cases the window around an assessment will include all dates from the midpoints between the target day and that of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w) +1.

For parameters which are not scheduled to be assessed at particular visits, the all-inclusive assessment windows will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

Prior to visit slotting, assessments are first assigned to a study Phase (screening, induction, maintenance, extension, sub-study screening, SC injection, return to gluteal injection, or Long Term Follow Up) based on the tables in Section 14.4.1 and treatment state based on Section 14.4.2.

Induction Phase and Maintenance Phase assessments are assigned based on the Induction Phase Study Day and Maintenance Phase Study Day, respectively, as shown in Table 14 and Table 15. The analysis visits from Week 4 to Week 100 should be only applied to the assessments that are already assigned to Maintenance Phase (on-treatment).

Extension Phase assessments are assigned based on the Maintenance Phase Study day for participants continuing Q4W IM dosing into the Extension Phase and based on the Extension Phase Study Day for participants switching from the control arm to Q4W IM dosing for the Extension Phase as shown in Table 16. The analysis visits from Week 104 (except for Follow-up) in the Extension Phase should be only applied to the assessments that are already assigned to Extension Phase (on-treatment).

Assessment windows at key analysis time points for the snapshot efficacy data are shown in Table 17.

The sub-study assessments other than health outcome, PK and HIV-1 RNA are assigned analysis visits based on Study Day as shown in Table A. The assessment visit windows for HIV-1 RNA data are defined in Table B, and the snapshot windows for visits up to Sub-study Week 12 are defined in Table C.Long-term Follow-up Phase assessments are assigned based on the LTFU study day as shown in Table 20. See Section 14.6.1 for derivation of Induction, Maintenance, Extension and LTFU Study Day.

# 14.3.2. Definitions of Assessment Windows for Data Other than Health Outcomes and PK

Table 14 Assessment Windows for Screening and Induction Phase Data

| Analysis Set | Parameter | Target | Analysis Window | Analysis Timepoint |
|---|---|---|---|---|
| / Domain | | Study<br>Day | | |
| All | All | The day of earliest record | Induction Study Day ≤1 | Screening |
| | | 1 | Last available recorded value up to<br>and including the date of first<br>Induction Phase dose of IP | Induction<br>Baseline (Week -20) |
| | | 29 | 2 ≤ Induction Study Day ≤ 42 | Week -16 |
| | | 57 | 43 ≤ Induction Study Day ≤ 70 | Week -12 |
| | | 85 | 71 ≤ Induction Study Day ≤ 98 | Week -8 |
| | | 113 | 99 ≤ Induction Study Day ≤ 126 | Week -4 |
| | | 141 | 127 ≤ Induction Study Day ≤ Induction ART Stop Day[a] + 1 | Day 1 |
| | | | For Participants not continuing into Maintenance Phase: Induction Study Day > (Induction | Follow-up |
| | | | ART Stop Day[a] +1) | |

#### NOTES:

- For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings.
- a. ABC/DTG/3TC stop day: the last permanently stop day among all ARTs taken during Induction Phase.

 Table 15
 Assessment Windows Maintenance Phase Data

| All Parameters expect where noted <sup>f</sup> | Analysis Window | Target<br>Study Day | Analysis<br>Timepoint |
|---|---|---|---|
| | Last available recorded value up to and including the date of first Maintenance Phase dose of IP | 1 | Maintenance<br>Baseline (Day 1) |
| ECG, CD8, CD4/CD8 ratio | 2 ≤ Study Day ≤ 70<br>2 ≤ Study Day ≤ 42 | 29 | Week 4 |
| | 43 ≤ Study Day ≤ 70 | 57 | Week 8 |
| | 71 ≤ Study Day ≤ 98 | 85 | Week 12 |
| | 99 ≤ Study Day ≤ 126 | 113 | Week 16 |
| | 127 ≤ Study Day ≤ 154 | 141 | Week 20 |
| CD8, CD4/CD8 ratio | 155 ≤ Study Day ≤ 210 | | |
| , | 155 ≤ Study Day ≤ 182 | 169 | Week 24 |
| | 183 ≤ Study Day ≤ 210 | 197 | Week 28 |
| | 211 ≤ Study Day ≤ 238 | 225 | Week 32 |
| | 239 ≤ Study Day ≤ 266 | 253 | Week 36 |
| | 267 ≤ Study Day ≤ 294 | 281 | Week 40 |
| | 295 ≤ Study Day ≤ 322 | 309 | Week 44 |
| ECG, CD8, CD4/CD8 ratio, Urinalysis [c], Renal and Bone marker analytes [d], Lipids [e], Weight, Height, Vital Signs | 323 ≤ Study Day ≤ 378 | 337 | Week 48 |
| | 323 ≤ Study Day ≤ 350 | | |
| | 351 ≤ Study Day ≤ 378 | 365 | Week 52 |
| | 379 ≤ Study Day ≤ 406 | 393 | Week 56 |
| | 407 ≤ Study Day ≤ 434 | 421 | Week 60 |
| | 435 ≤ Study Day ≤ 476 | 449 | Week 64 |
| | 477 ≤ Study Day ≤ 532 | 505 | Week 72 |
| | 533 ≤ Study Day ≤ 588 | 561 | Week 80 |
| | 589 ≤ Study Day ≤ 644 | 617 | Week 88 |
| ECG, CD4, CD8, CD4/CD8 ratio,<br>Urinalysis <sup>[c]</sup> ,<br>Renal and Bone marker analytes <sup>[d]</sup> ,<br>Lipids <sup>[e]</sup> , Weight, Height, Vital Signs | 645 ≤ Study Day ≤ 714 | 673 | Week 96 |
| | 645 ≤ Study Day ≤ 686 | | |

| All Parameters expect where noted <sup>f</sup> | Analysis Window | Target<br>Study Day | Analysis<br>Timepoint |
|---|---|---|---|
| ECG, CD4, CD8, CD4/CD8 ratio, Urinalysis <sup>[c]</sup> , Renal and Bone marker analytes <sup>[d]</sup> , Lipids <sup>[e]</sup> , Weight, Height, Vital Signs | For 'ABC/DTG/3TC' arm: 715 ≤ Study Day ≤ Maintenance ABC/DTG/3TCStop Day <sup>[b]</sup> + 1 For 'Q4W' arm: 715 ≤ Study Day ≤ Max (Day of Last Q4W IM Dose + 35, Last Oral dose Day + 1) [a] | 701 | Week 100 |
| | For 'ABC/DTG/3TC' arm: 687 ≤ Study Day ≤ Maintenance ABC/DTG/3TCStop Day <sup>[b]</sup> + 1 For 'Q4W' arm: 687 ≤ Study Day ≤ Max (Day of Last Q4W IM Dose + 35, Last Oral dose Day + 1) [a] | 701 | Week 100 |
| | a) For participants who discontinued from oral lead-in during Maintenance Phase: Study Day > (Day of last oral lead-in dose+1) b) For participants who are not continuing into the extension phase and who received at least one CAB/RPV injection: Study Day > Max (Day of Last Q4W IM Dose + 35, Last Oral dose Day + 1) For 'ABC/DTG/3TC' arm: Participants discontinued from ABC/DTG/3TC' and not continuing into the Extension Phase: Study Day > (Maintenance ABC/DTG/3TC Stop Day <sup>[b]</sup> +1) | | Follow-up |

- For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot).
- a. Last Q4W IM / last oral dose is only applied to participants who permanently discontinue from study treatment
- b. ABC/DTG/3TCstop day: the last permanently stop day among all ARTs taken during Maintenance Phase.
- c. **Urinalysis**: All parameters provided by the central laboratory under the category of urinalysis, including Urine Albumin/Creatinine, Urine Creatinine, Urine Ph, Urine Protein/Creatinine, Urine Erythrocytes, Urine Specific Gravity, Urine Leukocytes, Urine Retinol Binding Protein, Urine Phosphate, Urine Creatinine.
- d. **Bone Marker**: Bone Specific Alkaline Phosphatase, Osteocalcin, Procollagen 1 N-Terminal Propeptide, Vitamin D, Type I C-Telopeptides. **Renal marker**: Cystatin C, Retinol Binding Protein.
- e. **Lipids**: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
- f. Analysis windows for parameters with sparse collection are noted.

#### Table 16 Assessment Windows for Extension Phase Data

| All Parameters expect where noted <sup>b</sup> | Analysis Window | Target<br>Extension<br>Phase<br>Study<br>Day | Target<br>Study<br>Day | Analysis<br>Timepoint |
|---|---|---|---|---|
| | Participants Continuing Randomiz | ed Q4W IM Re | gimen | |
| Adverse Events [c] | Study day of Nominal Week 100<br>visit ≤ Study Day ≤ 742 | | | |
| Urinalysis [a] | Study day of Nominal Week 100<br>visit < Study Day ≤ 770 | | 729 | Week 104 |
| | Study day of Nominal Week 100<br>visit < Study Day ≤ 742 | | | |
| | 743≤ Study Day ≤770 | | 757 | Week 108 |
| | 771≤ Study Day ≤826 | | 785 | Week 112 |
| | (7*w - 41)<br>$\leq$ Study Day $\leq$ $(7*w + 42)$ | | 7*w + 1 | Week w<br>w = 124,136,<br>148, |
| | For participants who permanently discontinue extension phase study treatment: Study Day > Max (Day of Last Q4W IM Dose + 35, Day of Last Oral Dose Day + 1) | | | Follow-up |
| Participants Switching to Q4W IM Dosing | | | | |
| | Last available recorded value up to<br>and including the date of first<br>Extension Phase dose of IP | 1 | | Extension Baseline<br>(W100) |
| ECG, CD4, CD8,<br>CD4/CD8 ratio, | 2 ≤ Extension Study Day ≤ 70 | 29 | | Week 104 |

| All Parameters expect where noted <sup>b</sup> | Analysis Window | Target<br>Extension<br>Phase<br>Study<br>Day | Target<br>Study<br>Day | Analysis<br>Timepoint |
|---|---|---|---|---|
| Urinalysis [a], | | | | |
| Weight, Vital Signs | | | | |
| | 2 ≤ Extension Study Day ≤ 42 | | | |
| Excluding: ECG, CD4,<br>CD8, CD4/CD8 ratio,<br>Urinalysis [a], Weight,<br>Vital Signs | 43 ≤ Extension Study Day ≤ 70 | 57 | | Week 108 |
| | 71 ≤ Extension Study Day ≤ 98 | 85 | | Week 112 |
| | 99 ≤ Extension Study Day ≤ 126 | 113 | | Week 116 |
| | 127 ≤ Extension Study Day ≤ 154 | 141 | | Week 120 |
| | 155 ≤ Extension Study Day ≤ 210 | 169 | | Week 124 |
| | 211 ≤ Extension Study Day ≤ 294 | 253 | | Week 136 |
| | (7*(w-100) - 41)<br>$\leq$ Study Day $\leq$ $(7*(w-100) + 42)$ | 7*(w-100) +<br>1 | | Week w<br>w = 148, 160, |
| | For participants who permanently discontinue extension phase study treatment: Study Day > Max (Day of Last Q4W IM Dose + 35, Day of Last Oral Dose Day + 1) | | | Follow-up |

- For parameters which are not scheduled to be assessed at particular visits, the all-inclusive windows defined will still be used. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well as algorithms that make use of additional data (e.g., Snapshot).
- Nominal Week 100 visit is the original visit from eCRF (i.e., the VISIT variable as opposed to AVISIT)
- a. **Urinalysis**: All parameters provided by the central laboratory under the category of urinalysis, including Urine Albumin/Creatinine, Urine Creatinine, Urine pH, Urine Protein/Creatinine, Urine Erythrocytes, Urine Specific Gravity, Urine Leukocytes, Urine Retinol Binding Protein, Urine Phosphate, Urine Creatinine.
- b. Analysis windows for parameters with sparse collection are noted.
- c. For ISR specific displays, ISRs will be assigned to analysis timepoints based on onset date to the most recent planned IM injection visit prior or equal to the AE onset date.

Table 17 Assessment Windows for Summary of Snapshot Data — Data assigned to Maintenance Phase Only

| Snapshot Analy (if no viral load data in default window | | |
|---|---|---|
| Default (midpoint between planned visits) <sup>a</sup> | Expanded +6 Week upper window | Analysis<br>Timepoint |
| Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Maintenance<br>Baseline (Day 1) |
| 2 ≤ Study Day ≤ 42 | 2 ≤ Study Day ≤ 70 | Week 4 |
| 43 ≤ Study Day ≤ 70 | 43 ≤ Study Day ≤ 98 | Week 8 |
| 71 ≤ Study Day ≤ 98 | 71 ≤ Study Day ≤ 126 | Week 12 |
| 99 ≤ Study Day ≤ 126 | 99 ≤ Study Day ≤ 154 | Week 16 |
| 127 ≤ Study Day ≤ 154 | 127 ≤ Study Day ≤ 182 | Week 20 |
| 155 ≤ Study Day ≤ 182 | 155 ≤ Study Day ≤ 210 | Week 24 |
| 183 ≤ Study Day ≤ 210 | 183 ≤ Study Day ≤ 238 | Week 28 |
| 211 ≤ Study Day ≤ 238 | 211 ≤ Study Day ≤ 266 | Week 32 |
| 239 ≤ Study Day ≤ 266 | 239 ≤ Study Day ≤ 294 | Week 36 |
| 267 ≤ Study Day ≤ 294 | 267 ≤ Study Day ≤ 322 | Week 40 |
| 295 ≤ Study Day ≤ 322 | 295 ≤ Study Day ≤ 350 | Week 44 |
| 295 ≤ Study Day ≤ 378 | 295 ≤ Study Day ≤ 378 | Week 48 |
| 379 ≤ Study Day ≤ 406 | $379 \le \text{Study Day} \le 434$ | Week 56 |
| 407 ≤ Study Day ≤ 434 | 407 ≤ Study Day ≤ 462 | Week 60 |
| 435 ≤ Study Day ≤ 476 | 435 ≤ Study Day ≤ 490 | Week 64 |
| 477 ≤ Study Day ≤ 532 | 477 ≤ Study Day ≤ 546 | Week 72 |
| 533 ≤ Study Day ≤ 588 | 533 ≤ Study Day ≤ 602 | Week 80 |
| 589 ≤ Study Day ≤ 644 | 589 ≤ Study Day ≤ 658 | Week 88 |
| 631 ≤ Study Day ≤ 714 | 631 ≤ Study Day ≤ 714 | Week 96 |

Apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 30) within the Maintenance Phase (Per Table 25)

a.  $\pm$  6 Week window always used at key analysis timepoints (Week 48 and Week 96)

Table 18 For W124 Analysis: Extension Switch Population Assessment Windows for Snapshot Viral Load Data up to Week 124 — Data assigned to Extension Phase Only

| Snapshot Anal<br>(if no viral load data in default window | | |
|---|---|---|
| Default (midpoint between planned visits) <sup>a</sup> | Analysis<br>Timepoint | |
| Last available recorded value up to and including the date of first Extension Phase dose of IP (oral lead-in or injection, whichever occurs first) | Last available recorded value up to and including the date of first Extension Phase dose of IP (oral lead-in or injection, whichever occurs first) | Extension<br>Baseline (Week<br>100) |
| 2 ≤ Extension Study Day ≤ 42 | 2 ≤ Extension Study Day ≤ 70 | Week 104 |
| 43 ≤ Extension Study Day ≤ 70 | 43 ≤ Extension Study Day ≤ 98 | Week 108 |
| 71 ≤ Extension Study Day ≤ 98 | 71 ≤ Extension Study Day ≤ 126 | Week 112 |
| 99 ≤ Extension Study Day ≤ 126 | 99 ≤ Extension Study Day ≤ 154 | Week 116 |
| 127 ≤ Extension Study Day ≤ 154 | 127 ≤ Extension Study Day ≤ 182 | Week 120 |
| 127 ≤ Extension Study Day ≤ 210 | 127 ≤ Extension Study Day ≤ 210 | Week 124 |
| For participants who permanently discontinue extension phase study treatment: Extension Study Day > Max (Day of Last Q4W IM Dose + 35, Day of Last Oral Dose Day + 1) | | Follow-up |

Apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 30) within the Extension Phase (Per Table 25)

a.  $\pm$  6 Week window always used at key analysis timepoints (Week 124)

Table 19 For W124 Analysis: ITT-E (Randomized Q4W arm) Assessment Windows for Snapshot Viral Load Data up to Week 124 — Data assigned to Maintenance and Extension Phase

| Snapshot Anal (if no viral load data in default window | • | |
|---|---|---|
| Default (midpoint between planned visits) <sup>a</sup> | Expanded +6 Week upper window | Analysis<br>Timepoint |
| Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Maintenance<br>Baseline (Day 1) |
| 2 ≤ Study Day ≤ 42 | 2 ≤ Study Day ≤ 70 | Week 4 |
| 43 ≤ Study Day ≤ 70 | $43 \le \text{Study Day} \le 98$ | Week 8 |
| 71 ≤ Study Day ≤ 98 | 71 ≤ Study Day ≤ 126 | Week 12 |
| 99 ≤ Study Day ≤ 126 | 99 ≤ Study Day ≤ 154 | Week 16 |
| 127 ≤ Study Day ≤ 154 | 127 ≤ Study Day ≤ 182 | Week 20 |
| 155 ≤ Study Day ≤ 182 | 155 ≤ Study Day ≤ 210 | Week 24 |
| 183 ≤ Study Day ≤ 210 | 183 ≤ Study Day ≤ 238 | Week 28 |
| 211 ≤ Study Day ≤ 238 | 211 ≤ Study Day ≤ 266 | Week 32 |
| 239 ≤ Study Day ≤ 266 | 239 ≤ Study Day ≤ 294 | Week 36 |
| 267 ≤ Study Day ≤ 294 | 267 ≤ Study Day ≤ 322 | Week 40 |
| 295 ≤ Study Day ≤ 322 | 295 ≤ Study Day ≤ 350 | Week 44 |
| 295 ≤ Study Day ≤ 378 | 295 ≤ Study Day ≤ 378 | Week 48 |
| 379 ≤ Study Day ≤ 406 | 379 ≤ Study Day ≤ 434 | Week 56 |
| 407 ≤ Study Day ≤ 434 | 407 ≤ Study Day ≤ 462 | Week 60 |
| 435 ≤ Study Day ≤ 476 | 435 ≤ Study Day ≤ 490 | Week 64 |
| 477 ≤ Study Day ≤ 532 | 477 ≤ Study Day ≤ 546 | Week 72 |
| 533 ≤ Study Day ≤ 588 | 533 ≤ Study Day ≤ 602 | Week 80 |
| 589 ≤ Study Day ≤ 644 | 589 ≤ Study Day ≤ 658 | Week 88 |
| 631 ≤ Study Day ≤ 714 | 631 ≤ Study Day ≤ 714 | Week 96 |
| 715 ≤ Study Day ≤ 770 | 715 ≤ Study Day ≤ 798 | Week 108 |
| 771 ≤ Study Day ≤ 826 | 771 ≤ Study Day ≤ 826 | Week 112 |
| 827 ≤ Study Day ≤ 910 | 827 ≤ Study Day ≤ 910 | Week 124 |
| NOTES: | | |

Apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 30) within the Maintenance Phase and Extension Phases (Per Table 25)

Table A Assessment Windows for Sub-study Baseline, SC Injection Phase and Return to Gluteal Injection Phase Data (Excluding HIV-1 RNA Data)

| All Parameters<br>except for where<br>noted <sup>[a]</sup> | Target<br>Study Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| | First Sub-<br>study record | Study Day <7*w + 1 | Sub-study<br>Screening |
| All except ECG,<br>Labs, Vitals | 7*w + 1 | Study Day = 7*w + 1 | Sub-study Day 1 |

a.  $\pm$  6 Week window always used at key analysis timepoints (Week 48 and Week 96)

| All Parameters except for where | Target | | |
|---|---|---|---|
| noted <sup>[a]</sup> | Study Day | Analysis Window | Analysis Timepoint |
| ECG, Labs, Vitals | 7*w + 1 | Last available recorded value up to and including the date of first SC injection. | Sub-study<br>Baseline <sup>[b]</sup> |
| | 7*(w+1) +1 | $7*w + 2 \le Study Day \le 7*(w+2)$ | Sub-study Week 1 |
| Labs,CD4 | 7*(w+4) +1 | $7*(w + 2) + 1 \le \text{Study Day} \le 7*(w+4) + 1$<br>$7*w + 2 \le \text{Study Day} \le 7*(w+6)$ | Sub-study Week 4 |
| | 7*(w+5) +1 | $7*(w + 4) + 2 \le Study Day \le 7*(w+6)$ | Sub-study Week 5 |
| Labs, CD4 | 7*(w+8) +1 | $7^*(w + 6) + 1 \le \text{Study Day} \le 7^*(w+8) + 1$<br>$7^*(w + 6) + 1 \le \text{Study Day} \le 7^*(w+10)$ | Sub-study Week 8 |
| | 7*(w+9) +1 | $7*(w + 8) + 2 \le Study Day \le 7*(w+10)$ | Sub-study Week 9 |
| | | $7*(w + 10) + 1 \le Study Day \le 7*(w+12) + 1$ | |
| Labs, CD4 | | $7*(w + 10) + 1 \le Study Day \le 7*(w+14)$ | |
| ECG, Weight, CD8,<br>CD4/CD8 ratio<br>Urinalysis, Fasting<br>labs/lipids | 7*(w+12) +1 | 7*w + 2 ≤ Study Day | Sub-study Week 12 |
| | 7*(w+13) +1 | $7*(w + 12) + 2 \le Study Day \le 7*(w+14)$ | Sub-study Week 13 |
| Laka OD4 | 7*(w+16) +1 | $7*(w + 14) + 1 \le \text{Study Day} \le 7*(w+16) + 1$ | Sub-study Week 16 |
| Labs, CD4 | 7*/47\4 | $7*(w + 14) + 1 \le Study Day \le 7*(w+18)$ | Out atual Made 47 |
| | 7*(w+17) +1 | $7*(w + 16) + 2 \le Study Day \le 7*(w+18)$ | Sub-study Week 17 |
| | 7*(w+20) +1 | $7*(w+18) + 1 \le Study Day$ | Sub-study Week 20 |
| <u> </u> | t a participant i | permanently discontinued study treatment | : |
| | | Date > max (Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Date of Last Injection + 35) | Follow-up |

- The "w" in the target study day calculation refers to the week number within the Sub-study, starting with Week 0. For example, the Sub-study Day 1 Analysis Timepoint would have a "w" of 0, to allow for a Target Study Day of 1.
- Follow-up will be derived only for participants who permanently discontinued study treatment.
- Sub-study Day 1 (Post Dose), Sub-study Week 4 and Sub-study Week 8 visits are SC Injection phase visits, Sub-study Week 12 and Week 16 are Return to Gluteal Injection phase visits.

[a] Analysis windows for parameters with sparse collection are noted.

[b] The values considered for deriving Sub-study Baseline value include both Extension phase and sub-study data.

# Table B Assessment Windows for Sub-study Baseline, SC Injection Phase and Return to Gluteal Injection Phase HIV-1 RNA Data

| Phase | Target Study ase Day Analysis Window | | Analysis Timepoint |
|---|---|---|---|
| Sub-study Screening | 7*w + 1 | Last available recorded value up to<br>and including the date of first SC<br>injection | Sub-study Baseline |
| SC Injection | 7*(w+4) + 1 | $7*w + 2 \le Study Day \le 7*(w+6)$ | Sub-study Week 4 |
| SC Injection | 7*(w+8) + 1 | $7*(w+6) + 1 \le Study Day \le 7*(w+10)$ | Sub-study Week 8 |
| Return to Gluteal | 7*(w+12) + 1 | $7*(w+10) + 1 \le Study Day \le 7*(w+14)$ | Sub-study Week 12 |
| Injection | 7*(w+16) + 1 | $7*(w+14) + 1 \le Study Day \le 7*(w+18)$ | Sub-study Week 16 |
| If a | participant per | manently discontinued study treatment | |
| | | Date > max (Date of Last Dose of Oral<br>Study Treatment (CAB+RPV or SOC<br>Bridging) + 1, Date of Last Injection +<br>35) | Follow-up |

- The "w" in the target study day calculation refers to the week number within the Sub-study, starting with Week 0, Day 0 being the day prior to the first SC injection. For example, the Sub-study Day 1 Analysis Timepoint would have a "w" of 0, to allow for a Target Study Day of 1.
- Follow-up will be derived only for participants who permanently discontinued study treatment.

Table C Assessment Windows for Summary of Snapshot Data Up to Week 12 in Sub-study— Data Assigned to SC Injection Phase

| Snapshot A (If no on-treatment viral load da w | | |
|---|---|---|
| Default | Analysis Timepoint | |
| Last available recorded value up to<br>and including the date of first SC<br>injection | Last available recorded value up to and including the date of first SC injection | Sub-study Baseline |
| $7*w + 2 \le Study Day \le 7*(w+6)$ | $7*w + 2 \le Study Day \le 7*(w+10)$ | Sub-study Week 4 |
| $7*(w+6) + 1 \le Study Day \le 7*(w+10)$ | $7^*(w+6) + 1 \le Study Day \le 7^*(w+14)$ | Sub-study Week 8 |
| 7*(w+10) + 1 ≤ Study Day ≤<br>min( 7*(w+14), Day of First Return to<br>Gluteal IM Injection) | 7*(w+10) + 1 ≤ Study Day ≤ min(7*(w+18),<br>Day of First Return to Gluteal IM Injection) | Sub-study Week 12 |

#### NOTES:

- The "w" in the target study day calculation refers to the week number within the Sub-study, starting with Week 0, Day 0 being the day prior to the first SC injection. For example, the Sub-study Day 1 Analysis Timepoint would have a "w" of 0, to allow for a Target Study Day of 1.
- For post-baseline visits (i.e., Week 4 and afterwards), apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 30) within the SC Injection Phase (per Table 24).
- An on-treatment viral load assessment may be assigned to more than one snapshot analysis window, e.g., on-treatment assessment taken on 7\*(w+14) will be in both Sub-study Week 8 and Sub-study Week 12 visits.
- ± 6 Week window is always used at the key analysis timepoint, Sub-study Week 12 visit with the
  exclusion of HIV-1 RNA values collected on or after resuming IM injections. Only results collected while
  on SC injections will be considered.

Table 20 Assessment Windows for Summaries of Long-Term Follow Up
Phase Data for Participants Who Received At least One Injection of
CAB+RPV and Permanently Discontinued from Study Treatment

| Day of Assessment | Assessment<br>Window | Target Study Day of Window |
|---|---|---|
| 1 ≤ LTFU Study Day ≤ 60 | LTFU Month 1 | 30 |
| 61 ≤ LTFU Study Day ≤ 135 | LTFU Month 3 | 90 |
| 136 ≤ LTFU Study Day ≤ 225 | LTFU Month 6 | 180 |
| 226 ≤ LTFU Study Day ≤ 315 | LTFU Month 9 | 270 |
| 316 ≤ LTFU Study Day ≤ 405 | LTFU Month 12 | 360 |
| (30*m - 44) ≤ LTFU Study Day≤ (30*m + 45) | LTFU Month m<br>m = 15, 18, 21, | 30*m |
| NOTES: • An assessment may be slotted to both LTFU and Mainter | nance /Extension Phase | |

## 14.3.3. Assessment Window for Study Conclusion

The study conclusion and Phase conclusion records in disposition data will be slotted based on Table 14 (for Induction Phase conclusion records), Table 15 (for Maintenance Phase conclusion records) and Table 16 (for extension Phase conclusion records). However, if the discontinuation date is post-treatment (based on Table 30), then the discontinuation will be slotted to the participants the last attained on-treatment analysis visit across all assessments (e.g., analysis visit corresponding to the last on-treatment lab assessment), rather than follow up.

#### 14.3.4. Assessment Window for Health Outcome Data

#### 14.3.4.1. NRS

NRS questionnaire assessments are assigned to analysis visits based on the windows defined in Table 21.

Table 21 Assessment Windows for Maintenance Phase NRS Questionnaire Data

| Domain | Parameter | Target Date | Analysis Window | Analysis |
|---|---|---|---|---|
| | | | | Timepoint |
| NRS | All | Date of 1st<br>Injection | Assessment Date ≤ Date of 1st injection + 2 | Week 4B |
| | | Date of 1st<br>injection+7 | Date of 1 <sup>st</sup> injection +3 ≤ Assessment Date ≤ Date of 1 <sup>st</sup> injection + 42 | Week 5 |
| | | Date of W40<br>Injection | If participant received Week 40 injection: Date of WK40 injection - 42 ≤ Assessment Date ≤ Date of W40 Injection + 2 | |
| | | Date of 1 <sup>st</sup><br>Injection +<br>252 | If participant did not receive Week 40 injection: Date of 1st injection + 210 ≤ Assessment Date ≤ Date of 1st injection + 280 | Week 40 |
| | | Date of W40<br>Injection + 7 | If participant received Week 40 injection: Date of W40 Injection + 3 ≤ Assessment Date ≤ Date of W40 Injection + 28 | Week 41 |
| | | Date of 1 <sup>st</sup><br>Injection +<br>644 | Date of 1st Injection + 602 < Assessment Date ≤ Date of 1st Injection + 686 | Week 96 |

Note: Apply NRS analysis windows only to assessments that are on-treatment (per Table 30) within the Maintenance Phase (Per Table 25)

#### 14.3.4.2. PIN/HATQoL/SF-12/HIVTSQs/HIVTSQc/ACCEPT/Treatment Preference

PIN, HATQoL, SF-12, HIVTSQs, HIVTSQc, ACCEPT, and Treatment Preference questionnaire assessments will be assigned to analysis visits as follows:

- 1. Maintenance Baseline (Day 1) will be defined as last available recorded value up to and including the date of first Maintenance Phase dose of study treatment (expected to be collected at Day 1).
- 2. If the nominal visit identifier as captured in the source dataset corresponds to a scheduled collection per the Time and Events Schedule (see Section 14.2 and Table 22) and the assessment is collected in the Maintenance Phase (per Table 25), then the nominal visit identifier will be kept as the analysis visit (excluding Day 1 which will normally be assigned to Maintenance Baseline (Day 1).
- 3. If the nominal visit identifier is unscheduled or withdrawal, then the following procedure will be used:
  - a) Assign the assessment to a study Phase according to Table 25. Proceed to step b if the assessment is assigned to the Maintenance Phase.
  - b) Identify the 'last nominal visit' with the HO assessment performed prior to the unscheduled/withdrawal visit to be slotted.
  - c) The unscheduled/withdrawal visit will be slotted to the planned nominal visit subsequent to the 'last nominal visit'. If the 'last nominal visits' does

not exist (e.g., no records originate from a planned nominal visit), then the unscheduled/withdrawal visit will be slot to the first planned nominal visit after Day 1.

Example 1, for HATQoL, the planned nominal visits are Week 24, 48, and 96. If a participant has the 'last nominal visit' (with HATQoL assessment) at Week 24 prior to withdrawal at Week 36, the withdrawal assessment will be slotted to the subsequent planned nominal visit of Week 48.

Example 2, for HATQoL, if there is unscheduled visit between Week 24 and Week 48. This unscheduled visit will be slotted to Week 48 per the rule. In this case, there are two assessments with analysis visit equal to Week 48 (i.e., the slotted value and the value at original nominal week 48 visit). The original nominal value will be selected for summary per the rule below for multiple records—see Section 14.3.6.

Table 22 Planned Nominal Visit of Health Outcome Data

| Endpoints | Day1 | W4b | W5 | W8 | W24 | W40 | W41 | W44 | W48 | W52 | W96 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| PIN (Q4W) | | | Χ | | | | Χ | | Χ | | Χ |
| HATQoL | Х | | | | Χ | | | | Χ | | Χ |
| SF-12 | Х | | | | Χ | | | | Χ | | Χ |
| HIVTSQs | Х | x<br>(Q4W<br>arm<br>only) | | | Х | | | Х | | | Х |
| HIVTSQc | | | | | | | | | Χ | | |
| ACCEPT | Х | | | Х | Χ | | | | Х | | Χ |
| NRS (Q4W) | | Х | Χ | | | Χ | Χ | | | | Χ |
| Treatment preference (Q4W) | | | | | | | | | Х | | |

#### 14.3.4.3. Evaluable Criteria for Observed Case Displays — NRS and PIN

Post the visit slotting as described above, data that is assessed outside of 5-9 days post injection (relative to date of injection at Week 4b/40, respectively) at Week 5/41 for NRS/PIN, and data at Week 4b/40 for NRS that is not assessed on the same day as CAB+RPV injections (at Week 4b/40, respectively) are received will be excluded from Observed Case Displays (see Table 23). However, these data will still be used for LOCF displays.

| Endpoints | W4b | W5 | W40 | W41 | W96 |
|---|---|---|---|---|---|
| PIN | | Within Day | | Within Day 5-9 | |
| (Q4W) | | 5-9 post W4b | | post W40 | |
| | | injection | | injection | |
| NRS | On the same | Within Day | On the same | Within Day 5-9 | On the same day |
| (Q4W) | Day of W4b | 5-9 post W4b | day of W40 | post W40 | of W96 injection |
| | injection | injection | injection | injection | - |

Table 23 Evaluable Time Windows for Observed Cases Summary Tables

# 14.3.4.4. HIVTSQs/HIVTSQc/PIN/Preference/Reason for Switch/Interest in Substudy

HIVTSQs, HIVTSQc, PIN, Preference SC Injection vs Gluteal Injection, Reason for Switch, and Interest questionnaire assessments will be assigned to analysis visits as follows:

- 1. Sub-study Baseline will be defined as last available recorded value prior to the date of first SC injection. Baseline is not applicable for HIVTSQc, Preference SC Injection vs Gluteal Injection, Reason for Switch, or Interest assessments as they are not planned to be collected during the Sub-study Baseline.
- 2. For post-baseline visits, if the nominal visit identifier as captured in the source dataset corresponds to a scheduled collection per the Time and Events Schedule (see Section 14.2.2) and the assessment is collected in the planned phase (per Table 24, visits at/before Sub-study Week 12 belong to SC Injection phase, and visits after Sub-study Week 12 belong to Return to Gluteal Injection phase), then the nominal visit identifier will be kept as the analysis visit.
- 3. For post-baseline visits, if the nominal visit identifier is unscheduled or it is scheduled however not conducted in the planned phase (e.g., the sub-study Week 9 HIVTSQs assessment is conducted after the Week 12 gluteal injection and therefore belong to Return to Gluteal Injection phase), then this visit will be assigned to the planned visit in the same phase.

## 14.3.4.5. Tolerability of Injections (NRS) in Sub-study

After assigning the phases per Table 24, the NRS assessments will be slotted to analysis visits per Table D.

| Table D Assessment Window 1 | for | NRS | Data |
|-----------------------------|-----|-----|------|
|-----------------------------|-----|-----|------|

| Phase | Assessment Window | Visit |
|---|---|---|
| Sub-study | Q4W: post-dose and on the Week -4 injection date | Sub-study Week -4 |
| Screening | Q4W: (Week -4 injection date+1, Week -4 injection | Sub-study Week -3 |
| | date+14), inclusive | - |
| SC | Post-dose and on the Day 1 injection date | Sub-study Day 1 |
| Injection | (Day 1 injection date+1, Day 1 injection date+14), | Sub-study Week 1 |
| | inclusive | - |
| | Post-dose and on the Week 8 injection date | Sub-study Week 8 |

| Phase | Assessment Window | Visit |
|---|---|---|
| | (Week 8 injection date+1, Week 8 injection date+14), | Sub-study Week 9 |
| | inclusive | |
| Return to | Post-dose and on the Week 12 injection date | Sub-study Week 12 |
| Gluteal | (Week 12 injection date+1, Week 12 injection | Sub-study Week 13 |
| | date+14), inclusive | - |

#### 14.3.5. Assessment Window for PK concentration Data

#### 14.3.5.1. Maintenance/Extension Phase Assessments

For PK concentration data at a nominal withdrawal/unscheduled/LTFU Month1 visits during Maintenance or Extension Phase (after assignment to study phase according to Table 25), the visit will be slotting to the analysis visit per the following steps:

- 1. Identify the 'last nominal PK visit' with the PK assessment performed prior to the visit to be slotted during the same study Phase
- 2. The unscheduled/withdrawal/LTFU Month1 visit will be slotted to the earliest nominal visit from the following:
  - nominal visit corresponding to the next planned pre-dose PK assessment visit (excluding timepoints with storage PK collection in which samples have not been analysed for all participants), that is subsequent to the 'last nominal PK visit' during the same study phase.
  - nominal visit of the next planned injection visit within the study phase occurring on or after the date of the PK assessment.

During the Maintenance or Extension Phase, the planned nominal visits for PK Pre-dose are Week 4b, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 80, 88, 96, 100 for the Q4W arm; and Week 100 (direct to inject group), Week 101 (direct to inject group), Week 104a (direct to inject group), and Week 104b (oral lead-in group) for the Switch Q4W IM group. Planned Injection visits are Week 4, Week 8, continuing every 4 weeks for the Q4W arm and every 4 weeks for the ABC/DTG/3TC arm starting at Week 100 (for direct to inject group) and Week 104b for oral lead-in group.

There will be no slotting for planned nominal visits (i.e., analysis visit =visit).

Example 1: If a participant has the 'last nominal PK visit' at Week 24 and then withdraws (around Week 28) with a Maintenance Phase PK assessment labelled as 'LTFU Month 1' Phase, this assessment will be slotted to the subsequent planned PK assessment visit of Week 28.

Example 2: If a participant has the 'last nominal PK visit' at Week 60 and then withdraws (around Week 88, with last injection at W84) with a Maintenance Phase PK assessment labelled as 'LTFU Month 1', then this assessment will be slotted the subsequent planned injection visit of Week 88 (next injection visit).

## 14.3.5.2. Long-Term Follow-up Phase Assessments:

PK concentration data at nominal visits other than LTFU MONTH 1/LTFU MONTH 3/LTFU MONTH 6/LTFU MONTH 9/LTFU MONTH 12/LIVER EVENT which have been assigned to the Long-Term Follow-up phase (according to according to Table 27) will be slotting to analysis visits per the following steps:

- Identify the 'last nominal PK visit' with the PK assessment performed prior to the visit to be slotted during the LTFU phase;
- The unscheduled/withdrawal visit will be slotted to the nominal visit corresponding to the next planned LTFU PK assessment visit that is subsequent to the 'last nominal PK visit' during the LTFU phase.

There will be no slotting for planned PK nominal visits (i.e., analysis visit =visit): LTFU Month 1, LTFU Month 3, LTFU Month 6, LTFU Month 9 and LTFU Month 12.

### 14.3.5.3. Sub-study Assessments

PK concentration plots based on Sub-Study Day as appropriate for each phase where concentration data is collected. Unscheduled sub-study assessments will not be slotted to any analysis visit, however, will be displayed based on Sub-Study Day in individual PK plots. There will be no slotting for planned nominal visits (i.e., analysis visit=visit). Unscheduled assessments will not be summarized outside of individual plots, however, will be listed.

## 14.3.6. Multiple assessments within an Analysis Window

If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

For data other than health outcome/PK concentration:

- the assessment closest to the window target Study Day.
- if there are multiple assessments equidistant from the target Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean.

NRS questionnaire health outcomes assessments:

- the assessment closest to the window target Study Day will be used.
- if there are multiple assessments equidistant from the target Day, then the earliest assessment will be used.

Other health outcome assessments (i.e., apart from NRS) and PK concentration data:

- if there are multiple assessments assigned to the same analysis visit, the assessment from the original planned nominal visit will be used for summary statistics.
- if there are multiple assessments assigned to the same analysis visit and none originate from a planned nominal visit (e.g., two unscheduled/withdrawal nominal visits), then
  - a. the assessment closest to the window target Study Day will be used;

b. if there are multiple assessments equidistant from the target Study Day, then the earliest assessment will be used.

Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, all applicable assessments, irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g., snapshot algorithm or LOCF).

## 14.4. Appendix 4: Study Phases and Treatment State

## 14.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the Treatment Start Date defined in Section 14.6.1.

AEs will be assigned to study Phases as defined in Table 24. For example, adverse events prior to start of Extension Phase IP/LTFU ART will be assigned to the Maintenance Phase.

Laboratory data (efficacy, safety, and virology), HIV associated/ AIDS-defining conditions, health outcomes assessments, vital signs, PK, and ECGs will be assigned to study phases as defined as in Table 25. For example, assessments/events occurring up to and including start of extension phase IP/LTFU ART will be assigned to the Maintenance Phase.

Assessments/events are assigned to study phases sequentially, starting from the top of each table, except for the assessments/events occurring after returning to Extension phase from the sub-study participation.

Table 24 Assignment of Study Phases for AEs

| Study Phase | Date range |
|---|---|
| Screen | Date < Induction Treatment Start Date |
| Induction | For participants continuing into Maintenance Phase: |
| | Induction Treatment Start Date ≤ Date < Maintenance Treatment Start Date |
| | For participants not continuing into Maintenance Phase: |
| | Date ≥Induction Treatment Start Date |
| Maintenance | DTG/ABC/3TC Arm: For participants continuing into Extension Phase: Maintenance Treatment Start Date ≤ Date < min (Start Date of Extension Phase with Oral lead-in of CAB + RPV, Date of first CAB/RPV injection) |
| | For participants not continuing into Extension Phase: |
| | Date ≥Maintenance Treatment Start Date |

| Study Phase | Date range |
|---|---|
| | Q4W IM Arm: |
| | F |
| | For participants continuing into Extension Phase: |
| | Maintenance Treatment Start Date ≤ <b>Date</b> < Date of Nominal Week 100 Visit |
| | For participants not continuing into Extension Phase: |
| | Maintenance Treatment Start Date ≤ Date < LTFU ART Start Date |

| Study Phase | Date range |
|---|---|
| Extension | For participants continuing into the Extension Phase and not entering |
| | the Sub-study: |
| | - Participants continuing into LTFU Phase: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W: |
| | min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) ≤ <b>Date</b> < LTFU ART Start Date |
| | - Participants continuing maintenance Q4W into Extension Phase: |
| | Date of Nominal Week 100 Visit ≤ <b>Date</b> < LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and |
| | did not withdraw the study for safety related reasons: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W |
| | IM: |
| | Min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) ≤ Date < Date of end of study +35 days |
| | - Participants continuing maintenance Q4W IM into Extension Phase: |
| | Date of Nominal Week 100 Visit ≤ <b>Date</b> < Date of end of study +35 days |
| | For participants continuing into the Extension Phase autoring the Sub |
| | For participants continuing into the Extension Phase, entering the Sub- |
| | study but not returning to the Extension Phase: - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W |
| | IM: |
| | Min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) ≤ <b>Date</b> < Date of First Sub-study Record |
| | - Participants continuing maintenance Q4W IM into Extension Phase: |
| | Date of Nominal Week 100 Visit ≤ <b>Date</b> < Date of First Sub-study Record |
| | Date of Horimal Wook 100 Visit = Date of First out study Notoria |
| | For participants continuing into the Extension Phase, entering the Sub- |
| | study and returning to the Extension Phase: |
| | - Before the sub-study: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W |
| | IM: |
| | Min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) ≤ Date < Date of First Sub-study Record |
| | - Participants continuing maintenance Q4W IM into Extension Phase: |
| | Date of Nominal Week 100 Visit ≤ Date < Date of First Sub-study Record |
| | After the sub-study: |
| | - Participants continuing into LTFU Phase after return to extension |
| | phase: |
| | End of sub-study date ≤ <b>Date</b> < LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and |
| | did not withdraw the study for safety related reasons: |
| | End of sub-study date ≤ <b>Date</b> < Date of end of study +35 days |

| Study Phase | Date range |
|---|---|
| Sub-study | For participants entering the sub-study and not receiving any SC |
| Screening | injection: |
| | If participants continued into Extension Phase after the sub-study, then |
| | Date of First sub-study record ≤ Date ≤ End of Sub-study Date |
| | For participants entering the sub-study and receiving SC injection(s): |
| | Date of First sub-study record ≤ Date < Date of First SC Injection |
| SC Injection | For participants continuing into Return to Gluteal Injection Phase: |
| | Date of First SC Injection ≤ Date < Date of Nominal Sub-study Week 12 Visit |
| | For participants not continuing into Return to Gluteal Injection Phase: |
| | - Participants continued into Extension Phase after the sub-study: |
| | Date of First SC Injection ≤ Date ≤ End of Sub-study Date |
| | - Participants continuing into LTFU Phase after the sub-study: |
| | Date of First SC Injection ≤ Date < LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and |
| | did not withdraw the study for safety related reasons: |
| | Date of First SC Injection ≤ Date ≤ End of Sub-study Date +35 days |
| Return to | For participants continuing into Extension Phase after the sub-study: |
| Gluteal | Date of Nominal Sub-study Week 12 Visit ≤ Date ≤ End of Sub-study Date |
| Injection | For participants not continuing into Extension Phase after the sub- |
| | study: |
| | - Participants continuing into LTFU Phase after the sub-study: |
| | Date of Nominal Sub-study Week 12 Visit ≤ Date < LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and |
| | did not withdraw the study for safety related reasons: |
| | Date of Nominal Sub-study Week 12 Visit ≤ Date ≤ End of Sub-study Date |
| | +35 days |

- Date = AE Start date
- Maintenance Treatment Start Date: refer to Treatment Start Date in Section 14.6.1
- End of Sub-study Date and nominal Week 12 Visit Date are defined in Section 14.6.1.

Table 25 Assignment of Study Phases for Lab assessments, ECG, Vital Signs, PK, Health Outcomes, PDs, and HIV associated/AIDS-defining conditions

| Study Phase | Date range |
|---|---|
| Screen | Date ≤ Induction Treatment Start Date |
| Induction | For participants continuing into Maintenance Phase: |
| | Induction Treatment Start Date < Date ≤ Maintenance Treatment Start Date |
| | induction freatment otal bate - bate - maintenance freatment otal bate |
| | For participants not continuing into Maintenance Phase: |
| | Date > Induction Treatment Start Date |

| Study Phase | Date range |
|---|---|
| Maintenance | DTG/ABC/3TC Arm: |
| | For participants continuing into Extension Phase: Maintenance Treatment Start Date < Date ≤ min (Start Date of Extension Phase Oral lead in of CAB + RPV, Date of first CAB/RPV injection) (expected to be nominal Week 100) |
| | For participants <u>not</u> continuing into Extension Phase: Date >Maintenance Treatment Start Date |
| | Q4W IM Arm: |
| | For participants continuing into Extension Phase: Maintenance Treatment Start Date < Date ≤ Date of Nominal Week 100 visit |
| | For participants <u>not</u> continuing into Extension Phase: Maintenance Treatment Start Date < Date ≤ LTFU ART Start Date |

| Study Phase | Date range |
|---|---|
| Extension | For participants continuing into the Extension Phase and not entering |
| Extension | the Sub-study: |
| | - Participants continuing into LTFU Phase: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W: |
| | min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) < <b>Date</b> ≤ LTFU ART Start Date |
| | - Participants continuing maintenance Q4W into Extension Phase: |
| | Date of Nominal Week 100 Visit < <b>Date</b> ≤ LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and |
| | did not withdraw the study for safety related reasons: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W |
| | IM: |
| | Min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) < <b>Date</b> ≤ Date of end of study +35 days |
| | - Participants continuing maintenance Q4W IM into Extension Phase: |
| | Date of Nominal Week 100 Visit < <b>Date</b> ≤ Date of end of study +35 days |
| | Date of Hellimia Freek 100 Field Date = Date of ond of olday of days |
| | For participants continuing into the Extension Phase, entering the Sub- |
| | study but not returning to the Extension Phase: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W |
| | IM: |
| | Min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) < Date ≤ Date of First Sub-study Record |
| | - Participants continuing maintenance Q4W IM into Extension Phase: |
| | Date of Nominal Week 100 Visit < <b>Date</b> ≤ Date of First Sub-study Record |
| | , and the second |
| | For participants continuing into the Extension Phase, entering the Sub- |
| | study and returning to the Extension Phase: |
| | - Before the sub-study: |
| | - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W |
| | IM: |
| | Min (Start Date of Extension Phase Oral lead-in of CAB + RPV, Date of first |
| | CAB/RPV injection) < <b>Date</b> ≤ Date of First Sub-study Record |
| | - Participants continuing maintenance Q4W IM into Extension Phase: |
| | Date of Nominal Week 100 Visit < <b>Date</b> ≤ Date of First Sub-study Record |
| | After the sub-study: |
| | - Participants continuing into LTFU Phase after return to extension |
| | phase: |
| | End of sub-study date < Date ≤ LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and |
| | did not withdraw the study for safety related reasons: |
| | End of sub-study date < <b>Date</b> ≤ Date of end of study +35 days |
| L | l |

| Study Phase | Date range |
|---|---|
| Sub-study<br>Screening | For participants entering the sub-study and not receiving any SC injection: If participants continued into Extension Phase after the sub-study, then Date of First sub-study record < Date ≤ End of Sub-study Date For participants entering the sub-study and receiving SC injection(s): Date of First sub-study record < Date ≤ Date of First SC Injection |
| SC Injection | For participants continuing into Return to Gluteal Injection Phase: Date of First SC Injection < Date ≤ Date of Nominal Sub-study Week 12 Visit For participants not continuing into Return to Gluteal Injection Phase: - Participants continued into Extension Phase after the sub-study: Date of First SC Injection < Date ≤ End of Sub-study Date - Participants continuing into LTFU Phase after the sub-study: Date of First SC Injection < Date LTFU ART Start Date - Participants transitioning to marketed product/alternative HAART and did not withdraw the study for safety related reasons: Date of First SC Injection < Date ≤ Date of end of Sub-study +35 days |
| Return to<br>Gluteal<br>Injection | For participants continuing into Extension Phase after the sub-study: Date of Nominal Sub-study Week 12 Visit < Date ≤ End of Sub-study Date For participants continuing into LTFU Phase after the sub-study: Date of Nominal Sub-Study Week 12 Visit < Date ≤ LTFU ART Start Date For Participants transitioning to marketed product/alternative HAART and did not withdraw the study for safety related reasons: Date of Nominal Sub-Study Week 12 Visit < Date ≤ Date of end of Sub-study +35 days |

- Date = start or assessment date
- Maintenance Treatment Start Date: refer to Treatment Start Date in Section 14.6.1
- End of Sub-study Date and nominal Week 12 Visit Date are defined in Section 14.6.1.
- The post-dose assessments (e.g., 2-hour post-dose PK and NRS) taken on the date of first SC injection will be assigned SC Injection Phase, instead of Sub-study Screening Phase.
- The post-dose assessment (e.g., NRS) taken on the date of Sub-study Week 12 injection will be assigned Return to Gluteal Injection Phase, instead of SC Injection Phase.

Table 26 Assignment of Study Phases for Concomitant medication/ART

| Concomitant during: | Date range |
|---------------------|---------------------------------------------------|
| Prior | Medication Taken < Induction Treatment Start Date |

| Concomitant during: | Date range |
|---|---|
| Induction | For participants continuing into Maintenance Phase: |
| | Induction Treatment Start Date ≤ <b>Medication Taken</b> < Maintenance Treatment Start Date |
| | For participants not continuing into Maintenance Phase: |
| | <b>Medication Taken</b> ≥ Induction Treatment Start Date |
| | Note: ART stopped on the start date of Induction Treatment will be considered Prior ART and will not be considered concomitant during the Induction Phase. |
| Maintenance | DTG/ABC/3TC Arm: For participants continuing into Extension Phase: Maintenance Treatment Start Date ≤ Medication Taken < Start Date of Extension Phase CAB + RPV (expected to be WK100) |
| | For participants not continuing into Extension Phase: |
| | <b>Medication Taken</b> ≥ Maintenance Treatment Start Date |
| | Note: ART stopped on the start date of Maintenance Treatment will be considered concomitant during the Induction Phase and will not be considered concomitant during the Maintenance Phase. |
| | Q4W IM Arms: |
| | For participants continuing into Extension Phase: Maintenance Treatment Start Date ≤ Medication Taken < Date of Nominal Week 100 visit |
| | For participants <u>not</u> continuing into Extension Phase: Maintenance Treatment Start Date ≤ Medication Taken < LTFU ART Start Date |
| | Note: ART stopped on the start date of Maintenance Treatment will be considered concomitant during the Induction Phase and will not be considered concomitant during the Maintenance Phase. |

#### Extension

For Participants continuing into the Extension Phase and not entering the Sub-study:

- Participants continuing into LTFU Phase:
  - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W IM:

Start Date of Extension Phase CAB +  $RPV^{[a]} \le Medication Taken < LTFU ART Start Date$ 

- Participants continuing maintenance Q4W IM into Extension Phase:

Date of Nominal Week 100 Visit<sup>[b]</sup> ≤ **Medication Taken** < LTFU ART Start Date

- Participants transitioning to marketed product/alternative HAART and did not withdraw the study for safety related reasons:
  - Participants Switching from Maintenance DTG/ACB/3TC Arm to Q4W IM:

Start Date of Extension Phase CAB +  $RPV^{[a]} \le Medication Taken < Date of end of study +35 days$ 

-Participants continuing maintenance Q4W IM into Extension Phase:

Date of Nominal Week 100 Visit<sup>[b]</sup>  $\leq$  **Medication Taken** < Date of end of study +35 days

For participants continuing into the Extension Phase, entering the Sub-study but not returning to the Extension Phase:

- Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W IM:

Start Date of Extension Phase CAB +  $RPV^{[a]} \le Medication Taken < Date of First Sub-study Record$ 

- Participants continuing maintenance Q4W IM into Extension Phase:

Date of Nominal Week 100  $Visit^{[b]} \le$  **Medication Taken** < Date of First Sub-study Record

For participants continuing into the Extension Phase, entering the Sub-study and returning to the Extension Phase:

- Before the sub-study:
  - Participants Switching from Maintenance DTG/ABC/3TC Arm to Q4W IM:

Start Date of Extension Phase CAB +RPV<sup>[a]</sup>  $\leq$  Medication Taken < Date of First Sub-study Record

- Participants continuing maintenance Q4W IM into Extension Phase:

Date of Nominal Week 100  $Visit^{[b]} \le$  **Medication Taken** < Date of First Sub-study Record

## After the sub-study:

| Concomitant during: | Date range |
|---|---|
| , | - Participants continuing into LTFU Phase after return to extension phase: |
| | End of sub-study date <sup>[c]</sup> ≤ Medication Taken < LTFU ART Start Date - Participants transitioning to marketed product/alternative HAART and did not withdraw the study for safety related reasons: End of sub-study date <sup>[c]</sup> ≤ Medication Taken < Date of end of study |
| | +35 days |
| Long-Term Follow-Up | For participants who received at least one CAB and/or RPV Injection: |
| | Medication Taken ≥ LTFU ART Start Date |
| Sub-study Screening | For participants entering the sub-study and not receiving any SC injection: |
| | If participants continued into Extension Phase after the sub-study, then Date of First sub-study record <sup>[d]</sup> ≤ <b>Medication Start Date</b> < End of Substudy Date |
| | For participants entering the sub-study and receiving SC injection(s): |
| | Date of First sub-study record <sup>[d]</sup> ≤ <b>Medication Start Date</b> < Date of First SC Injection |
| SC Injection | For participants continuing into Return to Gluteal Injection Phase: Date of First SC Injection <sup>[e]</sup> ≤ Medication Start Date < Date of Nominal Sub-study Week 12 Visit |
| | For participants not continuing into Return to Gluteal Injection Phase: |
| | - Participants continued into Extension Phase after the Sub-study: Date of First SC Injection <sup>[e]</sup> ≤ Medication Start Date < End of Substudy Date |
| | - Participants continuing into LTFU Phase after the sub-study: Date of First SC injection <sup>[e]</sup> ≤ Medication Start Date < LTFU ART Start Date |
| | - Participants transitioning to marketed product/alternative HAART and did not withdraw the study for safety related reasons: Date of First SC Injection <sup>[e]</sup> ≤ Medication Start Date < Date of end of |
| Return to Gluteal | Sub-Study +35 days |
| Injection | For participants continuing into Extension Phase after the substudy: |
| | Date of Nominal Sub-study Week 12 Visit <sup>[f]</sup> ≤ <b>Medication Start Date</b> < End of Sub-study Date |
| | For participants continuing into LTFU Phase after the sub-study: Date of Nominal Sub-study Week 12 Visit <sup>[f]</sup> ≤ Medication Start Date < LTFU ART Start Date |
| | For participants transitioning to marketed product/alternative HAART and did not withdraw the study for safety related reasons: Date of Nominal Sub-study Week 12 Visit <sup>[f]</sup> ≤ Medication Start Date < Date of end of Sub-study +35 days |

- [a] ART stopped on the start date of Extension Phase CAB + RPV will not be assigned to the Extension Phase.
- [b] ART taken stopped on the date of nominal Week 100 visit will be considered concomitant during the Maintenance Phase and will not be considered concomitant during the Extension Phase.
- [c] ART taken stopped on the end of Sub-study date will be considered concomitant during the previous sub-Study Phase and will not be considered concomitant during the Extension Phase.
- [d] ART stopped on the date of first Sub-study record not be assigned to the Sub-study Screening Phase.
- [e] ART stopped on the date of first SC Injection will not be assigned to the SC Injection Phase.
- [f] ART stopped on the date of Nominal Sub-study Week 12 Visit will not be assigned to the Return to Gluteal Injection Phase.

If a partial date for medication/ART is recorded in the eCRF, the following convention will be used to assign the medication:

- if the partial date is a start date, a '01' will be used for missing days and 'Jan' will be used for missing months;
- if the partial date is a stop date, a '28/29/30/31' will be used for the missing day (dependent on the month and year) and 'Dec' will be used for the missing month; for medications recorded separately in the eCRF as prior ART, the earlier of this imputed date or the day before IP start will be used.

The recorded partial date will be displayed in listings.

Table 27 Assignment to Long-Term Follow-Up Phase

| Study Phase | Date range |
|---|---|
| Long-Term | Date > max (Last IM Injection Date, Last Oral Bridging End Date) |
| Follow-Up | |

• Date = Assessment/Start Date

Note that the long-term follow-up Phase and maintenance/extension Phases are not necessarily mutually exclusive and are to be defined with separate Phase variables in the datasets. For example, an Q4W IM participant who has Week 44 injection and withdrawal at Week 48 without receiving Week 48 injection, the "Week 48 withdrawal visit" belongs to both the Maintenance Phase and long-term follow-up Phase.

### 14.4.1.1. Study Periods

Certain displays will be produced for data collected during the oral-lead-in and during the first 52 weeks of the Maintenance Phase, respectively. These period variables are defined in Table 28 and Table 29 and will be reflected in the datasets in separate variables.

Table 28 Assignment of Study Period for AE Data

| Study Period | Date range |
|--------------|------------|
|--------------|------------|
| Maintenance ABC/DTG/3TC Arm: | | | |
|---|---|--|--|
| Phase up to<br>Week 52 | For participants continuing beyond Week 52: Maintenance Treatment Start Date ≤ Date < Date of Study Day 378 (Upper Assessment Window for Week 52) | | |
| | For participants <u>not</u> continuing beyond Week 52: | | |
| | Date ≥ Maintenance Treatment Start Date | | |
| | Q4W IM Arm: | | |
| | For participants continuing beyond Week 52: Maintenance Treatment Start Date ≤ Date < Date of Study Day 378 (Upper Assessment Window for Week 52) | | |
| | For participants <u>not</u> continuing beyond Week 52: Maintenance Treatment Start Date ≤ Date < LTFU ART Start Date | | |
| Maintenance<br>Phase Oral | Q4W IM Arm: | | |
| lead-in | For participants receiving at least one Maintenance Phase Injection: Maintenance Treatment Start Date ≤ Date < Date of First IM injection | | |
| | For participants withdrawing prior to first Maintenance Phase Injection: Date ≥ Maintenance Treatment Start Date | | |
| Extension<br>Phase Oral | Switch Q4W (Oral Lead-In Arm): | | |
| lead-in | For participants receiving at least one Extension Phase Injection:<br>Extension Oral CAB/RPV Start Date ≤ Date < Date of First IM injection | | |
| | For participants withdrawing prior to first Extension Phase Injection: Date ≥ Extension Oral CAB/RPV Start Date | | |

# Table 29 Assignment of Study Period for Lab assessments:

| Period | Date range |
|---|---|
| Maintenance up to Week 52 | ABC/DTG/3TC Arm: |
| [Note: this is derived for | For participants continuing beyond Week 52: |
| LAB assessments only] | Maintenance Treatment Start Date < <b>Date</b> ≤ Date of Study Day 378 (Upper Assessment Window for Week 52) |
| | For participants <u>not</u> continuing beyond Week 52: Date >Maintenance Treatment Start Date |

| | A (14/ 154 A |
|---|---|
| | Q4W IM Arm: |
| | For participants continuing beyond Week 52: Maintenance Treatment Start Date < Date ≤ Date of Study Day 378 (Upper Assessment Window for Week 52) |
| | For participants <u>not</u> continuing beyond Week 52:<br>Maintenance Treatment Start Date < Date ≤ LTFU ART Start Date |
| Maintenance Oral lead-in [Note: this is derived for | Q4W IM Arm: |
| LAB assessments only] | For participants receiving at least one Maintenance Phase Injection: |
| | Maintenance Treatment Start Date < <b>Date</b> ≤ Date of First IM injection |
| | For participants withdrawing prior to first Maintenance Phase Injection: |
| | Date >Maintenance Treatment Start Date |
| Extension Phase Oral lead-in | Switch Q4W (Oral Lead-In) Arm: |
| [Note: this is derived for LAB assessments only] | For participants receiving at least one Extension Phase Injection: |
| | Extension Oral CAB/RPV Start Date < <b>Date</b> ≤ Date of First IM injection |
| | For participants withdrawing prior to first Extension Phase Injection: |
| | Date > Extension Oral CAB/RPV Start Date |

### 14.4.2. Treatment State

Within each treatment study Phase (i.e., Induction, Maintenance and Extension—based on assignment of study Phase described in Section 14.4.1), only those assessments which occur within the ranges shown in Table 30 will be considered 'on-treatment' for the given Phase.

Table 30 Treatment State within Study Phases

| Study Phase <sup>a</sup> | Treatment State | Date Range |
|---|---|---|
| Screen | Pre-treatment | All assessments/events within Phase |
| Induction | On-treatment | Date ≤ Induction Treatment Stop Date + 1 |

| | Post-treatment | Date > Induction Treatment Stop Date + 1 |
|---|---|---|
| Maintenance | On-treatment | ABC/DTG/3TC ART arm: |
| | | Date ≤ Maintenance ART Stop Date + 1 |
| | | IM Q4W arm: |
| | | Date ≤ max (Date of Last Q4W IM Dose + 35,<br>Last Oral Dose Date + 1) |
| | Post-treatment | ABC/DTG/3TC arm: |
| | | Date > ABC/DTG/3TC Stop Date + 1 |
| | | IM Q4W arm: |
| | | Date > max (Date of Last Q4W IM Dose + 35,<br>Last Oral Dose Date + 1) |
| Extension | On-treatment | Date ≤ max (Date of Last Q4W IM Dose + 35,<br>Last Oral Dose Date + 1) |
| | Post-treatment | Date > Date of Last Q4W IM Dose + 35, Last<br>Oral Dose Date + 1) |
| Long-Term<br>Follow-up | On-treatment | Date ≤ min (LTFU ART start date, max (Last Injection Date + 35, Last Oral Dose Date + 1)) |
| | Post-treatment | Date > min (LTFU ART start date, max (Last Injection Date + 35, Last Oral Dose Date + 1)) |

Note1: Treatment State is determined after data has been assigned to the study Phases as defined in Section 14.4.1

Note2: Last Q4W IM / last oral dose / Induction Treatment stop date/Maintenance ART Stop Date is only applied to participants who permanently discontinue from study treatment Note3: Date = Assessment/Start Date.

 For Sub-study Screening, SC Injection and Return to Gluteal Injection phases, the same ontreatment and post-treatment algorithms as those in Extension Phase will be applied.

### 14.4.2.1. Treatment States for AE Data

For adverse events, partial AE start date will use imputation as described in Section 14.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment at Maintenance Phase unless an end date for the AE is provided which is before start of study treatment at Maintenance Phase; in such a case the AE is assigned as Pre-treatment.

Within each treatment study Phase, only those AE with onset date within the ranges shown in Table 30 will be considered 'on-treatment' for the given Phase. The onset date will be derived based on Table 31.

Table 31 AE onset date, AE duration and relation to study treatment

| | Definition |
|---|---|
| Onset date/study day | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date |
| Since 1st Dose<br>of each study<br>Phase (Days) | If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| Duration<br>(Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

 Onset date/study day will be derived for each study Phase, respectively (refer to Section 14.6.1)

### 14.4.3. Combining Treatment Phases and States

On-treatment and Post-treatment assessments and events will be classified as occurring during the Induction, Maintenance Phase, Extension, or Long-term follow up Phase.

# 14.5. Appendix 5: Data Display Standards & Handling Conventions

### 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently set 1. | upported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Area | \ARPROD\GSK1265744\mid201584\primary_01 (W48 analysis) \ARPROD\GSK1265744\mid201584\primary_07 (W96 analysis) \ARPROD\GSK1265744\mid201584\primary_09 (Day 1 Japan PK analysis) \ARPROD\GSK1265744\mid201584\primary_17 (Week 124 analysis) |
| QC Spreadsheet | : \ARWORK\GSK1265744\mid201584\documents\qc\ |
| <b>Analysis Datasets</b> | Analysis Datasets |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 &amp;<br/>AdaM IG Version 1.0).</li> </ul> | |
| <ul> <li>For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will<br/>be implemented for conversion from SI to SDTM.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for every reporting effort described in the RAP. | |

### 14.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

• Reporting for tables, figures and formal statistical analyses:

- Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject listings displays.

### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 14.3.2.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points
  and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 14.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| Descriptive Summary | Refer to IDSL PK Display Standards. |
| Statistics, Graphical Displays and Listings | Refer to IDSL Statistical Principle 6.06.1. |
| | NQ concentration values will be assigned a numeric value equal to the low limit of quantification (LLQ) (Refer to GUI_51487 for further details) for descriptive summary statistics/analysis and summarized graphical displays only. |
| | For Japan Day 1 PK concentrations, refer to the standard operating procedure, SOP-CPK-0001 and R&D Guideline: Non-Compartmental Analysis of Pharmacokinetic Data, GUI_51487 (3.0), for more information regarding the handling of plasma concentrations below the assay's lower limit of quantification (LLQ). Geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be reported. $CV_b (\%) = \sqrt{(exp(SD^2) - 1) * 100}, SD = SD \text{ of log transformed data}$ |
| | $\circ$ CV <sub>b</sub> (%) = $\vee$ (exp(SD <sup>2</sup> ) - 1) * 100, SD = SD of log transformed data) |

### 14.6. Appendix 6: Derived and Transformed Data

#### 14.6.1. General

### **Multiple Measurements at One Time Point**

- If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:
  - the assessment closest to the window target Study Day;
  - if there are multiple assessments equidistant from the target Study Day, then for continuous variables the mean of these values will be used and for categorical variables the worse assessment. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean
- Assessments not chosen for use in summary statistics by this algorithm will still appear in
  the associated listings. Also, such valid assessments will be used when determining values
  of potential clinical concern for the 'any time On-treatment' time point, and for any algorithm
  that has specific rules for which observation to use (e.g., Snapshot).

#### **Treatment Start Date**

Treatment start date is defined by Phase as follows:

#### Induction Phase

Start date of DTG regimen entered onto the Induction Phase IP exposure CRF

#### Maintenance Phase

- For participants randomised to Q4W IM, maintenance treatment start date is the date of oral lead-in of CAB+RPV entered onto the Maintenance Phase IP exposure CRF
- For participants randomised to ABC/DTG/3TC, maintenance treatment start is DTG regimen start date entered onto the Maintenance Phase IP exposure CRF

#### **Extension Phase**

 For participants randomised to Q4W IM, extension treatment start date is the date of Nominal Week 100 injection date.

For participants randomised to ABC/DTG/3TC, extension treatment start date is the start date of oral lead-in of CAB+RPV entered onto the Extension Phase IP exposure CRF.

#### SC Sub-Study

- For participants enrolled in the SC sub-study, treatment start date is the date of their screening injection. For purposes of exposure calculations, the date of the first SC injection will be used.
- For participants who received Sub-study Week 12 injection, nominal Sub-study Week 12 visit date is defined by the Sub-study Week 12 injection date. Otherwise, nominal Sub-study Week 12 visit date is defined by the date of latest Sub-study Week 12 assessment.
- For participants who continued into Return to Gluteal Injection Phase however missed Sub-study Week 12 visit, nominal Sub-study Week 12 visit date is defined by the end of SC Injection Phase date (i.e., date for the SC Injection Phase conclusion record in the SDTM DS domain) for the analysis purpose.

For sub-study screen failures, the end of sub-study date is defined by the date they
failed to meet the inclusion/exclusion criteria in the sub-study. For other sub-study
participants, the end of sub-study date is defined by the date of completion or
withdrawal available in the sub-study conclusion eCRF form or the Week 20 visit date,
whichever comes first.

### **Induction Phase Study Day**

The Induction Phase Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the initial start date of DTG in the Induction Phase as follows:

if date of event ≥ start date of Induction Phase DTG, then

Induction Phase Study Day = date of event - start date of Induction phase IP + 1

if date of event < start date of Induction Phase DTG, then

Induction Phase Study Day = date of event - start date of Induction phase IP

if date of event > start date of Maintenance Phase DTG, then

Induction Phase Study Day will not be derived (i.e., will be set to missing).

Note that the initial start date of Induction Phase DTG is considered to be on Induction Phase Study Day 1 and the day before this is Induction Phase Study Day -1; i.e., there is no Induction Phase Study Day 0.

### Study Day

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the start date of study treatment on Maintenance Phase as follows:

if date of event ≥ start date of study treatment, then

• Study Day = Date of Event – Start Date of Maintenance Phase IP + 1

if date of event < start date of study treatment, then

Study Day = Date of Event – Start Date of Maintenance Phase IP

Note that the start date of study treatment on Maintenance Phase is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Extension Phase Study Day

The Extension Phase Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the initial start date of Extension Phase IP as follows:

if date of event ≥ start date of extension Phase IP, then

Extension Phase Study Day = date of event - start date of Extension phase IP + 1

if date of event < start date of Extension Phase IP, then

Extension Phase Study Day = date of event - start date of Extension phase IP

Note that the start date of Extension Phase IP is considered to be on Extension Phase Study Day 1 and the day before this is Extension Phase Study Day -1; i.e., there is no Extension Phase Study Day 0.

### Long-Term Follow Up Study Day

The Long-Term Follow Up (LTFU) Study Day of an event (e.g., lab assessment, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the end of IP treatment [i.e., max (Last IM Injection Date, Last Oral Bridging End Date)]

as follows:

If the onset of event falls in Long-term Follow up Phase, then

• LTFU Study Day = date of event - end date of IP

### **Sub-study Phase Study Day**

Each phase Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the reference date for each phase of the sub-study as follows:

if date of event ≥ reference date, then

Study Day=date of event - reference date + 1

if date of event < reference date, then

Study Day=date of event - reference date

The reference dates for each Phase are as follows:

- SC Injection Phase: Date of first SC injection
- Return to Gluteal Injection Phase: Date of the nominal sub-study Week 12 visit date

The SC injection date will serve as the reference date for the overall study day.

#### Study treatment/drugs

 Refers to either investigation product (CAB+RPV oral /CAB+ RPV LA) or ABC/DTG/3TC or DTG plus alternate NRTIs.

### 14.6.2. Study Population

### **Demographics**

### Age

- Age, in whole years, will be calculated with respect to the participant's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied.
   Consequently, the age of the participant will not be calculated and will remain missing.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / Height (m)<sup>2</sup>, using Height collected at Day 1.

### **Hepatitis B Status**

A participant will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen (i.e., "REACTIVE") and/or detectable HBV DNA ("HBV DNA DETECTED" or HBV DNA ≥ 116 copies/mL, with "HBV DNA DETECTED" taking precedence over HBV DNA reported as <116 copies/mL). If DNA result is available, then this will be used to qualify as positive or negative; otherwise, Hepatitis B status will be determined using the surface antigen result.</li>

### **Hepatitis C Status**

- Hepatitis C status will be determined using antibody (IgM or IgG) and/or hepatitis C virus (HCV) RNA assessments performed during screening or during the conduct of the study.
- If both antibody and virus RNA assessments are available, then the latter will take
  precedence and positive/negative status will be based on whether HCV RNA is ≥15
  IU/mL. In the absence of an HBV RNA result, Hepatitis C antibody of "REACTIVE" or
  "BORDERLINE" will qualify as Hep C positive.

### **Lipid-modifying Agents**

- The following ATC codes correspond to lipid-modifying agents:
  - ATC Level 2: C10
  - ATC Level 3: C10A, C10B (if Level 2 is not available)
  - ATC Level 4: C10AA, C10AB, C10AC, C10AD, C10AX, C10BA, C10BX (if level 2, 3 are not available)
- Participants are considered to have used a lipid-modifying agent at baseline if they are taking the medication at the time of their baseline lipid testing date.
- Participants are also considered to have used a lipid-modifying agent at baseline if they stopped their lipid modifying medication within 12 weeks prior to their baseline lipid testing date.

#### Framingham Risk Equation

• The predicted probability,  $\hat{p}$ , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino, 2008] is

### for females:

 $\hat{p}_F = 1 - S_0(t) \exp\{2.32888 \times \log(\text{age}) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBPu) + 2.82263 \times \log(SBPt) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 1.76157 \times \log(SBPu) + 1.20904 \times \log(TC) + 1.2090$ 

### **Demographics**

$$0.52873 \times I_s + 0.69154 \times I_d - 26.1931$$

#### for males:

$$\hat{p}_{M} = 1 - S_{0}(t) \exp\{3.06117 \times \log(\text{age}) + 1.12370 \times \log(\text{TC}) - 0.93263 \times \log(\text{HDL}) + 1.93303 \times \log(\text{SBPu}) + 1.99881 \times \log(\text{SBPt}) + 1.99881 \times \log(\text{SBPt})$$

$$0.65451 \times I_s + 0.57367 \times I_d - 23.9802$$

#### where

$$S_0(t) = \begin{cases} 0.95012, \text{ females} \\ 0.88936, \text{ males} \end{cases}$$

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL),

SBPu = systolic blood pressure (mmHg) if participant is not treated for high blood pressure (note that if a participant is treated for high blood pressure, then log(SBPu) = 0)
SBPt = systolic blood pressure (mmHg) if participant is treated for high blood pressure (note that if a participant is not treated for high blood pressure, then log(SBPt) = 0)

$$I_{s} = \begin{cases} 1, \ current \ smo \ ker \\ 0, \ otherwise \end{cases}$$
 
$$I_{d} = \begin{cases} 1, \ diabetic \\ 0, \ otherwise \end{cases}$$

- A participant will be considered as treated for high blood pressure if during screening it has specified that is suffering from hypertension.
- A participant is classified as diabetic if current or past is indicated in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or if baseline fasting glucose ≥7.00 mmol/L (126 mg/dL).
- Smoking status is collected in the eCRF at Induction Baseline (Week -20). A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used tobacco products within the previous 6 months.
- This calculation will not be performed for participants who have indicated current or past
  myocardial infarction conditions on the eCRF. These participants will not be included in
  summary statistics of risk but will be counted in the highest category of risk in the
  summary by category.

 Exposure to CAB+RPV (oral lead-in), CAB LA+RPV LA, ABC/DTG/3TC (or DTG if alternate NRTI is used) will be calculated from the IP eCRF pages.

| alternate Wiff is used) will be calculated from the in contributes. | |
|---|---|
| Maintenance Phase: Q4W IM arm | |
| Exposure to CAB + RPV (oral lead-in) = | Oral lead-in CAB/RPV Stop Date – Oral lead-in CAB/RPV Start Date +1 |
| Exposure to CAB LA + RPV LA = | Number of IP injections received during Maintenance Phase (up to but not including Injections administered at Week 100) |
| Overall Exposure to IP = | min [Date of latest Maintenance Phase visit up to and including Week 100, max (Date of last IP injection +35 [a], Date of last oral CAB/RPV [a])] – Oral lead-in CAB/RPV Start Date +1 |
| Maintenance + Extension Phase: Q4V | V IM arm |
| Exposure to CAB LA + RPV LA = | Number of IP injections received during Maintenance Phase + Extension Phase |
| Overall Exposure to IP = | min [Min(Date of Last Study Contact, Long Term Follow Up HAART Start Date), max (Date of last IP injection +35 [a], Date of last oral CAB/RPV [a])] – Oral lead-in CAB/RPV Start Date +1 |
| a. Last Q4W IM / last oral dose is only applied | a. Last Q4W IM / last oral dose is only applied to participants who permanently discontinue from study |
| Maintenance Phase: ABC/DTG/3TC a | rm |
| Exposure = Min (Date of latest Maintenance Phase visit up to and including Week 100, Maintenance Phase Treatment Stop Date, Date of Maintenance Phase Discontinuation) – Maintenance Treatment Start Date + 1 | |
| Extension Phase: Switch Q4W IM gro | up (Extension Switch Population only) |
| Exposure to CAB + RPV (oral lead-in) = | min (Date of Last Study Contact, Long Term Follow Up HAART Start Date, Oral lead-in CAB/RPV Stop Date) – Oral lead-in CAB/RPV Start Date +1 |
| Exposure to CAB LA + RPV LA = | Number of IP injections received during Extension Phase |
| Overall Exposure to CAB + RPV = | min [min(Date of Last Study Contact, Long Term Follow Up HAART Start Date), max (Date of last IP injection +35 [a], Date of last oral CAB/RPV [a]) ] – min(Oral lead-in CAB/RPV Start Date, Date of First IP Injection) +1 |
| a. Last Q4W IM / last oral dose is only applied to participants who permanently discontinue from study | |
| E | |

 Duration of dosing in subject years will be calculated as the sum of subject duration of dosing in days (across all participants)/365.25

 Participants who were randomised to CAB LA+RPV LA but did not report an IP start date will be categorised as having zero days of exposure.

### SC Sub-study

- For SC Injection Phase
  - Exposure to CAB LA + RPV LA = Number of IP injection visits received during SC Injection Phase. Note that the planned Sub-study Week 12 injections belong to Return to Gluteal Injection Phase.
  - The SOC or CAB+RPV oral bridging are not allowed in this phase.
  - Overall exposure to IP:

min [Date of Latest SC Injection Phase Visit up to the Nominal Sub-study Week 12 Visit Date, max (Date of Last Injection + 35<sup>[a]</sup>, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] – Date of First SC Injection) + 1

Note that the Nominal Sub-study Week 12 visit date is defined in Section 14.6.1.

- Overall exposure to IP = Overall exposure to Study Treatment.
- For SC Injection + Return to Gluteal Injection Phase
  - Exposure to CAB LA + RPV LA = Number of IP injection visits received during SC Injection or Return to Gluteal Injection Phase. Note that the injections received on the date of Sub-study Week 20 visit belong to the Extension Phase in main study.
  - The SOC or CAB+RPV oral bridging are not allowed in these two phases.
  - Overall exposure to IP: min [End of Sub-study Date, max (Date of Last Injection + 35<sup>[a]</sup>, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] – Date of First SC Injection) + 1 Note that the End of Sub-study Date is defined in Section 14.6.1.
  - Overall exposure to IP = Overall exposure to Study Treatment.

[a] Last Injection/ last oral dose is only applied to participants who permanently discontinue the study.

#### Adherence to CAB/RPV Injection Schedule

For participants in the randomized Q4W arm, Timeliness of Injections Relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from Week 4b".

For participants in the Switch Q4W Oral Lead-in group, Timeliness of Injections Relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from Week 104b".

For participants in the Switch Q4W Direct to Inject group, timeliness of Injections Relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from Week 100".

For participants in the Sub-Study, timeliness of Injections Relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from Sub-study Week -4".

Each injection visit is counted only once. Individual CAB and RPV injections administered at the same visit are not counted twice. "Extra" unscheduled injections are excluded from all derivations. For example, if during a scheduled visit a participant receives 1 ml of injection instead of 2 ml due to a dosing error but returns one week later for the remaining 1 ml injection, then the additional visit is excluded. If a participant receives an extra injection at an unscheduled visit by mistake, this visit will also be excluded.

The categories of Timeliness of Injections Relative to Date of Projected Dosing Visits for summary are listed below:

< -14 days

-14 to -8 days

-7 to -4 days

-3 to -2 days -1

0 day

1

2 to 3 days

4 to 7 days

8 to 14 days

>14 days

Missed Injection without Oral Bridging

Missed Injection with Oral Bridging

#### **Corrected QTC**

When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

If RR interval (in msec) is provided, then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{RR/1000}} \qquad \qquad QTcF = \frac{QT}{\sqrt[3]{RR/1000}}$$

where uncorrected QT interval is also measured in msec.

If RR interval is not provided directly and one of QTcB or QTcF has been entered, then RR interval can be obtained from the above formulas and used to calculate the other correction method value; i.e.,

$$QTcB = \sqrt{\frac{QTcF^3}{QT}} \qquad \qquad QTcF = \sqrt[3]{QT \cdot QTcB^2}$$

### 14.6.3. Safety

### Adverse Events- DAIDS Grading

 Clinical adverse events will be graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, November 2014, as specified in the protocol Appendix 12.2.

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

### Estimate of Glomerular Filtration Rate (GFR) (Levey, 2012)

 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey, 2012]. be used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m2, as follows:

$$GFR = 141 \times \min \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{\alpha} \times \max \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{-1.209} \times 0.993^{Age} \times [1.018 \text{ if Female}] \times [1.159 \text{ if Black}]$$

where age (in years) is at time of assessment,  $\kappa$  = 0.7 if female or 0.9 if male,  $\alpha$  = -0.329 if female and -0.411 if male, min() indicates the minimum of CRT/ $\kappa$  or 1, max() indicates the maximum of CRT/ $\kappa$  or 1, and CRTmg/dL is serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRTmg/dL =0.0113x CRT $\mu$ mol/L.

• The CKD-EPI GFR will also be calculated using Cystatin C, as follows

133 X min(Scys/0.8, 1) -0.499 X max (Scys/0.8, 1)-1.328 X 0.996 Age X[0.932 if female]

Where Scys is serum cystatin C mg/Liter, min indicates the minimum of Scr/0.8 or 1, and max indicates the maximum of Scys/0.8 or 1

- Lab Toxicities DAIDS Grading based on Version 2.0, November 2014, as specified in the protocol of Appendix 12.2
- Toxicities will be based on the Division of AIDS (DAIDS) grading system, Version 2.0, November 2014, as specified in the protocol of Appendix 12.2. Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint for those ≥Grade 1 | Above Midpoint for those ≥Grade 1 |
|---|---|---|
| Fasted glucose | Hypoglycemia | Hyperglycemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

### National Cholesterol Education Program (NCEP) Lipid Categories

 In addition to DAIDS toxicity grades (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001]

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |

| | 5.18 to <6.21 | 200 to <240 | Borderline High |
|-----------------|---------------|-------------|--------------------|
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

### Total Cholesterol / HDL Cholesterol Ratio

When both total cholesterol and HDL cholesterol results are available from the same date
for a participant, then the ratio will be calculated by dividing the total cholesterol result by the
HDL cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------|--------------|
| Total Cholesterol | < 3.5 |
| / HDL Ratio | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥ 5 |

| D | ا ـ ـ ـ ـ ـ ا | L | £ 1: | : |
|---------|---------------|-------|--------|------|
| Percent | tage c | nange | tor II | pias |

| The percentage | change from | Maintenance | Raseline | (Day 1 | ) is calculated as: |
|---|---|---|---|---|---|

| % Change from Maintenance BL | Value at Week 48/Week 96 – Maintenance BL | X 100 % |
|---|---|---|
| = | value | |
| _ | Maintenance BL value | <del>_</del> |

The percentage change from Extension Baseline (Week 100) is calculated as:

| % Change from Maintenance BL | Value at Week 104 – Extension BL value | X 100 % |
|---|---|---|
| = | Extension BL value | |

### **Other Safety Endpoints**

### Columbia Suicide Severity Rating Scale (C-SSRS) (Posner, 2007)

Missing data will not have any imputation performed (Nilsson, 2013)

### 14.6.4. Efficacy

### Snapshot

• The Snapshot algorithm is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy. 'HIV-1 RNA <50 c/mL' or 'HIV-1 RNA ≥50 c/mL' within an analysis window (see Table 17) is determined by the last available HIV-1 RNA measurement in that window while the participant is On-treatment in the applicable phase(s), e.g., Maintenance Phase (as assigned based on Table 30).

### Snapshot

- When no HIV-1 RNA data is available within a window, a participant cannot be assigned to the category of 'HIV-1 RNA < 50 c/mL'. Depending on the reason for lack of data, the participant will be classified as a 'HIV-1 RNA≥50' or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a participant withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a participant withdraw for reasons other than AE and was not suppressed at the time, they will be a 'HIV-1 RNA≥50 c/mL'.</p>
- Full details of the algorithm, including the handling of special cases, are included in Section 14 11

### Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL.
   For the purposes of summary statistics, such values will be replaced by the next value beyond the limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data listings will show the censored values as provided.

### Target Detected / Target Non- Detected/Super low viral load testing

- When a measurement of plasma HIV-1 RNA is below the limit of quantification (i.e., 40 c/mL) and is qualitatively observable that will be denoted as a "Target Detected" measure, while HIV-1 RNA below the limit of quantification that is not qualitatively observable that will be denoted as "Target Not Detected". Any measurements <40 c/mL characterised as "Target Not Detected" or "Target Detected" will be captured in the database.</li>
- Super low viral load will also be tested by BioMNTR lab for Viral loads below the limit of quantification (i.e., <2 c/mL) at some visits (e.g., Week 48).</li>

### Treatment (TRDF) and Efficacy Related (ERDF) Discontinuation = Failure

- The analysis of time to confirmed virologic failure (CVF) or discontinuation due to treatment related reasons (i.e., drug-related AE, intolerability of injections, protocol defined safety stopping criteria, or lack of efficacy) will censor participants who, at the end of the Week 48 analysis window per Table 15 (i.e., study day 350), have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment. This will be the Treatment Related Discontinuation = Failure (TRDF) data.
- Participants who, at the end of the Week 48 analysis window per Table 15 (i.e., study day 350), have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than lack of efficacy, will be censored in the analysis of the Efficacy Related Discontinuation = Failure (ERDF) data.
- Proportion of Participants without virologic (ERDF) or tolerability (TRDF) failure will be
  estimated using the Kaplan-Meier nonparametric method based on the time to ERDF or
  TRDF. The estimated proportion at Week 48 (i.e., study day 350) will be presented by
  treatment group, along with estimated difference in proportions between treatment groups

### Snapshot

and its associated two-sided 95% CI. The estimate of the standard error used to derive confidence intervals will be based on Greenwood's formula [Kalbfleisch, 1980].

See Appendix 1: Variables Defined for Time to Event Analysis

### Observed Case Viral Load (HIV-1 RNA) Category by Visit Summary Tables

- For each visit with scheduled viral load collection (per time and events schedule in the protocol), the Observed Case proportion is defined using available data, with no imputation for missing values.
- Week 48 and Week 96:
  - Numerator: Number of participants with on-treatment HIV-1 RNA in the respective category (e.g., < 50 c/mL) based on the last viral load assessment collected within the analysis Snapshot window for Week 48 and Week 96, respectively. (i.e., Week 48 ±6 weeks and Week 96 ±6 weeks).
  - Denominator: Number of participants with on-treatment HIV-1 within the analysis Snapshot window for Week 48 and Week 96, respectively. (i.e., Week 48 ±6 weeks and Week 96 ±6 weeks).
- Other Visits:
  - Numerator: Number of participants with on-treatment HIV-1 RNA in the respective category (e.g., < 50 c/mL) based on the last viral load assessment collected within the default analysis visit windows for Maintenance phase assessments (Table 15).
  - Denominator: Number of participants with on-treatment HIV-1 RNA collected within the default analysis visit windows for Maintenance phase assessments (Table 15).
- Observed case proportions will be derived for the following HIV-1 RNA categories: RNA
   40, 40 <= RNA <50, RNA < 40 & Target Detected, RNA <40 & Target Not Detected.</li>
- For Maintenance Baseline (Day 1), the last viral load collected prior to or equal to the date of first Maintenance Phase study treatment dose will be selected for determining the observed case proportion at this timepoint.

### Confirmed Virologic Failure (CVF)

 The definition of CVF is provided in the Protocol, Section 5.4.4 – Definition of Virologic Failure

### **HIV-1** Disease progression Stage

- Categories:
  - CDC Stage I at Maintenance Baseline (Day 1) to CDC Stage II;
  - CDC Stage I at Maintenance Baseline (Day 1) to CDC Stage III;
  - CDC Stage II at Maintenance Baseline (Day 1) to CDC Stage III;
  - CDC Stage III at Maintenance Baseline (Day 1) to new CDC Stage III event;
  - CDC Stage I, II, III at Maintenance Baseline (Day 1) to Death.

Please refer to Protocol (Appendix 4: CDC Classification for HIV-1 Infection) for defining Stage.

For the purpose of analysis, the CDC at Maintenance Baseline (Day 1) and at post-Day 1

#### **Snapshot**

during Maintenance Phase will be derived as below:

- At Baseline (Week -20), the 'Baseline CDC stage' for each participant was assessed by investigator and recorded in the eCRF. However, for the analysis, Maintenance Baseline (Day 1) CDC stage will be derived based on Maintenance Baseline (Day 1) CD4+ values as well as whether any HIV-associated/AIDS-defining conditions present on the start date of maintenance treatment (i.e., started/stopped on Study Day 1 or ongoing through Study Day 1) per the Criteria's thresholds (Appendix 4 in Protocol).
- To analyse disease progression, the most advanced Maintenance CDC stage will be derived based on the occurrences of new AIDs-defining conditions (please refer to Appendix 4 in Protocol for the list of AIDs-defining Conditions) as well as the nadir value of Maintenance Phase CD4+.
- For example, If a participant with CDC 'Stage I' at Maintenance Baseline (Day 1) had the lowest Maintenance Phase CD4+ =120 cell/mm3 without new AIDs-defining conditions, then HIV disease progression for this participant would be considered as 'CDC stage I at Maintenance Baseline (Day 1) to CDC stage III'. If a participant with CDC 'Stage II' at Maintenance Baseline (Day 1) had the lowest Maintenance Phase CD4+ =220 cell/mm3 AND had at least one new AIDs-defining condition, then HIV disease progression for this participant would be considered as 'CDC stage II at Maintenance Baseline (Day 1) to CDC stage III'.

### **Delay in IP Injection**

IM dosing is expected to occur every 4 weeks from Week 4b onwards (for the Q4W arm). The Delay in IP injection (days) will be calculated as:

• Delay in IP injection(days) = Injection date - date of preceding injection - 28 days

Delay in IP injection will be grouped into: ≤1, 2-3, 4-7, >7 days.

The proportion of participants with HIV-1 RNA≥50 c/mL at Week 48 (Snapshot) will be summarized by last delay in IP Injection. The last delay in IP injection will be the delay in IP injection at Week 48, or the delay in last IP injection prior to Week 48 if a participant does not receive Week 48 injection (i.e., missing visit or withdrawal).

#### 14.6.5. Pharmacokinetic

This document is intended for planning analysis of PK concentration data only. Population pharmacokinetics and identification of important determinants of variability will be described in a separate document.

### Plasma CAB and RPV concentration-time data

Plasma samples for determination of CAB and RPV concentration will be collected throughout the Maintenance and Extension Phases of the study. Additional samples will be collected for storage during the Long-Term Follow-Up Phase.

#### Plasma CAB and RPV concentration-time data

PK analysis of the plasma CAB concentration-time data on Day 1 and Week 4b for Japan participants will be conducted using non-compartmental methods with WinNonlin (Version 5.2 or higher). Actual sampling and dosing times as recorded in the eCRF will be used for analysis.

#### **Evaluable concentration**

PK concentration will be summarized in two ways: 'all data' without regard to timing relative to scheduled time and 'evaluable data'.

The 'evaluable data' are from the samples that met sample collection window criteria, excluding samples affected by dosing errors/oral bridging. Sampling windows are determined relative to the previous dose as follows:

- 1-5 hours for 2-hour post dose samples;
- ± 3-10 days post last injection for 1-week post injection visits;
- ±4 day for pre-dose sample.
- Samples affected by dosing errors (e.g., wrong dose) or oral bridging will also be excluded.

| Timepoint | Evaluable window | For Programming: |
|---|---|---|
| PRE-DOSE:<br>WK4b/104b<br>only | 20-28 hrs after last oral dose taken and the last 3 oral doses administered properly | 20 hrs ≤ Days Since Last Oral Dose ≤ 28 hrs and the last 3 oral doses administered on the three consecutive days prior to WK4b/104b. |
| 2-HR-POST: | 1-5 hrs | 1 hr ≤ Hours Since Last Injection Dose ≤ 5 hrs |
| 1-WK-POST: | 3-10 days post last injection | 3 d ≤ Days Since Last Dose ≤ 10 d |
| PRE-DOSE: | ±4 days | 24 d ≤ Days Since Last Dose ≤ 32d |

Relative Time is calculated relative to the date and time of last previous dose. For example, if the time of the last previous dose (e.g., oral lead-in/oral-bridging) is missing, then the relative time for pre-dose PK sample will be set to missing and the sample will not be considered 'evaluable'.

If a pre-dose sample is collected on the same day as the first dose of oral bridging, and the time of the first dose (not recorded in eCRF) is confirmed to be 'after' the collection of pre-dose sample (by medical monitor or Data querying), then this PK sample will not be impacted by the oral bridging.

At Week 4b/104b, the evaluable window and relative time for 2-HR-POST will be derived based on last injection dose (not the last oral dose). The timing of last oral dose will not affect 'evaluable' status with the exception of the last oral dose taken after the 1st injection, i.e., if a participant took the last oral dose after the 1st injection, the 2-HR-POST will not be considered 'evaluable', because of the deviation from the IP administration sequence per protocol.

The time-deviation (hours) from the targeted timepoint will be calculated for the following timepoints:

#### Plasma CAB and RPV concentration-time data

Time\_deviation (hrs) for '1-Week-POST' =Sample date.time-last previous injection date.time - 7\*24 hours

Time\_deviation (hrs) for '1-HR-POST' =Sample date.time-last previous injection date.time -1 hours

Time\_deviation (hrs) for '2-HR-POST' =Sample date.time-last previous injection date.time -2 hours

Time\_deviation (hrs) for '4-HR-POST' =Sample date.time-last previous injection date.time -4 hours

Time\_deviation (hrs) for '5-HR-POST' =Sample date.time-last previous injection date.time -5 hours Time\_deviation (hrs) for '8-HR-POST' =Sample date.time-last previous injection date.time -8 hours

Time\_deviation (hrs) for '24-HR-POST' =Sample date.time-last previous injection date.time -24 hours

### For Long-term Follow-up Phase PK concentrations:

LTFU RPV concentrations for participants receiving oral RPV during the LTFU phase will be excluded from LTFU PK summary tables and mean/median concentration plot but will be included in data listings and PK concentration-time profiles plots (with footnotes indicate which participants were receiving oral RPV). Participants receiving inducers during the LTFU phase may also be excluded.

The following windows are for defining 'evaluable' Long-term Follow-up Phase PK concentrations.

| TIMEPOINT | EVALUABLE WINDOW | FOR PROGRAMMING: |
|---------------|------------------|-----------------------------------------|
| LTFU MONTH 1 | ± 4 days | 24d ≤ Days Since Last Injection ≤ 32d |
| LTFU MONTH 3 | ± 1 Week | 77d ≤ Days Since Last Injection ≤ 91d |
| LTFU MONTH 6 | ± 2 Week | 154d ≤ Days Since Last Injection ≤ 182d |
| LTFU MONTH 9 | ± 2 Week | 238d ≤ Days Since Last Injection ≤ 266d |
| LTFU MONTH 12 | ± 2 Week | 322d ≤ Days Since Last Injection ≤ 350d |

### **Pharmacokinetic Parameters**

 Population pharmacokinetics and identify important determinants of variability will be described in a separate document.

#### 14.6.6. Health Outcome



#### **Treatment Satisfaction Score**

- Total Treatment Satisfaction Score is computed with items 1-11. Items 1-11 are summed to produce a score with a possible range of 0 to 66.
- Item 12 will not be included in Total Treatment Satisfaction Score. Instead, it will be treated as a stand-alone item only.
- Higher scores represent greater treatment satisfaction as compared to the past few weeks.
- A maximum of 5 items can be missing, which can be imputed to reflect the mean of the completed item scores. If 6 or more items are missing, then the treatment satisfaction scale score should not be computed and instead be imputed using LOCF.

### **Individual Item Scores**

- Items are rated as 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied, inconvenient, inflexible, etc.).
- Higher scores represent greater satisfaction with each aspect of treatment
- For individual item scores outputs, missing scores will not be computed (according to Page 7 of the [HIVTSQ User Guidelines, 2016]) and instead be imputed using LOCF.



### **Treatment Satisfaction Score (change)**

- Total Treatment Satisfaction Score is computed with items 1-11. Items 1-11 are summed to produce a score with a possible range of -33 to 33
- Item 12 will be computed as an individual item only.
- The higher the score, the greater the <u>improvement</u> in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represents no change.
- A maximum of 5 items can be missing, the missing scores will be imputed with the mean of the completed item scores. If 6 or more items are missing, then the overall treatment satisfaction scale score should not be computed and will remain missing.

### **Individual Treatment Change Item Scores**

- Items are rated as +3 ('much more satisfied', 'much more convenient', 'much more flexible', etc.) to -3 ('much less satisfied', 'much less convenient', 'much less flexible', etc.).
- The higher the score, the greater the improvement in satisfaction with each aspect of treatment and the lower the score, the greater the deterioration in satisfaction with each aspect of treatment.



- The score of a domain is calculated as the mean of all items with the domain. Higher scores represent worse perception of injection.
- A maximum of <50% items can be missing within a domain, which can be imputed to reflect the
  mean of the completed item scores within the domain. Thus, if the number of missing items is
  ≥3 (Bother from injection site reactions), ≥2 (Leg movement/Sleep), ≥1 (Acceptability), then the
  total score for the domain should not be computed and instead be imputed using LOCF
  (Section 14.7.2.2)</li>
- LOCF will not be used for the SC sub-study

#### **Individual Item Scores**

- Items are rated on a 5-point scale, ranging from 1(very satisfied, not at all, etc.) to 5 (very dissatisfied, extremely, etc.).
- Higher scores represent worse perception of injection
- For individual item scores outputs, missing scores will not be computed and instead be imputed using LOCF (Section 14.7.2.2). Observed values will be used in the SC Sub-study.

### **SF-12**



CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

#### **Dimension Score**

- Changes from Baseline at Week 48 in health-related quality of life (using SF-12) for the physical component summary (PCS) and the mental component summary (MCS) were assessed for the two treatment groups. Scores are created according to the manual [SF-12 (v2) Health Survey 1994, 2002 Medical Outcomes Trust and QualityMetric Incorporated] and the component scores were calculated using computer software purchased from QualityMetric.(http://www.qualitymetric.com/)
- Missing component scores will be imputed using LOCF (Section 14.7.2.2).

### **Individual Item Scores**

- Items are rated as 5 except for Question 2. Question 2a and 2b are rated as 3
- Individual item missing scores will be imputed using LOCF (Section 14.7.2.2).

### HATQoL (Holmes, 1999)





### Tolerability of Injection (NRS)

### Questionnaire with one single question for Q4W IM arm only

- Maximum level of pain experienced with the most recent injections. Ranking from no pain (0) to extreme pain (10).
- Missing scores will be imputed using LOCF (Section 14.7.2.2). Observed values will be used in the SC Sub-study

#### Preference question

### Questionnaire with one single dichotomous preference question at Week 48 (Q4W IM arm)

- Assess the treatment preference: Months injection vs daily oral current ART at Week 48 for 'Q4W IM' arm
- Any missing values will remain missing (i.e., no imputation)
- A preference questionnaire will also be administered to sub-study participants. It asks participants to state their preference between IM and SC injections and to check off potential reasons why.

#### **Reasons for Switch Questionnaire**

Reason for Switch questionnaire is collected for sub-study participants and asks the reasons they agreed to switch to SC injections.

Any missing values will remain missing (i.e., no imputation).

### Interest Questionnaire

The Interest questionnaire is collected for sub-study participants and asks how interested they would be to switch to SC injections at home on a 5 point scale ranging from 'Not at all interested' to 'Extremely interested.'.

Any missing values will remain missing (i.e., no imputation).

### 14.6.7. Viral Genotype and Phenotype

### Genotype

### **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest.

### **Representation of Amino Acid Changes**

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' |
| | (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### **Resistance Associated Mutations**

 Known INI mutations associated with the development of resistance to Integrase Strand Transfer Inhibitors:

| Amino Acids in | H51Y, <b>T66</b> A/I/K, L68V/I, L74I/M, <b>E92Q</b> /V/G, Q95K, T97A, <b>G118R</b> , <b>F121Y/C</b> , |
|---|---|
| HIV Integrase for | E138A/D/K/T, <b>G140</b> A/C/ <b>R</b> /S, <b>Y143C/H/R</b> /K/S/G/A, P145S, Q146P, <b>S147G</b> , |
| Analysis | <b>Q148H/K/R</b> /N, V151/IL/A, S153F/Y, <b>N155H</b> /S/T, E157Q, G163R/K, G193E, |
| | S230R, <b>R263K</b> |

#### NOTES:

- Draft listing; may be modified in case of additional substantive data availability.
- Based on the IAS-USA list of mutations associated with resistance to Bictegravir, Cabotegravir, Dolutegravir, Elvitegravir, or Raltegravir (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019): T66A/I/K, L74M, E92Q/G, T97A, G118R, F121Y, E138A/K/T, G140A/C/R/S, Y143C/H/R, S147G, Q148H/K/R, S153F/Y, N155H, R263K) and observed mutations during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (study ING112574): H51Y, L74I, L68V/I, E92V, Q95K, E138D, Y143K/S/G/A, P145S, Q146P, V151I/L/A, N155S/T, E157Q, G163R/K, G193E, S230R.
- Major USA-IAS mutations associated with resistance to INSTI are bolded.
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis [Wensing, 2019].

| Genotype | |
|---|---|
| Class | Mutations |
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, |
| | Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L |
| Pls | D30N, V32I, M46I/L, I47A/V, G48V, I50V/L, I54V/M/L, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S, L90M |

Note: List generated from IAS\_USA Guideline, [Wensing, 2019]

### Treatment-Emergent Mutations Relative to Induction Baseline (Week -20)

 Treatment-emergent genotypic mutations are defined as mutations that appear between Induction Baseline (Week -20), i.e., prior to the start of Induction Phase study drug (inclusive), and an on-treatment assessment (e.g., at time of confirmed virologic failure). Note: If Monogram is not able to produce genotype at Week -20, then treatment-emergent will be determined relative to the screening genotype provided by the central laboratory.

### Phenotypic Susceptibility

- Phenotypic susceptibility to all licensed antiretroviral drugs and CAB will be determined using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change (FC) in IC50 relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.
- Since the maximum assay limit for FC for each ART varies from assay to assay, FC values that are greater than the maximum assay limit (e.g., '>100') will be interpreted as having a value equal to the smallest maximum assay limit for that ART in the study population for data analysis. Censored values will be presented 'as is' in the listings. Phenotypic susceptibilities will be categorized according to FC as shown below (based on Monogram PhenoSense assay). Clinical cutoffs (where available) or biological cutoffs by PhenoSense will be used to define the phenotypic susceptibility of ART therapy by Monogram.
- Replication capacity is generated as part of standard phenotypic assays

### PhenoSense Algorithm

| Drug | Abbreviation | Class | PhenoSense cutoff |
|---------------|--------------|-------|--------------------------|
| Abacavir | ABC | NRTI | (4.5 - 6.5) <sup>a</sup> |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF (TAF) | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |

| Genotype | | | |
|-----------------|-------|-------|--------------|
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Cabotegravir | CAB | INI | 2.5 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |

a. clinical cutoff (lower cutoff – higher cutoff).

Phenotypic susceptibility to each drug in a participant's background regimen is determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold resistance as below:

### **Full Sensitivity**

| Fold Change | Interpretation |
|--------------------------------------------|----------------|
| > clinical lower cutoff or biologic cutoff | resistance |
| ≤ clinical lower cutoff or biologic cutoff | sensitive |

### **Partial Sensitivity**

| Fold Change | Interpretation |
|------------------------------------------------------|---------------------|
| > clinical higher cutoff | resistance |
| ≤ clinical higher cutoff and > clinical lower cutoff | partially sensitive |
| ≤ clinical lower cutoff | sensitive |

PHENOTYP dataset from Monogram contains the phenotypic susceptibility for each drug derived from the cutoff listed above. Thus, phenotypic susceptibility (i.e., full sensitivity and partial sensitivity) will not be re-derived for our analysis.

### **Genotypic and Net Assessment Susceptibility**

Genotypic and Net assessment susceptibility to all licensed antiretroviral drugs and CAB will be
determined from Monogram Inc. and will be reported with the categories of 'resistance',
'partially sensitive', and 'sensitive' as what will be performed for phenotypic susceptibility.
Genotypic and Net assessment susceptibility will be assessed at time of CVF using plasma
sample, Genotypic susceptibility may be assessed at baseline using PBMC.

### Induction Baseline (Week -20) HIV-1 Subtype

 For participants without confirmed virologic failure: Screening visit subtype from Q SQUARED, unless a subtype from MONOGRAM is available on the same date.

# Genotype

 For participants with confirmed virologic failure: Select last pre-treatment subtype (expected to be the Week -20 result from MONOGRAM).

# 14.7. Appendix 7: Reporting Standards for Missing Data

# 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e., as specified in the protocol) was defined as: <ul> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including the Nominal Week 100 visit, and did not enter the Extension Phase;</li> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including the Nominal Week 100 visit, and entered and completed the Extension Phase (defined as remaining on study until commercial supplies of CAB LA + RPV LA become locally available, or development of CAB LA + RPV LA is terminated).</li> </ul> </li> </ul> |
| | · |

# 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be desumented along with the reason for evaluation in the clinical study report. |
| | be documented along with the reason for exclusion in the clinical study report. |

# 14.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment State.</li> <li>Missing Stop Day: Last day of the month will be used unless this is after the last contact date; in this case the last contact date will be used.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> </li> </ul> |
| Concomitant<br>Medications/<br>Medical History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>For medications recorded in the eCRF as prior ART, the earlier of this imputed date or the day before Screening date will be used.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Health outcomes | <ul> <li>For the health outcomes questionnaire data, please refer to Section 14.6.6.</li> <li>For the summary of individual item scores outputs, missing scores will not be computed.</li> </ul> |
| | For the SC Sub-study going forward, missing data for all HO assessments will not be imputed using the LOCF technique. Observed values will be used unless otherwise specified. |

# 14.7.2.2. Handling of Missing data for Statistical Analysis

| Element | Re | porting Detail | |
|---|---|---|--|
| Snapshot | • | In the Snapshot dataset, participants without HIV-1 RNA data in the assessment window for the visit of interest (due to missing data or discontinuation of IP prior to the visit window) do not belong to 'HIV-1 RNA < 50 c/mL (or <200 c/mL)'. The nature of this missing data will be further classified in Snapshot summaries as either 'HIV-1 RNA≥50' or 'No Virologic Data at Week X'; Appendix 11: Snapshot Algorithm Details for full details. | |
| LOCF | • | In the LOCF dataset, missing values will be carried forward from the previous, non-missing on-treatment assessment. | |
| Lipid LOCF | 1. | Maintenance (both arms) and Maintenance + Extension Phase (randomized Q4W arm only): | |
| | | <ul> <li>Maintenance Baseline (Day 1) for Lipids LOCF Analyses:</li> <li>Last evaluable lipids assessment up to and including the start of Maintenance Phase IP, where 'evaluable' is defined as: Lipid modifying agents not taken within 12 weeks of the date of assessment and Lipids are collected in a fasting state. Participants with unevaluable Maintenance Baseline (Day 1) for Lipids (as defined above) will be excluded from the analysis of Maintenance phase values and Maintenance + Extension phase values (Randomized Q4W arm).</li> </ul> | |
| | | <ul> <li>During Maintenance + Extension phases</li> <li>If participants initiate serum lipid-lowering agents during the Maintenance + Extension Phase, then the last available fasted On-treatment lipid values prior to the initiation will be used in place of future, observed On-treatment values.</li> <li>Imputation at visits with observed on-treatment values will continue even if the participant discontinues the lipid-lowering agent. Missing assessments will not be imputed.</li> </ul> | |
| | | <ul> <li>Analyses Evaluated with Lipid LOCF dataset:</li> <li>This dataset will be used to summarize fasting lipids parameters in the following displays: <ul> <li>Summary of Chemistry Values by visit</li> <li>Summary of Chemistry Change from Maintenance Baseline (Day 1) by visit</li> <li>Summary of Fasting TC/HDL Ratio Change from Maintenance Baseline (Day 1)</li> </ul> </li> </ul> | |
| | | All other displays of lipids (i.e., toxicity tables and NCEP tables) will use observed fasting data, without LOCF imputation. | |
| | 2. | Extension Phase (Q4W Switch IM group): | |
| | | Extension Baseline (Week 100) for Lipids LOCF Analyses: Last evaluable lipids assessment up to and including the first dose of Extension phase CAB and/or RPV, where 'evaluable' is defined as: Lipid modifying agents not taken within 12 weeks of the date of assessment and | |
| Element | Reporting Detail |
|---|---|
| | Lipids are collected in a fasting state. Participants with unevaluable Extension Baseline (Week 100) for Lipids (as defined above) will be excluded from the analysis of Extension phase values (Extension Switch population). |
| | <ul> <li>During Extension phase</li> <li>If participants initiate serum lipid-lowering agents during the Extension Phase, then the last available fasted On-treatment lipid values prior to the initiation will be used in place of future, observed On-treatment values. </li> <li>Imputation at visits with observed on-treatment values will continue even if the participant discontinues the lipid-lowering agent. Missing assessments will not be imputed.</li> </ul> |
| | Baseline for Lipids LOCF Analyses in sub-study: Last evaluable lipids assessment up to and including the start of SC injection, where 'evaluable' is defined as: Lipid-modifying agents not taken within 12 weeks of the date of assessment and Lipids are collected in a fasting state. |
| | <ul> <li>During the SC Injection or Return to Gluteal Injection Phase:</li> <li>If participants initiate serum lipid-modifying agents during the SC injection or Return to Gluteal Injection Phase, then the last available fasted on-treatment lipid values prior to the initiation will be used in place of future, observed ontreatment values in sub-study.</li> <li>Imputation at planned visits will continue even if the participant discontinues the lipid-modifying agent. Missing assessments will not be imputed if there is no last available fasting on-treatment lipid value prior to the initiation of serum lipid-modifying agent.</li> <li>If participants take lipid modifying agents within 12 weeks prior to the start of the SC injection, all the post-baseline values in sub-study will be missing.</li> </ul> |
| | <ul> <li>Analyses Evaluated with Lipid LOCF dataset:</li> <li>This dataset will be used to summarize fasting lipids parameters in the following displays: <ul> <li>Summary of Chemistry Values by Visit (Extension Switch population)</li> <li>Summary of Chemistry Change from Extension Baseline (Week 100) by Visit</li> <li>Summary of Fasting TC/HDL Ratio Change from Extension Baseline (Week 100)</li> <li>Summary of Chemistry Changes from Sub-study Baseline by Visit (SC Injection + Return to Gluteal Injection Phase)</li> <li>Summary of Chemistry Values by Visit (SC Injection + Return to Gluteal Injection Phase)</li> </ul> </li> <li>All other displays of lipids (i.e., toxicity tables and NCEP tables) will use</li> </ul> |
| | observed fasting data, without LOCF imputation. |

# 14.8. Appendix 8: Values of Potential Clinical Importance

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values and<br>Adverse<br>Events | The central laboratory will flag lab parameter toxicities directly in the provided datasets based on Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.0, November 2014. |

# 14.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

PopPK will be described in a separate document.

# 14.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

PK/PD dataset specification and methodology will be described in a separate document.

### 14.11. Appendix 11: Snapshot Algorithm Details

#### **Detailed Algorithm Steps**

- Consider an analysis visit window for Week X (e.g., Week4, ...Week 24, Week 48 et al). The Window for Week 24/48 visit is defined in Table 17 (e.g., window for Week 48 is ± 6 Week: 295 ≤ Study Day ≤ 378) and in Table 15 for other visits through to Nominal Week 52 at Maintenance Phase. The Snapshot Analysis at post Maintenance Phase will not be appropriate because a large portion of responders will be switched to other studies and not all participants would have the chance to reach same timepoint.
- The HIV1-RNA threshold of 50, 200 copies/mL will be analysed, respectively, in this study
- The analysis window 'Week 48' and HIV1-RNA threshold of '50 copies/mL' are used for the purpose of illustration. A participant's Snapshot response and reason at Week 48 are categorized as below.
  - HIV1-RNA < 50 copies/mL
  - HIV1-RNA ≥ 50 copies/mL

Data in window not below 50 Discontinued for lack of efficacy Discontinued for other reason while not below 50 Change in background therapy\*

No Virologic Data at Week 48 Window
 Discontinued study due to AE or death
 Discontinued study for other reasons
 On study but missing data in window

 The steps in determining response and reasons are indicated in Table below, in the order stated.

| Detailed steps | | |
|---|---|---|
| Please note that the following scenarios will NOT be penalized Per Snapshot algorithm (i.e., please excluding these scenarios from Condition 1-4). | | |
| Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients) | | |
| Condition ('Week 48' indicates Week 48 window) | Response | Reasons |
| If non-permitted change in background therapy prior to<br>Week 48 | HIV1-RNA ≥ 50 | Change in background therapy |

<sup>\*</sup> Note: since changes in ART are not permitted in this protocol, all such participants who change ART during the Maintenance Phase will be considered 'HIV1-RNA ≥ 50 copies/mL'. if the change in ART is made prior to an analysis timepoint. Participants with protocol permitted oral bridging treatment will not be considered 'HIV1-RNA ≥ 50 copies/mL' due to 'change in ART'.

| 2. If permitted change[a] in background therapy prior to Week 48 AND the latest on-treatment VL prior to/on the date of change is ≥ 50 c/m (NA to this study) | HIV1-RNA ≥ 50 | Change in background therapy |
|---|---|---|
| 3: If non-permitted change in background therapy during Week 48 | | |
| <ul> <li>Last on-treatment VL during Week 48 prior to/on<br/>the date of change ≥ 50 c/mL</li> </ul> | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| <ul> <li>Last on-treatment VL during Week 48 prior to/on<br/>the date of change &lt;50 c/mL</li> </ul> | HIV1-RNA <<br>50 | |
| No VL during Week 48 prior to/on the date of change | HIV1-RNA ≥ 50 | Change in background therapy |
| 4: If permitted change[a] in background therapy during Week 48 AND the last on-treatment VL prior to/on the date of change is ≥ 50 c/mL (NA to this study) | | |
| 4.1 this last on-treatment VL occurs prior to Week 48 | HIV1-RNA ≥ 50 | Change in background therapy |
| 4. 2 this last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| 5: If none of the above conditions met | | |
| 5.1 VL available during Week 48 | | |
| <ul> <li>Last on-treatment VL during Week 48 ≥ 50 c/mL</li> </ul> | HIV1-RNA ≥ 50 | Data in window<br>not below 50 |
| Last on-treatment VL during Week 48 <50 c/mL | HIV1-RNA <<br>50 | |
| 5.2 No VL during Week 48 | | |
| 5.2.1 if participants still on study i.e. the upper bound of analysis snapshot window is prior to the following date: | No virologic<br>data at Week<br>48 Window | On study but<br>missing data in<br>window |
| For ABC/DTG/3TC arm: Min (ABC/DTG/3TC Stop Date + 1, withdrawal date) | | |

| | | Ţ |
|---|---|---|
| For Q4W arm: Min[max(Date of last Q4W IM Dose + 35, Date of last oral dose+1), withdrawal date] | | |
| 5.2.2 If participants withdraw before/during Week 48 due to | | |
| 5.2.2.1 Safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria et al, as recorded in eCRF Conclusion form) | No virologic<br>data at Week<br>48 Window | Disc due to<br>AE/death |
| 5.2.2.2 Non-safety related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion et al, as recorded in eCRF Conclusion Form) | | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL OR no on-<br/>treatment VL available during study</li> </ul> | No virologic<br>Data at Week<br>48 Window | Disc for other reasons |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to Lack of efficacy</li> </ul> | HIV1-RNA ≥<br>50 | Disc. for lack of efficacy |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND<br/>withdrawal due to all other non-safety related<br/>reasons</li> </ul> | HIV1-RNA ≥ 50 | Dis. for other reason while not below 50 |

a: Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result

#### **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

 HIV-RNA = 580 copies/mL at Day 336, HIV-RNA below 50 copies/mL on Day 350. This should be categorized as HIV-RNA below 50 copies/mL.

#### 2.No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as Discontinued due to AE or Death (as appropriate), regardless of the HIV-RNA result, even if the HIV-RNA is below 50 copies/mL at the time of discontinuation.
- However, if a patient has an HIV-RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response.
   This is the Virology First hierarchy:

- a. HIV-RNA below 50 copies/mL at Day 336 and discontinues because of AE or even dies on Day 360 — this person is categorized as having HIV-RNA below 50 copies/mL.
- b. HIV-RNA is 552 copies/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-RNA greater than or equal to 50 copies/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as Discontinued for Other Reasons.
- If a patient discontinues the study before the time window because of lack of efficacy, then the patient should be included in the HIV-RNA greater than or equal to 50 row and not in the Discontinued for Other Reasons row.
- If a patient discontinues because of participant withdrew consent and his or her HIV-1 RNA result at the time of discontinuation was equal to or above 50 copies/mL, then he or she should be categorized as HIV-RNA greater than or equal to 50 and NOT as Discontinued for Other Reasons.
- If a patient discontinued because of Lost to Follow-Up and the last HIV-RNA result was 49 copies/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment not permitted by protocol— they should be captured in the HIV-RNA greater than or equal to 50 copies/mL row.

#### 3.On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-RNA below 50 copies/mL on Day 380, this patient should be considered On Study but Missing Data in Window.
- If there are no data during Days 294 to 377, but there is an HIV-RNA equal to or above 50 copies/mL on Day 280, this patient also should be classified as On Study but Missing Data in Window.

#### 14.12. Appendix 12: AESI identification

G) (G) (T) ... | D) ... | 1 ... | G) (G) G ... | 200000007

SMQ and PT codes based on MedDRA dictionary version 22.0 for Week 96 CSR.

### 14.12.1. Hepatic Safety Profile

Medical concept of hepatic failure and hepatitis. Sub- SMQs (1) 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions' and (2) 'Hepatitis, non-infectious', both of parent SMQ 'Hepatic Disorders'; only narrow terms selected from sub-SMQs. Some preferred terms e.g. PT 'hepatitis fulminant' are duplicated.

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 | |
|---|---|
| Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and othe conditions' | er liver damage-related |
| Category: A | |
| Scope: Narrow | |
| Preferred Term | PT Code |
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |

SMQ: 'Hepatic Disorders'; SMQ Code: 20000005

Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related

conditions'
Category: A
Scope: Narrow

| Scope: Narrow | |
|------------------------------------|----------|
| Preferred Term | PT Code |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |

SMQ: 'Hepatic Disorders'; SMQ Code: 20000005

Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related

conditions'
Category: A
Scope: Narrow

| Scope: Narrow | |
|--------------------------------------|----------|
| Preferred Term | PT Code |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver injury | 10067125 |
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Nonalcoholic fatty liver disease | 10082249 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |

SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions' Category: A Scope: Narrow Preferred Term PT Code Primary biliary cholangitis 10080429 10080679 Regenerative siderotic hepatic nodule Renal and liver transplant 10052279 Retrograde portal vein flow 10067338 Reye's syndrome 10039012 10070953 Reynold's syndrome Splenic varices 10067823 Splenic varices haemorrhage 10068662 Steatohepatitis 10076331 Subacute hepatic failure 10056956 Varices oesophageal 10056091 Varicose veins of abdominal wall 10072284 10078438 White nipple sign SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 Sub-SMQ: 'Hepatitis, non-infectious' Category: A Scope: Narrow Preferred Term PT Code Acute graft versus host disease in liver 10066263 Allergic hepatitis 10071198 Alloimmune hepatitis 10080576 10003827 Autoimmune hepatitis Chronic graft versus host disease in liver 10072160 Chronic hepatitis 10008909 Graft versus host disease in liver 10064676 Hepatitis 10019717

10076331

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 | |
|---|---|
| Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-reconditions' Category: A Scope: Narrow | elated |
| Preferred Term | PT Code |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |

### 14.12.2. Hypersensitivity Reactions

Steatohepatitis

Medical concept of hypersensitivity reactions/DRESS. Only narrow terms selected from Category A of SMQ 'Drug reaction with eosinophilia and systemic symptoms syndrome'. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms) and a pre-requisite for any combination in algorithmic search. Overlap of some preferred terms with SMQ 'Severe Cutaneous Adverse Reactions'. Plus, additional preferred terms selected from HGLT 'Allergic conditions' under SOC 'Immune system disorders.

| SMQ: Drug reaction with eosinophilia and systemic symptoms syndrome SMQ Code: 20000225 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |

| SMQ: Drug reaction with eosinophilia and systemic symptoms syndrome SMQ Code: 20000225 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Additional preferred terms selected from HLGT 'Allergic conditions' under SOC 'Immune system disorders' | |
| Preferred Term | PT Code |
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |

## 14.12.3. Rash including severe cutaneous adverse reactions

Medical concept of rash including severe cutaneous adverse reactions. Only narrow terms from SMQ 'Severe cutaneous adverse reactions' selected. Plus several additional preferred terms selected from HLTs 'Rashes, eruptions and exanthems NEC', 'Pruritus

NEC', 'Pustular conditions', 'Dermatitis ascribed to specific agent' all under SOC 'Skin and subcutaneous tissue disorders'.

| SMQ: Severe Cutaneous Adverse Reactions<br>SMQ Code: 20000020<br>Category: A<br>Scope: Narrow | |
|---|---|
| SMQ | PT Code |
| Acute generalised exanthematous pustulosis | 10048799 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Exfoliative rash | 10064579 |
| Oculomucocutaneous syndrome | 10030081 |
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Target skin lesion | 10081998 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Additional preferred terms selected from HLTs 'Rashes, eruptions and exanthems NEC', 'Pruritus NEC', 'Pustular conditions', 'Dermatitis ascribed to specific agent' all under SOC 'Skin and subcutaneous tissue disorders'. | |
| Preferred Term | PT Code |
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |

| SMQ: Severe Cutaneous Adverse Reactions<br>SMQ Code: 20000020<br>Category: A<br>Scope: Narrow | |
|---|---|
| SMQ | PT Code |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

# 14.12.4. Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses

Notes: Medical concept of QT prolongation and complications. Only narrow terms from SMQ 'Torsade de pointes/QT prolongation' selected plus one additional PT under HLT 'ECG investigations'.

| SMQ: Torsade de pointes/QT prolongation<br>SMQ Code: 20000001<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |

| Electrocardiogram QT interval abnormal | 10063748 |
|---|---|
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |
| Additional preferred terms selected from HGLT 'ECG investigations' under SOC 'Investigations'. | |
| Preferred Term | PT Code |
| Electrocardiogram repolarisation abnormality | 10052464 |

#### 14.12.5. Suicidal Ideation/Behaviour

Medical concept of suicidal ideation and behaviour. Sub-SMQ 'Suicide/self-injury' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury'. Only narrow terms from the sub-SMQ selected.

| SMQ: 'Depression and Suicide/Self Injury' SMQ Code: 20000035 Sub-SMQ: 'Suicide/self-injury' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |

| Suicidal ideation | 10042458 |
|---------------------------|----------|
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide | 10082458 |
| Suspected suicide attempt | 10081704 |

## 14.12.6. Depression

Medical concept of Depression. Sub-SMQ 'Depression (excl suicide and self injury)' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury'. Only narrow terms from the sub-SMQ selected.

| SMQ: "Depression and Suicide/Self Injury" SMQ Code: 20000035 Sub-SMQ: 'Depression (excl suicide and self injury)' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |

| SMQ: "Depression and Suicide/Self Injury" SMQ Code: 20000035 Sub-SMQ: 'Depression (excl suicide and self injury)' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

## 14.12.7. Bipolar Disorder

Medical concept of bipolar disorder. All preferred terms from HLGT 'Manic and Bipolar mood disorders and disturbances' under SOC 'Psychiatric disorders'.

| Preferred Term | PT Code |
|----------------------|----------|
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |

## 14.12.8. Psychosis

Medical concept of psychosis. Only narrow terms from SMQ 'Psychosis and psychotic disorders' selected.

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acute psychosis | 10001022 |
| Alcoholic psychosis | 10001632 |
| Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder with marked stressors | 10048549 |
| Brief psychotic disorder without marked stressors | 10056395 |
| Brief psychotic disorder, with postpartum onset | 10006362 |
| Charles Bonnet syndrome | 10063354 |
| Childhood psychosis | 10061040 |
| Clang associations | 10009232 |
| Cotard's syndrome | 10059591 |
| Delusion | 10012239 |
| Delusion of grandeur | 10012241 |
| Delusion of reference | 10012244 |
| Delusion of replacement | 10012245 |
| Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, jealous type | 10012251 |
| Delusional disorder, mixed type | 10012252 |
| Delusional disorder, persecutory type | 10053195 |
| Delusional disorder, somatic type | 10012254 |
| Delusional disorder, unspecified type | 10012255 |
| Delusional perception | 10012258 |

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Dementia of the Alzheimer's type, with delusions | 10012295 |
| Depressive delusion | 10063033 |
| Derailment | 10012411 |
| Epileptic psychosis | 10059232 |
| Erotomanic delusion | 10015134 |
| Flight of ideas | 10016777 |
| Hallucination | 10019063 |
| Hallucination, auditory | 10019070 |
| Hallucination, gustatory | 10019071 |
| Hallucination, olfactory | 10019072 |
| Hallucination, synaesthetic | 10062824 |
| Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hysterical psychosis | 10062645 |
| Ideas of reference | 10021212 |
| Illusion | 10021403 |
| Jealous delusion | 10023164 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10028916 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10033864 |

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Paranoid personality disorder | 10033869 |
| Parkinson's disease psychosis | 10074835 |
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis | 10070669 |
| Post-injection delirium sedation syndrome | 10072851 |
| Posturing | 10036437 |
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |

## 14.12.9. Mood Disorders

Medical concept of mood disorders. All preferred terms from HLGT 'Mood disorders and disturbances NEC', under SOC 'Psychiatric disorders'.

| Preferred Term | PT Code |
|----------------------------------|----------|
| Affect lability | 10054196 |
| Affective ambivalence | 10077173 |
| Affective disorder | 10001443 |
| Alexithymia | 10077719 |
| Anger | 10002368 |
| Apathy | 10002942 |
| Blunted affect | 10005885 |
| Boredom | 10048909 |
| Constricted affect | 10010778 |
| Crying | 10011469 |
| Diencephalic syndrome of infancy | 10012774 |
| Dysphoria | 10013954 |
| Emotional disorder | 10014551 |
| Emotional distress | 10049119 |

| Preferred Term | PT Code |
|--------------------------------------------------|----------|
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Flat affect | 10016759 |
| Frustration tolerance decreased | 10077753 |
| Inappropriate affect | 10021588 |
| Irritability | 10022998 |
| Laziness | 10051602 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Moaning | 10027783 |
| Mood altered | 10027940 |
| Mood disorder due to a general medical condition | 10027944 |
| Mood swings | 10027951 |
| Morose | 10027977 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Premenstrual dysphoric disorder | 10051537 |
| Premenstrual syndrome | 10036618 |
| Screaming | 10039740 |
| Seasonal affective disorder | 10039775 |
| Steroid withdrawal syndrome | 10042028 |
| Substance-induced mood disorder | 10072387 |

## 14.12.10. Anxiety

Notes: Medical concept of anxiety disorders. All preferred terms from HLGT "Anxiety disorders and symptoms", under SOC "Psychiatric disorders".

| Preferred Terms | PT Code |
|-----------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |

| Preferred Terms | PT Code |
|-----------------------------------------------------|----------|
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |
| Anxiety disorder due to a general medical condition | 10002859 |
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Catastrophic reaction | 10082329 |
| Cibophobia | 10082413 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |

| Preferred Terms | PT Code |
|---------------------------------------|----------|
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |
| Herpetophobia | 10081809 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |

| Preferred Terms | PT Code |
|---|---|
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders associated with streptococcal infection | 10072147 |
| Panic attack | 10033664 |
| Panic disorder | 10033666 |
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Postpartum anxiety | 10082233 |
| Postpartum neurosis | 10036419 |
| Postpartum stress disorder | 10056394 |

| Preferred Terms | PT Code |
|--------------------------------|----------|
| Post-traumatic stress disorder | 10036316 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |
| Trichotillomania | 10044629 |

## 14.12.11. Sleep Disorders

Medical concept of sleep disorders. All preferred terms from (1) HLGT 'Sleep Disorders and Disturbances', 'Psychiatric disorders' SOC plus (2) HLGT 'Sleep disturbances (including subtypes)', 'Nervous system' SOC. Numerous duplicated preferred terms e.g. middle insomnia.

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Cataplexy | 10007737 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Exploding head syndrome | 10080684 |
| Hypersomnia | 10020765 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Insomnia related to another mental condition | 10022443 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Nightmare | 10029412 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Parasomnia | 10061910 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-------------------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep attacks | 10040981 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, parasomnia type | 10040988 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |
| HLGT Sleep disturbances (incl subtypes), HLGT code 10040998 | |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Central-alveolar hypoventilation | 10007982 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Hypersomnia | 10020765 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Microsleep | 10076954 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Sleep apnoea syndrome | 10040979 |
| Sleep deficit | 10080881 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Sudden onset of sleep | 10050014 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |

# 14.12.12. Injection site Reactions

Use eCRF terms for ISR.

#### 14.12.13. Seizures

Medical concept of seizures. Only narrow terms from SMQ 'Convulsions' selected plus selected PTs of possible seizure events from HLT 'Disturbances in consciousness NEC' under SOC 'Nervous systems disorders' and HLT 'Confusion and disorientation' under SOC 'Psychiatric disorders'.

| SMQ: 'Convulsions' SMQ Code: 20000079 Category: A Scope: Narrow | |
|-----------------------------------------------------------------|----------|
| Preferred Term | PT Code |
| 1p36 deletion syndrome | 10082398 |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Convulsion in childhood | 10052391 |
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |

| SMQ: 'Convulsions' SMQ Code: 20000079 Category: A Scope: Narrow | |
|-----------------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Generalised non-convulsive epilepsy | 10018090 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| Grey matter heterotopia | 10082084 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |

| Lafora's myoclonic epilepsy 1005 Lennox-Gastaut syndrome 1004 Migraine-triggered seizure 1007 Molybdenum cofactor deficiency 1006 Multiple subpial transection 1007 Myoclonic epilepsy 1005 Myoclonic epilepsy and ragged-red fibres 1006 Neonatal epileptic seizure 1008 Neonatal seizure 1008 Partial seizures 1006 Partial seizures 1006 Petit mal epilepsy 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal pychosis 1007 Post-traumatic epilepsy 1003 Schizencephaly 1003 Scizure 1007 Scizure 1007 Scizure 1007 | |
|---|---|
| Lafora's myoclonic epilepsy 1005 Lennox-Gastaut syndrome 1004 Migraine-triggered seizure 1007 Molybdenum cofactor deficiency 1006 Multiple subpial transection 1007 Myoclonic epilepsy 1005 Myoclonic epilepsy and ragged-red fibres 1006 Neonatal epileptic seizure 1008 Neonatal seizure 1008 Partial seizures 1006 Partial seizures with secondary generalisation 1005 Petit mal epilepsy 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal pychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1003 Scizure 1000 | Code |
| Lennox-Gastaut syndrome Migraine-triggered seizure 1007 Molybdenum cofactor deficiency 1006 Multiple subpial transection 1007 Myoclonic epilepsy 1005 Myoclonic epilepsy and ragged-red fibres 1006 Neonatal epileptic seizure 1008 Neonatal seizure 1008 Partial seizures 1006 Partial seizures with secondary generalisation 1005 Petit mal epilepsy 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1007 Postictal state 1008 Postictal state 1009 Schizencephaly 1003 Schizencephaly 1003 | 71082 |
| Migraine-triggered seizure 1007 Molybdenum cofactor deficiency 1006 Multiple subpial transection 1007 Myoclonic epilepsy 1005 Myoclonic epilepsy and ragged-red fibres 1006 Neonatal epileptic seizure 1008 Neonatal seizure 1008 Partial seizures 1006 Partial seizures 1006 Partial seizures with secondary generalisation 1005 Petit mal epilepsy 1003 Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Post ictal paralysis 1005 Postictal paralysis 1005 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1003 Schizencephaly 1003 Seizure 1003 | 54030 |
| Molybdenum cofactor deficiency Multiple subpial transection Myoclonic epilepsy Myoclonic epilepsy and ragged-red fibres Neonatal epileptic seizure Neonatal seizure Partial seizures Partial seizures with secondary generalisation Petit mal epilepsy Post stroke epilepsy Post stroke seizure Postictal headache Postictal paralysis Postictal psychosis Postictal state Post-traumatic epilepsy Seizure 1003 1004 1005 1006 1007 | 18816 |
| Multiple subpial transection Myoclonic epilepsy Myoclonic epilepsy and ragged-red fibres Neonatal epileptic seizure Neonatal seizure Partial seizures Partial seizures with secondary generalisation Petit mal epilepsy Polymicrogyria Post stroke epilepsy Post stroke seizure 1007 Post ctal headache Postictal paralysis Postictal prachysis Postictal state Post-traumatic epilepsy Seizure 1003 Seizure 1006 1006 1007 1008 1008 1009 1007 | 76676 |
| Myoclonic epilepsy1005Myoclonic epilepsy and ragged-red fibres1006Neonatal epileptic seizure1008Neonatal seizures1006Partial seizures with secondary generalisation1005Petit mal epilepsy1003Polymicrogyria1007Post stroke epilepsy1007Post stroke seizure1007Postictal headache1005Postictal paralysis1005Postictal state1004Post-traumatic epilepsy1003Schizencephaly1007Seizure1003 | 59687 |
| Myoclonic epilepsy and ragged-red fibres Neonatal epileptic seizure 1008 Neonatal seizure 1006 Partial seizures 1006 Partial seizures with secondary generalisation Petit mal epilepsy 1003 Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1006 Postictal headache 1007 Postictal paralysis 1005 Postictal pychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1007 Seizure 1007 | 79825 |
| Neonatal epileptic seizure1008Neonatal seizures1006Partial seizures with secondary generalisation1005Petit mal epilepsy1003Polymicrogyria1007Post stroke epilepsy1007Post stroke seizure1007Postictal headache1005Postictal paralysis1005Postictal state1004Post-traumatic epilepsy1003Schizencephaly1007Seizure1003 | 54859 |
| Neonatal seizure 1008 Partial seizures 1006 Partial seizures with secondary generalisation 1005 Petit mal epilepsy 1003 Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1003 Seizure 1003 | 59825 |
| Partial seizures 1006 Partial seizures with secondary generalisation 1005 Petit mal epilepsy 1003 Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1003 Seizure 1003 | 32068 |
| Partial seizures with secondary generalisation Petit mal epilepsy 1003 Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1003 | 32067 |
| Petit mal epilepsy 1003 Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1000 | 51334 |
| Polymicrogyria 1007 Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1007 | 56209 |
| Post stroke epilepsy 1007 Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1008 | 34759 |
| Post stroke seizure 1007 Postictal headache 1005 Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1000 | 73489 |
| Postictal headache Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1008 | 76982 |
| Postictal paralysis 1005 Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1003 | 76981 |
| Postictal psychosis 1007 Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1003 | 52470 |
| Postictal state 1004 Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1003 | 52469 |
| Post-traumatic epilepsy 1003 Schizencephaly 1007 Seizure 1003 | 70669 |
| Schizencephaly 1007 Seizure 1003 | 18727 |
| Seizure 1003 | 36312 |
| | 73487 |
| Saigura anavia | 39906 |
| Seizure anoxic 1005 | 39907 |
| Seizure cluster 1007 | 71350 |

| SMQ: 'Convulsions' SMQ Code: 20000079 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |
| Additional selected preferred terms from HLT 'Disturbances in consciousness NEC' under SOC 'Nervous systems disorders' and HLT 'Confusion and disorientation' under SOC 'Psychiatric disorders'. | |
| Preferred Term | PT Code |
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10001854 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |
#### 14.12.14. Weight Gain

Medical concept of weight gain. Selected PTs from HLT 'General nutritional disorders NEC', under SOC 'Metabolism and nutrition disorders', and HLT 'Physical examination procedures and organ system status', under SOC 'Investigations' and HLT 'General signs and symptoms NEC', under SOC 'General disorders and administration site conditions'.

| Preferred Term | PT Code |
|-------------------------------|----------|
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |
| Weight abnormal | 10056814 |
| Weight increased | 10047899 |
| Waist circumference increased | 10064863 |
| Body mass index abnormal | 10074506 |
| Body mass index increased | 10005897 |
| Fat tissue increased | 10016251 |

### 14.12.15. Rhabdomyolysis

Medical concept of rhabdomyolysis. Only narrow terms only for SMQ 'Rhabdomyolysis/myopathy' plus 2 additional preferred terms selected from HGLT 'muscle disorders' under SOC 'Musculoskeletal and connective tissue disorders'

| SMQ: 'Rhabdomyolysis/myopathy' SMQ Code: 20000002 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present | 10028631 |
| Myoglobinaemia | 10058735 |

| SMQ: 'Rhabdomyolysis/myopathy' SMQ Code: 20000002 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |
| Additional selected preferred terms from HLGT 'muscle disorders' under SOC 'Musculoskeletal and connective tissue disorders' | |
| Preferred Term | PT Code |
| Myalgia | 10028411 |
| Myositis | 10028653 |

### 14.12.16. Pancreatitis

Medical concept of acute pancreatitis. Only narrow terms of SMQ 'Acute pancreatitis' selected. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms).

| SMQ: 'Acute pancreatitis' SMQ Code: 20000022 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Hereditary pancreatitis | 10056976 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |

| SMQ: 'Acute pancreatitis' SMQ Code: 20000022 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Pancreatic abscess | 10048984 |
| Pancreatic cyst drainage | 10082531 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic necrosis | 10058096 |
| Pancreatic phlegmon | 10056975 |
| Pancreatic pseudoaneurysm | 10081762 |
| Pancreatic pseudocyst | 10033635 |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatitis | 10033645 |
| Pancreatitis acute | 10033647 |
| Pancreatitis haemorrhagic | 10033650 |
| Pancreatitis necrotising | 10033654 |
| Pancreatitis relapsing | 10033657 |
| Pancreatorenal syndrome | 10056277 |

### 14.12.17. Impact on Creatinine

Medical concept of worsening renal function/renal failure in the context of impact on creatinine. Only narrow terms from SMQ 'Acute renal failure' plus all PTs from HLT 'Renal failure and impairment', under SOC 'Renal and urinary disorders'. Numerous duplicated preferred terms e.g. renal failure

| SMQ: 'Acute renal failure' SMQ Code: 20000003 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |

| SMQ: 'Acute renal failure'<br>SMQ Code: 20000003<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment | 10078987 |
| Haemodialysis | 10018875 |
| Haemofiltration | 10053090 |
| Neonatal anuria | 10049778 |
| Nephropathy toxic | 10029155 |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |
| Prerenal failure | 10072370 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Subactute kidney injury | 10081980 |

| SMQ: 'Acute renal failure'<br>SMQ Code: 20000003<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Plus, all PTs from HLT 'Renal failure and impairment' under SOC 'Renal and urinary disorders' | |
| Preferred Term | PT Code |
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Foetal renal impairment | 10078987 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Nail-patella syndrome | 10063431 |
| Neonatal anuria | 10049778 |
| Oliguria | 10030302 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Prerenal failure | 10072370 |
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |

| SMQ: 'Acute renal failure' SMQ Code: 20000003 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Renal impairment | 10062237 |

| SMQ: 'Acute renal failure' SMQ Code: 20000003 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Renal impairment neonatal | 10049776 |
| Renal injury | 10061481 |
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |

# 14.12.18. Safety During Pregnancy

Use AE terms co-reported in pregnancy exposures to CAB.

# 14.13. Appendix 13: Abbreviations & Trade Marks

## 14.13.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| BMD | Bone Mineral Density |
| BMI | Body Mass Index |
| CAB | Cabotegravir |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CMH | Cochran-Mantel-Haenszel |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTR | Clinical Trial Register |
| CVb | Coefficient of Variation (Between) |
| CVb / CVw | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| CVD | Cardiovascular Disease |
| CVF | Confirmed Virologic Failure |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Place |
| DTG | Dolutegravir |
| eCRF | Electronic Case Record Form |
| eGFR | Estimated Glomerular Filtration Rate |
| EMA | European Medicines Agency |
| ERDF | Efficacy Related Discontinuation Failure |
| ES | Extension Switch Population |
| FDA | Food and Drug Administration |
| FSFV | First Subject First Visit |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HIV | Human Immunodeficiency Virus |
| HSR | Hypersensitivity Reaction |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| INI | Integrase Inhibitors |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| ITT-E | Intent-To-Treat Exposed |
| LOCF | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| NCEP | National Cholesterol Education Program |
| NNRTI | Non-Nucleoside Reverse Transcriptase Inhibitors |
| NQ | Non Quantifiable |
| NRTI | Nucleoside Reverse Transcriptase Inhibitors |
| OC | Observed Case |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PI | Protease Inhibitors |
| PK | Pharmacokinetic |
| PopPK | Population PK |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAMOS | Randomisation & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| RPV | Rilpivirine |
| SAE | Serious Adverse Event |
| SAC | Statistical Analysis Complete |
| SD | Standard Deviation |
| SDAC | Statistics Data Analysis Centre |
| SDTM | Study Data Tabulation Model |
| SMQ | Standardized MedDRA Queries |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation Failure |

## 14.13.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| Dolutegravir |
| Triumeq |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|
| NONMEM |
| Rilpivirine |
| SAS |
| WinNonlin |

### 14.14. Appendix 14: List of Data Displays for Week 48/Week 96

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

## 14.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-----------------------------------|-------------|-------------|
| Study Population | 1.01 to 1.n | 1.01 to 1.n |
| Efficacy | 2.01 to 2.n | 2.01 to 2.n |
| Safety | 3.01 to 3.n | 3.01 to 3.n |
| Pharmacokinetic | 4.01 to 4.n | 4.01 to 4.n |
| Pharmacokinetic / Pharmacodynamic | 5.01 to 5.n | 5.01 to 5.n |
| Health Outcomes | 6.01 to 6.n | 6.01 to 6.n |
| Virology | 7.01 to 7.n | 7.01 to 7.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

### 14.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided a separate document.

#### 14.14.3. Deliverables

| Delivery [1] | Description |
|--------------|---------------------|
| HL | Headline at Week 48 |
| W48 | Week 48 |
| W96 | Week 96 |
| EOS | End of study |

#### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 14.14.4. Study Population Tables

| oludy | Population Ta | l | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Subje | ct Disposition | | | | |
| 1.1. | All Subjects<br>Screened | SA1 | Summary of Study Populations | CS CORE For W96: add column for 'Switch Q4W' | HL, W48,<br>W96, EOS |
| 1.2. | All Subjects<br>Screened | Shell TSP1 | Summary of Subjects by Country and Investigator | For W96: add column for 'Switch Q4W' | W48, W96,<br>EOS |
| 1.3. | All Subjects<br>Screened | ES6 | Summary of Screening Status and Reasons for Screening Failures | CS CORE | W48, W96,<br>EOS |
| 1.4. | All Enrolled | EudraCT age | Summary of Age Categories | CS CORE | W48, W96,<br>EOS |
| 1.5. | ITT-E | ES1 | Summary of Subject Accountability: Study Conclusion Record | ICH E3, GSK CTR, FDAAA,<br>EudraCT<br>For W96: add column for 'Switch<br>Q4W' | W48, W96,<br>EOS |
| 1.6. | ITT-E | ES1 | Summary of Study Drug Discontinuation | CS CORE For W96: add column for 'Switch Q4W' | W48, W96,<br>EOS |
| 1.7. | ITT-E | ES1 | Summary of Subject Accountability: Maintenance Phase Conclusion Record | ICH E3, GSK CTR, FDAAA,<br>EudraCT | HL, W48,<br>W96 |
| 1.8. | LTFU | ES1 | Summary of Subject Accountability: Long-term follow up Phase Conclusion Record | ICH E3, GSK CTR, FDAAA,<br>EudraCT<br>For W96: add column for 'Switch<br>Q4W' | W48, W96,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.9. | ITT-E | HIV_ES1 | Summary of Subject Accountability: Withdrawals by Visit - Maintenance Phase | | W48, W96 |
| 1.10. | ITT-E | ES1 | Summary of Subject Accountability: Maintenance and Extension Phase Conclusion Record (Randomized Q4W) | For Randomized Q4W arm only Add the following subcategories under subject status: a) Completed Maintenance and did not enter Extension b) Completed Extension c) Withdrawn from Maintenance d) Withdrawn from Extension. | W96, EOS |
| 1.11. | ITT-E | HIV_ES1 | Summary of Subject Accountability: Withdrawals by Visit – Maintenance and Extension Phase (Randomized Q4W) | For Randomized Q4W arm only | W96, EOS |
| 1.12. | ES | ES1 | Summary of Subject Accountability: Extension Phase Conclusion Record (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 1.13. | ES | HIV_ES1 | Summary of Subject Accountability: Withdrawals by Visit – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 1.14. | All<br>Participants<br>Enrolled | ES4 | Summary of Subject Disposition at Each Study Epoch | See Mid200056//wk96cdisc/Table 6.1006 For W96: add column for 'Switch Q4W' | W48, W96,<br>EOS |
| 1.15. | All<br>Participants<br>Enrolled | ES5 | Summary of Reasons for Withdrawal at Each Epoch | See Mid200056//wk96cdisc/Table 6.1007 For W96: add column for 'Switch Q4W' | W48, W96,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.16. | ITT-E | DV1a | Summary of Important Protocol Deviations (Maintenance Phase) | CS CORE | W48, W96 |
| 1.17. | ITT-E | DV1a | Summary of Important Protocol Deviations -<br>Maintenance and Extension Phase (Randomized<br>Q4W) | CS CORE<br>For Randomized Q4W arm only | W96, EOS |
| 1.18. | ES | DV1a | Summary of Important Protocol Deviations – Extension Phase (Extension Switch Population) | CS CORE<br>Switch Q4W IM group only | W96, EOS |
| 1.19. | ITT-E | SP2 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population (Week X Analysis) [X =Week 48 or Week 96, depending on the deliverable)] | CS CORE Exclude deviations occurring during the Extension phase | W48, W96 |
| 1.20. | ITT-E | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | W48, W96,<br>EOS |
| 1.21. | All<br>Participants<br>Enrolled | ES1 | Summary of Subject Accountability: Induction Phase Conclusion Record | ICH E3, GSK CTR, FDAAA,<br>EudraCT | W48 |
| Demo | graphy and Ba | seline | | | |
| 1.22. | ITT-E | Shell TSP2 | Summary of Demographic Characteristics | See also DM1 in IDSL Age categorization will include: <=18, 19-64, >=65 (FDAAA requirement) 18-64, 65-84, >=85 (EMA requirement) | HL, W48,<br>W96, EOS |
| 1.23. | ITT-E | DM5 | Summary of Race and Racial Combinations | CS CORE | W48, W96,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.24. | ITT-E | DM6 | Summary of Race and Racial Combinations Details | CS CORE | W48, W96,<br>EOS |
| 1.25. | ITT-E | Shell TSP3 | Summary of Hepatitis Status at Induction Baseline (Week -20) | | W48, W96,<br>EOS |
| 1.26. | ITT-E | CDC1 | Summary of Derived CDC Stages of HIV Infection at Maintenance Baseline (Day 1) | | W48, W96,<br>EOS |
| 1.27. | ITT-E | Shell TSP4 | Summary of Induction Baseline (Week -20) Cardiovascular Risk Assessments | | W48, W96,<br>EOS |
| 1.28. | ITT-E | Shell TSP5 | Distribution of CD4+ Cell Count Results at Maintenance Baseline (Day 1) | Same presentation as shown in the mock shell for induction baseline. | W48, W96,<br>EOS |
| 1.29. | ITT-E | Shell TSP5 | Distribution of Quantitative Plasma HIV-1 RNA and CD4+ Cell Count Results at Screening and Induction Baseline (Week -20) | | W48, W96,<br>EOS |
| Medic | al Conditions, | Concomitant M | edications & Antiretroviral Therapy | | |
| 1.30. | ITT-E | MH1 | Summary of Current Medical Conditions | CS CORE | W48, W96,<br>EOS |
| 1.31. | ITT-E | MH1 | Summary of Past Medical Conditions | CS CORE | W48, W96,<br>EOS |
| 1.32. | ITT-E | MH4 | Summary of Current Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal and<br>Urinary, Nervous System Conditions, and<br>Hepatobiliary disorders | | W48, W96,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.33. | ITT-E | MH4 | Summary of Past Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal and<br>Urinary, Nervous System Conditions, and<br>Hepatobiliary disorders | | W48, W96,<br>EOS |
| 1.34. | ITT-E | CM8 | Summary of Concomitant Medication Ingredient Combinations (Maintenance Phase) | | W48, W96 |
| 1.35. | ITT-E | CM8 | Summary of Concomitant Medication Ingredient<br>Combinations - Maintenance and Extension Phase<br>(Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 1.36. | ES | CM8 | Summary of Concomitant Medication Ingredient<br>Combinations – Extension Phase (Extension Switch<br>Population) | Switch Q4W IM group only | W96, EOS |
| 1.37. | ITT-E | Shell TSP11 | Summary of Alternate Background NRTI Therapy at End of Induction Phase | | W48, W96,<br>EOS |
| 1.38. | ITT-E | Shell TSP9 | Summary of Lipid Modifying Agent Use at Maintenance Baseline (Day 1) | taken during the 12 weeks before<br>the first Maintenance Phase dose<br>of study drug | W48, W96,<br>EOS |
| 1.39. | ITT-E | Shell TSP10 | Summary of Lipid Modifying Agent Use Started During Maintenance | | W48, W96,<br>EOS |
| 1.40. | ITT-E | SU1 | Summary of Substance Use at Entry | | W48, W96,<br>EOS |
| 1.41. | ITT-E | Shell TSP12 | Summary of HIV Risk Factor | | W48, W96,<br>EOS |
| 1.42. | ITT-E | Shell TSP13 | Summary of Time from First HIV-1 RNA < 50 copies/mL until Initiation of Maintenance Phase Treatment | | W48, W96,<br>EOS |
| 1.43. | ITT-E | Shell CLAD1 | Summary of the Prevalence of HIV-1 Subtype | | W48, W96 |

# 14.14.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Primary Efficacy Analyses | | | | | |
| 2.1. | ITT-E | Shell TPEF1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-<br>1 RNA ≥50 c/mL at Week 48 (Maintenance Phase) – Snapshot<br>Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |
| 2.2. | Per-Protocol | Shell TPEF1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-<br>1 RNA ≥50 c/mL at Week 48 (Maintenance Phase) – Snapshot<br>Analysis (Per-Protocol Population) | For W96 deliverable, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |
| 2.3. | ITT-E | Shell TPEF2 | Summary of Study Outcomes (50 c/mL cut-off) at Week 48 (Maintenance Phase) – Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |
| 2.4. | ITT-E | Shell TPEF3 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL at Week 48 (Maintenance Phase) - Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |
| 2.5. | ITT-E | Shell TPEF4 | Summary of Analysis for Proportion of Subjects with Plasma HIV-<br>1 RNA ≥50 c/mL at Week 48 by Subgroup (Maintenance Phase) -<br>Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48, W96 |
| 2.6. | ITT-E | Shell TPEF5 | Summary of Study Outcomes (50 c/mL cut-off) at Week 48 by Subgroup (Maintenance Phase) – Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48, W96 |
| Second | dary Efficacy A | nalyses | | | |
| 2.7. | ITT-E | Shell TPEF1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |
| 2.8. | Per-Protocol | Shell TPEF1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis (Per-Protocol Population) | For W96 deliverable, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.9. | ITT-E | Shell TPEF3 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) - Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48, W96 |
| 2.10. | ITT-E | Shell TPEF4 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 by Subgroup (Maintenance Phase) - Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48, W96 |
| 2.11. | ITT-E | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.12. | ITT-E | Shell TSEF2.1 | Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL by Subgroup and Visit (Maintenance Phase) – Snapshot Analysis | | W48 |
| 2.13. | ITT-E | Shell TSEF7.0 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 48 - Treatment Related Discontinuation = Failure | For W96 deliverable, replace 'Week 52' with 'Week 100' | W48, W96 |
| 2.14. | ITT-E | Shell TSEF7.1 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 48 - Efficacy Related Discontinuation = Failure | For W96 deliverable, replace 'Week 52' with 'Week 100' | W48, W96 |
| 2.15. | ITT-E | Shell TSEF2.1 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.16. | ITT-E | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.17. | ITT-E | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA <200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.18. | ITT-E | Shell TSEF9 | Proportion of Subjects with HIV-1 RNA≥50 c/mL at Week 48 (Snapshot) by Last Delay in IP Injection (Maintenance Phase) | For Q4W IM arm only. The last delay in IP injection is the delay in IP injection at Week 48, or delay in last IP injection prior to Week 48 if a subject has no injection at WK48 (e.g., missing visit or early withdrawal) | W48 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.19. | ITT-E | Shell TSEF8 | Summary of Plasma HIV-1 RNA (log10 c/mL) by Visit (Maintenance Phase) | | W48, W96<br>EOS |
| 2.20. | ITT-E | Shell TSEF8 | Summary of Change from Maintenance Baseline (Day 1) in Plasma HIV-1 RNA (log10 c/mL) by Visit (Maintenance Phase) | | W96, EOS |
| 2.21. | ITT-E | Shell TSEF3 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria by Visit During the Maintenance Phase (Up to Week 52) | For Week 96 deliverable, show all visit up to Week 100. | HL, W48,<br>W96 |
| 2.22. | ITT-E | Shell TSEF3.1 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria During the Maintenance Phase | | HL, W48,<br>W96 |
| 2.23. | ITT-E | Shell TSEF3.1 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria During the Maintenance and Extension Phase (Randomized Q4W) | For Randomized Q4W arm only | W96, EOS |
| 2.24. | ES | Shell TSEF3.1 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria During the Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 2.25. | CVF | Shell TSEF4 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure – Maintenance Phase | | W48, W96 |
| 2.26. | ITT-E | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD4+Cell Count (cells/mm^3) by Visit -Maintenance Phase | Visits starting from Maintenance<br>Baseline (Day 1), Week 4, | W48, W96 |
| 2.27. | ITT-E | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD4+<br>Cell Count (cells/mm^3) by Visit - Maintenance and Extension<br>Phase (Randomized Q4W) | Visits starting from Maintenance<br>Baseline (Day 1), Week 4, | EOS |
| 2.28. | ES | Shell TSEF5 | Summary of Change from Extension Baseline (Week 100) in CD4+ Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | | EOS |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.29. | ITT-E | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD4+<br>Cell Count (cells/mm^3) at Week 48 by Subgroup (Maintenance<br>Phase) | Visits starting from Maintenance<br>Baseline (Day 1), Week 4,<br>For W96 deliverable, replace 'Week<br>48' with 'Week 96' | W48, W96 |
| 2.30. | ITT-E | Shell TSEF5 | Summary of CD4+ Cell Count (cells/mm^3) by Visit– Induction and Maintenance Phase | Visits starting from Induction<br>Baseline (Week -20), Week -16, | W48, W96,<br>EOS |
| 2.31. | ITT-E | Shell TSEF5 | Summary of CD4+ Cell Count (cells/mm^3) by Visit – Maintenance and Extension Phase (Randomized Q4W) | Visits starting from Induction<br>Baseline (Week -20), Week -16, | EOS |
| 2.32. | ES | Shell TSEF5 | Summary of CD4+ Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | | EOS |
| 2.33. | ITT-E | Shell TSEF5 | Summary of CD8+ Cell Count (cells/mm^3) by Visit – Induction + Maintenance Phase | Visits starting from Induction<br>Baseline (Week -20), Week -16, | W48, W96,<br>EOS |
| 2.34. | ITT-E | Shell TSEF5 | Summary of CD8+ Cell Count (cells/mm^3) by Visit – Maintenance and Extension Phase (Randomized Q4W) | Visits starting from Induction<br>Baseline (Week -20), Week -16, | EOS |
| 2.35. | ES | Shell TSEF5 | Summary of CD8+ Cell Count (cells/mm^3) by Visit– Extension Phase (Extension Switch Population) | | EOS |
| 2.36. | ITT-E | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD8+Cell Count (cells/mm^3) by Visit – Maintenance Phase) | Visits starting from Induction Maintenance Baseline, Week 4, | W48, W96, |
| 2.37. | ITT-E | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD8+<br>Cell Count (cells/mm^3) by Visit – Maintenance and Extension<br>Phase (Randomized Q4W) | Visits starting from Maintenance<br>Baseline (Day 1), Week 4, | EOS |
| 2.38. | ES | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD8+<br>Cell Count (cells/mm^3) by Visit – Extension Phase (Extension<br>Switch Population) | | EOS |
| 2.39. | ITT-E | Shell TSEF5 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit – Induction and Maintenance Phase | While both CD4+ and CD8+ are available on the same date | W48, W96 |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.40. | ITT-E | Shell TSEF5 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit – Induction, Maintenance and Extension Phase (Randomized Q4W) | For Randomized Q4W arm only | EOS |
| 2.41. | ES | Shell TSEF5 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | | EOS |
| 2.42. | ITT-E | HIV1/Shell<br>TSEF 6.0 | Summary of Maintenance Phase HIV-1 Associated Conditions Including Recurrences | | W48, W96 |
| 2.43. | ITT-E | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Including Recurrences - Maintenance and Extension Phase (Randomized Q4W) | For Randomized Q4W arm only | EOS |
| 2.44. | ES | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Including Recurrences – Extension Phase (Extension Switch Population) | | EOS |
| 2.45. | ITT-E | HIV1/Shell<br>TSEF 6.0 | Summary of Maintenance Phase HIV-1 Associated Conditions Excluding Recurrences | | W48, W96 |
| 2.46. | ITT-E | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Excluding Recurrences - Maintenance and Extension Phase (Randomized Q4W) | For Randomized Q4W arm only | EOS |
| 2.47. | ES | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Excluding Recurrences – Extension Phase (Extension Switch Population) | | EOS |
| 2.48. | ITT-E | HIV2/Shell<br>TSEF6.1 | Summary of HIV-1 Disease Progression and/or Deaths (Maintenance Phase) | | W48, W96 |
| 2.49. | ITT-E | HIV2/Shell<br>TSEF6.1 | Summary of HIV-1 Disease Progressions and/or Deaths - Maintenance and Extension Phase (Randomized Q4W) | For Randomized Q4W arm only | EOS |
| 2.50. | ES | HIV2/Shell<br>TSEF6.1 | Summary of HIV-1 Disease Progressions – Extension Phase (Extension Switch Population) | | EOS |
| 2.51. | ITT-E | TSEF12 | Proportion of Subjects with Plasma HIV-1 RNA <2 copies/mL by Visit - Observed Case Analysis (Maintenance Phase) | | W48, W96 |
| 2.52. | ITT-E | Shell TPEF2 | Summary of Study Outcomes (200 c/mL) at Week 48 (Maintenance Phase) – Snapshot Analysis | For W96 analysis, replace 'Week 48' with 'Week 96' | W48, W96 |
| 2.53. | ITT-E | Shell TSEF11 | Summary of Subjects per Viral Load Category by Visit – Maintenance Phase) | | W48, W96 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.54. | All<br>Participants<br>Enrolled | | | Induction Baseline (Week -20),<br>Week -16, Week -8, Week -4 and<br>Day 1. Single arm for Induction<br>ABC/DTG/3TC | W48 |

# 14.14.6. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primar | / Efficacy Anal | yses | | | |
| 2.1. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.2. | ITT - E | Shell FPEF2 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL at Week 48 by Subgroup – Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48, W96 |
| 2.3. | ITT-E | SNAPSHOT9B | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA >= 50 c/mL at Week 96 by Selected Demographic Subgroups (Maintenance Phase) - Snapshot Analysis | Include: Overall, Gender at Birth (Female, Male), Age (<35, 35-<50, >=50), Induction Baseline (Week - 20) BMI (<30, >=30), Region (Western/Central Europe and North America, Russian Federation, Japan, South Africa). | W96 |

| Effica | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | ITT-E | SNAPSHOT9B | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA >= 50 c/mL at Week 96 by Selected HIV Disease Characteristic Subgroups (Maintenance Phase) - Snapshot Analysis | Include: Overall, Induction BL<br>(Week -20) HIV-1 RNA (<100,000,<br>>=100,000), Induction BL (Week -<br>20) CD4+ cell count (<200, 200 to<br><350, 350 to <500, >=500), HIV-1<br>Subtype (A, A1, AE, Ag, B, C,<br>Other) | W96 |
| Secon | dary Efficacy A | nalyses | | | |
| 2.5. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.6. | ITT-E | SNAPSHOT9B | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA < 50 c/mL at Week 96 by Selected Demographic Subgroups (Maintenance Phase) - Snapshot Analysis | Include: Overall, Gender at Birth (Female, Male), Age (<35, 35-<50, >=50), Induction Baseline (Week - 20) BMI (<30, >=30), Region (Western/Central Europe and North America, Russian Federation, Japan, South Africa). | W96 |
| 2.7. | ITT-E | SNAPSHOT9B | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA < 50 c/mL at Week 96 by Selected HIV Disease Characteristic Subgroups (Maintenance Phase) - Snapshot Analysis | Include: Overall, Induction BL<br>(Week -20) HIV-1 RNA (<100,000,<br>>=100,000), Induction BL (Week -<br>20) CD4+ cell count (<200, 200 to<br><350, 350 to <500, >=500), HIV-1<br>Subtype (A, A1, AE, Ag, B, C,<br>Other) | W96 |
| 2.8. | ITT - E | Shell FPEF2 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week 48 by Subgroup – Snapshot Analysis | For W96 analysis, replace 'Week 48' with 'Week 96' | W48, W96 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.9. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA <200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.10. | ITT-E | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA (log10 copies/mL) Profiles by Visit– for CVF subjects (Randomized Q4W) | The first vertical line indicates start of Induction phase investigational product (ABC/DTG/3TC or DTG). The second vertical line indicates start of Maintenance phase investigational product (oral CAB + oral RPV). The third vertical reference line indicates last ontreatment study day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB+RPV+1), day of LTFU HAART start date). This line is only for participants who withdraw from the Maintenance/Extension phase. | HL, W48,<br>W96, EOS |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.11. | ITT-E | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA (log10 copies/mL) Profiles by Visit – for CVF subjects (Randomized ABC/DTG/3TC arm) | The first vertical line indicates start of Induction phase investigational product (ABC/DTG/3TC or DTG). The second vertical line indicates start of Maintenance phase investigational product (continuation of ABC/DTG/3TC or DTG). The third vertical reference line indicates last Maintenance phase on-treatment study day, i.e. day of last ABC/DTG/3TC (or DTG) dose + 1. This line is only for participants who withdraw or complete the Maintenance phase. The fourth vertical reference line indicates last Extension Phase ontreatment study day, i.e. min (max (day of last IP injection dose+35 days, day of last oral CAB+RPV+1), day of LTFU HAART start date). This line is only for participants who withdraw from the Extension phase. | HL, W48,<br>W96, EOS |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.12. | ITT - E | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA for subjects who are in the category of 'HIV-1 RNA ≥50 c/mL' at Week 48 per Snapshot algorithm (Randomized Q4W arm) | The first vertical line indicates start of Induction phase investigational product (ABC/DTG/3TC or DTG). The second vertical line indicates start of Maintenance phase investigational product (oral CAB + oral RPV). The third vertical reference line indicates last ontreatment study day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB+RPV+1), day of LTFU HAART start date). This line is only for participants who withdraw from the Maintenance/Extension phase. For W96 analysis, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.13. | ITT - E | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA for subjects who are in the category of 'viral load ≥50 c/mL' at Week 48 per Snapshot algorithm (Randomized ABC/DTG/3TC arm) | The first vertical line indicates start of Induction phase investigational product (ABC/DTG/3TC or DTG). The second vertical line indicates start of Maintenance phase investigational product (continuation of ABC/DTG/3TC or DTG). The third vertical reference line indicates last Maintenance phase on-treatment study day, i.e. day of last ABC/DTG/3TC (or DTG) dose + 1. This line is only for participants who withdraw or complete the Maintenance phase. The fourth vertical reference line indicates last Extension Phase ontreatment study day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB+RPV+1), day of LTFU HAART start date). This line is only for participants who withdraw from the Extension phase. For W96 analysis, replace 'Week 48' with 'Week 96' | HL, W48,<br>W96 |
| 2.14. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA >=200 c/mL by Visit – Snapshot Analysis | | W48, W96 |

# 14.14.7. Safety Tables

| Safety | Tables (Display | ys will be for both tr | eatment arms, unless specified) | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | sure | • | | | |
| 3.1. | Safety | Shell TS1.1 | Summary of Extent of Exposure to Investigational Product – Maintenance Phase | CS Core | W48, W96,<br>EOS |
| 3.2. | Safety | Shell TS1.1 | Summary of Extent of Exposure to Investigational Product – Maintenance Phase and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |
| 3.3. | ES | Shell TS1.1 | Summary of Extent of Exposure to Investigational Product – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | W96, EOS |
| 3.4. | Safety | Study 201584<br>(primary_02):<br>Table 3.114 | Summary of Categorized Needle Length and Gauge for CAB Injection - Maintenance Phase | Randomized Q4W arm only | W48, W96 |
| 3.5. | Safety | Study 201584<br>(primary_02):<br>Table 3.115 | Summary of Categorized Needle Length and Gauge for RPV Injection - Maintenance Phase | Randomized Q4W arm only | W48, W96 |
| 3.6. | Safety | Shell TS1.3 | Summary of Adherence to Q4W IM Dosing Schedule - Maintenance Phase | (only for randomized Q4W arm) please refer to Section 14.6.2 Adherence to CAB/RPV Injection Schedule | W48, W96 |
| Adver | se Events | | | | |
| 3.7. | Safety | AE1 | Summary of All Adverse Events by System Organ Class – Maintenance Phase | CS Core | W48, W96 |
| 3.8. | Safety | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Maintenance Phase | CS Core | HL, W48, W96 |
| 3.9. | Safety | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | ES | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | W96, EOS |
| 3.11. | Safety | AE5B | Summary of All On-treatment Adverse Events by System<br>Organ Class and Maximum Toxicity – Maintenance Phase | CS Core | W48, W96 |
| 3.12. | LTFU | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Long-term Follow-up Phase | CS Core | EOS |
| 3.13. | Safety | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Oral Lead-in Period at Maintenance Phase | CS Core<br>Randomized Q4W arm only | HL, W48 |
| 3.14. | Safety | AE3 | Summary of Common Adverse Events (>=5%) by Overall Frequency – Maintenance Phase | CS Core | W48, W96 |
| 3.15. | Safety | AE3 | Summary of Common Grade 2-5 Adverse Events (>=1%) by Overall Frequency – Maintenance Phase | | W48, W96 |
| 3.16. | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class– Maintenance Phase | | W48, W96 |
| 3.17. | Safety | AE5B | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Toxicity – Maintenance Phase | CS Core | HL, W48, W96 |
| 3.18. | Safety | AE5B | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |
| 3.19. | ES | AE5B | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | W96, EOS |
| 3.20. | Safety | AE3 | Summary of All Drug-Related Grade 2-5 Adverse Events by Overall Frequency – Maintenance Phase | | W48, W96 |
| Seriou | s and Other Sig | gnificant Adverse | Events | | |
| 3.21. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class – Maintenance Phase | CS Core | HL, W48, W96 |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.22. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |
| 3.23. | ES | AE1 | Summary of Serious Adverse Events by System Organ Class – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | W96, EOS |
| 3.24. | LTFU | AE1 | Summary of Serious Adverse Events by System Organ Class – Long term follow up | CS Core | W48, W96,<br>EOS |
| 3.25. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class — Oral Lead-in Period at Maintenance Phase | CS Core<br>Randomized Q4W arm only | HL, W48 |
| 3.26. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class – Maintenance Phase | CS Core | W48, W96 |
| 3.27. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |
| 3.28. | ES | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM only | W96, EOS |
| 3.29. | Safety | AE3 | Summary of Non-Fatal Serious Adverse Events by Overall Frequency – Maintenance Phase | | W48, W96 |
| 3.30. | Safety | AE3 | Summary of Drug-Related Non-Fatal Serious Adverse Events by Overall Frequency – Maintenance Phase | | W48, W96 |
| 3.31. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class – Maintenance Phase | CS Core | HL, W48, W96 |
| 3.32. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by SOC – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |

| Safety | Tables (Display | s will be for both tr | eatment arms, unless specified) | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.33. | ES | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by SOC – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | W96, EOS |
| 3.34. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by SOC – Oral Lead-in Period at Maintenance Phase | CS Core<br>Randomized Q4W arm only | W48, W96 |
| 3.35. | Safety | AE3 | Summary of Common (>=5%) Non-Serious Adverse Events by Overall Frequency – Maintenance Phase | CS Core | W48, W96 |
| 3.36. | Safety | EudraCT Non-<br>serious AE<br>AE15 | Summary of Subjects and Number of Occurrences of Common (>=5%) Non-Serious Adverse Events by System Organ Class – Maintenance Phase | CS Core for FDAAA and EMA disclosure requirements. EudraCT Use macro TD_AE4VCTR for New Data Disclosure HARP Reporting Tools | W48, W96 |
| 3.37. | Safety | EudraCT SAE<br>AE16 | Summary of Subjects and Number of Occurrences of SAEs,<br>Fatal SAEs, and Drug-related SAEs – Maintenance Phase | CS Core for FDAAA and EMA disclosure requirements. EudraCT | W48, W96 |
| 3.38. | Safety | Shell TS2.1 | Summary of Cumulative Adverse Events by Visit – Maintenance Phase | Please note this table only display AEs occurring >=5% subjects during Maintenance Phase | W48, W96 |
| 3.39. | All<br>Participants<br>Enrolled | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class – Induction Phase | CS Core | W48 |
| Injection | on Site Reaction | n Adverse Events | | | |
| 3.40. | Safety | Shell TS2.2 | Summary of Injection Site Reaction Adverse Events (Event-<br>Level Summary) – Maintenance Phase | Randomized Q4W arm only | HL, W48, W96 |
| 3.41. | Safety | Shell TS2.2 | Summary of Injection Site Reaction Adverse Events (Event-<br>Level Summary) – Maintenance and Extension Phase<br>(Randomized Q4W) | Randomized Q4W arm only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.42. | ES | Shell TS2.2 | Summary of Injection Site Reaction Adverse Events (Event-<br>Level Summary) – Extension Phase (Extension Switch<br>Population) | Switch Q4W IM group only | W96, EOS |
| 3.43. | Safety | Shell TS2.3 | Summary of Subject-Level Characteristics of Injection Site<br>Reaction Adverse Events (Overall and Common) –<br>Maintenance Phase | Common ISR includes pain,<br>induration, nodules and any other<br>ISR with ≥5% subjects (for<br>randomized Q4W arm only) | W48, W96 |
| 3.44. | Safety | Shell TS2.3 | Summary of Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Maintenance and Extension Phase (Randomized Q4W) | Common ISR includes pain,<br>induration, nodules and any other<br>ISR with ≥5% subjects (for<br>randomized Q4W arm only) | W96, EOS |
| 3.45. | ES | Shell TS2.3 | Summary of Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (Switch Q4W IM group only) | W96, EOS |
| 3.46. | Safety | Shell TS2.4 | Summary of Injection Site Reaction Adverse Events by Visit and Maximum Severity (Overall and Common) – Maintenance Phase | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for randomized Q4W arm only) | W48, W96 |
| 3.47. | Safety | Shell TS2.2 | Summary of CAB Drug-Related Injection Site Reaction<br>Adverse Events (Event-Level Summary) – Maintenance Phase | Randomized Q4W arm only | W48, W96 |
| 3.48. | Safety | Shell TS2.3 | Summary of CAB Drug-Related Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Maintenance Phase | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for Q4W arm only) | W48, W96 |
| 3.49. | Safety | Shell TS2.4 | Summary of CAB Drug-Related Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity (Overall and<br>Common) – Maintenance Phase | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for Q4W arm only) | W48, W96 |

| | | IDSL / TST ID / | | | Deliverable |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | [Priority] |
| 3.50. | Safety | Shell TS2.5 | Summary of Maximum CAB Drug-Related Injection Site<br>Reaction Adverse Event Grade by Needle Length (Common<br>ISRs) – Maintenance Phase | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for randomized Q4W arm only) | W48, W96 |
| 3.51. | Safety | Shell TS2.2 | Summary of RPV Drug-Related Injection Site Reaction<br>Adverse Events (Event-Level Summary) – Maintenance Phase | | W48, W96 |
| 3.52. | Safety | Shell TS2.3 | Summary of RPV Drug-Related Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Maintenance Phase | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for randomized Q4W arm only) | W48, W96 |
| 3.53. | Safety | Shell TS2.4 | Summary of RPV Drug-Related Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity (Overall and<br>Common) – Maintenance Phase | | W48, W96 |
| 3.54. | Safety | Shell TS2.5 | Summary of Maximum RPV Drug-Related Injection Site<br>Reaction Adverse Event Grade by Needle Length (Common<br>ISRs) – Maintenance Phase | Common ISR includes pain,<br>induration, nodules and any other<br>ISR with ≥5% subjects (for Q4W<br>arm only) | W48, W96 |
| Labora | atory: Chemisti | ry, Hematology and | d Renal Markers | | |
| 3.55. | Safety | LB1 | Summary of Chemistry Changes from Maintenance Baseline (Day 1) by Visit – Maintenance Phase | CS Core (include lipids and glucose in Conventional Units, renal markers of Retinol Binding Protein, Cystatin C, and CKD-EP1 GFR using Creatinine, and CKD-EP1 using Cystatin C et al | W48, W96 |

| Safety | Tables (Display | s will be for both tre | eatment arms, unless specified) | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.56. | Safety | LB1 | Summary of Chemistry Changes from Maintenance Baseline (Day 1) by Visit – Maintenance and Extension Phase (Randomized Q4W) | CS Core (include lipids and glucose in Conventional Units, renal markers of Retinol Binding Protein, Cystatin C, and CKD-EP1 GFR using Creatinine, and CKD-EP1 using Cystatin C et al) Randomized Q4W arm only | EOS |
| 3.57. | ES | LB1 | Summary of Chemistry Changes from Extension Baseline (Week 100) by Visit – Extension Phase (Extension Switch Population) | CS Core (include lipids and glucose in Conventional Units, renal markers of Retinol Binding Protein, Cystatin C, and CKD-EP1 GFR using Creatinine, and CKD-EP1 using Cystatin C et al) Switch Q4W IM group only | EOS |
| 3.58. | Safety | LB1 | Summary of Chemistry Values by Visit – Maintenance Phase | (include lipids and glucose in<br>Conventional Units, renal markers<br>of Retinol Binding Protein, Beta-2<br>Microglobulin, Cystatin C, et al) | W48, W96,<br>EOS |
| 3.59. | Safety | LB1 | Summary of Chemistry Values by Visit – Maintenance and Extension Phase (Randomized Q4W) | (include lipids and glucose in<br>Conventional Units, renal markers<br>of Retinol Binding Protein, Beta-2<br>Microglobulin, Cystatin C, et al) | EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.60. | ES | LB1 | Summary of Chemistry Values by Visit – Extension Phase (Extension Switch Population) | (include lipids and glucose in<br>Conventional Units, renal markers<br>of Retinol Binding Protein, Beta-2<br>Microglobulin, Cystatin C, et al) | EOS |
| 3.61. | Safety | LB1 | Summary of Hematology Changes from Maintenance Baseline (Day 1) by Visit – Maintenance Phase | Switch Q4W IM group only CS Core | W48, 96, EOS |
| 3.62. | Safety | LB1 | Summary of Hematology Changes from Maintenance Baseline (Day 1) by Visit – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | EOS |
| 3.63. | ES | LB1 | Summary of Hematology Changes from Maintenance Baseline (Day 1) by Visit – Extension Phase (Extension Switch Population) | CS Core | EOS |
| 3.64. | Safety | LB1 | Summary of Hematology Values by Visit – Maintenance Phase | CS Core | W48, W96,<br>EOS |
| 3.65. | Safety | LB1 | Summary of Hematology Values by Visit – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | EOS |
| 3.66. | ES | LB1 | Summary of Hematology Values by Visit – Extension Phase (Extension Switch Population) | CS Core | EOS |
| 3.67. | Safety | Shell TS9.1 | Summary of Maximum Maintenance Phase Emergent Chemistry Toxicities | CS Core | W48, W96 |
| 3.68. | Safety | Shell TS9.2 | Summary of Maximum Maintenance and Extension Phase Emergent Chemistry Toxicities (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |
| 3.69. | ES | Shell TS9.3 | Summary of Maximum Extension Phase Emergent Chemistry Toxicities – Extension Switch Population | CS Core<br>Switch Q4W IM group only | W96, EOS |

| Safety | Tables (Display | ys will be for both tr | eatment arms, unless specified) | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.70. | Safety<br>(Q4W IM<br>only) | Shell TS9.2 | Summary of Maximum Maintenance Phase Emergent<br>Chemistry Toxicities – Maintenance Phase Oral Lead-in<br>Period | CS Core<br>Randomized Q4W arm only | W48 |
| 3.71. | Safety | Shell TS9.1 | Summary of Maximum Maintenance Phase Emergent Hematology Toxicities | CS Core | W48, W96 |
| 3.72. | Safety | Shell TS9.2 | Summary of Maximum Maintenance and Extension Phase Emergent Hematology Toxicities (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | W96, EOS |
| 3.73. | ES | Shell TS9.3 | Summary of Maximum Extension Phase Emergent Hematology Toxicities – Extension Switch Population | CS Core (for ABC/DTG/3TC arm only | W96, EOS |
| 3.74. | Safety<br>(Q4W IM<br>only) | Shell TS9.2 | Summary of Maximum Maintenance Phase Emergent<br>Hematology Toxicities – Maintenance Phase Oral Lead-in<br>Period | CS Core<br>Randomized Q4W arm only | W48 |
| 3.75. | Safety | Shell TS16 | Summary of Fasting Lipids Percentage Changes from<br>Maintenance Baseline (Day 1) by Visit (Lipid LOCF) –<br>Maintenance Phase | | W48, W96 |
| Labora | atory: Urinalysi | is | | | |
| 3.76. | Safety | UR3 or SHELL<br>TS3 | Summary of Urinalysis Dipstick Results by Visit – Maintenance Phase (Randomized Q4W) | | W48, W96,<br>EOS |
| 3.77. | Safety | UR3 or SHELL<br>TS3 | Summary of Urinalysis Dipstick Results by Visit – Maintenance and Extension Phase (Randomized Q4W) | CS Core<br>Randomized Q4W arm only | EOS |
| 3.78. | ES | UR3 or SHELL<br>TS3 | Summary of Urinalysis Dipstick Results by Visit – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | EOS |
| 3.79. | Safety | LB1 | Summary of Urine Concentrations Changes from Maintenance<br>Baseline (Day 1) by Visit – Maintenance Phase | CS Core | W48, W96,<br>EOS |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.80. | Safety | LB1 | Summary of Urine Concentrations Changes from Maintenance<br>Baseline (Day 1) by Visit – Maintenance and Extension Phase<br>(Randomized Q4W) | CS Core<br>Randomized Q4W arm only | EOS |
| 3.81. | ES | LB1 | Summary of Urine Concentrations Changes from Maintenance<br>Baseline (Day 1) by Visit – Extension Phase (Extension Switch<br>Population) | CS Core | EOS |
| 3.82. | Safety | Shell TS4 | Summary of Changes in Proteinuria Maintenance Baseline (Day 1) Laboratory Result to Maximum Maintenance Phase Laboratory Result – Maintenance Phase | | W48, W96 |
| Safety Tables (Displays will be for both treatment arms, unless specified) | | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| Labora | atory: NCEP Lip | pid and Markers | | | | |
| 3.83. | Safety | Shell TS5 | Summary of Changes in Maintenance Baseline (Day 1) NCEP Fasting Lipid Category to Maximum Maintenance Phase Category – Triglycerides | | W48, W96 | |
| 3.84. | Safety | Shell TS5 | Summary of Changes in Maintenance Baseline (Day 1) NCEP Fasting Lipid Category to Maximum Maintenance Phase Category – Total Cholesterol | | W48, W96 | |
| 3.85. | Safety | Shell TS5 | Summary of Changes in Maintenance Baseline (Day 1) NCEP<br>Fasting Lipid Category to Minimum Maintenance Phase<br>Category – HDL Cholesterol | | W48, W96 | |
| 3.86. | Safety | Shell TS5 | Summary of Changes in Maintenance Baseline (Day 1) NCEP Fasting Lipid Category to Maximum Maintenance Phase Category – LDL Cholesterol | | W48, W96 | |
| 3.87. | Safety | Shell TS6 | Summary of Fasting TC/HDL Ratio Changes from<br>Maintenance Baseline (Day 1) (Maintenance Phase) – Lipids<br>LOCF | | W48, W96 | |
| 3.88. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Maximum Extension Phase Category – Triglycerides (Extension Switch Population) | Switch Q4W IM (Oral Lead-In) group only | EOS | |
| 3.89. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Maximum Extension Phase Category – Total Cholesterol (Extension Switch Population) | Switch Q4W IM (Oral Lead-In) group only | EOS | |
| 3.90. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Minimum Extension Phase Category – HDL Cholesterol (Extension Switch Population) | Switch Q4W IM (Oral Lead-In) group only | EOS | |
| 3.91. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Maximum Extension Phase Category – LDL Cholesterol (Extension Switch Population) | Switch Q4W IM (Oral Lead-In) group only | EOS | |

| Safety | Tables (Display | ys will be for both tr | eatment arms, unless specified) | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.92. | ES | Shell TS6 | Summary of Fasting TC/HDL Ratio Changes from Extension Baseline (Week 100) (Extension Phase) – Lipids LOCF (Extension Switch Population) | Switch Q4W IM (Oral Lead-In) group only | EOS |
| 3.93. | Safety | Shell TS7 | Summary of Bone Markers Changes from Maintenance Baseline (Day 1) – Maintenance Phase | | W48, W96 |
| 3.94. | Safety | Shell TS7 | Summary of Bone Markers Values – Maintenance Phase | | W48, W96 |
| 3.95. | Safety | Shell TS8 | Statistical Analysis of Log-Transformed Ratio to Maintenance<br>Baseline (Day 1) in Bone Markers at Week 48 – Observed<br>Case | For W96, replace Week 48 with W96. | W48, W96 |
| Labora | tory: Hepatobi | iliary (Liver) | | | |
| 3.96. | Safety | Liver1 /Shell<br>TS11 | Summary of Liver Monitoring/Stopping Event Reporting - Maintenance Phase | | W48, W96 |
| 3.97. | Safety | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria - Maintenance Phase | | W48, W96 |
| 3.98. | Safety | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria - Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.99. | ES | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM group only | W96, EOS |
| 3.100. | Safety<br>(Q4W arm<br>only) | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality<br>Criteria – Maintenance Phase Oral Lead-in Period | Randomized Q4W arm only | WK48 |
| ECG | | | | | |
| 3.101. | Safety | EG1 | Summary of ECG Findings – Maintenance Phase | | W48, W96 |
| 3.102. | ES | EG1 | Summary of ECG Findings – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | EOS |

| Safety | Tables (Display | ys will be for both tro | eatment arms, unless specified) | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.103. | Safety | EG2 | Summary of Change from Maintenance Baseline (Day 1) in ECG Values by Visit -Maintenance Phase | | WK48, W96,<br>EOS |
| 3.104. | ES | EG2 | Summary of Change from Extension Baseline (Week 100) in ECG Values by Visit – Extension Phase (Extension Switch Population) | Switch Q4W IM (Oral Lead-In) group only | EOS |
| 3.105. | Safety | EG10 | Summary of QTc Values by Category – Maintenance Phase | Mid200056/wk48idsl/Table 8.1043 | W48, W96 |
| 3.106. | ES | EG10 | Summary of QTc Values by Category – Extension Phase (Extension Switch Population) | Mid200056/wk48idsl/Table 8.1043<br>Switch Q4W IM (Oral Lead-In)<br>group only | EOS |
| 3.107. | Safety | EG10 | Summary of Change from Maintenance Baseline (Day 1) QTc Values by Category – Maintenance Phase | Mid200056/wk48idsl/Table 8.1044 | W48, W96 |
| 3.108. | ES | EG10 | Summary of Change from Extension Baseline (Week 100)<br>QTc Values by Category – Extension Phase (Extension Switch<br>Population) | Mid200056/wk48idsl/Table 8.1044 Switch Q4W IM (Oral Lead-in) group only | EOS |
| eC-SSF | R and Others | | | | |
| 3.109. | Safety | VS1 | Summary of Change from Maintenance Baseline (Day 1) in Vital Signs by Visit – Maintenance Phase | CS Core | W48, W96 |
| 3.110. | ES | VS1 | Summary of Change from Extension Baseline (Week 100) in Vital Signs by Visit – Extension Phase (Extension Switch Population) | CS Core<br>Switch Q4W IM (Oral Lead-in)<br>group only | EOS |
| 3.111. | Safety | Shell TS14 | Summary of Subjects with eC-SSRS Suicidal Ideation or Behaviour During the Maintenance Phase | | W48, W96 |
| 3.112. | Safety | VS1 | Summary of Change from Induction Baseline (Week -20) in Weight and BMI by Visit – Maintenance Phase | CS Core | W48, W96 |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.113. | Safety | See Safety<br>Table 1.16 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Shift in BMI Categories at Week 96 | | W96 |
| 3.114. | Safety | See Safety<br>Table 1.17 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Shift in BMI from Induction Baseline (Week -20) to Maximum Post-baseline Category – Maintenance Phase | | W96 |
| 3.115. | ES | VS1 | Summary of Change from Extension Baseline (Week 100) in Weight and BMI by Visit – Extension Phase (Extension Switch Population) | CS Core Switch Q4W IM (Oral Lead-in) group only | EOS |
| 3.116. | Safety | AE5B | Summary of All Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Maintenance Phase | CS Core | HL, W48, W96 |
| 3.117. | Safety | AE5B | Summary of All Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | CS Core Randomized Q4W arm only | EOS |
| 3.118. | ES | AE5B | Summary of All Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | CS Core Switch Q4W IM group only | EOS |
| 3.119. | Safety | AE5B | Summary of All Drug-Related Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Maintenance Phase | CS Core | HL, W48, W96 |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.120. | Safety | AE5B | Summary of All Drug-Related Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.121. | ES | AE5B | Summary of All Drug-Related Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | CS Core Switch Q4W IM group only | EOS |
| Advers | e Events of Sp | ecial Interest | | | • |
| 3.122. | Safety | See Safety<br>Table 3.44 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Depression Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.123. | Safety | See Safety<br>Table 3.44 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Depression Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.124. | ES | See Safety<br>Table 3.44 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Depression Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |

| Safety Tables (Displays will be for both treatment arms, unless specified) | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.125. | Safety | See Safety Table 3.48 in reporting effort: gsk1265744/mid 209522/iss_01 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.126. | Safety | See Safety<br>Table 3.48 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.127. | ES | See Safety<br>Table 3.48 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.128. | Safety | See Safety<br>Table 3.43 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Suicidal Ideation/Behaviour Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.129. | Safety | See Safety Table 3.43 in reporting effort: gsk1265744/mid 209522/iss_01 | Summary of Suicidal Ideation/Behaviour Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.130. | ES | See Safety Table 3.43 in reporting effort: gsk1265744/mid 209522/iss_01 | Summary of Suicidal Ideation/Behaviour Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.131. | Safety | Shell TS14.1 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety and Suicidal Ideation/Behaviour at Screening — Maintenance Phase | For W96 and EOS: include additional stratification by 'any history' vs. 'no history'. | W48, W96,<br>EOS |
| 3.132. | Safety | Shell TS14.1 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety and Suicidal Ideation/Behaviour at Screening — Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only For W96 and EOS: include additional stratification by 'any history' vs. 'no history' | W96, EOS |
| 3.133. | ES | Shell TS14.1 | Summary of Depression, Anxiety and Suicidal and Self-Injury<br>Adverse Events by System Organ Class, Maximum DAIDS<br>Toxicity Grade, and History of Depression, Anxiety and<br>Suicidal Ideation/Behaviour at Screening – Extension Phase<br>(Extension Switch Population) | Switch Q4W IM group only For W96 and EOS: include additional stratification by 'any history' vs. 'no history' | W96, EOS |
| 3.134. | Safety | See Safety<br>Table 3.38 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Seizure Adverse Events of Special Interest by<br>System Organ Class and Preferred Term (Number of Subjects<br>and Occurrences) – Maintenance Phase | | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.135. | Safety | See Safety<br>Table 3.38 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Seizure Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.136. | ES | See Safety<br>Table 3.38 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Seizure Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.137. | Safety | See Safety<br>Table 3.39 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.138. | Safety | See Safety<br>Table 3.39 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.139. | ES | See Safety<br>Table 3.39 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.140. | Safety | See Safety Table 3.40 in reporting effort: gsk1265744/mid 209522/iss_01 | Summary of Hypersensitivity Reaction (HSR) Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.141. | Safety | See Safety<br>Table 3.40 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hypersensitivity Reaction (HSR) Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.142. | ES | See Safety<br>Table 3.40 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hypersensitivity Reaction (HSR) Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.143. | Safety | See Safety<br>Table 3.41 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rash Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.144. | Safety | See Safety<br>Table 3.41 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rash Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.145. | ES | See Safety<br>Table 3.41 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rash Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.146. | Safety | See Safety<br>Table 3.42 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.147. | Safety | See Safety<br>Table 3.42 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.148. | ES | See Safety<br>Table 3.42 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.149. | Safety | See Safety<br>Table 3.45 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.150. | Safety | See Safety<br>Table 3.45 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.151. | ES | See Safety<br>Table 3.45 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.152. | Safety | See Safety<br>Table 3.46 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Psychosis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.153. | Safety | See Safety<br>Table 3.46 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Psychosis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.154. | ES | See Safety<br>Table 3.46 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Psychosis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.155. | Safety | See Safety<br>Table 3.47 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Mood Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.156. | Safety | See Safety<br>Table 3.47 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Mood Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.157. | ES | See Safety<br>Table 3.47 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Mood Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.158. | Safety | See Safety<br>Table 3.49 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Sleep Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.159. | Safety | See Safety<br>Table 3.49 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Sleep Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.160. | ES | See Safety<br>Table 3.49 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Sleep Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.161. | Safety | See Safety<br>Table 3.51 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Weight Gain Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.162. | Safety | See Safety<br>Table 3.51 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Weight Gain Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Maintenance and Extension<br>Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.163. | ES | See Safety<br>Table 3.51 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Weight Gain Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Extension Phase (Extension<br>Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.164. | Safety | See Safety<br>Table 3.52 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.165. | Safety | See Safety<br>Table 3.52 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.166. | ES | See Safety<br>Table 3.52 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.167. | Safety | See Safety<br>Table 3.53 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Pancreatitis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.168. | Safety | See Safety<br>Table 3.53 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Pancreatitis Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Maintenance and Extension<br>Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.169. | ES | See Safety<br>Table 3.53 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Pancreatitis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.170. | Safety | See Safety<br>Table 3.54 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.171. | Safety | See Safety<br>Table 3.54 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |
| 3.172. | ES | See Safety<br>Table 3.54 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |
| 3.173. | Safety | See Safety<br>Table 3.55 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance Phase | | W96, EOS |
| 3.174. | Safety | See Safety<br>Table 3.55 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | Randomized Q4W arm only | W96, EOS |

| Safety | Safety Tables (Displays will be for both treatment arms, unless specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.175. | ES | See Safety<br>Table 3.55 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | Switch Q4W IM group only | W96, EOS |

# 14.14.8. Safety Figures

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | |
| 3.1. | Safety | AE10 | Plot of Common Maintenance Phase Adverse Events and Relative Risk (Excluding ISRs) – Q4W vs ABC/DTG/3TC | CS CORE | HL, W48, W96 |
| 3.2. | Safety | LIVER9 | Scatter Plot of Maximum vs. Maintenance Baseline (Day 1) for ALT – Maintenance Phase | CS CORE | HL, W48, W96 |
| 3.3. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – Maintenance Phase | CS CORE | HL, W48, W96 |
| 3.4. | Safety | Shell FS2 | Matrix Plot of Maximum Liver Chemistries – Maintenance Phase | CS CORE | HL, W48, W96 |
| 3.5. | Safety | LIVER9 | Scatter Plot of Maximum vs. Maintenance Baseline (Day 1) for ALT – Maintenance and Extension Phase | CS CORE<br>Randomized Q4W arm only | EOS |
| 3.6. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – Maintenance and Extension Phase | CS CORE<br>Randomized Q4W arm only | EOS |
| 3.7. | Safety | Shell FS2 | Matrix Plot of Maximum Liver Chemistries – Maintenance and Extension Phase | CS CORE<br>Randomized Q4W arm only | EOS |
| 3.8. | ES | LIVER9 | Scatter Plot of Maximum vs. Extension Baseline (Week 100) for ALT – Extension Phase (Extension Switch Population) | CS CORE<br>Switch Q4W IM group only | W96, EOS |
| 3.9. | ES | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – Extension Phase (Extension Switch Population) | CS CORE<br>Switch Q4W IM group only | W96, EOS |
| 3.10. | ES | Shell FS2 | Matrix Plot of Maximum Liver Chemistries – Extension Phase (Extension Switch Population) | CS CORE<br>Switch Q4W IM group only | W96, EOS |
| 3.11. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance Phase Injection Site Reaction AEs by Maximum Grade — CAB and/or RPV | Randomized Q4W arm only | W48, W96 |

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – CAB | Randomized Q4W arm only | W48, W96 |
| 3.13. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – RPV | Randomized Q4W arm only | W48, W96 |
| 3.14. | Safety | Shell FS4 | Plot of Incidence of Maintenance Phase Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) – CAB and/or<br>RPV | Randomized Q4W arm only | W48, W96 |
| 3.15. | Safety | Shell FS4 | Plot of Incidence of Maintenance Phase Drug-Related Injection<br>Site Reaction Adverse Events by Visit (Overall and Common) –<br>CAB | Randomized Q4W arm only | W48, W96 |
| 3.16. | Safety | Shell FS4 | Plot of Incidence of Maintenance Phase Drug-Related Injection<br>Site Reaction Adverse Events by Visit (Overall and Common) –<br>RPV | Randomized Q4W arm only | W48, W96 |
| 3.17. | Safety | Shell FS4/ | Plot of Incidence of Grade 3-5 Maintenance Phase Injection<br>Site Reaction Adverse Events by Visit (Overall and Common)<br>— CAB and/or RPV | Randomized Q4W arm only | W48, W96 |
| 3.18. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance and Extension Phase Injection Site Reaction AEs by Maximum Grade – CAB and/or RPV (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.19. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance and Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – CAB (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.20. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance and Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – RPV (Randomized Q4W) | Randomized Q4W arm only | EOS |

| Safety | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.21. | Safety | Shell FS4 | Plot of Incidence of Maintenance and Extension Phase Injection Site Reaction Adverse Events by Visit (Overall and Common) – CAB and/or RPV (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.22. | Safety | Shell FS4 | Plot of Incidence of Maintenance and Extension Phase Drug-<br>Related Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) – CAB (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.23. | Safety | Shell FS4 | Plot of Incidence of Maintenance and Extension Phase Drug-<br>Related Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) – RPV (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.24. | Safety | Shell FS4 | Plot of Incidence of Grade 3-5 Maintenance and Extension Phase Injection Site Reaction Adverse Events by Visit (Overall and Common) — CAB and/or RPV (Randomized Q4W) | Randomized Q4W arm only | EOS |
| 3.25. | ES | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – CAB (Extension Switch Population) | Switch Q4W IM group only | EOS |
| 3.26. | ES | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – RPV (Extension Switch Population) | Switch Q4W IM group only | EOS |
| 3.27. | ES | Shell FS4 | Plot of Incidence of Extension Phase Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) – CAB and/or<br>RPV (Extension Switch Population) | Switch Q4W IM group only | EOS |
| 3.28. | ES | Shell FS4 | Plot of Incidence of Extension Phase Drug-Related Injection<br>Site Reaction Adverse Events by Visit (Overall and Common) –<br>CAB (Extension Switch Population) | Switch Q4W IM group only | EOS |
| 3.29. | ES | Shell FS4 | Plot of Incidence of Extension Phase Drug-Related Injection<br>Site Reaction Adverse Events by Visit (Overall and Common) –<br>RPV (Extension Switch Population) | Switch Q4W IM group only | EOS |

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.30. | ES | Shell FS4/ | Plot of Incidence of Grade 3-5 Extension Phase Injection Site Reaction Adverse Events by Visit (Overall and Common) — CAB and/or RPV (Extension Switch Population) | Switch Q4W IM group only | EOS |
| 3.31. | Safety | Shell FS1 | Bar Chart of Fasting Lipid NCEP Categories at Week 48 vs. Maintenance Baseline (Day 1) – Triglycerides, Total Cholesterol, LDL Cholesterol | For W96, replace W48 with W96 Example: arenv/arprod/gsk3365791/mid_dori _ph3/week48/outputs/Figure 3.062 | W48, W96 |
| 3.32. | Safety | Shell FS1 | Bar Chart of Fasting Lipid NCEP Categories at Week 48 vs. Maintenance Baseline (Day 1) - HDL Cholesterol | For W96, replace W48 with W96 Example: arenv/arprod/gsk3365791/mid_dori _ph3/week48/outputs/Figure 3.062 | W48, W96 |

### 14.14.9. Pharmacokinetic Tables

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes The similar outputs below from study 200056 (week48idsl), unless otherwise specified | Deliverable<br>[Priority] |
| PK | | | | | |
| 14.1. | PK | PKCT1 | Summary of Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit (Maintenance Phase) – Included Log-transformed Statistics | Table 10.1010 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.2. | PK | PKCT1 | Summary of Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Maintenance Phase) – Included Log-transformed Statistics | Table 10.1011 Visits up to W48 for the W48 deliverable. | W48, W96 |

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes The similar outputs below from study 200056 (week48idsl), unless otherwise specified | Deliverable<br>[Priority] |
| 14.3. | PK | PKCT1 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL)-Time Data by Treatment and Visit (Maintenance Phase) – Included Log-transformed Statistics | Table 10.1012 Visits up to W48 for the W48 deliverable. | W48, W96 |
| 14.4. | PK | PKCT1 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Maintenance Phase) – Included Log-transformed Statistics | Table 10.1013 Visits up to W48 for the W48 deliverable. | W48, W96 |
| 14.5. | PK | Shell TPK01 | Summary of Results of Steady State Assessment (Maintenance Phase) | Table 10.1005 Visits up to W48 for the W48 deliverable. | W48 |
| 14.6. | PK | Shell TPK01 | Summary of Results of Steady State Assessment (Maintenance Phase) - Evaluable concentration | Table 10.1009 Visits up to W48 for the W48 deliverable. | W48 |
| 14.7. | PK | PKCT1 | Summary of Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit (Maintenance Phase) – Included Log-transformed Statistics by Hepatitis C Status at Induction Baseline | | W96 |
| 14.8. | PK | PKCT1 | Summary of Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Maintenance Phase) – Included Log-transformed Statistics by Hepatitis C Status at Induction Baseline | | W96 |
| 14.9. | ES | PKCT1 | Summary of Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit (Included Log-transformed Statistics) – Extension Phase (Extension Switch Population) | | EOS |
| 14.10. | ES | PKCT1 | Summary of Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Included Log-transformed Statistics) – Extension Phase (Extension Switch Population) | | EOS |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes The similar outputs below from study 200056 (week48idsl), unless otherwise specified | Deliverable<br>[Priority] |
| 14.11. | ES | PKCT1 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL)-Time Data by Treatment and Visit (Included Log-transformed Statistics) – Extension Phase (Extension Switch Population) | | EOS |
| 14.12. | ES | PKCT1 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit (Included Log-transformed Statistics) – Extension Phase (Extension Switch Population) | | EOS |
| 14.13. | LTFU | PKCT1 | Summary of Long-Term Follow-up Phase Plasma CAB PK<br>Concentration (ug/mL) -Time Data by Treatment and Visit -<br>Included Log-transformed Statistics | Table 10.1001 (WK96CDISC); For 'Total' treatment group (combining Q4W and Switch Q4W groups) | W96, EOS |
| 14.14. | LTFU | PKCT1 | Summary of Long-Term Follow-up Phase Plasma RPV PK<br>Concentration (ng/mL) -Time Data by Treatment and Visit -<br>Included Log-transformed Statistics | Table 10.1002 (WK96CDISC) For 'Total' treatment group (combining Q4W and Switch Q4W groups) | W96, EOS |

## 14.14.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. Population IDSL / TST ID / Example Shell Title Title Title Programming Notes The mock-up below from study 200056 (week48idsl) Deliverable [Priority] | | | | | |
| PK | | | | | |
| 14.1. | PK | PKCF1 | Individual Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1001 Visits up to W52 for the W48 deliverable. | W48, W96 |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes The mock-up below from study 200056 (week48idsl) | Deliverable<br>[Priority] |
| 14.2. | PK | PKCF1 | Individual Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1002 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.3. | PK | PKCF2 | Mean (SD) Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1003 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.4. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Plasma CAB Concentration-<br>Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1004 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.5. | PK | PKCF2 | Mean (SD) Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1005 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.6. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Plasma RPV Concentration-<br>Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1006 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.7. | PK | PKCF2 | Mean (SD) Evaluable Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1007 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.8. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Evaluable Plasma CAB<br>Concentration-Time Plots (Linear and Semi-Log) –<br>Maintenance Phase | Figure 10.1008 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.9. | PK | PKCF2 | Mean (SD) Evaluable Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Maintenance Phase | Figure 10.1009 Visits up to W52 for the W48 deliverable. | W48, W96 |
| 14.10. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Evaluable Plasma RPV<br>Concentration-Time Plots (Linear and Semi-Log) –<br>Maintenance Phase | Figure 10.1010 Visits up to W52 for the W48 deliverable | W48, W96 |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes The mock-up below from study 200056 (week48idsl) | Deliverable<br>[Priority] |
| 14.11. | PK | PKCF2 | Mean (SD) Evaluable Plasma CAB Concentration-Time Plots (Semi-Log) – Maintenance Phase | Figure 10.1011<br>Visits up to W52 for the W48<br>deliverable | W48, W96 |
| 14.12. | PK | PKCF2 | Mean (SD) Evaluable Plasma RPV Concentration-Time Plots (Semi-Log) – Maintenance Phase | Figure 10.1012 Visits up to W52 for the W48 deliverable | W48, W96 |
| 14.13. | LTFU | PKCF6 | Individual Plasma CAB and RPV Concentration-Time Plots (Semi-Log) Post Last Injection for Subjects in LTFU | Overlay all subjects, across arms; use actual relative time since last injection as the x-variable, labelled as "Time post last injection (Weeks)"; one graph each for CAB and RPV, respectively, on the same page. Mark subjects who are receiving oral RPV during LTFU. | W96, EOS |

### 14.14.11. Pharmacokinetic / Pharmacodynamic Tables

| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Last T | rough/ Nominal | Week 8 Trough CAE | B/RPV Concentration and efficacy measures | | |
| 5.1. | PK | Shell<br>TPK03/Table<br>11.1007 (see<br>applicable<br>subgroups in<br>Section 5.4.2) | Logistic Regression Analysis of Snapshot 'HIV-1 RNA≥50 c/mL' at Week 48 by Trough PK Concentration and subgroup –univariable analysis | Last Trough Concentration and Nominal Week-8 trough PK concentration will be treated both as continuous variable and as a categorical subgroup. For W96 delivery, replace Week 48 with Week 96. For W96: This analysis will not be performed if no CVF cases have occurred since Week 48 (for the Q4W arm). | W48, W96 |
| 5.2. | PK | Shell<br>TPK03/Table<br>11.1008 | Multivariable Logistic Regression Analysis of Predictors of Snapshot 'HIV-1 RNA≥50 c/mL' at Week 48 | For W96 delivery, replace Week 48 with Week 96; For W96: This analysis will not be performed if no CVF cases have occurred since Week 48 (for the Q4W arm). | W48, W96 |

| Pharm | Pharmacokinetic / Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.3. | PK | Shell TPK02 | Summary of Last trough CAB PK concentration by<br>Snapshot Virologic Response at Week 48– Included Log-<br>transformed Statistics | The Virologic Response include: WK48 Snapshot HIV-1 RNA>=50 (Yes/No) For W96 delivery, replace Week 48 with Week 96 | W48 |
| 5.4. | PK | Shell TPK02 | Summary of Last trough RPV PK concentration by<br>Snapshot Virologic Response at Week 48 – Included Log-<br>transformed Statistics | Same as above | W48 |
| 5.5. | PK | Shell TPK02 | Summary of Week 8 trough CAB PK concentration by Virologic Response at Maintenance– Included Log-transformed Statistics | The Virologic Response include: WK48 Snapshot HIV-1 RNA>=50 (Yes/No) For W96 delivery, replace Week 48 with Week 96; For W96: this summary will not be produced if no CVF cases have occurred since Week 48 (for the Q4W arm). | W48, W96 |

| Pharmacokinetic / Pharmacodynamic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.6. | PK | Shell TPK02 | Summary of Week 8 trough RPV PK concentration by Virologic Response at Maintenance– Included Log-transformed Statistics | For W96: this summary will not be performed if no CVF cases have occurred since Week 48 (for the Q4W arm). | W48, W96 |

## 14.14.12. Pharmacokinetic / Pharmacodynamic Figures

| Pharm | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| Last tr | ough/Nominal W | eek 8 trough CAB/I | RPV concentration/parameters and efficacy measures | | |
| 5.1. | PK | Shell<br>FPK01/Figure<br>11.1004 | Scatter Plot of Last Trough CAB PK Concentration by Snapshot HIV-1 RNA ≥50c/mL (yes vs. no) at Week 48 | | W48 |
| 5.2. | PK | Shell<br>FPK01/Figure<br>11.1005 | Scatter Plot of Last Trough RPV PK Concentration by Snapshot HIV-1 RNA≥50 c/mL (yes vs. no) at Week 48 | | W48 |
| 5.3. | PK | Shell<br>FPK01/Figure<br>11.1004 | Scatter Plot of Week 8 Trough CAB PK Concentration by Snapshot 'HIV-1 RNA≥50 c/mL' (yes vs. no) at Week 48 | | W48 |
| 5.4. | PK | Shell<br>FPK01/Figure<br>11.1005 | Scatter Plot of Week 8 Trough RPV PK Concentration by Snapshot HIV-1 RNA≥50 c/mL (yes vs. no) at Week 48 | | W48 |
| 5.5. | PK | Figure 11.1006 | Scatter Plot of Delay in last IP injection by Last Trough CAB Concentration at Week 48 at Maintenance Phase | Different symbols for Snapshot<br>Non- 'HIV-1 RNA≥50' and 'HIV-1<br>RNA≥50'. X axis represents last<br>trough CAB concentration, Y axis<br>indicates Delay in last IP injection<br>(Days) | W48 |

| Pharm | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.6. | PK | Figure 11.1006 | Scatter Plot of Delay in last IP injection by Last Trough RPV Concentration at Week 48 at Maintenance Phase | Different symbols for Snapshot<br>Non- 'HIV-1 RNA≥50' and 'HIV-1<br>RNA≥50' . X axis represents last<br>trough RPV concentration, Y axis<br>indicates Delay in last IP injection<br>(Days) | W48 |
| 5.7. | PK | Figure 11.1002 | Individual CAB trough concentration-time Profiles for subjects with Snapshot HIV-1 RNA≥50 c/mL at Week 48 with Median, 5th & 95th percentile of CAB Conc-Time Profiles for other subjects (Semi-Log) | For W96 delivery, replace Week 48 with Week 96 | W48, W96 |
| 5.8. | PK | Figure 11.1003 | Individual RPV trough concentration-time Profiles for subjects with Snapshot HIV-1 RNA≥50 c/mL at Week 48 with Median, 5th & 95th CAB Conc-Time Profiles for other subjects (Semi-Log) | For W96 delivery, replace Week 48 with Week 96 | W48, W96 |
| 5.9. | PK | Shell FPK02 | Scatter plot of Last Trough Concentration of CAB and RPV in relation to occurrence of Snapshot 'HIV-1 RNA≥50 c/mL' at Week 48 | Quartiles of CAB and RPV last trough concentration will be marked with vertical and horizontal lines. Induction Baseline BMI category will also be marked For W96 delivery, replace Week 48 with Week 96 | W48 |

| Pharma | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.10. | PK | Shell FPK02 | Scatter plot of Week 8 Trough Concentration of CAB and RPV in relation to occurrence of Snapshot 'HIV-1 RNA≥50 c/mL' at Week 48 | Same as above. For W96: this figure will not be produced if no CVF cases have occurred since Week 48 (for the Q4W arm). | W48, W96 |
| PK Cor | ncentration and s | afety measures | | | |
| 5.11. | PK | shell FPK03 | Scatter Plot of Change from Maintenance Baseline (Day 1) in 2-Hr QTc versus CAB 2-Hr Post-dose PK Concentrations at Week X [Week 4b and Week 48 for Week 48 delivery, Week 96 for W96 delivery] | For each visit (i.e. wk4b, 48, 96), produce separate plots of 2-Hr PK concentration vs QTcF and 'overall'. Missing QTcB/QTcF will be derived using RR, if RR is available. For 'overall' plot, if QTcF remains missing with derivation from RR, then other QTc parameters will be used in the order of QTcB, QTc-unspecified, with different colours to differentiate each parameter. (2hr post dose PK concentration at WK4b, week 48 vs CFB in QTc at these two visits) For W96 delivery, produce plot for Week 96 only | W48, W96 |

| Pharm | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.12. | PK | Shell FPK03 | Scatter Plot of Change from Maintenance Baseline (Day 1) in 2-Hr QTc versus RPV 2-Hr Post-dose PK Concentrations at Week X [Week4b and Week 48 for W48 delivery, Week 96 for W96 delivery] | Similar to the above for CAB | W48, W96 |
| 5.13. | PK | shell FPK04 | Scatter Plot of Maximum Change from Maintenance<br>Baseline (Day 1) in ALT versus Last Trough CAB PK<br>Concentrations during the Maintenance Phase | Last Trough CAB/RPV PK concentration is defined as the most recent trough PK concentration prior or equal to the date of ALT assessment with maximum CFB, at Maintenance Phase | W48 |
| 5.14. | PK | shell FPK04 | Scatter Plot of Maximum Change from Maintenance Baseline (Day 1) in ALT versus Last Trough RPV PK Concentrations during the Maintenance Phase | Same as above for CAB | W48 |
| 5.15. | PK | shell FPK04 | Scatter Plot of Maximum Change from Maintenance Baseline (Day 1) in Total Bilirubin versus Last Trough CAB PK Concentrations during the Maintenance Phase | Last Trough CAB/RPV PK concentration is defined as the most recent trough PK concentration prior or equal to the date of Total Bili assessment with maximum CFB, at Maintenance Phase | W48 |
| 5.16. | PK | shell FPK04 | Scatter Plot of Maximum Change from Maintenance Baseline (Day 1) in Total Bilirubin versus Last Trough RPV PK Concentrations during the Maintenance Phase | Same as above for CAB | W48 |

| Pharma | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>The similar<br>outputs below<br>from study<br>200056<br>(week48idsl) | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.17. | PK | shell FPK05 | Box Plot of Maximum Toxicity Grades of Most Frequently Reported non-ISR AEs (e.g. Headache, Fever, Fatigue, Nausea, Dizziness) versus Last Trough CAB PK Concentrations during the Maintenance Phase | The AEs for this analysis should be the top 5 in incidence of non-ISR AEs within the Q4W arm during the Maintenance Phase. Last Trough CAB/RPV PK concentration is defined as the most recent trough PK concentration prior or equal to the onset date of the most frequently reported AE with maximum toxicity grade during the Maintenance Phase. If a subject has no AE most commonly reported, then the last trough value at Maintenance Phase will be used for the plot | W48 |
| 5.18. | PK | shell FPK05 | Box Plot of Maximum Toxicity Grades of Most Frequently Reported AEs (e.g. Headache, Fever, Fatigue, Nausea, Dizziness) versus Last Trough RPV PK Concentrations during the Maintenance Phase | The same as above | W48 |

### 14.14.13. Health Outcomes Tables

| Health Outcomes: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable |
| Percept | ion of Injection | Questionnaire ( | PIN) | | • |
| 6.1. | ITT-E | THO2 | Proportion of Subjects with each individual item score in PIN by Visit – LOCF (Maintenance Phase) | | W48, W96 |
| 6.2. | ITT-E | THO1 | Summary of PIN in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit (Maintenance Phase) | | W48, W96 |
| 6.3. | ITT-E | THO10 | Summary and Statistical Analysis of PIN in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit - LOCF (Maintenance Phase) | Wilcoxon Signed -rank test for analysis (acceptance score only) | W48, W96 |
| 6.4. | ITT-E | THO1 | Summary of PIN Change from Week 5 in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit (Maintenance Phase) | | W48, W96 |
| 6.5. | ITT-E | THO1 | Summary of PIN Change from Week 5 in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit – LOCF (Maintenance Phase) | | W48, W96 |
| Health-r | related quality | of Life (HATQoL) | | | |
| 6.6. | ITT-E | THO2 | Proportion of Subjects with each Individual Questionnaire Item Score in HATQoL by Visit - LOCF (Maintenance Phase) | | W48, W96 |

| Health | Outcomes: T | ables | | | |
|---|---|---|---|---|---|
| 6.7. | ITT-E | THO1 | Summary of Quality of Life (HATQoL) Score in Life<br>Satisfaction, HIV Medication, and Disclosure worries by Visit<br>(Maintenance Phase) | | W48, W96 |
| 6.8. | ITT-E | THO1 | Summary of Quality of Life (HATQoL) Score in Life<br>Satisfaction, HIV medication, and Disclosure worries by Visit -<br>LOCF (Maintenance Phase) | | W48, W96 |
| 6.9. | ITT-E | THO1 | Summary of Quality of Life Score (HATQoL) – Change from Maintenance Baseline (Day 1) in Life Satisfaction, HIV Medication, and Disclosure Worries by Visit (Maintenance Phase) | | W48, W96 |
| 6.10. | ITT-E | THO1 | Summary of Quality of Life Score (HATQoL) – Change from Maintenance Baseline (Day 1) in Life Satisfaction, HIV Medication, and Disclosure Worries by Visit - LOCF (Maintenance Phase) | | W48, W96 |
| 6.11. | ITT-E | Shell THO3 | Statistical Analysis of Quality of Life Score (HATQoL) – Change from Maintenance Baseline (Day 1) in Life Satisfaction, HIV medication, and Disclosure Worries by Visit – LOCF (Maintenance Phase) | ANCOVA for analysis | W48, W96 |
| Health | Status:12-ite | m short form surv | ey (SF-12) | | |
| 6.12. | ITT-E | THO2 | Proportion of Subjects with SF-12 Individual Item Scores by Visit - LOCF (Maintenance Phase) | | W48, W96 |
| 6.13. | ITT-E | THO1 | Summary of SF-12 (MCS and PCS Scores) by Visit (Maintenance Phase) | | W48, W96 |
| 6.14. | ITT-E | THO1 | Summary of SF-12 (MCS and PCS Scores) by Visit - LOCF (Maintenance Phase) | | W48, W96 |
| 6.15. | ITT-E | THO1 | Summary of Change from Maintenance Baseline (Day 1) in SF-<br>12 (MCS and PCS Scores) by Visit (Maintenance Phase) | | W48, W96 |
| 6.16. | ITT-E | THO1 | Summary of Change from Maintenance Baseline (Day 1) in SF-<br>12 (MCS and PCS Scores) by Visit - LOCF (Maintenance<br>Phase) | | W48, W96 |

| Health | Health Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| 6.17. | ITT-E | Shell THO3 | Statistical Analysis of SF-12 Change from Maintenance Baseline (Day 1) in MCS, and PCS Score by Visit – LOCF (Maintenance Phase) | ANCOVA for analysis | W48, W96 |
| Treatm | ent Satisfactior | n (HIVTSQs) | | | |
| 6.18. | ITT-E | Shell THO2 | Proportion of Subjects with HIVTSQs – Treatment Satisfaction Individual Item Scores by Visit - LOCF) (Maintenance Phase) | | W48, W96 |
| 6.19. | ITT-E | Shell THO2 | Proportion of Subjects with HIVTSQs – Treatment Satisfaction Individual Item Scores by Visit and Subgroup - LOCF) (Maintenance Phase) | Subgroups: Induction Baseline (Week -20) HIV-1 RNA (<100,000, ≥100,000 c/mL), gender at birth, age (<35; 35-<50; ≥50), Maintenance Baseline (Day 1) CD4+ cell count (<200; 200 to <350; 350 to <500; ≥ 500 cells/mm3), and race (i.e. white, non-white). | W48, W96 |
| 6.20. | ITT-E | Shell THO1 | Summary of HIVTSQs - Total Treatment Satisfaction Score by Visit) (Maintenance Phase) | | W48, W96 |
| 6.21. | ITT-E | Shell THO1 | Summary of HIVTSQs - Total Treatment Satisfaction Score by Visit - LOCF) (Maintenance Phase) | | W48, W96 |
| 6.22. | ITT-E | Shell THO1 | Summary of HIVTSQs - Change from Maintenance Baseline (Day 1) in Total Treatment Satisfaction Score by Visit (Maintenance Phase) | | W48, W96 |
| 6.23. | ITT-E | Shell THO1 | Summary of HIVTSQs - Change from Maintenance Baseline (Day 1) in Total Treatment Satisfaction Score by Visit – LOCF (Maintenance Phase) | | W48, W96 |
| 6.24. | ITT-E | Shell THO3 | Statistical Analysis of HIVTSQs - Change from Maintenance Baseline (Day 1) in Total Treatment Satisfaction Score by Visit - LOCF) (Maintenance Phase) | ANCOVA for analysis | W48, W96 |

| Health Outcomes: Tables | | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| 6.25. | ITT-E | See Table<br>6.40 in<br>reporting<br>effort:<br>gsk1265744/2<br>01584/primary<br>_02 | Summary of HIVTSQs - Change from Maintenance Baseline (Day 1) in Individual Item Score by Visit - LOCF (Maintenance Phase) | | W96 | | | |
| Treatme | ent Satisfaction | n (HIVTSQc) | | | | | | |
| 6.26. | ITT-E | Shell THO2 | Proportion of Subjects with HIV-Treatment Satisfaction<br>Questionnaire Individual Item Scores change) (Maintenance<br>Phase) | | W48 | | | |
| 6.27. | ITT-E | Shell THO1 | Summary of HIV-Treatment Satisfaction Questionnaire in Treatment Satisfaction Score Change) (Maintenance Phase) | | W48 | | | |
| 6.28. | ITT-E | Shell THO5 | Statistical Analysis of HIV-Treatment Satisfaction Questionnaire in Treatment Satisfaction Score Change at Week 48 (Maintenance Phase) | ANOVA for analysis | W48 | | | |
| Treatme | ent Acceptance | (ACCEPT) | | | | | | |
| 6.29. | ITT-E | Shell THO2 | Proportion of Subjects with Treatment Acceptance<br>Questionnaire (ACCEPT) Individual Item Scores by Visit -<br>LOCF) (Maintenance Phase) | | W48, W96 | | | |
| 6.30. | ITT-E | Shell THO1 | Summary of Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit (Maintenance Phase) | | W48, W96 | | | |
| 6.31. | ITT-E | Shell THO1 | Summary of Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit – LOCF (Maintenance Phase) | | W48, W96 | | | |
| 6.32. | ITT-E | Shell THO1 | Summary of Change from Maintenance Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit (Maintenance Phase) | | W48, W96 | | | |
| 6.33. | ITT-E | Shell THO1 | Summary of Change from Maintenance Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit – LOCF (Maintenance Phase) | | W48, W96 | | | |
| Health ( | Health Outcomes: Tables | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| 6.34. | ITT-E | Shell THO3 | Statistical Analysis of Change from Maintenance Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit – LOCF (Maintenance Phase) | ANCOVA for analysis | W48, W96 | | | | |
| Tolerab | ility of Injection | n, NRS (for Q4W | IM) | | | | | | |
| 6.35. | ITT-E | Shell THO2 | Proportion of Subjects with Tolerability of Injection (NRS) Individual item scores by Visit – LOCF (Maintenance Phase) | | W48, W96 | | | | |
| 6.36. | ITT-E | Shell THO9 | Summary of Tolerability of Injection (NRS) scores by Visit (Maintenance Phase) | | W48, W96 | | | | |
| 6.37. | ITT-E | Shell THO9 | Summary of Tolerability of Injection (NRS) scores by Visit – LOCF (Maintenance Phase) | | W48, W96 | | | | |
| 6.38. | ITT-E | Shell THO9 | Summary of Tolerability of Injection (NRS) by Visit – Change from Week 4b Scores (Maintenance Phase) | | W48, W96 | | | | |
| 6.39. | ITT-E | Shell THO9 | Summary of Tolerability of Injection (NRS) by Visit – Change from Week 4b Scores - LOCF (Maintenance Phase) | | W48, W96 | | | | |
| Prefere | Preferences (Dichotomous preference question) (for Q4W IM) | | | | | | | | |
| 6.40. | ITT-E | Shell THO8 | Treatment Preference at Week 48 (Maintenance Phase) | | W48 | | | | |

## 14.14.14. Health Outcomes Figures

| Healt | Health Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 6.1. | ITT-E | Shell FHO1 | Line Plot of Adjusted Mean (95% CI) Change from<br>Maintenance Baseline (Day 1) in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) – LOCF | | W48, W96 |
| 6.2. | ITT-E | Shell FHO2 | Line Plot of Difference (95% CI) in Adjusted Mean Change from Maintenance Baseline (Day 1) in HIVTSQs Total Treatment Satisfaction Score over Time (ANCOVA) – LOCF | | W48, W96 |
| 6.3. | ITT-E | Shell FHO1 | Line Plot of Adjusted Mean (95% CI) Change from Maintenance Baseline (Day 1) in SF-12 (MCS and PCS subscale) Score over Time (ANCOVA) – LOCF | | W48, W96 |
| 6.4. | ITT-E | Shell FHO2 | Line Plot of Difference (95% CI) in Adjusted Mean Change from Maintenance Baseline (Day 1) in SF-12 (MCS and PCS subscale) Score over Time (ANCOVA) – LOCF | | W48, W96 |
| 6.5. | ITT-E | Shell FHO1 | Line Plot of Adjusted Mean (95% CI) Change from Maintenance Baseline (Day 1) in HATQoL (Life Satisfaction, HIV medication, and Disclosure Worries) by Visit (ANCOVA) – LOCF | | W48, W96 |
| 6.6. | ITT-E | Shell FHO2 | Line Plot of Difference in Adjusted Mean (95% CI) Change from Maintenance Baseline (Day 1) in HATQoL (Life Satisfaction, HIV Medication, and Disclosure Worries) by Visit (ANCOVA) – LOCF | | W48, W96 |

## 14.14.15. Virology Tables

| Virology: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>(mock up<br>below from<br>study<br>200056\wk48id<br>sl) | Title | Programming Notes | Deliverable |
| Genoty | rpe | | | | |
| 7.1. | CVF | Table 9.1001 | Summary of the Prevalence of Known INI Resistance<br>Mutations at time of CVF (Maintenance Phase) – Plasma<br>Sample | Known INI resistance mutation per<br>Section 14.6.6. Need to add small<br>'n' for actual no. of subjects<br>included in the analysis. The % will<br>be based on 'n' rather than 'N' | W48, W96 |
| 7.2. | CVF | Table 9.1002 | Summary of the Prevalence of Treatment Emergent Known INI Resistance Mutations at time of CVF (Maintenance Phase) – Plasma Sample | Known INI resistance mutation per<br>Section 14.6.6. Need to add small<br>'n' for actual no. of subjects<br>included in the analysis. The % will<br>be based on 'n' rather than 'N' | W48, W96 |
| 7.3. | CVF | Table 9.1003<br>(modify region<br>to class) | Summary of the Prevalence of Major Resistance Mutations of NRTI, NNRTI and PI Class at time of CVF (Maintenance Phase) Plasma Sample | Major Mutation of NRTI, NNRTI, PI class per Section 14.6.6. Need to add small 'n' for actual no. of subjects included in the analysis. The % will be based on 'n' rather than 'N' (programming for defining class: can refer to arenv/arprod/gsk1349572/mid2003 04/week24/drivers/t_adpf_4001.sas | W48, W96 |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>(mock up<br>below from<br>study<br>200056\wk48id<br>sl) | Title | Programming Notes | Deliverable |
| 7.4. | CVF | | Summary of the Prevalence of Treatment-Emergent Major<br>Resistance Mutations of NRTI, NNRTI and PI Class at time of<br>CVF (Maintenance Phase) Plasma Sample | Major Mutation of NRTI, NNRTI, PI class per Section 14.6.6. Need to add small 'n' for actual no. of subjects included in the analysis. The % will be based on 'n' rather than 'N' (programming for defining class: can refer to arenv/arprod/gsk1349572/mid2003 04/week24/drivers/t_adpf_4001.sas | W48, W96 |
| 7.5. | ITT-E | | Summary of the Prevalence of Major Resistance Mutations of NRTI, NNRTI and PI Class at Induction Baseline (Week -20) Plasma Sample | Major Mutation of NRTI, NNRTI, PI class per Section 14.6.6. Need to add small 'n' for actual no. of subjects included in the analysis. The % will be based on 'n' rather than 'N' (programming for defining class: can refer to arenv/arprod/gsk1349572/mid2003 04/week24/drivers/t_adpf_4001.sas | W48, W96 |
| Phenot | уре | | | | |
| 7.6. | CVF | Table 9.1005 | Summary of Phenotype by Phenotypic Cutoff at time of CVF (Maintenance Phase) Plasma Sample | | W48, W96 |
| 7.7. | CVF | Table 9.1005 | Summary of Genotypic Susceptibility at time of CVF (Maintenance Phase) Plasma Sample | | W48, W96 |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>(mock up<br>below from<br>study<br>200056\wk48id<br>sl) | Title | Programming Notes | Deliverable |
| 7.8. | CVF | Table 9.1005 | Summary of Net Assessment at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.9. | CVF | Table 9.1006 | Summary of Phenotype: Number of Drugs to Which Subject are Resistant at Time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.10. | CVF | Table 9.1007 | Summary of Fold Change to CAB, RPV and DTG at Induction Baseline (Week -20) and Time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.11. | CVF | Table 9.1008 | Summary of Change from Induction Baseline (Week -20) in Fold Change to CAB, RPV, and DTG (Maintenance Period) | | W48, W96 |
| 7.12. | CVF | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria During the Maintenance Phase – Induction Baseline (Week -20) and Time of CVF | | HL, W48, W96 |
| 7.13. | CVF | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure During the Maintenance and Extension Phase – Induction Baseline (Week -20) and Time of CVF (Randomized Q4W arm) | Randomized Q4W arm only | W96, EOS |
| 7.14. | CVF | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria During the Extension Phase – Induction Baseline (Week -20) and Time of CVF (Switch Q4W IM) | Switch Q4W IM group only | W96, EOS |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>(mock up<br>below from<br>study<br>200056\wk48id<br>sl) | Title | Programming Notes | Deliverable |
| 7.15. | ITT-E | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects | May include genotypic and phenotypic data on the last ontreatment isolates for participants with HIV-1 RNA ≥200 c/mL Include columns for phase, phase treatment, phase day. | W48, W96,<br>EOS |

# 14.14.16. ICH Listings

| ICH: Li | ICH: Listings (Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study | Study Population | | | | |
| 1. | Randomised | Shell LSP1 | Listing of Subjects Randomised But Not Treated | CS CORE (related to 'Listing for exclusion from any population) | W48, W96, EOS |
| 2. | Randomised | TA1 | Listing of Randomised and Actual Strata and Treatment Assignment | CS CORE | W48, W96, EOS |
| 3. | All Subjects<br>Screened | ES7 | Listing of Reasons for Screen Failure | CS CORE | W48, W96, EOS |

| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | CS CORE | HL, W48, W96,<br>EOS |
| 5. | ITT-E | ES2 | Listing of Reasons for Study Drug Discontinuation | CS CORE | W48, W96, EOS |
| 6. | All Enrolled | DV2 | Listing of Important Protocol Deviations | CS CORE | W48, W96, EOS |
| 7. | ITT-E | DV2 | Listing of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | CS CORE | HL, W48, W96,<br>EOS |
| 8. | All Enrolled | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | CS CORE | W48, W96, EOS |
| 9. | ITT-E | DM2 | Listing of Demographic Characteristics | CS CORE | W48, W96, EOS |
| 10. | ITT-E | DM9 | Listing of Race | CS CORE | W48, W96, EOS |
| Prima | ry Efficacy | | | | |
| 11. | All Enrolled | Study 201584 (primary_02):<br>Listing 33 | Listing of All Plasma HIV-1 RNA Data | | W96, EOS |
| 12. | ITT-E | Shell LPEF1 | Listing of Study Outcome (50 c/mL) at Week 48 – Snapshot Analysis | | HL, W48, W96,<br>EOS |
| Expos | sure | | | | |
| 13. | Safety | HIV_IP5 | Listing of Investigational Product Exposure Data | CS CORE | W48, W96, EOS |
| Adver | se Events | | | | |
| 14. | All Enrolled | AE8 | Listing of All Adverse Events | CS CORE,<br>Include LTFU AEs. | W96, EOS |
| 15. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | CS CORE | W48, W96, EOS |
| 16. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | CS CORE | W48, W96, EOS |

| N. | Damulatian | IDSL / TST ID | Title | Dua manusia a Nata a | Deliverable |
|---|---|---|---|---|---|
| No. | Population | / Example<br>Shell | Title | Programming Notes | [Priority] |
| 17. | Safety | AE8 | Listing of Fatal Adverse Events | CS CORE | W48, W96, EOS |
| 18. | All Enrolled | AE8 | Listing of Non-Fatal Serious Adverse Events (Induction Phase) | CS CORE | W48, W96, EOS |
| 19. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | CS CORE | W48, W96, EOS |
| 20. | All Enrolled | AE8 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product (Induction Phase) | CS CORE | W48, W96, EOS |
| 21. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | CS CORE | HL, W48, W96,<br>EOS |
| 22. | Safety | AE8 | Listing of Changes in Intensity/Grades of Injection Site Related AE | Based on AE details inform page for changes in intensity of the same event. | W48, W96, EOS |
| 23. | Safety | PREG1a | Listing of Subjects Who Became Pregnant During the Study (Maintenance +Extension Phase) | | W48, W96, EOS |
| Labor | | | | | |
| Hepat | obiliary (Liver) | 1.440 | | 1 | T |
| 24. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver stopping<br>Events | | W48, W96, EOS |
| 25. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | W48, W96, EOS |
| ECG 8 | & Vital Signs | | | | |
| 26. | Safety | EG3 | Listing of ECG Values for subjects with a value of potential clinical importance | | W48, W96, EOS |
| 27. | Safety | EG5 | Listing of ECG Findings | | W48, W96, EOS |
| eC-SS | RS | | | | |
| 28. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data:<br>Event and Description (Section 1-Section 2) | | W48, W96, EOS |
| 29. | Safety | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | | W48, W96, EOS |

| ICH: L | .istings (Global F | Programming Note | : Include columns for phase, phase treatment, phase day, where d | ata is collected in multiple phases | ). |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 30. | Safety | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | | W48, W96, EOS |
| 31. | Safety | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5-Section 8) | | W48, W96, EOS |
| PK | • | | , | | |
| 32. | PK | Study 200056<br>Listing<br>10.1001(wk48i<br>dsl) | Listing of Plasma CAB PK Concentration-Time Data | Add a variable of 'evaluable'<br>(Y/N) | W48, W96, EOS |
| 33. | PK | Study 200056<br>Listing<br>10.1002(wk48i<br>dsl) | Listing of Plasma RPV PK Concentration-Time Data | Add a variable of 'evaluable' (Y/N) | W48, W96, EOS |
| 34. | LTFU | Study 200056<br>Listing<br>10.1001(wk48i<br>dsl) | Listing of Plasma CAB PK Concentration-Time Data (LTFU Phase) | Add a variable of 'evaluable' (Y/N) | W96, EOS |
| 35. | LTFU | Study 200056<br>Listing<br>10.1002(wk48i<br>dsl) | Listing of Plasma RPV PK Concentration-Time Data (LTFU Phase) | Add a variable of 'evaluable' (Y/N) | W96, EOS |
| Other | | | | | |
| 36. | All Enrolled | CM2 | Listing of Concomitant Medications for Subjects with Confirmed Virologic Failure | | W96, EOS |

## 14.14.17. Non-ICH Listings

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| Study | Population | | | | |
| 37. | All Enrolled | ES2 | Listing of Reasons for Induction Phase Withdrawal | | W48, W96, EOS |
| 8. | ITT-E | ES2 | Listing of Reasons for Maintenance Phase Withdrawal | | W48, W96, EOS |
| 89. | ITT-E | ES2 | Listing of Reasons for Maintenance Phase Oral Lead-in Period Withdrawal | | W48, W96, EOS |
| ₩. | ITT-E | ES2 | Listing of Reasons for Extension Phase Withdrawal | | W96, EOS |
| 1. | LTFU | ES2 | Listing of Reasons for Long-term Follow Up Withdrawal | | W48, W96, EOS |
| 2. | All Enrolled | CA3 | Listing of Prior ART Medications | | W48, W96, EOS |
| 3. | All Enrolled | CA3 | Listing of Concomitant ART Medications Received during Induction Phase | | WK48, W96, EOS |
| 4. | ITT-E | CA3 | Listing of Concomitant ART Medications Received during Maintenance Phase | | W48, W96, EOS |
| 5. | ITT-E | CA3 | Listing of ART Medications Received during LTFU Phase | | W48, W96, EOS |
| 6. | ITT-E | CA3 | Listing of subjects with changes in Concomitant ARTs during Maintenance Phase | | W48, W96, EOS |
| 7. | ITT-E | Shell LSP11 | Listing of Investigational Product Accountability - Oral Regimens | | W48, W96, EOS |
| ·8. | ITT-E | MHSZE | Listing of Medical History of Seizure | | W48, W96, EOS |
| 9. | All Enrolled | | Listing of Subjects with Hepatitis C at Induction Baseline (Week -20) | | W96 |
| Seco | ndary Efficacy | | | | |
| 50. | All Enrolled | Shell LSEF3 | Listing of All Plasma HIV-1 RNA data for subjects with Confirmed Virologic Failure (Induction Phase) | | W48, W96, EOS |

| Non-I | Non-ICH: Listings (Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 51. | CVF | Shell LSEF3 | Listing of All Plasma HIV-1 RNA data for subjects with Confirmed Virologic Failure | | W48, W96, EOS |
| 52. | ITT-E | Shell LSEF1 | Listing of All Plasma HIV-1 RNA data for subjects with viral load >=50 c/mL at any time during the Maintenance Phase | | HL, W48, W96,<br>EOS |
| 53. | ITT-E | Shell LSEF1 | Listing of Plasma All HIV-1 RNA data for subjects with viral load >=50 c/mL during the Maintenance Oral lead-in Period | | W48 |
| 54. | ITT-E | Shell LSEF5 | Listing of HIV-1 Associated Conditions | | W48, W96, EOS |
| Safety | , | | | | |
| 55. | Safety | ABC_HSR<br>EXPO2 | Listing of Abacavir Hypersensitivity Reaction Record - Exposure to Abacavir | | W48, W96, EOS |
| 56. | Safety | ABC_HSR<br>DRUG2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject History of Drug Allergies | | W48, W96, EOS |
| 57. | Safety | ABC_HSR<br>COND2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject and Family Conditions | | W48, W96, EOS |
| 58. | Safety | ABC_HSR<br>_RASH2 | Listing of Abacavir Hypersensitivity Reaction Record - Skin Rash Details | | W48, W96, EOS |
| 59. | Safety | ABC_HSR<br>_SYMP4 | Listing of Abacavir Hypersensitivity Reaction Record - Symptoms | | W48, W96, EOS |
| 60. | Safety | VS4 | Listing of Abacavir Hypersensitivity Reaction Record - Vital Signs | | W48, W96, EOS |
| 61. | Safety | ABC_HSR<br>_SYMP6 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments (Excluding Other Symptoms) | | W48, W96, EOS |
| 62. | Safety | ABC_HSR<br>_SYMP7 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments (Other Symptoms) | | W48, W96, EOS |

| Non-I | JH: Listings (Gid | <u></u> | Note: Include columns for phase, phase treatment, phase day, whe | re data is collected in multiple phas | , |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 63. | Safety | See Listing 3 in<br>reporting effort:<br>gsk1265744/mi<br>d209522/iss_0<br>1 | Listing of all Subjects Meeting Liver Stopping Criteria | | W96, EOS |
| 64. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | W48, W96, EOS |
| 65. | Safety | LIVER6 | Listing of Liver Event Information for RUCAM Score | | W48, W96, EOS |
| 66. | Safety | LIVER7 | Listing of Liver Biopsy Details | | W48, W96, EOS |
| 67. | Safety | LIVER8 | Listing of Liver Imaging Details | | W48, W96, EOS |
| 68. | Safety | Liver13 | Listing Subjects Meeting Hepatobiliary Lab Criteria | Please also add those additional items shown in the summary of subjects meeting hepatobiliary lab criteria post-baseline (i.e. AST >3xULN and ALP <2xULN and BIL >=2xULN]; ALT+AST>=xx) | W48, W96, EOS |
| 69. | Safety | AE8 | Listing of Adverse Events Related to Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses | | W48, W96, EOS |
| 70. | Safety | EG3 | Listing of ECG Values for Subjects with Adverse Events Related to Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses | | W48, W96, EOS |
| 71. | Safety | Latte2<br>WK96CDISC<br>report | Listing of Each Subjects ALT, AST, Bilirubin (including total and direct Bilirubin), INR, and ALP for subject meeting Hepatobiliary Lab abnormality criteria | 8.1037 (add AST, ALP, INR, and direct Bilirubin to the listing and only for subject meeting Hepatobiliary Lab abnormality criteria) | HL, W48, W96,<br>EOS |

| Non-ICI | Non-ICH: Listings (Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 72. | Safety | Latte2<br>WK96CDISC<br>report | Listing of Investigational Product Exposure Data for Subject Receiving Oral Bridging | 8.1038 | W48, W96, EOS |
| 73. | Safety | DEV1 | Listing of Dosing Errors and IP Device Malfunctions | | W48, W96, EOS |
| Virolog | Virology (mock up below from study 200056\wk96cdisc), 'Study Phase' will be added as a column to the listing. | | | | |
| 74. | CVF | Listing 9.1005 | Listing of Replication Capacity in IN and PR/RT Region | | W48, W96, EOS |
| 75. | All Enrolled | Table 9.1009 | Listing of Genotypic Mutation Data at All Timepoints | | W96, EOS |

### 14.15. Appendix 15: List of Data Displays for Week 124

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

Unless stated otherwise, all Extension Switch population tables and figures will include treatment groups for direct to inject, oral lead-in and total.

#### 14.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.01 to 1.n | 1.01 to 1.n |
| Efficacy | 2.01 to 2.n | 2.01 to 2.n |
| Safety | 3.01 to 3.n | 3.01 to 3.n |
| Pharmacokinetic | 4.01 to 4.n | 4.01 to 4.n |
| Virology | 7.01 to 7.n | 7.01 to 7.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

### 14.15.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided a separate document.

#### 14.15.3. Deliverables

| Delivery | Description |
|----------|-----------------------|
| HL | Headline for Week 124 |
| Week 124 | Week 124 |

## 14.15.4. Study Population Tables

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Subje | ct Disposition | | | | |
| 1.1. | All Subjects<br>Screened | SA1 | Summary of Study Populations | | HL, W124 |
| 1.2. | All Subjects<br>Screened | Shell TSP1 | Summary of Subjects by Country and Investigator | | W124 |
| 1.3. | ITT-E | ES1 | Summary of Subject Accountability: Study Conclusion Record | | W124 |
| 1.4. | ITT-E | ES1 | Summary of Study Drug Discontinuation | | W124 |
| 1.5. | LTFU | ES1 | Summary of Subject Accountability: Long-term follow up Phase Conclusion Record | | W124 |
| 1.6. | ITT-E | ES1 | Summary of Subject Accountability: Maintenance and Extension Phase Conclusion Record (Randomized Q4W) | For Randomized Q4W arm only Add the following subcategories under subject status: a) Completed Maintenance and did not enter Extension b) Completed Extension c) Withdrawn from Maintenance d) Withdrawn from Extension. | W124 |
| 1.7. | ITT-E | HIV_ES1 | Summary of Subject Accountability: Withdrawals by Visit – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 1.8. | ES | ES1 | Summary of Subject Accountability: Extension Phase Conclusion Record (Extension Switch Population) | | HL, W124 |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.9. | ES | HIV_ES1 | Summary of Subject Accountability: Withdrawals by Visit – Extension Phase (Extension Switch Population) | | W124 |
| 1.10. | All<br>Participants<br>Enrolled | ES4 | Summary of Subject Disposition at Each Study Epoch | | W124 |
| 1.11. | All<br>Participants<br>Enrolled | ES5 | Summary of Reasons for Withdrawal at Each Epoch | | W124 |
| 1.12. | ITT-E | DV1a | Summary of Important Protocol Deviations -<br>Maintenance and Extension Phase (Randomized<br>Q4W) | | W124 |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.13. | ES | DV1a | Summary of Important Protocol Deviations –<br>Extension Phase (Extension Switch Population) | | W124 |
| Demo | graphy and Ba | seline | | | |
| 1.14. | ES | Shell TSP2 | Summary of Demographic Characteristics (Extension Switch Population) | See also DM1 in IDSL Age categorization will include: <=18, 19-64, >=65 (FDAAA requirement) 18-64, 65-84, >=85 (EMA requirement) | HL, W124 |
| 1.15. | ES | DM5 | Summary of Race and Racial Combinations (Extension Switch Population) | CS CORE | W124 |
| 1.16. | ES | DM6 | Summary of Race and Racial Combinations Details (Extension Switch Population) | CS CORE | W124 |
| 1.17. | ES | Shell TSP3 | Summary of Hepatitis Status at Induction Baseline (Week -20) – Extension Switch Population | | W124 |
| 1.18. | ES | CDC1 | Summary of Derived CDC Stages of HIV Infection at Extension Baseline (Week 100) | | W124 |
| 1.19. | ES | Shell TSP5 | Distribution of CD4+ Cell Count Results at Extension Baseline (Week 100) - Extension Switch Population | Same presentation as shown in the mock shell for induction baseline. | W124 |
| Medic | Medical Conditions, Concomitant Medications & Antiretroviral Therapy | | | | |
| 1.20. | ES | MH4 | Summary of Current Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal and<br>Urinary, Nervous System Conditions, and<br>Hepatobiliary disorders (Extension Switch Population) | | W124 |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.21. | ES | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, Nervous System Conditions, and Hepatobiliary disorders (Extension Switch Population) | | W124 |
| 1.22. | ITT-E | CM8 | Summary of Concomitant Medication Ingredient<br>Combinations - Maintenance and Extension Phase<br>(Randomized Q4W) | | W124 |
| 1.23. | ES | CM8 | Summary of Concomitant Medication Ingredient<br>Combinations – Extension Phase (Extension Switch<br>Population) | | W124 |
| 1.24. | ES | Shell TSP11 | Summary of Alternate Background NRTI Therapy at End of Maintenance Phase (Extension Switch Population) | | W124 |
| 1.25. | ES | Shell TSP9 | Summary of Lipid Modifying Agent Use at Extension Baseline (Week 100) – Extension Switch Population | | W124 |
| 1.26. | ES | Shell CLAD1 | Summary of the Prevalence of HIV-1 Subtype at Induction Baseline (Week -20) - Extension Switch Population | | W124 |

# 14.15.5. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Efficacy | Analyses | | | | |
| 2.1. | ES | Shell TPEF2 | Summary of Study Outcomes (50 c/mL cut-off) at Week 124 – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | HL, W124 |
| 2.2. | ES | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper- Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | HL, W124 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.3. | ES | Shell TSEF2.1 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper- Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | HL, W124 |
| 2.4. | ES | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA <200 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper- Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5. | ES | Shell TSEF3 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria by Visit During the Extension Phase (Up to Week 124) — Extension Switch Population | Oral Lead-In, Direct to Inject, Total show all planned extension phase visits up to Week 124. | HL, W124 |
| 2.6. | ES | Shell TSEF3.1 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria During the Extension Phase (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | HL, W124 |
| 2.7. | ES | Shell TSEF5 | Summary of CD4+ Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | W124 |
| 2.8. | ES | Shell TSEF5 | Summary of Change from Extension Baseline (Week 100) in CD4+ Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | W124 |
| 2.9. | ES | Shell TSEF5 | Summary of CD8+ Cell Count (cells/mm^3) by Visit– Extension Phase (Extension Switch Population) | Oral Lead-In | W124 |
| 2.10. | ES | Shell TSEF5 | Summary of Change from Extension Baseline (Week 100) in CD8+ Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | Oral Lead-In | W124 |
| 2.11. | ES | Shell TSEF5 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit – Extension Phase (Extension Switch Population) | Oral Lead-In | W124 |
| 2.12. | ES | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Including Recurrences – Extension Phase (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | W124 |
| 2.13. | ES | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Excluding Recurrences – Extension Phase (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | W124 |
| 2.14. | ES | HIV2/Shell<br>TSEF6.1 | Summary of HIV-1 Disease Progressions and/or Deaths – Extension Phase (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | W124 |
| 2.15. | ES | Shell TPEF2 | Summary of Study Outcomes (200 c/mL) at Week 124 – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total | W124 |
| 2.16. | ES | Shell TSEF11 | Summary of Subjects per Viral Load Category by Visit (Extension Phase) — Extension Switch Population | Oral Lead-In, Direct to Inject, Total | W124 |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.17. | ITT-E | Shell TPEF2 | Summary of Study Outcomes (50 c/mL cut-off) at Week 124 – Snapshot Analysis (Randomized Q4W) | | HL, W124 |
| 2.18. | ITT-E | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | | W124 |
| 2.19. | ITT-E | Shell TSEF2.1 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | | W124 |
| 2.20. | ITT-E | Shell TSEF2 | Proportion of Subjects with Plasma HIV-1 RNA <200 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | | W124 |
| 2.21. | ITT-E | Shell TSEF3 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria by Visit During the Maintenance and Extension Phase (Up to Week 124) — Randomized Q4W | show all visits up to Week 124 | W124 |
| 2.22. | ITT-E | Shell TSEF3.1 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria During the Maintenance and Extension Phase (Randomized Q4W) | | HL, W124 |
| 2.23. | ITT-E | Shell TSEF5 | Summary of Change from Maintenance Baseline (Day 1) in CD4+Cell Count (cells/mm^3) by Visit - Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 2.24. | ITT-E | Shell TSEF5 | Summary of CD4+ Cell Count (cells/mm^3) by Visit – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 2.25. | ITT-E | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Including Recurrences - Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 2.26. | ITT-E | HIV1/Shell<br>TSEF 6.0 | Summary of HIV-1 Associated Conditions Excluding Recurrences - Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 2.27. | ITT-E | HIV2/Shell<br>TSEF6.1 | Summary of HIV-1 Disease Progressions and/or Deaths - Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.28. | ITT-E | Shell TPEF2 | Summary of Study Outcomes (200 c/mL) at Week 124 (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | | W124 |
| 2.29. | ITT-E | | Summary of Subjects per Viral Load Category by Visit (Maintenance and Extension Phase) — Randomized Q4W | | W124 |

## 14.15.6. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.1. | ES | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | HL, W124 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.2. | ES | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA <50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | HL, W124 |
| 2.3. | ES | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA <200 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA <200 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |

| Efficac | fficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | ES | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA >=200 c/mL by Visit (Extension Phase) – Snapshot Analysis (Extension Switch Population) | Oral Lead-In, Direct to Inject, Total Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥200 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |
| 2.5. | ES | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA (log10 copies/mL) Profiles by Visit for CVF subjects (Extension Switch Population – Direct to Inject Group) | The first vertical line indicates extension phase day of first CAB/RPV injection. The second vertical reference line indicates last on-treatment extension phase day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB/RPV+1), day of LTFU HAART start date). This line is only for participants who discontinue from the Extension phase. | W124 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | ES | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA (log10 copies/mL) Profiles by Visit for CVF subjects (Extension Switch Population – Oral Lead-in Group) | The first vertical line indicates extension phase day for start of oral lead-in with oral CAB/RPV. The second vertical reference line indicates last on-treatment extension phase day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB/RPV+1), day of LTFU HAART start date). This line is only for participants who discontinue from the Extension phase. | W124 |
| 2.7. | ES | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA Profiles by Visit for subjects who are in the category of 'viral load ≥50 c/mL' at Week 124 per Snapshot algorithm (Extension Switch Population – Direct to Inject Group) | The first vertical line indicates extension phase day of first CAB/RPV injection. The second vertical reference line indicates last on-treatment extension phase day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB/RPV+1), day of LTFU HAART start date). This line is only for participants who discontinue from the Extension phase. | HL, W124 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ES | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA Profiles by Visit for subjects who are in the category of 'viral load ≥50 c/mL' at Week 124 per Snapshot algorithm (Extension Switch Population – Oral Leadin Group) | The first vertical line indicates extension phase day for start of oral lead-in with oral CAB/RPV. The second vertical reference line indicates last on-treatment extension phase day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB/RPV+1), day of LTFU HAART start date). This line is only for participants who discontinue from the Extension phase. | HL, W124 |
| 2.9. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA < 50c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |
| 2.11. | ITT - E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA <200 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA <200 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | ITT-E | Shell FPEF1 | Proportion (95% CI) of Subjects with HIV-1 RNA >=200 c/mL by Visit (Maintenance and Extension Phase) – Snapshot Analysis (Randomized Q4W) | Line plots, with 95% confidence intervals (Cls), for the proportion of participants with HIV-1 RNA ≥200 c/mL by treatment group at each visit. The 95% Cls will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation. | W124 |
| 2.13. | ITT-E | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA (log10 copies/mL) Profiles by Visit) – for CVF subjects (Randomized Q4W) | The first vertical line indicates start of Induction phase investigational product (ABC/DTG/3TC or DTG). The second vertical line indicates start of Maintenance phase investigational product (oral CAB + oral RPV). The third vertical reference line indicates last ontreatment study day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB+RPV+1), day of LTFU HAART start date). This line is only for participants who withdraw from the Maintenance/Extension phase. | W124 |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.14. | ITT - E | Mid200056//wk<br>96cdisc/Figure<br>7.1007 | Individual Plasma HIV-1 RNA Profiles by Visit for subjects who are in the category of 'HIV-1 RNA ≥50 c/mL' at Week 124 per Snapshot algorithm (Randomized Q4W arm) | The first vertical line indicates start of Induction phase investigational product (ABC/DTG/3TC or DTG). The second vertical line indicates start of Maintenance phase investigational product (oral CAB + oral RPV). The third vertical reference line indicates last ontreatment study day, i.e. min (max(day of last IP injection dose+35 days, day of last oral CAB+RPV+1), day of LTFU HAART start date). This line is only for participants who withdraw from the Maintenance/Extension phase. | HL, W124 |

# 14.15.7. Safety Tables – Extension Switch Population

| All Tab | All Tables will have treatment columns for Oral lead-in, Direct-to-Inject and Total, unless otherwise specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | Exposure | | | | |
| 3.1. | ES | Shell TS1.1 | Summary of Extent of Exposure to Investigational Product – Extension Phase (Extension Switch Population) | | HL, W124 |
| 3.2. | ES | Study 201584<br>(primary_02):<br>Table 3.114 | Summary of Categorized Needle Length and Gauge for CAB Injection - Extension Phase (Extension Switch Population) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.3. | ES | Study 201584<br>(primary_02):<br>Table 3.115 | Summary of Categorized Needle Length and Gauge for RPV Injection - Extension Phase (Extension Switch Population) | | W124 |
| 3.4. | ES | Shell TS1.3 | Summary of Adherence to Q4W IM Dosing Schedule -<br>Extension Phase (Extension Switch Population) | Please refer to Section 14.6.2<br>Adherence to CAB/RPV Injection<br>Schedule | W124 |
| Adver | se Events | | | | |
| 3.5. | ES | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | | HL, W124 |
| 3.6. | ES | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Extension Phase Oral Lead-in Period (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.7. | ES | AE3 | Summary of Common Adverse Events (>=5%) by Overall Frequency – Extension Phase (Extension Switch Population) | | W124 |
| 3.8. | ES | AE3 | Summary of Common Grade 2-5 Adverse Events (>=1%) by Overall Frequency – Extension Phase (Extension Switch Population) | | W124 |
| 3.9. | ES | AE5B | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | | HL, W124 |
| 3.10. | ES | AE3 | Summary of All Drug-Related Grade 2-5 Adverse Events by Overall Frequency – Extension Phase (Extension Switch Population) | | W124 |
| Seriou | s and Other Si | gnificant Adverse | Events | | |
| 3.11. | ES | AE1 | Summary of Serious Adverse Events by System Organ Class – Extension Phase (Extension Switch Population) | | HL, W124 |

| All Tab | All Tables will have treatment columns for Oral lead-in, Direct-to-Inject and Total, unless otherwise specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | ES | AE1 | Summary of Serious Adverse Events by System Organ Class — Extension Phase Oral Lead-in Period (Extension Switch Population) | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| 3.13. | ES | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class – Extension Phase (Extension Switch Population) | | W124 |
| 3.14. | ES | AE3 | Summary of Non-Fatal Serious Adverse Events by Overall Frequency – Extension Phase (Extension Switch Population) | | W124 |
| 3.15. | ES | AE3 | Summary of Drug-Related Non-Fatal Serious Adverse Events by Overall Frequency – Extension Phase (Extension Switch Population) | | W124 |
| 3.16. | ES | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by SOC – Extension Phase (Extension Switch Population) | | HL, W124 |
| 3.17. | ES | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by SOC – Extension Phase Oral Lead-in Period (Extension Switch Population) | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| 3.18. | ES | AE3 | Summary of Common (>=5%) Non-Serious Adverse Events by Overall Frequency – Extension Phase (Extension Switch Population) | | W124 |
| 3.19. | ES | EudraCT Non-<br>serious AE<br>AE15 | Summary of Subjects and Number of Occurrences of Common (>=5%) Non-Serious Adverse Events by System Organ Class – Extension Phase (Extension Switch Population) | CS Core for FDAAA and EMA disclosure requirements. EudraCT Use macro TD_AE4VCTR for New Data Disclosure HARP Reporting Tools | W124 |
| 3.20. | ES | EudraCT SAE<br>AE16 | Summary of Subjects and Number of Occurrences of SAEs,<br>Fatal SAEs, and Drug-related SAEs – Extension Phase<br>(Extension Switch Population) | CS Core for FDAAA and EMA disclosure requirements. EudraCT | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.21. | ES | AE5B | Summary of All Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | | W124 |
| 3.22. | ES | AE5B | Summary of All Drug-Related Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Extension Phase (Extension Switch Population) | | W124 |
| njecti | on Site Reaction | n Adverse Events | | | |
| 3.23. | ES | Shell TS2.2 | Summary of Injection Site Reaction Adverse Events (Event-<br>Level Summary) – Extension Phase (Extension Switch<br>Population) | | HL, W124 |
| 3.24. | ES | Shell TS2.3 | Summary of Subject-Level Characteristics of Injection Site<br>Reaction Adverse Events (Overall and Common) – Extension<br>Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |
| 3.25. | ES | Shell TS2.4 | Summary of Injection Site Reaction Adverse Events by Visit and Maximum Severity (Overall and Common) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |
| 3.26. | ES | Shell TS2.2 | Summary of CAB Drug-Related Injection Site Reaction<br>Adverse Events (Event-Level Summary) – Extension Phase<br>(Extension Switch Population) | | W124 |
| 3.27. | ES | Shell TS2.3 | Summary of CAB Drug-Related Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |
| 3.28. | ES | Shell TS2.4 | Summary of CAB Drug-Related Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity (Overall and<br>Common) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.29. | ES | Shell TS2.5 | Summary of Maximum CAB Drug-Related Injection Site<br>Reaction Adverse Event Grade by Needle Length (Common<br>ISRs) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |
| 3.30. | ES | Shell TS2.2 | Summary of RPV Drug-Related Injection Site Reaction<br>Adverse Events (Event-Level Summary) – Extension Phase<br>(Extension Switch Population) | | W124 |
| 3.31. | ES | Shell TS2.3 | Summary of RPV Drug-Related Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |
| 3.32. | ES | Shell TS2.4 | Summary of RPV Drug-Related Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity (Overall and<br>Common) – Extension Phase (Extension Switch Population) | | W124 |
| 3.33. | ES | Shell TS2.5 | Summary of Maximum RPV Drug-Related Injection Site<br>Reaction Adverse Event Grade by Needle Length (Common<br>ISRs) – Extension Phase (Extension Switch Population) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects | W124 |
| Labora | tory: Chemistr | ry, Hematology an | d Renal Markers | | |
| 3.34. | ES | LB1 | Summary of Chemistry Values by Visit – Extension Phase (Extension Switch Population) | (include lipids and glucose in<br>Conventional Units, renal markers<br>of Retinol Binding Protein, Beta-2<br>Microglobulin, Cystatin C, et al) | W124 |
| 3.35. | ES | LB1 | Summary of Chemistry Changes from Extension Baseline (Week 100) by Visit – Extension Phase (Extension Switch Population) | CS Core (include lipids and glucose in Conventional Units, renal markers of Retinol Binding Protein, Cystatin C, and CKD-EP1 GFR using Creatinine, and CKD-EP1 using Cystatin C et al) | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.36. | ES | Shell TS9.3 | Summary of Maximum Extension Phase Emergent Chemistry Toxicities (Extension Switch Population) | | W124 |
| 3.37. | ES | Shell TS9.2 | Summary of Maximum Emergent Chemistry Toxicities – Extension Phase Oral Lead-in Period (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.38. | ES | LB1 | Summary of Hematology Values by Visit – Extension Phase (Extension Switch Population) | | W124 |
| 3.39. | ES | LB1 | Summary of Hematology Changes from Extension Baseline (Week 100) by Visit – Extension Phase (Extension Switch Population) | | W124 |
| 3.40. | ES | Shell TS9.3 | Summary of Maximum Extension Phase Emergent Hematology Toxicities (Extension Switch Population) | | W124 |
| 3.41. | ES | Shell TS9.2 | Summary of Maximum Emergent Hematology Toxicities – Extension Phase Oral Lead-in Period (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.42. | ES | Shell TS16 | Summary of Fasting Lipids Percentage Changes from Extension Baseline (Week 100) by Visit (Lipid LOCF) – Extension Phase (Extension Switch Population) | | W124 |
| Labora | atory: Urinalysi | S | | | |
| 3.43. | ES | UR3 or SHELL<br>TS3 | Summary of Urinalysis Dipstick Results by Visit – Extension Phase (Extension Switch Population) | | W124 |
| 3.44. | ES | LB1 | Summary of Urine Concentrations Changes from Extension Baseline (Week 100) by Visit – Extension Phase (Extension Switch Population) | | W124 |
| 3.45. | ES | Shell TS4 | Summary of Changes in Proteinuria Extension Baseline (Week 100) Laboratory Result to Maximum Extension Phase Laboratory Result – Extension Phase (Extension Switch Population) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.46. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Maximum Extension Phase Category – Triglycerides (Extension Switch Population) | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| 3.47. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Maximum Extension Phase Category – Total Cholesterol (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.48. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Minimum Extension Phase Category – HDL Cholesterol (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.49. | ES | Shell TS5 | Summary of Changes in Extension Baseline (Week 100) NCEP Fasting Lipid Category to Maximum Extension Phase Category – LDL Cholesterol (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.50. | ES | Shell TS6 | Summary of Extension Phase Fasting TC/HDL Ratio Changes from Extension Baseline (Week 100) – Lipids LOCF (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| abora | atory: Hepatobi | iliary (Liver) | | | |
| 3.51. | ES | Liver1 /Shell<br>TS11 | Summary of Liver Monitoring/Stopping Event Reporting – Extension Phase (Extension Switch Population) | | W124 |
| 3.52. | ES | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria – Extension Phase (Extension Switch Population) | | W124 |
| 3.53. | ES | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria – Extension Phase Oral Lead-in Period (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| ECG | | | | | |
| 3.54. | ES | EG1 | Summary of ECG Findings – Extension Phase (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.55. | ES | EG2 | Summary of Change from Extension Baseline (Week 100) in ECG Values by Visit – Extension Phase (Extension Switch Population) | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| | | | Oral lead-in, Direct-to-Inject and Total, unless otherwise specified | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.56. | ES | EG10 | Summary of QTc Values by Category – Extension Phase (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| 3.57. | ES | EG10 | Summary of Change from Extension Baseline (Week 100) in QTc Values by Category – Extension Phase (Extension Switch Population) | Switch Q4W Oral Lead-in Group Only | W124 |
| Others | ; | | | | |
| 3.58. | ES | VS1 | Summary of Change from Extension Baseline (Week 100) in Vital Signs by Visit – Extension Phase (Extension Switch Population) | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| 3.59. | ES | VS1 | Summary of Change from Extension Baseline (Week 100) in Weight and BMI by Visit – Extension Phase (Extension Switch Population) | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| 3.60. | ES | | Summary of Shift in BMI Categories at Week 104b | Switch Q4W Oral Lead-in Group Only | W124 |
| Advers | se Events of Sp | pecial Interest | | | |
| 3.61. | ES | See Safety<br>Table 3.44 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Depression Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.62. | ES | See Safety<br>Table 3.48 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |

| All Tab | les will have tre | atment columns for | Oral lead-in, Direct-to-Inject and Total, unless otherwise specified | ) | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.63. | ES | See Safety<br>Table 3.43 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Suicidal Ideation/Behaviour Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.64. | ES | Shell TS14.1 | Summary of Depression, Anxiety and Suicidal and Self-Injury Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety and Suicidal Ideation/Behaviour at Screening – Extension Phase (Extension Switch Population) | include additional stratification by 'any history' vs. 'no history' | W124 |
| 3.65. | ES | See Safety<br>Table 3.38 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Seizure Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.66. | ES | See Safety<br>Table 3.39 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatotoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.67. | ES | See Safety<br>Table 3.40 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hypersensitivity Reaction (HSR) Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |

| All Tab | All Tables will have treatment columns for Oral lead-in, Direct-to-Inject and Total, unless otherwise specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.68. | ES | See Safety<br>Table 3.41 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rash Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.69. | ES | See Safety<br>Table 3.42 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.70. | ES | See Safety<br>Table 3.45 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.71. | ES | See Safety<br>Table 3.46 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Psychosis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.72. | ES | See Safety<br>Table 3.47 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Mood Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |

| All Tab | All Tables will have treatment columns for Oral lead-in, Direct-to-Inject and Total, unless otherwise specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.73. | ES | See Safety<br>Table 3.49 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Sleep Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.74. | ES | See Safety<br>Table 3.51 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Weight Gain Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Extension Phase (Extension<br>Switch Population) | | W124 |
| 3.75. | ES | See Safety<br>Table 3.52 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |
| 3.76. | ES | See Safety<br>Table 3.53 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Pancreatitis Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Extension Phase (Extension<br>Switch Population) | | W124 |
| 3.77. | ES | See Safety<br>Table 3.54 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |

| All Tabl | All Tables will have treatment columns for Oral lead-in, Direct-to-Inject and Total, unless otherwise specified) | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.78. | ES | See Safety Table 3.55 in reporting effort: gsk1265744/mid 209522/iss_01 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Extension Phase (Extension Switch Population) | | W124 |

### 14.15.8. Safety Tables – Maintenance + Extension Phase (Randomized Q4W Only)

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| Expos | ure | | | | |
| 3.79. | Safety | Shell TS1.1 | Summary of Extent of Exposure to Investigational Product – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.80. | Safety | Study 201584<br>(primary_02):<br>Table 3.114 | Summary of Categorized Needle Length and Gauge for CAB Injection – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.81. | Safety | Study 201584<br>(primary_02):<br>Table 3.115 | Summary of Categorized Needle Length and Gauge for RPV Injection – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.82. | Safety | Shell TS1.3 | Summary of Adherence to Q4W IM Dosing Schedule – Maintenance and Extension Phase (Randomized Q4W) | please refer to Section 14.6.2<br>Adherence to CAB/RPV Injection<br>Schedule | W124 |
| Adver | se Events | | | | |
| 3.83. | Safety | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.84. | LTFU | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Long-term Follow-up Phase | | W124 |
| 3.85. | Safety | AE3 | Summary of Common Adverse Events (>=5%) by Overall Frequency – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.86. | Safety | AE3 | Summary of Common Grade 2-5 Adverse Events (>=1%) by Overall Frequency – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.87. | Safety | AE5B | Summary of All Drug-Related Adverse Events by System<br>Organ Class and Maximum Toxicity – Maintenance and<br>Extension Phase (Randomized Q4W) | | W124 |
| 3.88. | Safety | AE3 | Summary of All Drug-Related Grade 2-5 Adverse Events by<br>Overall Frequency – Maintenance and Extension Phase<br>(Randomized Q4W) | | W124 |
| Seriou | s and Other Si | gnificant Adverse | Events | | |
| 3.89. | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.90. | Safety | AE1 | Summary of Drug-Related Serious Adverse Events by System Organ Class – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.91. | Safety | AE3 | Summary of Non-Fatal Serious Adverse Events by Overall Frequency – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.92. | Safety | AE3 | Summary of Drug-Related Non-Fatal Serious Adverse Events by Overall Frequency – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.93. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.94. | Safety | AE3 | Summary of Common (>=5%) Non-Serious Adverse Events by Overall Frequency – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.95. | Safety | EudraCT Non-<br>serious AE<br>AE15 | Summary of Subjects and Number of Occurrences of Common (>=5%) Non-Serious Adverse Events by System Organ Class – Maintenance and Extension Phase (Randomized Q4W) | CS Core for FDAAA and EMA disclosure requirements. EudraCT Use macro TD_AE4VCTR for New Data Disclosure HARP Reporting Tools | W124 |
| 3.96. | Safety | EudraCT SAE<br>AE16 | Summary of Subjects and Number of Occurrences of SAEs,<br>Fatal SAEs, and Drug-related SAEs – Maintenance and<br>Extension Phase (Randomized Q4W) | CS Core for FDAAA and EMA disclosure requirements. EudraCT | W124 |
| Injectio | on Site Reaction | n Adverse Events | | | |
| 3.97. | Safety | Shell TS2.2 | Summary of Injection Site Reaction Adverse Events (Event-<br>Level Summary) – Maintenance and Extension Phase<br>(Randomized Q4W) | | W124 |
| 3.98. | Safety | Shell TS2.3 | Summary of Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Maintenance and Extension Phase (Randomized Q4W) | Common ISR includes pain,<br>induration, nodules and any other<br>ISR with ≥5% subjects (for<br>randomized Q4W arm only) | W124 |
| 3.99. | Safety | Shell TS2.4 | Summary of Injection Site Reaction Adverse Events by Visit and Maximum Severity (Overall and Common) – Maintenance and Extension Phase (Randomized Q4W) | Common ISR includes pain,<br>induration, nodules and any other<br>ISR with ≥5% subjects (for<br>randomized Q4W arm only) | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.100. | Safety | Shell TS2.2 | Summary of CAB Drug-Related Injection Site Reaction<br>Adverse Events (Event-Level Summary) – Maintenance and<br>Extension Phase (Randomized Q4W) | | W124 |
| 3.101. | Safety | Shell TS2.3 | Summary of CAB Drug-Related Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Maintenance and Extension Phase (Randomized Q4W) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for Q4W arm only) | W124 |
| 3.102. | Safety | Shell TS2.4 | Summary of CAB Drug-Related Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity (Overall and<br>Common) – Maintenance and Extension Phase (Randomized<br>Q4W) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for Q4W arm only) | W124 |
| 3.103. | Safety | Shell TS2.5 | Summary of Maximum CAB Drug-Related Injection Site<br>Reaction Adverse Event Grade by Needle Length (Common<br>ISRs) – Maintenance and Extension Phase (Randomized<br>Q4W) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for randomized Q4W arm only) | W124 |
| 3.104. | Safety | Shell TS2.2 | Summary of RPV Drug-Related Injection Site Reaction<br>Adverse Events (Event-Level Summary) – Maintenance and<br>Extension Phase (Randomized Q4W) | | W124 |
| 3.105. | Safety | Shell TS2.3 | Summary of RPV Drug-Related Subject-Level Characteristics of Injection Site Reaction Adverse Events (Overall and Common) – Maintenance and Extension Phase (Randomized Q4W) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for randomized Q4W arm only) | W124 |
| 3.106. | Safety | Shell TS2.4 | Summary of RPV Drug-Related Injection Site Reaction<br>Adverse Events by Visit and Maximum Severity (Overall and<br>Common) – Maintenance and Extension Phase (Randomized<br>Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.107. | Safety | Shell TS2.5 | Summary of Maximum RPV Drug-Related Injection Site<br>Reaction Adverse Event Grade by Needle Length (Common<br>ISRs) – Maintenance and Extension Phase (Randomized<br>Q4W) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for Q4W arm only) | W124 |
| 3.108. | Safety | AE5B | Summary of All Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.109. | Safety | AE5B | Summary of All Drug-Related Adverse Events Excluding Injection Site Reactions by System Organ Class and Maximum Toxicity – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| Labora | tory: Chemistr | y, Hematology and | d Renal Markers | | |
| 3.110. | Safety | LB1 | Summary of Chemistry Values by Visit – Maintenance and Extension Phase (Randomized Q4W) | (include lipids and glucose in<br>Conventional Units, renal markers<br>of Retinol Binding Protein, Beta-2<br>Microglobulin, Cystatin C, et al) | W124 |
| 3.111. | Safety | LB1 | Summary of Chemistry Changes from Maintenance Baseline (Day 1) by Visit – Maintenance and Extension Phase (Randomized Q4W) | CS Core (include lipids and glucose in Conventional Units, renal markers of Retinol Binding Protein, Cystatin C, and CKD-EP1 GFR using Creatinine, and CKD-EP1 using Cystatin C et al) | W124 |
| 3.112. | Safety | LB1 | Summary of Hematology Values by Visit – Maintenance and Extension Phase (Randomized Q4W) | , | W124 |
| 3.113. | Safety | LB1 | Summary of Hematology Changes from Maintenance Baseline (Day 1) by Visit – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.114. | Safety | Shell TS9.2 | Summary of Maximum Maintenance and Extension Phase<br>Emergent Chemistry Toxicities (Randomized Q4W) | | W124 |
| 3.115. | Safety | Shell TS9.2 | Summary of Maximum Maintenance and Extension Phase<br>Emergent Hematology Toxicities (Randomized Q4W) | | W124 |
| Labora | tory: Hepatobi | liary (Liver) | | | |
| 3.116. | Safety | Liver1 /Shell<br>TS11 | Summary of Liver Monitoring/Stopping Event Reporting – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.117. | Safety | liver10/Shell<br>TS12 | Summary of Subjects Meeting Hepatobiliary Abnormality<br>Criteria - Maintenance and Extension Phase (Randomized<br>Q4W) | | W124 |
| Urinaly | sis | | | | |
| 3.118. | Safety | UR3 or SHELL<br>TS3 | Summary of Urinalysis Dipstick Results by Visit – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.119. | Safety | LB1 | Summary of Urine Concentrations Changes from Maintenance<br>Baseline (Day 1) by Visit – Maintenance and Extension Phase<br>(Randomized Q4W) | | W124 |
| 3.120. | Safety | Shell TS4 | Summary of Changes in Proteinuria Maintenance Baseline (Day 1) Laboratory Result to Maximum Maintenance Phase Laboratory Result – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| AEs of | Special Interes | st | | | |
| 3.121. | Safety | See Safety<br>Table 3.44 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Depression Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 3.122. | Safety | See Safety<br>Table 3.48 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.123. | Safety | See Safety<br>Table 3.43 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Suicidal Ideation/Behaviour Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.124. | Safety | Shell TS14.1 | Summary of Depression, Anxiety and Suicidal and Self-Injury Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety and Suicidal Ideation/Behaviour at Screening – Maintenance and Extension Phase (Randomized Q4W) | include additional stratification by<br>'any history' vs. 'no history' | W124 |
| 3.125. | Safety | See Safety<br>Table 3.38 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Seizure Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.126. | Safety | See Safety<br>Table 3.39 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatotoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.127. | Safety | See Safety<br>Table 3.40 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Hypersensitivity Reaction (HSR) Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.128. | Safety | See Safety<br>Table 3.41 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rash Adverse Events of Special Interest by<br>System Organ Class and Preferred Term (Number of Subjects<br>and Occurrences) – Maintenance and Extension Phase<br>(Randomized Q4W) | | W124 |
| 3.129. | Safety | See Safety<br>Table 3.42 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.130. | Safety | See Safety<br>Table 3.45 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.131. | Safety | See Safety<br>Table 3.46 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Psychosis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.132. | Safety | See Safety<br>Table 3.47 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Mood Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.133. | Safety | See Safety<br>Table 3.49 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Sleep Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.134. | Safety | See Safety<br>Table 3.51 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Weight Gain Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Maintenance and Extension<br>Phase (Randomized Q4W) | | W124 |
| 3.135. | Safety | See Safety<br>Table 3.52 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.136. | Safety | See Safety<br>Table 3.53 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Pancreatitis Adverse Events of Special Interest<br>by System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) – Maintenance and Extension<br>Phase (Randomized Q4W) | | W124 |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.137. | Safety | See Safety<br>Table 3.54 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |
| 3.138. | Safety | See Safety<br>Table 3.55 in<br>reporting effort:<br>gsk1265744/mid<br>209522/iss_01 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) – Maintenance and Extension Phase (Randomized Q4W) | | W124 |

# 14.15.9. Safety Tables – Long Term Follow Up

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Exposu | ire | | | | |
| 3.139. | LTFU | AE1 | Summary of Serious Adverse Events by System Organ Class – Long Term Follow Up Phase | | W124 |

# 14.15.10. Safety Figures – Extension Switch Population

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adver | se Events | | | | |
| 3.1. | ES | LIVER9 | Scatter Plot of Maximum vs. Extension Baseline (Week 100) for ALT – Extension Phase (Extension Switch Population) | | W124 |
| 3.2. | ES | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – Extension Phase (Extension Switch Population) | | W124 |
| 3.3. | ES | Shell FS2 | Matrix Plot of Maximum Liver Chemistries – Extension Phase (Extension Switch Population) | | W124 |
| 3.4. | ES | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Extension Phase Injection Site Reaction AEs by Maximum Grade — CAB and/or RPV (Extension Switch Population) | | W124 |
| 3.5. | ES | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – CAB (Extension Switch Population) | | W124 |
| 3.6. | ES | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – RPV (Extension Switch Population) | | W124 |
| 3.7. | ES | Shell FS4 | Plot of Incidence of Extension Phase Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) – CAB and/or<br>RPV (Extension Switch Population) | | W124 |
| 3.8. | ES | Shell FS4 | Plot of Incidence of Extension Phase Drug-Related Injection<br>Site Reaction Adverse Events by Visit (Overall and Common) –<br>CAB (Extension Switch Population) | | W124 |
| 3.9. | ES | Shell FS4 | Plot of Incidence of Extension Phase Drug-Related Injection<br>Site Reaction Adverse Events by Visit (Overall and Common) –<br>RPV (Extension Switch Population) | | W124 |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | ES | Shell FS4/ | Plot of Incidence of Grade 3-5 Extension Phase Injection Site Reaction Adverse Events by Visit (Overall and Common) — CAB and/or RPV (Extension Switch Population) | | W124 |
| 3.11. | Safety | Shell FS1 | Bar Chart of Fasting Lipid NCEP Categories at Week W104 vs. Extension Baseline (Week 100) – Triglycerides, Total Cholesterol, LDL Cholesterol | Switch Q4W Oral Lead-in Group<br>Only | W124 |
| 3.12. | Safety | Shell FS1 | Bar Chart of Fasting Lipid NCEP Categories at Week 104 vs. Extension Baseline (Week 100) - HDL Cholesterol | Switch Q4W Oral Lead-in Group Only | W124 |

### 14.15.11. Safety Figures – Maintenance + Extension Phase (Randomized Q4W)

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | |
| 3.13. | Safety | LIVER9 | Scatter Plot of Maximum vs. Maintenance Baseline (Day 1) for ALT – Maintenance and Extension Phase | | W124 |
| 3.14. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin – Maintenance and Extension Phase | | W124 |
| 3.15. | Safety | Shell FS2 | Matrix Plot of Maximum Liver Chemistries – Maintenance and Extension Phase | | W124 |
| 3.16. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance and Extension Phase Injection Site Reaction AEs by Maximum Grade – CAB and/or RPV (Randomized Q4W) | | W124 |
| 3.17. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance and Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – CAB (Randomized Q4W) | | W124 |

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.18. | Safety | Shell FS3 | Plot of Onset, Duration, and Severity of Overall and Common Maintenance and Extension Phase Drug-Related Injection Site Reaction AEs by Maximum Grade – RPV (Randomized Q4W) | | W124 |
| 3.19. | Safety | Shell FS4 | Plot of Incidence of Maintenance and Extension Phase Injection Site Reaction Adverse Events by Visit (Overall and Common) – CAB and/or RPV (Randomized Q4W) | | W124 |
| 3.20. | Safety | Shell FS4 | Plot of Incidence of Maintenance and Extension Phase Drug-<br>Related Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) – CAB (Randomized Q4W) | | W124 |
| 3.21. | Safety | Shell FS4 | Plot of Incidence of Maintenance and Extension Phase Drug-<br>Related Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) – RPV (Randomized Q4W) | | W124 |
| 3.22. | Safety | Shell FS4 | Plot of Incidence of Grade 3-5 Maintenance and Extension Phase Injection Site Reaction Adverse Events by Visit (Overall and Common) — CAB and/or RPV (Randomized Q4W) | | W124 |

#### 14.15.12. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes The similar outputs below from study 200056 (week48idsl), unless otherwise specified | Deliverable<br>[Priority] |
| PK | | | | | |
| 4.1. | PK | PKCT1 | Summary of Extension Phase Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics (Extension Switch Population) | | W124 |

| Pharn | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes The similar outputs below from study 200056 (week48idsl), unless otherwise specified | Deliverable<br>[Priority] |
| 4.2. | PK | PKCT1 | Summary of Extension Phase Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics (Extension Switch Population) | | W124 |
| 4.3. | PK | PKCT1 | Summary of Evaluable Extension Phase Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics (Extension Switch Population) | | W124 |
| 4.4. | PK | PKCT1 | Summary of Evaluable Extension Phase Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics (Extension Switch Population) | | W124 |
| 4.5. | PK | PKCT1 | Summary of Extension Phase Plasma CAB PK Concentration (ug/mL) -Time Data by Visit and Hepatitis C Status at Induction Baseline – Including Log-transformed Statistics (Extension Switch Population) | | W124 |
| 4.6. | PK | PKCT1 | Summary of Extension Phase Plasma RPV PK Concentration (ng/mL) -Time Data by Visit and Hepatitis C Status at Induction Baseline – Including Log-transformed Statistics (Extension Switch Population) | | W124 |
| 4.7. | LTFU | PKCT1 | Summary of Long-Term Follow-up Phase Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit - Included Log-transformed Statistics | Table 10.1001 (WK96CDISC); For 'Total' treatment group (combining Q4W and Switch Q4W groups) | W124 |
| 4.8. | LTFU | PKCT1 | Summary of Long-Term Follow-up Phase Plasma RPV PK<br>Concentration (ng/mL) -Time Data by Visit (Excluding Subjects<br>Receiving Oral RPV in the LTFU Phase) - Including Log-<br>transformed Statistics | Table 10.1002 (WK96CDISC) For 'Total' treatment group (combining Q4W and Switch Q4W groups) | W124 |

### 14.15.13. Pharmacokinetic Figures

| | nacokinetic: Figu | | | Programming Notes | D |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | The mock-up below from study 200056 (week48idsl) | Deliverable<br>[Priority] |
| PK | | | | | |
| 4.1. | PK | PKCF1 | Individual Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.2. | PK | PKCF1 | Individual Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.3. | PK | PKCF2 | Mean (SD) Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.4. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Plasma CAB Concentration-<br>Time Plots (Linear and Semi-Log) – Extension Phase<br>(Extension Switch Population) | | W124 |
| 4.5. | PK | PKCF2 | Mean (SD) Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.6. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Plasma RPV Concentration-<br>Time Plots (Linear and Semi-Log) – Extension Phase<br>(Extension Switch Population) | | W124 |
| 4.7. | PK | PKCF2 | Mean (SD) Evaluable Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.8. | PK | PKCF3 | Median (5th and 95th percentile) Evaluable Plasma CAB<br>Concentration-Time Plots (Linear and Semi-Log) –<br>Extension Phase (Extension Switch Population) | | W124 |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes The mock-up below from study 200056 (week48idsl) | Deliverable<br>[Priority] |
| 4.9. | PK | PKCF2 | Mean (SD) Evaluable Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.10. | PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Evaluable Plasma RPV<br>Concentration-Time Plots (Linear and Semi-Log) –<br>Extension Phase (Extension Switch Population) | | W124 |
| 4.11. | PK | PKCF2 | Mean (SD) Evaluable Plasma CAB Concentration-Time<br>Plots (Semi-Log) – Extension Phase (Extension Switch<br>Population) | | W124 |
| 4.12. | PK | PKCF2 | Mean (SD) Evaluable Plasma RPV Concentration-Time Plots (Semi-Log) – Extension Phase (Extension Switch Population) | | W124 |
| 4.13. | LTFU | PKCF6 | Individual Plasma CAB and RPV Concentration-Time Plots (Semi-Log) Post Last Injection for Subjects in LTFU | Overlay all subjects, across arms; use actual relative time since last injection as the x-variable, labelled as "Time post last injection (Weeks)"; one graph each for CAB and RPV, respectively, on the same page. Mark subjects who are receiving oral RPV during LTFU. | W124 |

### 14.15.14. Virology Tables

| Virology: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>(mock up<br>below from<br>study<br>200056\wk48id<br>sl) | Title | Programming Notes | Deliverable |
| 7.1. | ES | | Summary of the Prevalence of Major Resistance Mutations of INI, NRTI, NNRTI and PI Class at Induction Baseline (Week - 20) Plasma Sample (Extension Switch Population) | Major Mutation of NRTI, NNRTI, PI class, and known INI resistance mutations, per Section 14.6.6. Need to add small 'n' for actual no. of subjects included in the analysis. The % will be based on 'n' rather than 'N' (programming for defining class: can refer to arenv/arprod/gsk1349572/mid2003 04/week24/drivers/t_adpf_4001.sas | W124 |
| 7.2. | CVF | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure During the Maintenance and Extension Phase – Induction Baseline (Week -20) and Time of CVF (Randomized Q4W arm) | Randomized Q4W arm only | W124 |
| 7.3. | CVF<br>(Extension<br>Switch) | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria During the Extension Phase – Induction Baseline (Week -20) and Time of CVF (Extension Switch Population) | Switch Q4W IM group only | HL, W124 |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell<br>(mock up<br>below from<br>study<br>200056\wk48id<br>sl) | Title | Programming Notes | Deliverable |
| 7.4. | ITT-E | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects (Randomized Q4W) | May include genotypic and phenotypic data on the last ontreatment isolates for participants with HIV-1 RNA ≥200 c/mL Include columns for phase, phase treatment, phase day. | W124 |
| 7.5. | ES | Shell TV1 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects (Extension Switch Population) | May include genotypic and phenotypic data on the last ontreatment isolates for participants with HIV-1 RNA ≥200 c/mL Include columns for phase, phase treatment, phase day. | W124 |

#### 14.15.15. ICH Listings

**ICH: Listings (**Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). Listings will present data for the Randomized Q4W arm (data collected in any study phase, where applicable) and the Extension Switch Q4W arm (data collected in the Extension and LTFU phases, where applicable).

| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Study | Population | • | | | |
| 1. | ITT-E | ES2 | Listing of Reasons for Study Withdrawal | | W124 |
| 2. | ITT-E | ES2 | Listing of Reasons for Study Drug Discontinuation | | W124 |
| 3. | ITT-E | DV2 | Listing of Important Protocol Deviations | Remove column for "Deviation Requires Exclusion from the Per Protocol Population". | |
| 4. | ITT-E | DM2 | Listing of Demographic Characteristics | sting of Demographic Characteristics | |
| 5. | ITT-E | DM9 | Listing of Race | | W124 |
| Prima | ry Efficacy | • | | | |
| 6. | ITT-E | Study 201584<br>(primary_02):<br>Listing 33 | Listing of All Plasma HIV-1 RNA Data | isting of All Plasma HIV-1 RNA Data | |
| 7. | ITT-E | Shell LPEF1 | Listing of Study Outcome (50 c/mL) at Week 124 – Snapshot Analysis | | HL, W124 |
| Expos | ure | | | | |
| 8. | Safety | HIV_IP5 | Listing of Investigational Product Exposure Data | | HL, W124 |
| Adver | se Events | | | | • |
| 9. | Safety | AE8 | Listing of All Adverse Events | | W124 |
| 10. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | W124 |
| 11. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | W124 |

**ICH: Listings (**Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). Listings will present data for the Randomized Q4W arm (data collected in any study phase, where applicable) and the Extension Switch Q4W arm (data collected in the Extension and LTFU phases, where applicable).

| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 12. | Safety | AE8 | Listing of Fatal Adverse Events | | W124 |
| 13. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | | W124 |
| 14. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | | HL, W124 |
| 15. | Safety | AE8 | Listing of Changes in Intensity/Grades of Injection Site Related AE | Based on AE details inform page for changes in intensity of the same event. | W124 |
| 16. | Safety | PREG1a | Listing of Subjects Who Became Pregnant During the Study | | W124 |
| Labor | | • | | | |
| Hepat | obiliary (Liver) | | | | |
| 17. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver stopping Events | | W124 |
| 18. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | | W124 |
| ECG 8 | & Vital Signs | <u>.</u> | | | |
| 19. | Safety | EG3 | Listing of ECG Values for subjects with a value of potential clinical importance | | W124 |
| 20. | Safety | EG5 | Listing of ECG Findings | | W124 |
| eC-SS | RS | • | | | |
| 21. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data:<br>Event and Description (Section 1-Section 2) | | W124 |
| 22. | Safety | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | | W124 |
| 23. | Safety | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | | W124 |

**ICH: Listings (**Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). Listings will present data for the Randomized Q4W arm (data collected in any study phase, where applicable) and the Extension Switch Q4W arm (data collected in the Extension and LTFU phases, where applicable).

| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 24. | Safety | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5-Section 8) | | W124 |
| PK | | | | | |
| 25. | PK | Study 200056<br>Listing<br>10.1001(wk48i<br>dsl) | Listing of Plasma CAB PK Concentration-Time Data | Add a variable of 'evaluable' (Y/N) | W124 |
| 26. | PK | Study 200056<br>Listing<br>10.1002(wk48i<br>dsl) | Listing of Plasma RPV PK Concentration-Time Data | Add a variable of 'evaluable' (Y/N) | W124 |
| 27. | LTFU | Study 200056<br>Listing<br>10.1001(wk48i<br>dsl) | Listing of Plasma CAB PK Concentration-Time Data (LTFU Phase) | Add a variable of 'evaluable' (Y/N) | W124 |
| 28. | LTFU | Study 200056<br>Listing<br>10.1002(wk48i<br>dsl) | Listing of Plasma RPV PK Concentration-Time Data (LTFU Phase) | Add a variable of 'evaluable' (Y/N) | W124 |
| Other | | | | | |
| 29. | ITT-E | CM2 | Listing of Concomitant Medications for Subjects with Confirmed Virologic Failure | | W124 |

#### 14.15.16. Non-ICH Listings

**Non-ICH: Listings (**Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). Listings will present data for the Randomized Q4W arm (data collected in any study phase, where applicable) and the Extension Switch Q4W arm (data collected in the Extension and LTFU phases, where applicable), unless otherwise stated in the programming notes.

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Study | Population | | | | |
| 30. | ITT-E | ES2 | Listing of Reasons for Maintenance Phase Withdrawal (Randomized Q4W) | | W124 |
| 31. | ITT-E | ES2 | Listing of Reasons for Extension Phase Withdrawal (Randomized Q4W) | | HL, W124 |
| 32. | ES | ES2 | Listing of Reasons for Extension Phase Withdrawal (Extension Switch Population) | | HL, W124 |
| 33. | LTFU | ES2 | Listing of Reasons for Long-term Follow Up Withdrawal | | W124 |
| 34. | ITT-E | CA3 | Listing of Concomitant ART Medications Received during the Maintenance and/or Extension Phase | | W124 |
| 35. | ITT-E | CA3 | Listing of Subjects with Changes in Concomitant ARTs during the Maintenance Phase and/or Extension Phase (Randomized Q4W) | | W124 |
| 36. | ES | CA3 | Listing of Subjects with Changes in Concomitant ARTs during the Extension Phase (Extension Switch Population) | | W124 |
| 37. | ITT-E | CA3 | Listing of ART Medications Received during LTFU Phase | | W124 |
| 38. | ES | Shell LSP11 | Listing of Investigational Product Accountability - Oral Regimens (Extension Switch Population) | | W124 |
| 39. | ITT-E | | Listing of Subjects with Hepatitis C at Induction Baseline (Week -20) | | W124 |
| Effica | су | | | | |
| 40. | CVF | Shell LSEF3 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | | W124 |

**Non-ICH: Listings** (Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). Listings will present data for the Randomized Q4W arm (data collected in any study phase, where applicable) and the Extension Switch Q4W arm (data collected in the Extension and LTFU phases, where applicable), unless otherwise stated in the programming notes.

| No. | · Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 41. | ITT-E | Shell LSEF1 | Listing of All Plasma HIV-1 RNA data for subjects with viral load >=50 c/mL at any time during the Maintenance and/or Extension Phase | | HL, W124 |
| 42. | ITT-E | Shell LSEF5 | Listing of HIV-1 Associated Conditions | | W124 |
| Safety | , | • | | | |
| 43. | Safety | See Listing 3 in<br>reporting effort:<br>gsk1265744/mi<br>d209522/iss_0<br>1 | Listing of all Subjects Meeting Liver Stopping Criteria | | W124 |
| 44. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | W124 |
| 45. | Safety | LIVER6 | Listing of Liver Event Information for RUCAM Score | | W124 |
| 46. | Safety | LIVER7 | Listing of Liver Biopsy Details | | W124 |
| 47. | Safety | LIVER8 | Listing of Liver Imaging Details | | W124 |
| 48. | Safety | Liver13 | Listing Subjects Meeting Hepatobiliary Lab Criteria | Please also add those additional items shown in the summary of subjects meeting hepatobiliary lab criteria post-baseline (i.e. AST >3xULN and ALP <2xULN and BIL >=2xULN]; ALT+AST>=xx) | W124 |
| 49. | Safety | AE8 | Listing of Adverse Events Related to Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses | | W124 |

**Non-ICH: Listings** (Global Programming Note: Include columns for phase, phase treatment, phase day, where data is collected in multiple phases). Listings will present data for the Randomized Q4W arm (data collected in any study phase, where applicable) and the Extension Switch Q4W arm (data collected in the Extension and LTFU phases, where applicable), unless otherwise stated in the programming notes.

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 50. | Safety | EG3 | Listing of ECG Values for Subjects with Adverse Events Related to Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses | | W124 |
| 51. | Safety | Latte2<br>WK96CDISC<br>report | Listing of Each Subjects ALT, AST, Bilirubin (including total and direct Bilirubin), INR, and ALP for subject meeting Hepatobiliary Lab abnormality criteria | 8.1037 (add AST, ALP, INR, and direct Bilirubin to the listing and only for subject meeting Hepatobiliary Lab abnormality criteria) | W124 |
| 52. | Safety | Latte2<br>WK96CDISC<br>report | Listing of Investigational Product Exposure Data for Subject Receiving Oral Bridging | 8.1038 | W124 |
| 53. | Safety | DEV1 | Listing of Dosing Errors and IP Device Malfunctions | | W124 |
| Virolo | gy (mock up bel | ow from study 200 | 0056\wk96cdisc), 'Study Phase' will be added as a column to t | he listing. | |
| 54. | CVF | Listing 9.1005 | Listing of Replication Capacity in IN and PR/RT Region | Show data in all phases for randomized Q4W IM and extension switch IM participants. | W124 |
| 55. | ITT-E | Table 9.1009 | Listing of Genotypic Mutation Data at All Timepoints | Show data in all phases for randomized Q4W IM and extension switch IM participants. | W124 |

#### 14.16. Appendix 16: IDMC

An IDMC was instituted to perform a triggered periodic review of the accumulating data based on confirmed virologic failures to ensure that subjects are not being sub-optimally treated. In addition, the IDMC will review a futility analysis when 50% of subjects will have reached their Week 24 visit. See full details of the analysis and decision criteria in the IDMC charter.

A list of outputs required for each IDMC analysis was provided in the IDMC Charter, Section 12.3, Appendix C.

Data handing methods and derived data definitions were provided in a separate critical components RAP.

#### 14.16.1. CVF Monitoring (Adhoc IDMC review)

The number of subjects meeting Confirmed Virologic Failure (CVF) Criterion per the protocol is being monitored and may result in adhoc IDMC data reviews.

The Statistics Data Analysis Centre (SDAC) is notified by the study virologist in writing every time a CVF occurs in either study. The SDAC will track the number of subjects past Week 4. The rate of CVF will be monitored against the thresholds specified in IDMC Charter Table 1 (See IDMC Charter, Section 3.5.2).

# 14.17. Appendix 17: Variables Defined for Time to Event Analysis

| Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| Participant met CVF event criteria during the Maintenance Phase (based on derived CVF) | CNSR=0 | EVNTDESC=CVF AVAL=Date of SVF* *immediately preceding CVF |
| 2. Participant with Maintenance Phase withdrawal due to 'Lack of Efficacy', 'Treatment related AE', 'intolerability due to injection', or 'protocol defined Safety stopping criteria' during Maintenance Phase Note: primary reason for discontinuation based on Maintenance Conclusion form in the eCRF. 'Treatment related AE' is defined as subjects that have primary reason for withdrawal = AE and that the participant has at least one AE considered drug related and leading to withdrawal/permanent discontinuation of investigational product. | CNSR=0 | EVNTDESC= terms in italic, respectively. For ABC/DTG/3TC arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, Study Day of Maintenance IP Stop Date + 1] For Q4W arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, max(Study Day of Last Q4W IM Dose + 35, Study Day of Last Oral CAB/RPV Dose + 1)] Note: Last Q4W IM / last oral dose/ Maintenance IP Stop Date is only applied to subjects who permanently discontinue from study treatment. Note: Date of Maintenance Phase discontinuation is from the Maintenance Phase Conclusion form in the eCRF. |
| If none of the above conditions met | | |
| Participant with Maintenance Phase withdrawal due to other reasons | CNSR=1 | EVNTDESC='Censored due to Study Discontinuation for Other Reasons' AVAL will be defined as the same as above 2 |
| Participant did not have premature withdrawal from the Maintenance Phase | CNSR=1 | EVNTDESC='Censored due to data cutoff for analysis' |

| Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| | | AVAL = Last on-treatment date during the Maintenance Phase, For ABC/DTG/3TC arm: min [Study Day of Week 100 Visit, Day of Last Contact at time of analysis, Study Day of Maintenance IP stop Date + 1] For Q4W arm min [Study Day of Week 100 Visit, Study Day of Starting LTFU HAART, Study Day of Last Contact Date at time of analysis, max(Study Day of Last Q4W IM Dose + 35, Study Day of Last oral CAB/RPV dose + 1)] |

Note: Last Q4W IM Dose & Last oral CAB/RPV dose is only applied to participants who permanently discontinue from study treatment.

The same approach as will be used to define 'ERDF', Efficacy-related discontinuation equals failure, except that the reason of withdrawal in Condition 2 will be restricted to 'Lack of Efficacy'.

### 14.18. Appendix 18: Japan-Specific Requirements

The following data displays will be produced to support reporting requirements for an expected regulatory submission in Japan.

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|---------------|---------------|
| Study Population | 11.01 to 11.n | 11.01 to 11.n |
| Efficacy | 12.01 to 12.n | 12.01 to 12.n |
| Safety | 13.01 to 13.n | 13.01 to 13.n |
| Pharmacokinetic | 14.01 to 14.n | 14.01 to 14.n |
| Health Outcomes | 15.01 to 15.n | 15.01 to 15.n |
| Section | Listings | |
| ICH Listings | 100 to y | |
| Other Listings | 200 to z | |

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided a separate document.

### 14.18.1. Study Population Tables - Japan

| Study Population Japan: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Demogr | aphy and Baseline | | | | |
| 11.1. | Intent-to-Treat<br>Exposed (Japan) | Shell TSP2 | Summary of Demographic Characteristics | See also DM1 in IDSL Age categorization will include: <=18, 19-64, >=65 (FDAAA requirement) 18-64, 65-84, >=85 (EMA requirement) | W48 Japan,<br>W96 Japan |

### 14.18.2. Efficacy Tables - Japan

| Efficacy Japan: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 12.1. | Intent-to-Treat<br>Exposed (Japan) | Shell TPEF1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48 Japan,<br>W96 Japan |
| 12.2. | Per-Protocol (Japan) | Shell TPEF1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA ≥50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis (Per-Protocol Population - Japan) | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48 Japan,<br>W96 Japan |

| Efficacy Japan: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 12.3. | Intent-to-Treat<br>Exposed (Japan) | Shell TPEF2 | Summary of Study Outcomes (50 c/mL cut-off) at Week 48 (Maintenance Phase) – Snapshot Analysis | For W96 deliverable, replace 'Week 48' with 'Week 96' | W48 Japan,<br>W96 Japan |

# 14.18.3. Safety Tables - Japan

| Safety Japan: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | se Events | | | | • |
| 13.1. | Safety (Japan) | AE1 | Summary of All Adverse Events by System<br>Organ Class – Maintenance Phase | CS Core | W48 Japan,<br>W96 Japan |
| 13.2. | Safety (Japan) | AE5B | Summary of All Adverse Events by System<br>Organ Class and Maximum Toxicity –<br>Maintenance Phase | CS Core | W48 Japan,<br>W96 Japan |
| 13.3. | Safety (Japan) | AE5B | Summary of All Adverse Events by System Organ Class and Maximum Toxicity – Oral Lead-in Period at Maintenance Phase | CS Core (for Q4W arm only) | W48 Japan,<br>W96 Japan |
| 13.4. | Safety (Japan) | AE3 | Summary of All Grade 3 or Higher Adverse<br>Events by Overall Frequency – Maintenance<br>Phase | | W48 Japan,<br>W96 Japan |
| 13.5. | Safety | AE3 | Summary of All Grade 3 or Higher Adverse<br>Events by Overall Frequency – Maintenance<br>Phase (Safety Population) | New | W48 Japan,<br>W96 Japan |

| Safety | Japan: Tables | | | | |
|---|---|---|---|---|---|
| 13.6. | Safety (Japan) | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class– Maintenance Phase | | W48 Japan,<br>W96 Japan |
| 13.7. | Safety (Japan) | AE5B | Summary of All Drug-Related Adverse Events by System Organ Class and Maximum Toxicity – Maintenance Phase | CS Core | W48 Japan,<br>W96 Japan |
| Serious | and Other Significan | t Adverse Ever | ts | | |
| 13.8. | Safety (Japan) | AE1 | Summary of Serious Adverse Events by<br>System Organ Class – Maintenance Phase | CS Core | W48 Japan,<br>W96 Japan |
| 13.9. | Safety (Japan) | AE1 | Summary of Drug-Related Serious Adverse<br>Events by System Organ Class – Maintenance<br>Phase | CS Core | W48 Japan,<br>W96 Japan |
| 13.10. | Safety (Japan) | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class– Maintenance Phase | CS Core | W48 Japan,<br>W96 Japan |
| Injectio | on Site Reaction Adve | rse Events | | | |
| 13.11. | Safety (Japan) | Shell TS2.2 | Summary of Injection Site Reaction Adverse<br>Events (Event-Level Summary) –Maintenance<br>Phase | (for Q4W arm only) | W48 Japan,<br>W96 Japan |
| 13.12. | Safety (Japan) | Shell TS2.3 | Summary of Subject-Level Characteristics of Injection Site Reaction Adverse Events – Overall and Common (Maintenance Phase) | Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects (for Q4W arm only) | W48 Japan,<br>W96 Japan |

### 14.18.4. Pharmacokinetic Tables - Japan

| Pharm | Pharmacokinetic Japan: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes The similar outputs below from study 200056 (week48idsl), unless otherwise specified | Deliverable<br>[Priority] |
| PK | | | | | |
| 14.1. | Japan PK | PKCT1 | Summary of Plasma CAB PK Concentrations (ug/mL) -Time Data (Q4W arm) – Day 1 | Day 1 (following first oral CAB dose during lead-in phase): Pre-dose, 1, 2, 3, 4, 8, and 24 hours post-dose | W48 Japan |
| 14.2. | Japan PK | PKCT1 | Summary of Plasma CAB PK Concentration (ug/mL) - Time Data by Visit (Q4W arm) – Week 4b to Week 48 | Table 10.1011 | Japan W48 |
| 14.3. | Japan PK | PKCT1 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL) -Time Data by Visit (Q4W arm) – Week 4b to Week 48 | Table 10.1011 | Japan W48 |
| 14.4. | Japan PK | PKCT1 | Summary of Plasma RPV PK Concentration (ng/mL) - Time Data by Visit (Q4W arm) – Week 4b to Week 48 | Table 10.1011 | Japan W48 |
| 14.5. | Japan PK | PKCT1 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Visit (Q4W arm) – Week 4b to Week 48 | Table 10.1011 | Japan W48 |
| 14.6. | Japan PK | PKPT4 | Summary of Derived Plasma CAB PK Parameters at Day 1 | GSK1265744/LAI117010,<br>Table 3.3 | |
### 14.18.5. Pharmacokinetic Figures - Japan

| Pharm | Pharmacokinetic Japan: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | | | | | |
| 14.1. | Japan PK | PKCF1P | Individual Plasma CAB Concentration-Time Plots by Subject (Linear and Semi-Log) – Day 1 | One plot per subject; Day 1 (following first oral CAB dose during lead-in phase): Predose, 1, 2, 3, 4, 8, and 24 hours post-dose | Japan W48 |
| 14.2. | Japan PK | PKCF1P | Individual Plasma CAB Concentration-Time Plots by Treatment (Linear and Semi-Log) – Day 1 | Overlay all subjects; Day 1 (following first oral CAB dose during lead-in phase): Predose, 1, 2, 3, 4, 8, and 24 hours post-dose | Japan W48 |
| 14.3. | Japan PK | PKCF1P | Individual Plasma CAB Concentration-Time Plots by Subject (Linear and Semi-Log) – Week 4b to Week 48 | One plot per subject | Japan W48 |
| 14.4. | Japan PK | PKCF1P | Individual Plasma CAB Concentration-Time Plots by Treatment (Linear and Semi-Log) – Week 4b to Week 48 | Overlay all subjects | Japan W48,<br>Japan W96 |
| 14.5. | Japan PK | PKCF1 | Individual Plasma RPV Concentration-Time Plots by Subject (Linear and Semi-Log) – Week 4b to Week 48 | One plot per subject | Japan W48,<br>Japan W96 |
| 14.6. | Japan PK | PKCF1 | Individual Plasma RPV Concentration-Time Plots by Treatment (Linear and Semi-Log) – Week 4b to Week 48 | Overlay all subjects | Japan W48,<br>Japan W96 |

| Pharma | Pharmacokinetic Japan: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 14.7. | Japan PK | PKCF2 | Mean (SD) Plasma CAB Concentration-Time<br>Plots (Linear and Semi-Log) – Day 1 | Figure 10.1003; Day 1 (following first oral CAB dose during lead-in phase): Predose, 1, 2, 3, 4, 8, and 24 hours post-dose | Japan W48, |
| 14.8. | Japan PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Plasma CAB<br>Concentration-Time Plots (Linear and Semi-Log)<br>– Day 1 | Figure 10.1004; Day 1 (following first oral CAB dose during lead-in phase): Predose, 1, 2, 3, 4, 8, and 24 hours post-dose | Japan W48 |
| 14.9. | Japan PK | PKCF2 | Mean (SD) Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Week 4b to Week 48 | Figure 10.1003 | Japan W48,<br>Japan W96 |
| 14.10. | Japan PK | PKCF3 | Median (5th and 95th percentile) Plasma CAB<br>Concentration-Time Plots (Linear and Semi-Log)<br>– Week 4b to Week 48 | Figure 10.1004 | Japan W48,<br>Japan W96 |
| 14.11. | Japan PK | PKCF2 | Mean (SD) Evaluable Plasma CAB Concentration-Time Plots (Linear and Semi-Log) – Week 4b to Week 48 | Figure 10.1003 | Japan W48,<br>Japan W96 |
| 14.12. | Japan PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Evaluable<br>Plasma CAB Concentration-Time Plots (Linear<br>and Semi-Log) – Week 4b to Week 48 | Figure 10.1004 | Japan W48,<br>Japan W96 |
| 14.13. | Japan PK | PKCF2 | Mean (SD) Plasma RPV Concentration-Time<br>Plots (Linear and Semi-Log) – Week 4b to Week<br>48 | Figure 10.1005 | Japan W48,<br>Japan W96 |
| 14.14. | Japan PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Plasma RPV<br>Concentration-Time Plots (Linear and Semi-Log)<br>– Week 4b to Week 48 | Figure 10.1006 | Japan W48,<br>Japan W96 |

| Pharma | Pharmacokinetic Japan: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 14.15. | Japan PK | PKCF2 | Mean (SD) Evaluable Plasma RPV Concentration-Time Plots (Linear and Semi-Log) – Week 4b to Week 48 | Figure 10.1007 Visits up to W52 for the W48 deliverable. | Japan W48,<br>Japan W96 |
| 14.16. | Japan PK | PKCF3 | Median (5 <sup>th</sup> and 95 <sup>th</sup> percentile) Evaluable<br>Plasma RPV Concentration-Time Plots (Linear<br>and Semi-Log) – Week 4b to Week 48 | Figure 10.1008 Visits up to W52 for the W48 deliverable. | Japan W48,<br>Japan W96 |

### 14.18.6. Health Outcomes Tables - Japan

| Health ( | Health Outcomes Japan: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable |
| Treatme | ent Satisfaction (HIV | TSQs) | | | |
| 15.1. | Intent-to-Treat<br>Exposed (Japan) | Shell THO2 | Proportion of Subjects with HIVTSQs – Treatment Satisfaction Individual Item Scores by Visit - LOCF) (Maintenance Phase) | | Japan W48,<br>Japan W96 |
| 15.2. | Intent-to-Treat<br>Exposed (Japan) | Shell THO1 | Summary of HIVTSQs - Total Treatment Satisfaction<br>Score by Visit - LOCF) (Maintenance Phase) | | Japan W48,<br>Japan W96 |
| 15.3. | Intent-to-Treat<br>Exposed (Japan) | Shell THO1 | Summary of HIVTSQs - Change from Maintenance<br>Baseline (Day 1) in Total Treatment Satisfaction<br>Score by Visit (Maintenance Phase) | | Japan W48,<br>Japan W96 |
| 15.4. | Intent-to-Treat<br>Exposed (Japan) | Shell THO1 | Summary of HIVTSQs - Change from Maintenance Baseline (Day 1) in Total Treatment Satisfaction Score by Visit - LOCF (Maintenance Phase) | | Japan W48,<br>Japan W96 |

| Health C | Health Outcomes Japan: Tables | | | |
|---|---|---|---|---|
| Treatme | ent Satisfaction (HIV | TSQc) | | |
| 15.5. | Intent-to-Treat<br>Exposed (Japan) | Shell THO2 | Proportion of Subjects with HIVTSQc – Treatment Satisfaction Individual Item Scores at Week 48 (Maintenance Phase) | Japan W48 |
| 15.6. | Intent-to-Treat<br>Exposed (Japan) | Shell THO1 | Summary of HIVTSQc - Total Treatment Satisfaction Score at Week 48 (Maintenance Phase) | Japan W48 |
| 15.7. | Intent-to-Treat<br>Exposed (Japan) | See Table 6.41 in<br>reporting effort:<br>gsk1265744/2015<br>84/primary_02 | Summary of HIVTSQc Individual Item Scores at Week 48 (Maintenance Phase) | Japan W48 |
| Preferer | Preferences (Dichotomous preference question) (for Q4W IM) | | | |
| 15.8. | Intent-to-Treat<br>Exposed (Japan) | Shell THO8 | Treatment Preference at Week 48 (Maintenance Phase) | Japan W48 |

### 14.18.7. ICH Listings - Japan

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic | | | | |
| 100. | All Enrolled (Japan) | AE8 | Listing of All Adverse Events (Induction + Maintenance Phase) | | Japan W48,<br>Japan W96 |
| 101. | All Enrolled (Japan) | Study 201584 (primary_02): Listing 33 | Listing of All Plasma HIV-1 RNA Data | | Japan W48,<br>Japan W96 |

### 14.18.8. Non-ICH Listings - Japan

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | Pharmacokinetic | | | | |
| 200. | Japan PK | PKPL1 | Listing of Derived Plasma CAB Pharmacokinetic Parameters – Day 1 | | Japan W48 |
| 201. | Japan PK | PKCL1 | Listing of Plasma CAB Pharmacokinetic Concentration Time Data | | Japan W48,<br>Japan W96 |
| 202. | Japan PK | PKCL1 | Listing of Plasma RPV Pharmacokinetic Concentration Time Data | | Japan W48,<br>Japan W96 |

# 14.19. Appendix 19: List of Data Displays for Subcutaneous Substudy Analysis

Unless otherwise specified, in sub-study analysis, age refers to the age at the sub-study screening, Baseline weight and Baseline BMI refer to the weight and BMI at the sub-study baseline respectively, and the listings will not be presented by prior exposure to CAB + RPV as the shell.

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology. The RAPIDO Data Viewer will be utilized in this study at SAC and will take the place of many previously produced listings.

#### 14.19.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.18 | |
| Efficacy | 2.1 to 2.20 | 2.1 to 2.4 |
| Safety | 3.1 to 3.75 | 3.1 to 3.13 |
| Pharmacokinetic | 4.1 to 4.12 | 4.1 to 4.8 |
| Health Outcomes | 6.1 to 6.21 | |
| Virology | 7.1 to 7.3 | |
| Section | Listings | |
| ICH Listings | 1 to 13 | |
| Other Listings | 14 to 20 | |

#### 14.19.2. Mock Example Shell Referencing

For all displays referring to A2M (207966), remove treatment arm distinction from all shells (i.e. Q4W vs. Q8W) unless otherwise specified.

#### 14.19.3. Deliverables

| Delivery [1] | Description |
|--------------|-----------------------------------|
| SS-ISR | Sub-study ISR Monitoring Interim |
| SS-Interim | Sub-study Week 9 Interim Analysis |
| SS-HL | Headline at Sub-study SAC |
| SS-SAC | Sub-study SAC |

### 14.19.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Subjec | Subject Disposition | | | | |
| 1.1 | Sub-study<br>Enrolled | 201584/primary_01/T1.2 | Summary of Sub-study Subjects Enrolled by Country and Site ID | Remove Induction Phase column. Do not include countries and sites without any subjects enrolled in the sub-study. | SS-Interim<br>SS-SAC |
| 1.2 | Sub-study<br>Screened | 207966/primary_46/T1.2 | Summary of Screening Status and Reasons for Sub-study Screening Failures | | SS-SAC |
| 1.3 | Sub-study<br>Screened | 201584/primary_01/T1.1 | Summary of Sub-study Populations | Remove Induction Phase column. Only include analysis populations used in the sub-study analysis | SS-SAC |
| 1.4 | Sub-study<br>Safety | 207966/primary_46/T1.3 | Summary of Subject Accountability: Substudy Conclusion Record | Include counts of those transitioned to marketed product | SS-SAC |
| 1.5 | Sub-study<br>Safety | 207966/primary_46/T1.4 | Summary of Subject Accountability: SC Injection Phase Conclusion Record | | SS-SAC |
| 1.6 | Sub-study<br>Safety | 207966/primary_46/T1.5 | Summary of Subject Accountability:<br>Return to Gluteal Injection Phase<br>Conclusion Record | | SS-SAC |
| 1.7 | Sub-study<br>Safety | 207966/primary_46/T1.6 | Summary of Subject Disposition at Each Study Phase | Replace Thigh Injection Phase with SC Injection Phase | SS-SAC |
| 1.8 | Sub-study<br>Safety | 207966/primary_46/T1.9 | Summary of Important Sub-study Protocol Deviations | | SS-SAC |
| 1.9 | Sub-study<br>Safety | 207966/primary_46/T1.10 | Summary of Important Sub-study Protocol Deviations (SC Injection Phase) | | SS-SAC |
| 1.10 | Sub-study<br>Safety | 207966/primary_46/T1.12 | Summary of Important COVID-19 Related Sub-study Protocol Deviations | | SS-SAC |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 1.11 | Sub-study<br>Safety | 207966/primary_46/T1.13 | Summary of Important Non-COVID-19<br>Related Sub-study Protocol Deviations | | SS-SAC |
| Demog | raphic and Baseli | ine Characteristics | | | |
| 1.12 | Sub-study<br>Safety | 207966/primary_46/T1.14 | Summary of Demographic Characteristics | After the continuous BMI parameter, add a categorical BMI parameter (BMI < 30 kg/m^2, >=30 kg/m^2) | SS-HL<br>SS-SAC |
| 1.13 | Sub-study<br>Safety | 207966/primary_46/T1.15 | Summary of Race and Racial Combinations | | SS-SAC |
| 1.14 | Sub-study<br>Safety | 207966/primary_46/T1.16 | Summary of Race and Racial Combinations Details | | SS-SAC |
| Medica | ations / Other | | | | |
| 1.15 | Sub-study<br>Safety | 207966/primary_46/T1.17 | Summary of Extent of Exposure to Study<br>Treatment including SOC Oral Bridging<br>Prior to the First SC Injection | Replace references to ATLAS/A2M with FLAIR. Include FLAIR Maintenance randomization assignments in the columns. | SS-SAC |
| 1.16 | Sub-study<br>Safety | 207966/primary_46/T1.18 | Summary of Concomitant Non-ART<br>Medication Ingredient Combinations by<br>Study Phase | Include columns for SC Phase, Return to Gluteal Phase, and Overall | SS-SAC |
| 1.17 | Sub-study<br>Safety | 207966/primary_46/T1.19 | Summary of Smoking Status at Sub-study Baseline | | SS-SAC |
| 1.18 | Sub-study<br>Safety | 207966/primary_46/T1.20 | Summary of COVID-19 Pandemic Visit Impacts in Sub-study | Only include visits in sub-study | SS-SAC |

#### 14.19.5. Efficacy Tables

Note: The following subgroups will be included in subgroup summaries: Age (<35; 35-<50; >=50), Sex at Birth (Female vs Male), Race/Ethnicity (White: Non-Hispanic, White: Hispanic, Black, Asian, Other), Sub-study Baseline BMI (<30, >=30).

| Efficac | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | Sub-study Safety | 207966/primary_46/T2.1 | Summary of Study Outcomes (50 c/mL Threshold) at Sub-study Week 12 – Snapshot Analysis | | SS-HL<br>SS-SAC |
| 2.2 | Sub-study Safety | 207966/primary_46/T2.2 | Summary of Study Outcomes (50 c/mL Threshold) at Sub-study Week 12 by Subgroup – Snapshot Analysis | | SS-SAC |
| 2.3 | Sub-study Safety | 207966/primary_46/T2.3 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Visit (SC Injection Phase) – Snapshot Analysis | Observed values to be displayed prior to Week 12 | SS-SAC |
| 2.4 | Sub-study Safety | 207966/primary_46/T2.4 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Subgroup and Visit (SC Injection Phase) – Snapshot Analysis | Observed values to be displayed prior to Week 12 | SS-SAC |
| 2.5 | Sub-study Safety | 207966/primary_46/T2.5 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (SC Injection Phase) – Snapshot Analysis | Observed values to be displayed prior to Week 12 | SS-SAC |
| 2.6 | Sub-study Safety | 207966/primary_46/T2.6 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit (SC Injection Phase) – Snapshot Analysis | Observed values to be displayed prior to Week 12 | SS-SAC |
| 2.7 | Sub-study Safety | 207966/primary_46/T2.7 | Summary of Change from Sub-study Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |
| 2.8 | Sub-study Safety | 207966/primary_46/T2.8 | Summary of Plasma HIV-1 RNA (log10 c/mL) by Visit (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |
| 2.9 | Sub-study Safety | 207966/primary_34/T2.25 | Cumulative Proportion of Subjects Meeting Confirmed Virology Failure Criteria by Visit (SC Injection + Return to Gluteal Injection Phase) | | SS-HL<br>SS-SAC |

| Efficac | y Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.10 | Sub-study Safety | 207966/primary_34/T2.27 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |
| 2.11 | Sub-study Safety | 207966/primary_46/T2.11 | Summary of Subjects per Viral Load Category by Visit (SC Injection Phase) | | SS-SAC |
| 2.12 | Sub-study Safety | 207966/primary_46/T2.12 | Summary of Change from Sub-study Baseline in CD4+<br>Cell Count (cells/mm^3) by Visit (SC Injection + Return<br>to Gluteal Injection Phase) | | SS-SAC |
| 2.13 | Sub-study Safety | 207966/primary_46/T2.13 | Summary of Change from Sub-study Baseline in CD4+<br>Cell Count (cells/mm^3) at Sub-study Week 12 by<br>Subgroup | | SS-SAC |
| 2.14 | Sub-study Safety | 207966/primary_46/T2.14 | Summary of CD4+ Cell Count (cells/mm^3) by Visit (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |
| 2.15 | Sub-study Safety | 207966/primary_46/T2.15 | Summary of Change from Sub-study Baseline in CD8+Cell Count (cells/mm^3) by Visit (SC Injection Phase) | | SS-SAC |
| 2.16 | Sub-study Safety | 207966/primary_46/T2.16 | Summary of CD8+ Cell Count (cells/mm^3) by Visit (SC Injection Phase) | | SS-SAC |
| 2.17 | Sub-study Safety | 207966/primary_46/T2.17 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit (SC Injection Phase) | | SS-SAC |
| 2.18 | Sub-study Safety | 207966/primary_46/T2.18 | Summary of HIV-1 Associated Conditions Including Recurrences (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |
| 2.19 | Sub-study Safety | 207966/primary_46/T2.19 | Summary of HIV-1 Associated Conditions Excluding Recurrences (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |

| Efficac | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.20 | Sub-study Safety | 207966/primary_46/T2.20 | Summary of HIV-1 Disease Progression from Sub-study<br>Baseline and/or Deaths (SC Injection + Return to<br>Gluteal Injection Phase) | | SS-SAC |

# 14.19.6. Efficacy Figures

| Efficacy | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | Sub-study Safety | 201584/primary_01/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (SC Injection Phase) – Snapshot Analysis | | SS-SAC |
| 2.2 | Sub-study Safety | 201584/primary_01/F2.3 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (SC Injection Phase) – Snapshot Analysis | | SS-SAC |
| 2.3 | Sub-study Safety | 201584/primary_01/F2.6 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Sub-study Visit – for CVF Subjects | Replace the first 2 footnotes with "First vertical reference line corresponds to the date of first SC injection." | SS-HL<br>SS-SAC |
| 2.4 | Sub-study Safety | 201584/primary_01/F2.8 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for Subjects Who are in the Category of 'HIV-1 RNA >=50 c/mL' at Sub-study Week 12 per Snapshot Algorithm | Replace the first 2 footnotes with "First vertical reference line corresponds to the date of first SC injection." | SS-SAC |

#### 14.19.7. Safety Tables

Note: The following subgroups will be included in subgroup summaries: Age (<35, 35-<50, >=50), Sex at Birth (Female vs Male), Race/Ethnicity (White: Non-Hispanic, White: Hispanic, Black, Asian, Other), Sub-study Baseline BMI (<30, >=30).

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Expos | sure | | , | | |
| 3.1 | Sub-study<br>Safety | 207966/primary_46/T3.1 | Summary of Extent of Exposure to Study<br>Treatment (SC Injection + Return to Gluteal<br>Injection Phase) | Add footnote: "Note: Overall exposure includes 35 days since the last Q4W injection." | SS-HL<br>SS-SAC |
| 3.2 | Sub-study<br>Safety | 207966/primary_46/T3.2 | Summary of Needle Length and Gauge for CAB Injection (SC Injection Phase) | | SS-SAC |
| 3.3 | Sub-study<br>Safety | 207966/primary_46/T3.3 | Summary of Needle Length and Gauge for RPV Injection (SC Injection Phase) | | SS-SAC |
| 3.4 | Sub-study<br>Safety | 207966/primary_34/T3.4 | Summary of Adherence to CAB/RPV<br>Injection Dosing Schedule (SC Injection<br>Phase) | | SS-SAC |
| 3.5 | Sub-study<br>Safety | 207966/primary_34/T3.5 | Summary of Adherence to CAB/RPV<br>Injection Dosing Schedule (SC Injection +<br>Return to Gluteal Injection Phase) | | SS-SAC |
| 3.6 | Sub-study<br>Safety | 207966/primary_34/T3.4 | Summary of Adherence to CAB/RPV<br>Injection Dosing Schedule by Subgroup<br>(SC Injection Phase) | Repeat Table 3.4 by subgroup | SS-SAC |
| Adver | rse Events | | | | |
| 3.7 | Sub-study<br>Safety | 213199/final_01/T3.9 | Adverse Event Overview by Study Phase and Overall | Do not include any LTFU information | SS-Interim<br>SS-HL<br>SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.8 | Sub-study<br>Safety | 213199/final_01/T3.11 | Summary of All Adverse Events by Study<br>Phase, System Organ Class, and<br>Maximum Toxicity | Repeat results for both study phases and overall. | SS-Interim<br>SS-HL<br>SS-SAC |
| 3.9 | Sub-study<br>Safety | 213199/final_01/T3.12 | Summary of All Adverse Events by Study<br>Phase, System Organ Class, and<br>Maximum Toxicity – Excluding Injection<br>Site Reactions | Repeat results for both study phases and overall. | SS-SAC |
| 3.10 | Sub-study<br>Safety | 213199/final_01/T3.11 | Summary of All Adverse Events by<br>Subgroup, System Organ Class, and<br>Maximum Toxicity | Repeat results for both study phases and overall. | SS-SAC |
| 3.11 | Sub-study<br>Safety | 213199/final_01/T3.15 | Summary of Common Adverse Events (>=5%) by Study Phase and Overall Frequency | Repeat results for both study phases and overall. | SS-SAC |
| 3.12 | Sub-study<br>Safety | 213199/final_01/T3.16 | Summary of Common Grade 2-5 Adverse<br>Events (>=1%) by Study Phase and Overall<br>Frequency | Repeat results for both study phases and overall. | SS-SAC |
| 3.13 | Sub-study<br>Safety | 213199/final_01/T3.19 | Summary of Drug-related Adverse Events by Study Phase, System Organ Class, and Maximum Toxicity | Repeat results for both study phases and overall. | SS-SAC |
| 3.14 | Sub-study<br>Safety | 213199/final_01/T3.22 | Summary of Drug-related Adverse Events<br>by Study Phase, System Organ Class, and<br>Maximum Toxicity – Excluding Injection<br>Site Reactions | Repeat results for both study phases and overall. | SS-SAC |
| 3.15 | Sub-study<br>Safety | 213199/final_01/T3.19 | Summary of Drug-related Adverse Events by Subgroup, System Organ Class, and Maximum Toxicity | Repeat results for both study phases and overall. | SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.16 | Sub-study<br>Safety | 213199/final_01/T3.24 | Summary of Common Grade 2-5 Drug-<br>Related Adverse Events (>=1%) by Study<br>Phase and Overall Frequency | Repeat results for both study phases and overall. | SS-SAC |
| 3.17 | Sub-study<br>Safety | 213199/final_01/T3.9 | Adverse Event Overview by Subgroup,<br>Study Phase and Overall | Repeat Table 3.7 by subgroup Do not include any LTFU information | SS-SAC |
| Seriou | us and Other S | Significant Adverse Events | | | |
| 3.18 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Serious Adverse Events by<br>Study Phase, System Organ Class, and<br>Maximum Grade | Repeat results for both study phases and overall. | SS-HL<br>SS-Interim<br>SS-SAC |
| 3.19 | Sub-study<br>Safety | 213199/final_01/T3.30 | Summary of Serious Adverse Events by<br>Study Phase, System Organ Class, and<br>Preferred Term (Number of Subjects and<br>Occurrences) | Repeat results for both study phases and overall. | SS-SAC |
| 3.20 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Serious Adverse Events by<br>Study Phase, System Organ Class, and<br>Maximum Grade – Excluding Injection Site<br>Reactions | Repeat results for both study phases and overall. | SS-SAC |
| 3.21 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Serious Adverse Events by<br>Subgroup, System Organ Class, and<br>Maximum Grade | Repeat results for both study phases and overall. | SS-SAC |
| 3.22 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Drug-related Serious Adverse<br>Events by Study Phase, System Organ<br>Class, and Preferred Term | Repeat results for both study phases and overall. | SS-SAC |
| 3.23 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by Study Phase, | Repeat results for both study phases and overall. | SS-HL<br>SS-Interim<br>SS-SAC |

| Safety | / Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | | | System Organ Class, and Maximum Grade | | |
| 3.24 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by Study Phase, System Organ Class, and Maximum Grade – Excluding Injection Site Reactions | Repeat results for both study phases and overall. | SS-SAC |
| 3.25 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Drug-related Serious Adverse Events by Subgroup, System Organ Class, and Preferred Term | Repeat results for both study phases and overall. | SS-SAC |
| 3.26 | Sub-study<br>Safety | 213199/final_01/T3.27 | Summary of Serious Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by Study Phase, System Organ Class, and Maximum Grade | Repeat results for both study phases and overall. | SS-SAC |
| 3.27 | Sub-study<br>Safety | 213199/final_01/T3.23 | Summary of Common (>=5%) Non-Serious<br>Adverse Events by Study Phase, System<br>Organ Class, and Preferred Term (Number<br>of Subjects and Occurrences) | Repeat results for both study phases and overall. | SS-SAC |
| Study | Drug Injection | Site Reaction Adverse Events | | | |
| 3.28 | Sub-study<br>Safety | 213199/final_01/T3.37 | Summary of Study Drug Injection Site<br>Reaction Adverse Events (Event-level<br>Summary) | Report Study Phase in the columns<br>Sort by CAB+RPV, CAB, RPV | SS-Interim<br>SS-HL<br>SS-SAC |
| 3.29 | Sub-study<br>Safety | 213199/final_01/T3.38 | Summary of Subject-level Characteristics of Study Drug Injection Site Reaction Adverse Events – Overall and Common | Report Study Phase in the columns<br>Sort by CAB+RPV, CAB, RPV<br>>=5% is common threshold | SS-Interim<br>SS-HL<br>SS-SAC |
| 3.30 | Sub-study | 213199/final_01/T3.39 | Summary of Study Drug Injection Site | Report Study Phase in the columns | SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Safety | | Reaction Adverse Events by Visit and Maximum Severity – Overall and Common in Sub-study | Sort by CAB+RPV, CAB, RPV >=5% is common threshold | |
| 3.31 | Sub-study<br>Safety | 213199/final_01/T3.37 | Summary of Study Drug Injection Site<br>Reaction Adverse Events by Subgroup<br>(Event-level Summary) - Overall and<br>Common | Report Study Phase in the columns Report only for CAB+RPV >=5% is common threshold | SS-SAC |
| 3.32 | Sub-study<br>Safety | 213199/final_01/T3.38 | Summary of Subject-level Characteristics of Study Drug Injection Site Reaction Adverse Events by Subgroup – Overall and Common | Report Study Phase in the columns Report only for CAB+RPV >=5% is common threshold | SS-SAC |
| 3.33 | Sub-study<br>Safety | 207966/primary_46/T3.27 | Summary of Maximum Study Drug Injection<br>Site Reaction Adverse Event Grade by<br>Needle Length & Categorical BMI (SC<br>Injection Phase) – Common (CAB) | Repeat results for each ISR, needle length, and BMI category within needle length (overall, >=30, <30) | SS-SAC |
| 3.34 | Sub-study<br>Safety | 207966/primary_46/T3.27 | Summary of Maximum Study Drug Injection<br>Site Reaction Adverse Event Grade by<br>Needle Length & Categorical BMI (SC<br>Injection Phase) – Common (RPV) | Repeat results for each ISR, needle length, and BMI category within needle length (overall, >=30, <30) | SS-SAC |
| 3.35 | Sub-study<br>Safety | 213199/final_01/T3.37 | Summary of High Impact Study Drug<br>Injection Site Reaction Adverse Events<br>(Event-level Summary) | Report Study Phase in the columns<br>Sort by CAB+RPV, CAB, RPV<br>Add footnote "Note: High Impact ISRs<br>include Grade 4 ISRs and Grade 3<br>ISRs of ulceration, secondary<br>infection, phlebitis, drainage, or sterile<br>abscess and may potentially lead to<br>pausing or stopping SC injections." | SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.36 | Sub-study<br>Safety | 213199/final_01/T3.38 | Summary of Subject-level Characteristics of High Impact Study Drug Injection Site Reaction Adverse Events | Report Study Phase in the columns Sort by CAB+RPV, CAB, RPV Add footnote "Note: High Impact ISRs include Grade 4 ISRs and Grade 3 ISRs of ulceration, secondary infection, phlebitis, drainage, or sterile abscess and may potentially lead to pausing or stopping SC injections." | SS-SAC |
| 3.37 | Sub-study<br>Safety | 213199/final_01/T1.15 | Summary of Dimensions of Select,<br>Measurable SC Injection Site Reaction<br>Adverse Events (Erythema, Redness,<br>Induration, & Swelling) | Report Study Phase in the columns<br>Sort by CAB+RPV, CAB, RPV<br>Report descriptive statistics of the<br>diameter and width (mm) of the ISRs. | SS-SAC |
| 3.38 | Sub-study<br>Safety | GSK3640254/208379/primary_01/T2.1 | Summary of the Posterior Probability that the True Rate of SC ISRs of Interest >0.05 after 50% of Subjects Initiate SC Injections | Keep the first and last statistical categories, use only one column for SC, update study info to align with FLAIR ISR monitoring criteria. | SS-ISR |
| Labor | atory: Chemis | stry and Hematology | | | |
| 3.39 | Sub-study<br>Safety | 207966/primary_46/T3.32 | Summary of Chemistry Changes from Substudy Baseline by Visit (SC Injection + Return to Gluteal Injection Phase) | Do not use lipid LOCF at interim, use actual values. Replace first footnote with "Note: Fasting data is shown for lipids and glucose." Use lipid LOCF at SS-SAC. | SS-Interim<br>SS-SAC |
| 3.40 | Sub-study<br>Safety | 207966/primary_46/T3.33 | Summary of Chemistry Values by Visit (SC Injection + Return to Gluteal Injection Phase) | Use Lipid LOCF at SS-SAC. | SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.41 | Sub-study<br>Safety | 207966/primary_46/T3.36 | Summary of Maximum Post Sub-study<br>Baseline Emergent Chemistry Toxicities<br>(SC Injection Phase) | | SS-SAC |
| 3.42 | Sub-study<br>Safety | 207966/primary_46/T3.34 | Summary of Hematology Changes from<br>Sub-study Baseline by Visit (SC Injection +<br>Return to Gluteal Injection Phase) | | SS-Interim<br>SS-SAC |
| 3.43 | Sub-study<br>Safety | 207966/primary_46/T3.35 | Summary of Hematology Values by Visit (SC Injection + Return to Gluteal Injection Phase) | | SS-SAC |
| 3.44 | Sub-study<br>Safety | 207966/primary_46/T3.37 | Summary of Maximum Post Sub-study<br>Baseline Emergent Hematology Toxicities<br>(SC Injection Phase) | | SS-SAC |
| Labor | atory: Urinalys | sis | | | |
| 3.45 | Sub-study<br>Safety | 207966/primary_46/T3.38 | Summary of Urinalysis Dipstick Results by Visit (SC Injection Phase) | | SS-SAC |
| 3.46 | Sub-study<br>Safety | 207966/primary_46/T3.39 | Summary of Urine Concentrations<br>Changes from Sub-study Baseline by Visit<br>(SC Injection Phase) | | SS-SAC |
| 3.47 | Sub-study<br>Safety | 207966/primary_46/T3.40 | Summary of Changes in Proteinuria Baseline Laboratory Result to Maximum Post Sub-study Baseline Laboratory Result (SC Injection Phase) | | SS-SAC |
| Labor | atory: Hepatol | piliary (Liver) | | | |
| 3.48 | Sub-study<br>Safety | 213199/final_01/T3.46 | Summary of Liver Stopping Event<br>Reporting (SC Injection Phase) | | SS-SAC |
| 3.49 | Sub-study | 207966/primary_46/T3.42 | Summary of Subjects Meeting | | SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| | Safety | | Hepatobiliary Abnormality Criteria (SC Injection Phase) | | |
| ECG | | | | | |
| 3.50 | Sub-study<br>Safety | 207966/primary_46/T3.43 | Summary of ECG Findings (SC Injection Phase) | | SS-SAC |
| 3.51 | Sub-study<br>Safety | 207966/primary_46/T3.44 | Summary of Change from Sub-study<br>Baseline in ECG values by Visit (SC<br>Injection Phase) | | SS-SAC |
| Vital S | Signs | | | | <u> </u> |
| 3.52 | Sub-study<br>Safety | 207966/primary_46/T3.47 | Summary of Change from Sub-study<br>Baseline in Vital Signs by Visit (SC<br>Injection Phase) | Include weight and BMI | SS-SAC |
| Adver | se Event of Sp | ecial Interest (AESI) | | | |
| 3.53 | Sub-study<br>Safety | 207966/primary_46/T3.48 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and Prior History of Depression, Anxiety and Suicidal Ideation at Screening (SC Injection Phase) | | SS-SAC |
| 3.54-<br>3.70 | Sub-study<br>Safety | 207966/primary_46/T3.50-3.66 | Summary of XXX Adverse Events of<br>Special Interest by System Organ Class<br>and Preferred Term (Number of Subjects<br>and Occurrence) – SC Injection Phase | | SS-SAC |
| 3.71 | Sub-study<br>Safety | 207966/primary_46/T3.67 | Summary of Characteristics of Adverse<br>Events of Special Interest – SC Injection<br>Phase | | SS-SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| COVIE | 0-19 Adverse | Event | | | |
| 3.72 | Sub-study<br>Safety | 213199/final_01/T3.11 | Summary of COVID-19 Adverse Events by Study Phase, System Organ Class, and Maximum Toxicity | Repeat results for both study phases and overall. | SS-SAC |
| 3.73 | Sub-study<br>Safety | 213199/final_01/T3.52 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | | SS-SAC |
| 3.74 | Sub-study<br>Safety | 213199/final_01/T3.53 | Summary of COVID-19 Additional<br>Assessments for Subjects with COVID-19<br>Adverse Events | | SS-SAC |
| 3.75 | Sub-study<br>Safety | 213199/final_01/T3.54 | Summary of COVID-19 Symptoms for<br>Subjects with COVID-19 Adverse Events | | SS-SAC |

# 14.19.8. Safety Figures

| Safety | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.1 | Sub-study<br>Safety | 207966/primary_34/F3.1 | Plot of Common Adverse Events and Relative Risk – SC vs. IM, Excluding Study Drug ISRs (SC Sub-study) | Only IM events occurring during the sub-study should be included. | SS-SAC |
| 3.2 | Sub-study<br>Safety | 207966/primary_34/F3.2 | Plot of Common Study Drug Injection Site Reaction<br>Adverse Events and Relative Risk – SC vs. IM (SC<br>Sub-study) | Only IM events occurring during the sub-study should be included. | SS-SAC |
| 3.3 | Sub-study<br>Safety | AE10 | Plot of Common Grade 1+ Injection Site Reaction<br>Adverse Events and Relative Risk Overall & by<br>Subgroup – SC vs. Pre-SC IM | Include ISRs from all SC injections and the first 3 IM injections of the parent study for each participant Report incidence rate ratios instead of risk ratios as mentioned in Section 8.6 | SS-SAC |
| 3.4 | Sub-study<br>Safety | AE10 | Plot of Common Grade 1+ Injection Site Reaction<br>Adverse Events and Relative Risk Overall & by<br>Subgroup – SC vs. Post-SC IM | Include ISRs from the first 2 SC injections and the 2 IM injections subsequent to SC dosing for each participant Report incidence rate ratios instead of risk ratios as mentioned in Section 8.6 | SS-SAC |
| 3.5 | Sub-study<br>Safety | AE10 | Plot of Common Grade 2+ Injection Site Reaction<br>Adverse Events and Relative Risk Overall & by<br>Subgroup – SC vs. Pre-SC IM | Include ISRs from all SC injections and the first 3 IM injections of the parent study for each participant Report incidence rate ratios instead of risk ratios as mentioned in Section 8.6 | SS-SAC |

| Safety F | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.6 | Sub-study<br>Safety | AE10 | Plot of Common Grade 2+ Injection Site Reaction<br>Adverse Events and Relative Risk Overall & by<br>Subgroup – SC vs. Post-SC IM | Include ISRs from the first 2 SC injections and the 2 IM injections subsequent to SC dosing for each participant Report incidence rate ratios instead of risk ratios as mentioned in Section 8.6 | SS-SAC |
| 3.7 | Sub-study<br>Safety | 207966/primary_34/F3.3 | Plot of Incidence of Sub-study Study Drug Injection Site Reaction Adverse Events by Visit (Overall and Common) – CAB and/or RPV | X-Axis timepoints to run from Screening to Week 20. Remove the second footnote. | SS-SAC |
| 3.8 | Sub-study<br>Safety | 207966/primary_34/F3.4 | Plot of Incidence of Sub-study Study Drug Injection Site Reaction Adverse Events by Visit (Overall and Common) – CAB X-Axis timepoints to run from Screening to Week 20. Remove the second footnote. | | SS-SAC |
| 3.9 | Sub-study<br>Safety | 207966/primary_34/F3.5 | Plot of Incidence of Sub-study Study Drug Injection Site Reaction Adverse Events by Visit (Overall and Common) – RPV | X-Axis timepoints to run from<br>Screening to Week 20.<br>Remove the second footnote. | SS-SAC |
| 3.10 | Sub-study<br>Safety | 207966/primary_34/F3.6 | Plot of Incidence of Sub-study Study Drug Injection Site Reaction Adverse Events by Subgroup and Visit – CAB and/or RPV | X-Axis timepoints to run from Screening to Week 20. Remove the second and third footnotes. | SS-SAC |
| 3.11 | Sub-study<br>Safety | 207966/primary_46/F3.2 | Scatter Plot of Maximum vs. Sub-study Baseline for ALT (SC Injection Phase) | | SS-SAC |
| 3.12 | Sub-study<br>Safety | 213199/final_01/F3.4 | Scatter Plot of Maximum Total Bilirubin vs. Maximum ALT – eDISH Plot (SC Injection Phase) | | SS-SAC |
| 3.13 | Sub-study<br>Safety | 207966/primary_46/F3.4 | Histogram of Timeliness of Injections (SC Injection Phase) | | SS-SAC |

#### 14.19.9. Pharmacokinetic Tables

Note: The following subgroups will be included in subgroup summaries: Age (<35; 35-<50; >=50), Sex at Birth (Female vs Male), Race/Ethnicity (White: Non-Hispanic, White: Hispanic, Black, Asian, Other), Sub-study Baseline BMI (<30, >=30).

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | Sub-study PK<br>Concentration | 208832/final_01/T4.3 | Summary of Sub-study Plasma Cabotegravir PK<br>Concentration (ug/mL)-Time Data by Study Phase and<br>Nominal Timepoint | | SS-Interim,<br>SS-SAC |
| 4.2 | Sub-study PK<br>Concentration | 208832/final_01/T4.4 | Summary of Sub-study Plasma Rilpivirine PK<br>Concentration (ng/mL)-Time Data by Study Phase and<br>Nominal Timepoint | | SS-Interim,<br>SS-SAC |
| 4.3 | Sub-study PK<br>Parameter | 207966/primary_46/T4.5 | Summary of Sub-study Derived Plasma CAB PK Parameters by Dosing Interval | Parameters included are AUC(0-Tau), CMax, TMax, and CTau. Dosing intervals will include Screening Gluteal injection, 1st SC injection, 2nd, SC injection, and last SC injection. CTau will be taken from concentration data at Day 1 (gluteal), Week 4, and Week 12 (SC) | SS-Interim,<br>SS-SAC |
| 4.4 | Sub-study PK<br>Parameter | 207966/primary_46/T4.6 | Summary of Sub-study Derived Plasma RPV PK Parameters by Dosing Interval | Same notes as 4.3. | SS-Interim,<br>SS-SAC |
| 4.5 | Sub-study PK<br>Concentration | 208832/final_01/T4.3 | Summary of Sub-study Plasma Cabotegravir PK<br>Concentration (ug/mL)-Time Data by Study Phase,<br>Subgroup, and Nominal Timepoint | Repeat 4.1 with subgroups | SS-SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.6 | Sub-study PK<br>Concentration | 208832/final_01/T4.4 | Summary of Sub-study Plasma Rilpivirine PK<br>Concentration (ng/mL)-Time Data by Study Phase,<br>Subgroup, and Nominal Timepoint | Repeat 4.2 with subgroups | SS-SAC |
| 4.7 | Sub-study PK<br>Parameter | 207966/primary_46/T4.5 | Summary of Sub-study Derived Plasma CAB PK Parameters by Subgroup & Dosing Interval | Repeat 4.3 with subgroups | SS-SAC |
| 4.8 | Sub-study PK<br>Parameter | 207966/primary_46/T4.6 | Summary of Sub-study Derived Plasma RPV PK Parameters by Subgroup & Dosing Interval | Repeat 4.4 with subgroups | SS-SAC |
| 4.9 | Sub-study PK<br>Parameter | 207966/primary_46/T4.7 | Statistical Analysis of Plasma CAB PK Parameters by Treatment in Sub-study | GMR will be calculated for AUC(0-Tau), CMax, and CTau for SC Injection 1 / Gluteal Injection, SC Injection 2 / Gluteal Injection and SC Injection 3 / Gluteal Injection Add footnote: "GMR taken from exponentiated log values output from an ANCOVA with fixed effects of Phase and Substudy Baseline BMI (<30, >=30) as a covariate and a random effect of subject." | SS-HL<br>SS-SAC |
| 4.10 | Sub-study PK<br>Parameter | 207966/primary_46/T4.8 | Statistical Analysis of Plasma RPV PK Parameters by Treatment in Sub-study | Same notes as 4.5. | SS-HL<br>SS-SAC |

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.11 | Sub-study PK<br>Concentration | GSK3739937/212548/final_01/T4.6 | Summary Results of SC Steady State CAB<br>Concentration Assessment | Model to begin with subcutaneous phase concentrations Day 1 – Week 12 | SS-SAC |
| 4.12 | Sub-study PK<br>Concentration | GSK3739937/212548/final_01/T4.6 | Summary Results of SC Steady State RPV Concentration Assessment | Same note as 4.7. | SS-SAC |

### 14.19.10. Pharmacokinetic Figures

| Pharmaco | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | Sub-study PK<br>Concentration | 207966/primary_46/F4.1 | Individual Plasma CAB Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Add to footnote: "The LLQ has been imputed for non-quantifiable values" | SS-SAC |
| 4.2 | Sub-study PK<br>Concentration | 207966/primary_46/F4.2 | Individual Plasma RPV Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Add to footnote: "The LLQ has been imputed for non-quantifiable values" | SS-SAC |
| 4.3 | Sub-study PK<br>Concentration | 207966/primary_46/F4.3 | Mean (SD) Evaluable Plasma CAB<br>Concentration-Time Plots (Linear and Semi-<br>Log) in Sub-study | Add to footnote: "The LLQ has been imputed for non-quantifiable values" | SS-Interim,<br>SS-SAC |
| 4.4 | Sub-study PK<br>Concentration | 207966/primary_46/F4.4 | Mean (SD) Evaluable Plasma RPV<br>Concentration-Time Plots (Linear and Semi-<br>Log) in Sub-study | Add to footnote: "The LLQ has been imputed for non-quantifiable values" | SS-Interim,<br>SS-SAC |
| 4.5 | Sub-study PK<br>Concentration | 207966/primary_46/F4.5 | Median (5th and 95th Percentile) Evaluable Plasma CAB Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Add to footnote: "The LLQ has been imputed for non-quantifiable values" | SS-Interim,<br>SS-SAC |
| 4.6 | Sub-study PK<br>Concentration | 207966/primary_46/F4.6 | Median (5th and 95th Percentile) Evaluable Plasma RPV Concentration-Time Plots (Linear and Semi-Log) in Sub-study | Add to footnote: "The LLQ has been imputed for non-quantifiable values" | SS-Interim,<br>SS-SAC |
| 4.7 | Sub-study PK<br>Parameter | 207966/primary_46/F4.7 | Geometric Mean Ratios and 90% Cls of<br>Plasma CAB PK Parameters in Sub-study by<br>Treatment and Comparison Type | The comparisons include First SC vs Gluteal, Second SC vs Gluteal and Last SC vs Gluteal. | SS-SAC |
| 4.8 | Sub-study PK<br>Parameter | 207966/primary_46/F4.8 | Geometric Mean Ratios and 90% Cls of<br>Plasma RPV PK Parameters in Sub-study by<br>Treatment and Comparison Type | Same notes as Figure 4.7. | SS-SAC |

#### 14.19.11. Health Outcomes Tables

Note: The following subgroups will be included in subgroup summaries: Age (<35; 35-<50; >=50), Sex at Birth (Female vs Male), Race/Ethnicity (White: Non-Hispanic, White: Hispanic, Black, Asian, Other), Sub-study Baseline BMI (<30, >=30).

Note: LOCF should not be used for any Health Outcomes table.

| Health ( | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| HIV Trea | HIV Treatment Satisfaction Questionnaire Status or Change Version (HIVTSQs, HIVTSQc) | | | | |
| 6.1 | Sub-study<br>Safety | 207966/primary_46/T6.1 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit in Sub-study | | SS-SAC |
| 6.2 | Sub-study<br>Safety | 207966/primary_46/T6.4 | Summary of HIVTSQs - Change in Individual Item Score in Sub-study | Replace Weeks 16 and 24/20 with 9 and 17 | SS-SAC |
| 6.3 | Sub-study<br>Safety | 207966/primary_46/T6.2 | Summary of HIVTSQs - Total Treatment Satisfaction Score by Visit in Sub-study | Replace Weeks 16 and 24/20 with 9 and 17 Add the footnote: "[1] Sub-study Week 9 and Sub-study Week 17 are compared with the Sub-study Baseline using Wilcoxon signed-rank test." | SS-SAC |
| 6.4 | Sub-study<br>Safety | 207966/primary_46/T6.3 | Summary of HIVTSQs - Change in Total Treatment Satisfaction Score in Sub-study | Replace Weeks 16 and 24/20 with 9 and 17. | SS-SAC |
| 6.5 | Sub-study<br>Safety | 207966/primary_46/T6.2 | Summary of HIVTSQs - Total Treatment<br>Satisfaction Score by Visit & Subgroup in Sub-<br>study | Repeat Table 6.3 by subgroup | SS-SAC |
| 6.6 | Sub-study<br>Safety | 207966/primary_46/T6.5 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Sub-study Week 9 (SC Injection Phase) | | SS-SAC |
| 6.7 | Sub-study<br>Safety | 207966/primary_46/T6.6 | Summary of HIVTSQc - Individual Item Change<br>Score at Sub-study Week 9 (SC Injection Phase) | Replace Week 16 with 9. | SS-SAC |

| Health ( | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.8 | Sub-study<br>Safety | 207966/primary_46/T6.7 | Summary of HIVTSQc - Total Treatment<br>Satisfaction Change Score at Sub-study Week 9<br>(SC Injection Phase) | Replace Week 16 with 9 | SS-SAC |
| Tolerab | ility of Injection | (NRS) | | | |
| 6.9 | Sub-study<br>Safety | 208832/final_01/T6.3 | Proportion of Subjects with Tolerability of Injection (NRS) Individual Item Scores by Visit in Sub-study | Replace Actual Relative Time values with Week -4, Week -3, Day 1, Week 1, Week 8, Week 9, Week 12, and Week 13 | SS-SAC |
| 6.10 | Sub-study<br>Safety | 208832/final_01/T6.4 | Summary of Tolerability of Injection (NRS) Scores by Visit in Sub-study | Replace Actual Relative Time values with same visits as Table 6.9 | SS-Interim<br>SS-SAC |
| 6.11 | Sub-study<br>Safety | 208832/final_01/T6.6 | Summary of Tolerability of Injection (NRS) Change from Baseline Scores by Visit in Sub-study | Replace Actual Relative Time values with same visits as Table 6.9 | SS-SAC |
| 6.12 | Sub-study<br>Safety | 208832/final_01/T6.4 | Summary of Tolerability of Injection (NRS) Scores by Visit & Subgroup in Sub-study | Repeat Table 6.10 by subgroup | SS-SAC |
| Percept | ion of Injection | (PIN) | | | |
| 6.13 | Sub-study<br>Safety | 208832/final_01/T6.2 | Proportion of Subjects with each individual item score in PIN by Visit and Item in Sub-study | Replace Day 8 with Week -3, Week 1, Week 9, and Week 13 | SS-SAC |
| 6.14 | Sub-study<br>Safety | 201584/primary_01/T6.2 | Summary of Perception of Injection (PIN) Questionnaire Results in Domain Scores and Individual Item Scores by Visit in Sub-study | Replace current visits with Week -3,<br>Week 1, Week 9, and Week 13<br>Remove p-value column | SS-SAC |
| 6.15 | Sub-study<br>Safety | 201584/primary_01/T6.4 | Summary of PIN Change from Baseline (Week -3) Results in Domain Scores and Individual Item Scores by visit in Sub-study | Replace current visits with Week -3, Week 1, Week 9, and Week 13 | SS-SAC |

| Health C | Health Outcomes Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 6.16 | Sub-study<br>Safety | 201584/primary_01/T6.2 | Summary of Perception of Injection (PIN) Questionnaire Results in Domain Scores and Individual Item Scores by Visit & Subgroup in Substudy | Questionnaire Results in Domain Scores and ndividual Item Scores by Visit & Subgroup in Sub- | |
| 6.17 | Sub-study<br>Safety | 201584/primary_01/T6.3 | Summary and Statistical Analysis of PIN in Domain Scores and Individual Item Scores by Visit in Substudy | Compare scores at Weeks 1, 9, and 13 to Baseline using the Wilcoxon Signed Rank test | SS-SAC |
| Preferer | nce | | | | |
| 6.18 | Sub-study<br>Safety | 207966/primary_46/T6.11 | Proportion of Subjects with Response to Each Individual Question in Preference SC Injection vs Gluteal Injection Questionnaire by Visit in Substudy | Replace Weeks 8/12 and 24/20 with 9 and 17. | SS-Interim<br>SS-HL<br>SS-SAC |
| 6.19 | Sub-study<br>Safety | 207966/primary_46/T6.11 | Proportion of Subjects with Response to Each Individual Question in Preference SC Injection vs Gluteal Injection Questionnaire by Visit & Subgroup in Sub-study | Repeat 6.18 by subgroup | SS-SAC |
| Reason | for Switch | | | | |
| 6.20 | Sub-study<br>Safety | 207966/primary_46/T6.11 | Proportion of Subjects with Response to Each Reason in the Reason for Switch to SC Questionnaire in Sub-study | Map question and responses based on questionnaire | SS-SAC |
| Interest | | | | | |
| 6.21 | Sub-study<br>Safety | 207966/primary_46/T6.11 | Proportion of Subjects with Each Response to the Interest in Home Administration Questionnaire in Sub-study | Map question and responses based on questionnaire | SS-SAC |

### 14.19.12. Virology Tables

If no data are available, Virology Tables will be displayed with "No data to report."

| Virology | Virology Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Genoty | pe & Phenotype | | | | 1 |
| 7.1 | Sub-study<br>Safety | 213199/final_01/T2.9 | Summary of the Prevalence of Treatment-Emergent Major Resistance Mutations of INI, NRTI, NNRTI and PI Class at time of CVF (SC Injection + Return to Gluteal Injection Phase) – Plasma Sample | | SS-SAC |
| 7.2 | Sub-study<br>Safety | 213199/final_01/T2.10 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the SC Injection or Return to Gluteal Injection Phase | | SS-SAC |
| 7.3 | Sub-study<br>Safety | 213199/final_01/T2.11 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Did Not Meet Confirmed Virologic Failure Criteria during the SC Injection or Return to Gluteal Injection Phase | | SS-SAC |

### 14.19.13. ICH Listings

| ICH Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | | | | |
| 1 | Sub-study<br>Screened | 207966/primary_46/L1 | Listing of Reasons for Screen Failure in Sub-study | | SS-SAC |
| 2 | Sub-study<br>Safety | 213199/final_01/L1 | Listing of Reasons for Sub-study<br>Withdrawal | | SS-SAC |
| 3 | Sub-study<br>Safety | 213199/final_01/L2 | Listing of Reasons for Study Drug<br>Discontinuation | | SS-SAC |
| 4 | Sub-study<br>Safety | 207966/primary_46/L4 | Listing of Important Protocol Deviations | | SS-SAC |
| 5 | Sub-study<br>Safety | 213199/final_01/L8 | Listing of Demographic Characteristics | | SS-SAC |
| Efficacy | 1 | | | | |
| 6 | Sub-study<br>Safety | 213199/final_01/L11 | Listing of Study Outcome (50 c/mL<br>Threshold) at Sub-study Week 12 –<br>Snapshot Analysis | | SS-SAC |
| Safety | | | | | |
| 7 | Sub-study<br>Safety | 207966/primary_46/L10 | Listing of Serious Adverse Events<br>and Reasons for Considering as a<br>Serious Adverse Event | | SS-SAC |
| 8 | Sub-study<br>Safety | 213199/final_01/L14 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | | SS-SAC |
| 9 | Sub-study | LB5A | Listing of all Laboratory Data for | | SS-SAC |

| ICH List | ICH Listings | | | | |
|---|---|---|---|---|---|
| | Safety | | Subjects with Any Value Outside<br>Normal Range | | |
| 10 | Sub-study<br>Safety | 207966/primary_46/L20 | Listing of ECG Values for Subjects with a Value of Potential Clinical Importance in Sub-study | | SS-SAC |
| 11 | Sub-study<br>Safety | 213199/final_01/L46 | Listing of All Vital Signs Results | Include Weight and BMI | SS-SAC |
| PK | | | | | |
| 12 | Sub-study PK<br>Concentration | 207966/primary_46/L21 | Listing of Plasma CAB PK<br>Concentration-Time Data | | SS-SAC |
| 13 | Sub-study PK<br>Concentration | 207966/primary_46/L22 | Listing of Plasma RPV PK<br>Concentration-Time Data | | SS-SAC |

### 14.19.14. Non-ICH Listings

| Non-ICH Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Study Population | | | | | |
| 14 | Sub-study<br>Safety | 213199/final_01/L31 | Listing of Concomitant ART Medications During the Sub-study | Only list ART medications that were concomitant at any time during the sub-study. | SS-SAC |
| 15 | Sub-study<br>Safety | 207966/primary_46/L30 | Listing of Transition to CAB + RPV LA Marketed Product Status | | SS-SAC |
| Efficacy | | | | | |
| 16 | Sub-study<br>Safety | 207966/primary_34/L35 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | | SS-SAC |
| Safety | | | | | |
| 17 | Sub-study<br>Safety | 207966/primary_34/L43 | Listing of Subjects Meeting Hepatobiliary Lab<br>Criteria (SC Injection + Return to Gluteal Injection<br>Phase) | Drop Treatment, Display by Phase | SS-SAC |
| PK | | | | | |
| 18 | Sub-study<br>PK<br>Parameter | 208832/final_01/L34 | Listing of Derived Plasma Cabotegravir PK Parameters by Sub-study Phase | Replace Treatment column with Phase/Dosing Interval | SS-SAC |
| 19 | Sub-study<br>PK<br>Parameter | 208832/final_01/L35 | Listing of Derived Plasma Rilpivirine PK Parameters by Sub-study Phase | Replace Treatment column with Phase/Dosing Interval | SS-SAC |

### 14.20. Appendix 20: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request.